# **Cover Page for Statistical Analysis Plan**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT03172494 |
| Sponsor trial ID: | NN9068-4148 |
| Official title of study: | A trial comparing the efficacy and safety of insulin degludec/liraglutide, insulin degludec, and liraglutide in Chinese subjects with type 2 diabetes inadequately controlled on oral antidiabetic drugs (OADs). |
| Document date: | 16 December 2019 |

IDegLira
Trial ID: NN9068-4148
Clinical Trial Report
Appendix 16.1.9

Date: 16 December 2019
Version: 1.0
Status: Final

# 16.1.9 Documentation of statistical methods

# List of contents

| Statistical analysis plan | Link |
|---------------------------|------|
| Statistical documentation | Link |

Redacted statistical analysis plan Includes redaction of personal identifiable information only.

Statistical Analysis Plan Trial ID: NN9068-4148 UTN: U1111-1154-6671 EudraCT No.: N/A


Date: Version: Status: Page:

23 September 2019 | Novo Nordisk Final

1 of 23

# **Statistical Analysis Plan**

**Trial ID: NN9068-4148** 

A trial comparing the efficacy and safety of insulin degludec/liraglutide, insulin degludec, and liraglutide in Chinese subjects with type 2 diabetes inadequately controlled on oral antidiabetic drugs (OADs)



This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.


Date: Version: Status: Page:

23 September 2019 | Novo Nordisk 1.0 Final 2 of 23

#### **Table of contents** Page

| Ta | ble of c | ontents | ••••• | | 2 |
|---|---|---|---|---|---|
| Li | st of ab | breviation | s | | 3 |
| 1 | Intro | Trial inf | formation | | 5 |
| | 1.2 | Scope o | f the statistical | al analysis plan | 5 |
| 2 | Statis | tical consi | derations | | 5 |
| | 2.1 | | | tion | |
| | 2.2 | Definiti | on of analysi | is sets | 7 |
| | 2.3 | | • | | |
| | | 2.3.1 | | y analysis | |
| | 2.4 | Seconda | | ts | |
| | | 2.4.1 | Confirma | atory secondary endpoints | 10 |
| | | 2.4.2 | | ve secondary endpoints | |
| | | | 2.4.2.1 | • • | |
| | | | 2.4.2.2 | Safety endpoints | 14 |
| | 2.5 | Pharma | cokinetic m | odelling | |
| 3 | Chan | ges to the | statistical an | nalyses planned in the protocol | 21 |
| 4 | Refer | ences | | | 23 |

Statistical Analysis Plan Trial ID: NN9068-4148 UTN: U1111-1154-6671 EudraCT No.: N/A


Date: Version: Status: Page:

23 September 2019 1.0

Final 3 of 23

Novo Nordisk

# List of abbreviations

ADA American Diabetes Association

AE adverse event

AGI α-glucosidase inhibitors ANCOVA analysis of covariance

BG blood glucose
BMI body mass index
CAS completer analysis set
CTR clinical trial report
CV coefficient of variation

DBL database lock
ECG electrocardiogram
EOT End of treatment
FAS full analysis set

FDA U.S. Food and Drug Administration

FPG fasting plasma glucose

FU follow-up

GLP-1 glucagon-like peptide-1 HbA<sub>1c</sub> glycosylated haemoglobin HDL high density lipoprotein

HOMA-β homeostatic model assessment IDegLira insulin degludec/liraglutide

IDeg insulin degludec

IDF International Diabetes Federation

ITT intention-to-treat
LDL low density lipoprotein
LLOQ lower limit of quantification

LOCF Last Observation Carried Forward MACE major adverse cardiovascular event

MAP modelling analysis plan MCMC Markov Chain Monte Carlo

MedDRA Medical Dictionary for Regulatory Activities
MMRM mixed model for repeated measurements

OAD oral antidiabetic drug PK pharmacokinetics PP per protocol

SAP statistical analysis plan SAS safety analysis set SD standard deviation

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 4 of 23 | |

SU sulphonylureas

T2DM type 2 diabetes mellitus

TEAEs treatment emergent adverse events

TTT treat-to-target
TZD thiazolidinedione
UNR upper normal range
UTN Universal Trial Number
VLDL very low density lipoprotein

Statistical Analysis Plan
Trial ID: NN9068-4148
UTN: U1111-1154-6671
EudraCT No.: N/A

Date: 23 September 2019
Version: 1.0
Status: Final


#### 1 Introduction

#### 1.1 Trial information

This is a 26 week, randomised, parallel three-arm, open-label, multi-centre, treat-to-target (TTT) confirmatory trial in Chinese subjects with T2DM inadequately controlled with metformin  $\pm$  one other OAD:  $\alpha$ -glucosidase inhibitors (AGI), sulphonylureas (SU), glinides and thiazolidinediones (TZD). The trial is comparing efficacy and safety of insulin degludec/liraglutide (IDegLira), insulin degludec (IDeg) and liraglutide, all in combination with Metformin. For further details please see the protocol.

#### 1.2 Scope of the statistical analysis plan

This Statistical Analysis Plan (SAP) is based on final Protocol version 5.0 (05-Dec-2016). The scope of this SAP is to add one sensitivity analysis for change from baseline in  $HbA_{1c}$  after 26 weeks of treatment and several sensitivity analyses for confirmatory secondary endpoints, and to perform other minor changes. For further details on the changes see section  $\underline{3}$ .

# 2 Statistical considerations

Novo Nordisk will analyse and report data from all sites together.

All analyses of efficacy and safety endpoints will be based on the full analysis set (FAS). The analysis of the primary endpoint and the confirmatory secondary endpoint, change from baseline in body weight after 26 weeks of treatment, will be repeated on the per-protocol (PP) analysis set and the completer analysis set (CAS) for sensitivity purposes. All efficacy endpoints will be summarised using the FAS and safety endpoints will be summarised using the safety analysis set (SAS).

The impact of protocol deviations and outliers may be investigated further in sensitivity analyses if deemed relevant.

Unless otherwise specified, all continuous measurements will be summarised descriptively at each visit by treatment using observed data. After 26 weeks of treatment, descriptive statistics will be presented based both on observed and last observation carried forward (LOCF) imputed data. Endpoints that are analysed untransformed and endpoints that are not formally analysed are summarised by the arithmetic mean, standard deviation (SD), median, and minimum and maximum value. Endpoints that are analysed log-transformed are summarised by the geometric mean and coefficient of variation (CV).

For measurements over time, mean values will be plotted to explore the trajectory over time. LOCF imputed data will be used as the basis for plotting data, if not otherwise specified. For endpoints that are analysed log-transformed, the geometric mean values will be plotted.

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 6 of 23 | |

A standard analysis of covariance (ANCOVA) model will be applied for the continuous primary and secondary endpoints. The model includes treatment and previous OAD treatment (metformin or metformin in combination with one other OAD) as fixed factors and the corresponding baseline value as covariate. In the following, this model will be referred to as the standard ANCOVA model.

Presentation of results from a statistical analysis will include the estimated mean treatment effects (Least Square Means [LSMeans]) for absolute values and change from baseline. In addition, estimated mean treatment difference (or ratio) will be presented together with the two-sided 95% confidence interval and corresponding two-sided p-value.

#### Handling of missing data

The expected percentage of missing data is around 15%. In accordance with industry guidance<sup>1</sup> endpoints will be assessed at frequent visits and also on subjects who withdraw prematurely. This will facilitate an analysis in accordance with ITT principles. Also, the combined information on frequent outcomes and information on reason for drop-out is assumed to account for the missing data anticipated.

If an assessment has been made both at screening (Visit 1) and randomisation (Visit 2), and if not otherwise specified, the value from the randomisation visit will be used as the baseline value. If the value measured at the randomisation visit is missing and the assessment also has been made at screening, then the screening value will be used as the baseline value.

Missing values (including intermittent missing values) will be imputed using the LOCF method. Subjects without data after randomisation will be included by carrying forward their baseline value. LOCF has been a standard approach in diabetes trials for many years, and was used as the primary analysis in both IDegLira and IDeg phase 3a trials. LOCF is considered to be an appropriate method in the context of TTT trials, where subjects after withdrawal typically continue their therapy using commercially available insulin. In previous TTT trials with IDegLira and IDeg, LOCF has generally provided similar results to alternative methods applied to handle missing data, such as repeated measures models and completer analyses. In this trial, similar sensitivity analyses will be made to examine the robustness of the LOCF method. The LOCF approach will also be used to impute missing values in CAS.

#### 2.1 Sample size calculation

The primary objective of this trial is to confirm the efficacy of IDegLira in controlling glycaemia as assessed by change from baseline in HbA<sub>1c</sub> after 26 weeks of treatment vs. IDeg and liraglutide, respectively. This is done by comparing the difference in change from baseline in HbA<sub>1c</sub> after 26 weeks of treatment to a non-inferiority margin of 0.4% for IDegLira vs. IDeg and to a superiority margin of 0.0% for IDegLira vs. liraglutide. The non-inferiority margin of 0.4% (absolute) was chosen in accordance with the FDA guidance<sup>1</sup>.

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 7 of 23 | |

A hierarchical testing procedure is applied. This is based on an a priori ordering of the null-hypotheses and testing them in this order using the two-sided 95% confidence interval approach until an insignificant result appears. Non-inferiority and superiority will thus be considered confirmed if the upper bound of the two-sided 95% confidence interval is below 0.4% and 0.0%, respectively. This is equivalent to using a one-sided test of size 2.5%, which means that the type 1 error rate is controlled at 2.5% (one-sided).

Formally, let D be the mean difference in change from baseline in  $HbA_{1c}$ . The null-hypotheses are given as:

- Non-inferiority:  $H_0$  D $\geq$ 0.40% against  $H_A$  D<0.40%, with an assumed mean difference in treatment of 0.0% and a standard deviation of 1.0%
- Superiority: H<sub>0</sub> D≥0.0% against H<sub>A</sub> D<0.0%, with an assumed mean difference in treatment of -0.3% and a standard deviation of 1.0%</li>

For evaluation of non-inferiority the PP-population is used for the sample size calculations, while the FAS is used for evaluation of superiority. It is assumed that 15% of the randomised subjects will be excluded from the PP analysis set. The above assumptions are based on experience from the phase 3a development programmes for IDegLira and IDeg. The sample size is determined using a t-statistic under the assumption of a one-sided test of size 2.5% for both the superiority and non-inferiority testing. Based on these assumptions a sample size of 720 patients results in a non-inferiority power of 98.1% and a superiority power of 90.7% i.e. the combined power for meeting the primary objective is 98.1% \* 90.7% = 89.0%. A sample size of 720 patients with a 15% drop-out rate and a 2:1:1 randomisation results in 306 PP patients in the IDegLira arm.

#### 2.2 Definition of analysis sets

The following analysis sets are defined in accordance with the ICH-E9 guidance<sup>2</sup>.

- Full Analysis Set (FAS): includes all randomised subjects. In exceptional cases, subjects may be eliminated from the full analysis set. In such cases the elimination will be justified and documented. The statistical evaluation of the FAS will follow the intention-to-treat (ITT) principle and subjects will contribute to the evaluation "as randomised".
- **Per-Protocol (PP) analysis set:** includes all subjects in the FAS who fulfils the following criteria:
  - Have not violated any inclusion criteria
  - Have not fulfilled any exclusion criteria
  - Have a non-missing HbA<sub>1c</sub> at screening or randomisation
  - Have at least one non-missing HbA<sub>1c</sub> after 12 weeks of exposure
  - Have at least 12 weeks of exposure

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 8 of 23 | |

Subjects will contribute to the evaluation "as treated".

- Safety Analysis Set (SAS): includes all subjects receiving at least one dose of the investigational product or comparator. Subjects in the safety set will contribute to the evaluation "as treated".
- Completer Analysis Set (CAS): includes all randomised subjects who have completed the trial. Subjects in the completer analysis set will contribute to the evaluation "as randomised".

Randomised subjects who are lost to follow up and where no exposure information of the investigational product or comparators is available after randomisation will be handled as unexposed.

Before data are released for statistical analysis, a review of all data will take place to identify protocol deviations that could potentially affect the results. Any decision to exclude any subject or observation from the statistical analysis is the joint responsibility of the members of the study group. The subjects or observations to be excluded, and the reasons for their exclusion must be documented and signed by those responsible before database lock. The subjects and observations excluded from analysis sets, and the reason for this, will be described in the clinical trial report.

## 2.3 Primary endpoint

The primary endpoint is defined as change from baseline in HbA<sub>1c</sub> after 26 weeks of treatment.

The change from baseline in  $HbA_{1c}$  after 26 weeks of treatment will be analysed using an ANCOVA model with treatment and previous OAD treatment (metformin  $\pm$  one other OAD) as fixed factors and baseline  $HbA_{1c}$  as covariate. Missing values after 26 weeks of treatment will be imputed applying LOCF using  $HbA_{1c}$  values at and after baseline.

Non-inferiority of IDegLira vs. IDeg will be considered as confirmed if the 95% confidence interval for the mean treatment difference lies entirely below 0.4%; equivalent to a one-sided test with significance level of 2.5%. Non-inferiority will be investigated on the FAS. Sensitivity analysis will be performed on the PP analysis set.

Superiority of IDegLira vs. liraglutide will be considered as confirmed if the 95% confidence interval for the mean treatment difference for change from baseline in  $HbA_{1c}$  lies entirely below 0.0%; equivalent to a one-sided test with significance level of 2.5%. Conclusion of superiority will be based on FAS. The primary objective will be fulfilled only if both non-inferiority of IDegLira vs. IDeg and superiority of IDegLira vs. liraglutide are confirmed.

In addition to the non-inferiority margin of 0.4% the upper bound of the confidence interval for the mean treatment difference of IDegLira vs. IDeg will also be compared to a 0.0% margin. This comparison is not part of the hierarchical testing procedure.

Statistical Analysis Plan
Trial ID: NN9068-4148
UTN: U1111-1154-6671
EudraCT No.: N/A

Date: 23 September 2019
Version: 1.0
Status: Final


#### 2.3.1 Sensitivity analysis

The primary analysis will be repeated on the PP analysis set and the CAS as sensitivity analysis. Furthermore, sensitivity analysis will be performed on FAS using the mixed model for repeated measurement (MMRM) to evaluate the sensitivity of using LOCF. All HbA<sub>1c</sub> values available post baseline at scheduled measurement times will be analysed in a linear mixed normal model using an unstructured residual covariance matrix for HbA<sub>1c</sub> measurements within the same subject. The model will include treatment, visit, and previous OAD treatment as fixed factors and baseline HbA<sub>1c</sub> as covariate. Interactions between visit and all factors and the covariate are also included in the model.

Further, a pattern mixture model approach, mimicking an ITT scenario will be applied. The imputation will follow the hypothesis being tested. i.e., when deriving the IDegLira vs. IDeg contrast the imputation in the IDegLira arm will be based on IDeg values, whereas for the IDegLira vs. liraglutide contrast the imputation in the IDegLira arm will be based on liraglutide values. Furthermore, 0.4% (absolute) will be added to the imputed values in the IDegLira arm for the non-inferiority comparison against IDeg to mimic a scenario where subjects discontinued from IDegLira treatment are assumed to be switched to a treatment inferior to IDeg. In other words: two imputation datasets will be made, one for IDegLira and IDeg and one for IDegLira and liraglutide. In the analyses, depending on the hypothesis being tested, the respective imputation dataset will be used and the third arm (from the other imputation dataset) will be kept in the model. The imputations for each hypothesis will be done as follows:

- In the first step intermittent missing values are imputed using a Markov Chain Monte Carlo (MCMC) method, in order to obtain a monotone missing data pattern. This imputation is done for each treatment group separately and 1000 copies of the dataset will be generated.
- In the second step, for each of the 1000 copies of the dataset, an analysis of variance model with previous OAD treatment as a fixed factor, and baseline HbA<sub>1c</sub> as a covariate is fitted to the change in HbA<sub>1c</sub> from baseline to 4 weeks (Visit 6) for a given comparator group only. The estimated parameters, and their variances, from this model are used to impute missing values at 4 weeks for subjects in the comparator and IDegLira treatment groups, based on previous OAD treatment and HbA<sub>1c</sub> at baseline.
- In the third step, for each of the 1000 copies of the dataset, missing HbA<sub>1c</sub> values at 8 weeks (Visit 10) are imputed in the same way as for 4 weeks. Now the imputations are based on an analysis of variance model with the same factors and the HbA<sub>1c</sub> values at baseline and 4 weeks as covariates, fitted to the comparator group.
- This stepwise procedure is then repeated sequentially over the available planned visits, adding one visit in each step until the last planned visit at 26 weeks (Visit 28).

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 10 of 23 | |

• For the comparison against IDeg, for each subject discontinued from treatment in the IDegLira treatment group, a value of 0.4% (absolute; the non-inferiority limit) is added to the change in HbA<sub>1c</sub> at 26 weeks.

For each of the complete data sets, the change from baseline to 26 weeks is analysed using an analysis of variance model with treatment and previous OAD treatment as fixed factors and baseline HbA<sub>1c</sub> value as a covariate.

The estimates and standard deviations for the 1000 data sets are pooled to one estimate and associated standard deviation using Rubin's rule<sup>3</sup>. From these pooled estimates the confidence interval for the treatment differences and the associated p-value are calculated.

The results of sensitivity analyses will be compared to the result of the standard ANCOVA method using LOCF for imputation of missing data. Any marked difference between the MMRM, the pattern mixture approach and ANCOVA LOCF approach regarding the estimated treatment difference will be commented upon in the CTR.

#### 2.4 Secondary endpoints

#### 2.4.1 Confirmatory secondary endpoints

The following two confirmatory endpoints will be tested for superiority of IDegLira vs. IDeg.

- Change from baseline in body weight after 26 weeks of treatment.
- Number of treatment emergent severe or BG confirmed hypoglycaemic episodes during 26 weeks of treatment.

The tests for superiority of the confirmatory secondary endpoints will be based on the FAS and will only be carried out if non-inferiority of IDegLira vs. IDeg and superiority of IDegLira vs. liraglutide with regards to the primary endpoint are confirmed.

In order to control the overall type I error on a 2-sided 5% level with regards to the secondary endpoints, a hierarchical testing procedure will be used. If superiority is confirmed with respect to change from baseline in body weight after 26 weeks of treatment the number of treatment emergent severe or BG confirmed hypoglycaemic episodes during 26 weeks of treatment will be tested for superiority.

Superiority for change from baseline in body weight will be considered confirmed if the upper bound of the two-sided 95% confidence interval for the estimated mean treatment difference (IDegLira minus IDeg) is strictly below zero or equivalently if the p-value for the one-sided test of

Statistical Analysis Plan
Trial ID: NN9068-4148
UTN: U1111-1154-6671
EudraCT No.: N/A

Date: 23 September 2019
Version: 1.0
Status: Final


is less than 2.5%, where D is the treatment difference.

The change from baseline in body weight after 26 weeks of treatment will be analysed using an ANCOVA model with treatment and previous OAD treatment (metformin  $\pm$  one other OAD) as fixed factors and baseline weight as covariate.

Similar sensitivity analyses as specified for the primary endpoint (ANCOVA on the PP analysis set and CAS; MMRM; the pattern mixture model similar to that described for HbA<sub>1c</sub>, but without added non-inferiority penalty) will be performed.

Superiority for hypoglycaemic episodes will be considered confirmed if the upper bound of the two-sided 95% confidence interval for the estimated mean treatment ratio (IDegLira vs. IDeg) is strictly below one or equivalently if the p-value for the one-sided test of

H0 RR≥1.0 against HA RR<1.0,

is less than 2.5%, where RR is the treatment rate ratio.

Number of treatment emergent severe or BG confirmed hypoglycaemic episodes during 26 weeks of treatment will be analysed using a negative binominal regression model with a log-link function and the logarithm of the time period in which a hypoglycaemic episode is considered treatment emergent as offset. The model will include treatment and previous OAD treatment as fixed factors.

As a sensitivity analysis, for withdrawn subjects, the number of episodes in the missing period (time of withdrawal to planned treatment emergent period [max of 27 weeks and longest treatment emergent time observed in the trial, in all 3 treatment arms]) will be imputed using a multiple imputation technique<sup>4</sup>. The first step (getting samples from the posterior distribution) is done once, for all three arms together. In the second step, the imputation will follow the hypothesis being tested. When deriving the IDegLira vs. IDeg treatment ratio the imputation will be based on an assumption that the event rates before and after withdrawal in both arms correspond to the event rate in the IDeg group. Similarly for the IDegLira vs liraglutide treatment ratio, the event rate before and after withdrawal is assumed to correspond to the event rate in the liraglutide arm. In other words: two imputation datasets will be made, one for IDegLira and IDeg and one for IDegLira and liraglutide. In the analyses, depending on the hypothesis being tested, the respective imputation dataset will be used and the third arm (from the other imputation dataset) will be kept in the model.

The imputation will be done as follows:

As a first step, a Bayes negative binomial model with the same fixed factors used in the original
confirmatory analysis model is fitted to the event rate data to obtain the posterior distribution of
model parameters.

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 12 of 23 | |

In the second step, based on the estimated parameters for comparator in this model, the number
of events in the missing period is imputed for all withdrawn subjects, i.e. pre and post
withdrawal event rates in the conditional distribution used for imputation are as for a given
comparator. Multiple copies (1000 copies) of a complete data set are generated by sampling
from the estimated distribution.

For each of the complete data sets, the number of events is analysed using a negative binomial model including the same fixed factors used in the original model.

The estimates and standard deviations for the 1000 data sets are pooled to one estimate and associated standard deviation using Rubin's rule<sup>3</sup>. From these pooled estimates the confidence interval for the treatment ratio and the associated p-value are calculated.

Subjects with missing exposure time will not contribute to the analysis.

#### 2.4.2 Supportive secondary endpoints

## 2.4.2.1 Efficacy endpoints

In the following the statistical models will be fitted to all data simultaneously (all treatment groups) and from this model the treatment differences for IDegLira vs. IDeg and IDegLira vs. liraglutide will be estimated. For insulin dose, the model will be fitted only to data from the IDegLira and IDeg treatment groups.

#### Insulin dose after 26 weeks of treatment

The actual daily insulin dose after 26 weeks of treatment will be analysed using an ANCOVA model including treatment and previous OAD treatment as fixed factors and baseline HbA<sub>1c</sub> value as covariate.

#### Responder for HbA<sub>1c</sub> after 26 weeks of treatment

Two dichotomous endpoints (responder/non-responder) will be defined based on whether a subject has met a specific target level after 26 weeks of treatment:

- ADA HbA<sub>1c</sub> target (HbA<sub>1c</sub> < 7.0%)
- International Diabetes Federation (IDF)  $HbA_{1c}$  target ( $HbA_{1c} \le 6.5\%$ )

Analysis of each of the two responder endpoints will be based on a logistic regression model with treatment and previous OAD treatment as fixed factors and baseline  $HbA_{1c}$  value as a covariate.

#### HbA<sub>1c</sub> responder endpoints without weight gain

Responder for  $HbA_{1c}$  without weight gain after 26 weeks of treatment will be defined as  $HbA_{1c} < 7.0\%$  or  $\le 6.5\%$  at end of treatment and change from baseline in body weight below or

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 13 of 23 | |

equal to zero. Analysis of each of the two responder endpoints will be based on a logistic regression model with treatment and previous OAD treatment as fixed factors and baseline  $HbA_{1c}$  and body weight values as covariates.

#### HbA<sub>1c</sub> responder endpoints without hypoglycaemic episodes

Responder for  $HbA_{1c}$  without hypoglycaemic episodes after 26 weeks of treatment will be defined as  $HbA_{1c} < 7.0\%$  or  $\le 6.5\%$  at end of treatment and without severe or BG confirmed episodes during the last 12 weeks of treatment. Analysis of each of the two responder endpoints will be based on a logistic regression model with treatment and previous OAD treatment as fixed factors and baseline  $HbA_{1c}$  values as a covariate.

#### HbA<sub>1c</sub> responder endpoints without hypoglycaemic episodes and weight gain

Responder for  $HbA_{1c}$  without hypoglycaemic episodes and weight gain after 26 weeks of treatment will be defined as  $HbA_{1c} < 7.0\%$  or  $\le 6.5\%$  at end of treatment, without severe or BG confirmed episodes during the last 12 weeks of treatment, and change from baseline in body weight below or equal to zero. Analysis of each of the two responder endpoints will be based on a logistic regression model with treatment and previous OAD treatment as fixed factors and baseline  $HbA_{1c}$  and body weight values as covariates.

## Fasting plasma glucose (FPG)

Change from baseline in FPG after 26 weeks of treatment will be analysed using the standard ANCOVA model.

#### Waist circumference

Change from baseline in waist circumference after 26 weeks of treatment will be analysed using the standard ANCOVA model.

#### Beta-cell function (fasting insulin, fasting C-peptide, fasting glucagon, and HOMA-β)

In addition to fasting insulin, fasting C-peptide, and fasting glucagon, one derived parameter will be calculated; beta-cell function (HOMA- $\beta$ ). The calculation of the HOMA endpoint will be done as follows:

• Beta-cell function (%) =  $20 \cdot \text{fasting insulin} \left[ \mu U/mL \right] / (FPG[mmol/L] - 3.5)$ 

These endpoints after 26 weeks of treatment will be analysed separately using the standard ANCOVA model. In these statistical analyses the endpoint will be log-transformed and so will the baseline covariate.

Statistical Analysis Plan
Trial ID: NN9068-4148
UTN: U1111-1154-6671
EudraCT No.: N/A

Date: 23 September 2019 Version: 1.0
Status: Final


### Fasting lipid profile

Cholesterol, LDL cholesterol, HDL cholesterol, VLDL cholesterol, triglycerides, and free fatty acids after 26 weeks of treatment will be analysed separately using the standard ANCOVA model. In these statistical analyses the endpoint will be log-transformed and so will the baseline covariate.

#### Self-measured plasma glucose 9-point profile

Three endpoints from the 9-point profile will be defined:

- 9-point profile
- Mean of the 9-point profile, defined as the area under the profile (calculated using the trapezoidal method) divided by the measurement time
- Post-prandial plasma glucose increments (from before meal to 90 min after for breakfast, lunch and dinner). The mean increment over all meals will be derived as the mean of all available meal increments

A mixed effect model will be fitted to the 9-point profile data. The model will include treatment, previous OAD treatment, time, interaction between treatment and time, and interaction between previous OAD treatment and time as fixed factors, and subject as random effect, where measurements within subjects will be assumed correlated with a compound symmetry covariance matrix. From the model mean profile by treatment and relevant treatment differences will be estimated and explored.

Change from baseline after 26 weeks of treatment in mean of the 9-point profile and post-prandial increment endpoints will be analysed separately using the standard ANCOVA model.

#### 2.4.2.2 Safety endpoints

#### Adverse events

AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) coding.

A treatment emergent adverse event (TEAE) is defined as an event that has onset date on or after the first day of exposure to randomised treatment and no later than seven days after the last day of randomised treatment. If the event has onset date before the first day of exposure on randomised treatment and increases in severity during the treatment period and until 7 days after the last drug date, then this event should also be considered as a TEAE. Major adverse cardiovascular events (MACEs, defined as all cardiovascular deaths, non-fatal myocardial infarctions and non-fatal strokes) are considered treatment-emergent until 30 calendar days after the last dose of trial product.

TEAEs are summarised descriptively, whereas non-TEAEs are presented in listings. TEAE data will be displayed in terms of the number of subjects with at least one event (N), the percentage of

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 15 of 23 | |

subjects with at least one event (%), the number of events (E) and the event rate per 100 years of exposure (R).

Summaries of TEAEs and of serious TEAEs will be presented as an overview including all AEs, AEs by seriousness, AEs by severity, AEs by relation to treatment, technical complaint AEs and AEs by outcome (including deaths).

Furthermore, summary tables based on system organ class and preferred terms are made for:

- All TEAEs
- TEAEs leading to withdrawal
- Serious TEAEs
- Possibly or probably related TEAEs
- Severe, moderate and mild TEAEs
- TEAEs reported by safety areas of interest
- TEAEs with preferred term that are experienced by at least 5% of the subjects in any treatment arm or by at least 5% of all subjects

A listing for non-TEAEs with onset date before the first day of exposure to randomised treatment will be presented. A listing will also be presented for non-TEAEs collected after the treatment emergent period according to the definition of TEAE.

#### Classification of Hypoglycaemia

**Treatment emergent:** hypoglycaemic episodes will be defined as treatment emergent if the onset of the episode occurs on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.

**Nocturnal hypoglycaemic episodes:** are episodes with time of onset between 00:01 and 05.59 both inclusive.

Hypoglycaemic episodes are classified according to the Novo Nordisk classification of hypoglycaemia (see <u>Figure 2–1</u>) and the ADA classification of hypoglycaemia (see <u>Figure 2–2</u>).

#### Novo Nordisk classification of hypoglycaemia

In normal physiology, symptoms of hypoglycaemia occur below a plasma glucose level of 3.1 mmol/L.<sup>5</sup> Therefore, Novo Nordisk has included hypoglycaemia with plasma glucose levels below this cut-off point in the definition of BG confirmed hypoglycaemia.

Novo Nordisk uses the following classification (see <u>Figure 2–1</u>) in addition to the ADA classification (see <u>Figure 2–2</u>):

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 16 of 23 | |

- Severe or BG confirmed symptomatic hypoglycaemia: An episode that is severe according to the ADA classification<sup>6</sup> or BG confirmed by a plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia.
- Severe or BG confirmed hypoglycaemia: An episode that is severe according to the ADA classification<sup>6</sup> or BG confirmed by a plasma glucose value <3.1 mmol/L with or without symptoms consistent with hypoglycaemia.



Note: Glucose measurements are performed with capillary blood calibrated to plasma equivalent glucose values

 $\operatorname{BG}$ : blood glucose  $\operatorname{PG}$ : plasma glucose  $\operatorname{SMPG}$ : Self-measured plasma glucose

Figure 2–1 Novo Nordisk classification of hypoglycaemia

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 17 of 23 | |

# ADA classification of hypoglycaemia<sup>6</sup>

- Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
- Asymptomatic hypoglycaemia: An episode not accompanied by typical symptoms of hypoglycaemia, but with a measured plasma glucose concentration ≤ 3.9 mmol/L.
- Documented symptomatic hypoglycaemia: An episode during which typical symptoms of hypoglycaemia are accompanied by a measured plasma glucose concentration ≤ 3.9 mmol/L.
- Pseudo-hypoglycaemia: An episode during which the person with diabetes reports any of the typical symptoms of hypoglycaemia with a measured plasma glucose concentration
   3.9 mmol/L but approaching that level.
- Probable symptomatic hypoglycaemia: An episode during which symptoms of hypoglycaemia are not accompanied by a plasma glucose determination but that was presumably caused by a plasma glucose concentration ≤ 3.9 mmol/L.



Note: Glucose measurements are performed with capillary blood calibrated to plasma equivalent glucose values PG: plasma glucose SMPG: Self-measured plasma glucose

Figure 2–2 ADA classification of hypoglycaemia

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 18 of 23 | |

Data on treatment emergent hypoglycaemic episodes are presented in terms of the number of subjects with at least one event (N), the percentage of subjects with at least one event (%), the number of events (E) and the event rate per 100 years (R).

Separate summaries are made for severe or BG confirmed hypoglycaemic episodes, severe or BG confirmed symptomatic hypoglycaemic episodes, nocturnal severe or BG confirmed hypoglycaemic episodes, nocturnal severe or BG confirmed symptomatic hypoglycaemic episodes and the ADA classification of hypoglycaemia.

The number of hypoglycaemic episodes during 26 weeks of treatment will be analysed separately for each endpoint using a negative binomial regression model with a log-link function and the logarithm of the time period in which a hypoglycaemic episode is considered treatment emergent as offset. The model will include treatment and previous OAD treatment at fixed factors.

#### **Pulse**

Change from baseline in pulse after 26 weeks of treatment will be analysed using the standard ANCOVA model

#### Systolic and diastolic blood pressure

Change from baseline in systolic and diastolic blood pressure after 26 weeks of treatment will be analysed using the standard ANCOVA model.

#### Clinical evaluations (physical examination, eye examination and ECG)

Eye examination (dilated fundoscopy/fundus photography) and ECG findings will be summarised descriptively, including:

- Summaries
- The change from baseline after 26 weeks of treatment

Any clinically significant deterioration of a pre-existing condition after the screening visit, as well as any new clinically significant findings will be recorded as adverse events.

#### Laboratory assessments

All laboratory parameters will be summarised descriptively. The following tables will be presented based on both observed and LOCF imputed data:

- Shift tables from baseline to after 26 weeks of treatment.
- Proportion of subjects with measurements outside reference range by treatment and week.

Laboratory values for lipase, amylase and calcitonin will be presented graphically as box plots by treatment and week.

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 19 of 23 | |

For each laboratory parameter, individual values outside the reference ranges (abnormal values) will be listed

For lipase and amylase the following rule applies in the evaluation of the result:

• If the amylase or lipase baseline (at screening) value is > 3xUNR the information will be recorded as medical history for that subject.

#### Calcitonin

The purpose of the calcitonin analysis is to evaluate longitudinal changes in calcitonin, with main focus on subjects who develop persistently high levels of calcitonin during the trial.

Calcitonin will be displayed in terms of the number of subjects (N), the percentage of subjects (%) and the event rate per 100 years of exposure (R). The following criteria are defined for tabulations:

#### • Persistent (all post baseline measurements)

- From < UNR to persistently  $\ge$  UNR
- From < UNR to persistently  $\ge 1.5$  UNR
- From < UNR to persistently  $\ge 20 \text{ ng/L}$
- From < UNR to persistently  $\ge 50 \text{ ng/L}$
- From < 20 ng/L to persistently  $\ge 20 \text{ ng/L}$
- From < 50 ng/L to persistently  $\ge 50 \text{ ng/L}$

# • Incidental (at least one post baseline measurements)

- From  $\leq$  UNR to  $\geq$  UNR
- From < UNR to  $\ge 1.5$  UNR
- From < UNR to  $\ge 20$  ng/L
- From < UNR to  $\ge 50$  ng/L
- From  $\leq 20 \text{ ng/L to} \geq 20 \text{ ng/L}$
- From  $< 50 \text{ ng/L to} \ge 50 \text{ ng/L}$

The distribution of all calcitonin measurements across treatment groups and time will be shown with box plots and corresponding cumulative plots for actual levels of calcitonin and change from baseline. The plots will be presented by treatment group at EOT using LOCF imputed values and within treatment group by week. Plots will be done by each gender, separately.

Summaries tables of calcitonin continuous measurements, will include number and percentage of observations < and  $\ge$  LLOQ, minimum, Q25, median, Q75 and maximum. Summaries will be presented for all subjects and by gender.

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 20 of 23 | |

Longitudinal changes for subjects with calcitonin levels  $\geq 20$  ng/l will be plotted (longitudinal plots). The plots will be done by treatment and gender. They will be done for subjects in the persistent and incidental categories, separately.

A listing of subjects with at least one post baseline value  $\geq 20$  ng/l will be done. The listing will include age, gender, calcitonin measurements over time and AE history (including preferred term, onset and stop dates).

#### Urinalysis

Categorical urinalysis parameters will be summarised descriptively by:

- Shift from baseline to EOT (using the number of subjects in the different categories).
- Subjects with at least one post baseline measurement outside reference range will be listed.

#### **Insulin and GLP-1 antibodies**

Insulin antibodies (IDeg specific, cross-reacting to human insulin and total) will be summarised with arithmetic mean, standard deviation (SD), median, and minimum and maximum value by treatment and treatment week, and their mean over time will be plotted. Correlations will be explored graphically as follows. Insulin antibodies (IDeg specific, cross-reacting to human insulin and total) will be plotted against  $HbA_{1c}$  after 26 weeks,  $HbA_{1c}$  change from baseline after 26 weeks, and dose after 26 weeks. Change from baseline to FU1 in insulin antibodies (IDeg specific, cross-reacting to human insulin and total) will be plotted against  $HbA_{1c}$  after 26 weeks,  $HbA_{1c}$  change from baseline after 26 weeks, and dose after 26 weeks.

GLP-1 antibodies (liraglutide specific, cross-reacting to native GLP-1, liraglutide *in vitro* neutralising and *in vitro* neutralising to native GLP-1) will be summarised by number of subjects (N) and percentage of subjects (%) with positive and negative samples.

#### 2.5 Pharmacokinetic modelling

#### Population pharmacokinetic analysis

The objective for this analysis is to compare the pharmacokinetics of IDegLira and its individual components at clinically relevant doses during 26 weeks of treatment. Furthermore, dose-proportionality of IDeg and liraglutide exposures following doses of IDegLira will be evaluated and the effects of pre-specified covariates on exposures of IDeg and liraglutide will be investigated. Pharmacokinetic samples for IDeg and liraglutide sampled at site visits will be included in the analysis. No pre-defined time of day is specified for the sampling, but the date and exact clock time of sampling will be recorded by the investigator. The subjects must be instructed to write in their

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 21 of 23 | |

diary the date, exact clock time, dose, and injection site of the previous three days of dosing as well as the dose on the day of the visit, if taken before PK blood sampling.

The population PK analysis will be performed by the Quantitative Clinical Pharmacology Department at Novo Nordisk. A more technical and detailed elaboration of the population PK analysis will be given in the modelling analysis plan (MAP) which will be finalised before DBL.

The pre-specified analysis will explore the effects of covariates on the IDeg and liraglutide exposure. The structural models and covariate relationships will be predefined in detail in the MAP. In brief, previously developed population PK models for IDeg and liraglutide will be used. For both PK models, the absorption rate constant (Ka) will be fixed and the apparent clearance (CL/F) and the apparent volume of distribution (Vd/F) will be estimated.

The covariates of interest will be evaluated using criteria which will be specified in the MAP.

The following covariates will be tested on the apparent clearance (CL/F):

- Dose
- Treatment (IDegLira, IDeg, liraglutide)
- Injection site area (Abdomen, Upper arm, Thigh)
- Body weight
- Age group ( $< 65, \ge 65$  years)
- Gender (Male/Female)

For the categorical variables, it is a requirement to have at least 20 subjects in each category.

#### **Exposure-response analysis**

The exposure-response relationship will be investigated for selected response variables, such as HbA<sub>1c</sub>. Individual drug concentration data will be tabulated in the CTR.

The population PK and exposure-response analyses will be reported in a separate modelling report, which will not be a part of the CTR.

# 3 Changes to the statistical analyses planned in the protocol

- Additional sensitivity analysis was added, using the pattern mixture model, in order to evaluate
  the sensitivity of using LOCF for primary endpoint, change from baseline in HbA<sub>1c</sub> after 26
  weeks of treatment.
- Sensitivity analyses for confirmatory secondary endpoint, change from baseline in body weight after 26 weeks of treatment, were added to evaluate the sensitivity of using LOCF.

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 22 of 23 | |

- Sensitivity analysis for confirmatory secondary endpoint, number of treatment emergent severe or BG confirmed hypoglycaemic episodes during 26 weeks of treatment, was added to evaluate the sensitivity of the analysis specified in the protocol.
- A minor correction regarding the analysis model for the supportive secondary endpoint of 9-point self-measured plasma glucose was made (baseline value was removed from the model and interaction between previous OAD and time was added).
- Box plots will only be presented for relevant laboratory assessments: lipase, amylase and calcitonin.
- Listings deemed unnecessary were removed: antibody measurements, physical examination findings.
- Minor editorial changes were made, and clarifications were added where considered relevant.

| Statistical Analysis Plan | Date: | 23 September 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.: N/A | Page: | 23 of 23 | |

# 4 References

- 1. Food and Drug Administration, CDER. Guidance for Industry. Diabetes Mellitus: Developing Drugs and Therapeutic Biologics for Treatment and Prevention, Draft Guidance. February 2008.
- 2. ICH Harmonised Tripartite Guideline. Statistical Principles for Clinical Trials E9, Current Step 4 version. 05 Feb 1998.
- 3. Little RJA, Rubin DB. Statistical analysis with missing data. New York: Wiley. 1987. xiv, 278 p.
- 4. Keene ON, Roger JH, Hartley BF, Kenward MG. Missing data sensitivity analysis for recurrent event data using controlled imputation. Pharmaceutical Statistics. 2014;13(4):258-64.
- 5. Schwartz NS, Clutter WE, Shah SD, Cryer PE. Glycemic thresholds for activation of glucose counterregulatory systems are higher than the threshold for symptoms. J Clin Invest. 1987;79(3):777-81.
- 6. Seaquist ER, Anderson J, Childs B, Cryer P, Dagogo-Jack S, Fish L, et al. Hypoglycemia and diabetes: a report of a workgroup of the American Diabetes Association and the Endocrine Society. Diabetes Care. 2013;36(5):1384-95.

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 1 of 412 | |

# **Table of contents**

| | Page |
|---|---|
| 1: Actual daily total insulin dose after 26 weeks of treatment - supportive statistical analysis - full analysis set | 3 |
| 2: HbA1c after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set | 5 |
| 3: HbA1c after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set | 15 |
| 4: HbA1c after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set | 25 |
| 5: HbA1c after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM full analysis set | |
| 6: HbA1c after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set | 59 |
| 7: HbA1c after 26 weeks of treatment – change from baseline – supportive statistical analysis – full analysis set | 87 |
| 8: Responder for HbA1c treatment target - supportive statistical analysis - full analysis set | 97 |
| 9: Responder for HbA1c treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes - supportive statistical analysis - full analysis set | 101 |
| 10: Responder for HbA1c treatment target without weight gain - supportive statistical analysis - full analysis set | 105 |
| 11: Responder for HbA1c treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes and weight gain - supportive statistical analysis - full analysis set | 109 |
| 12: Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis full analysis set | |
| 13: Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set | 123 |
| 14: Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set | 133 |
| 15: Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set | 143 |
| 16: Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set | 167 |
| 17: Waist circumference after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set | |
| 18: Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical | 200 |
| 19: 9-point self-measured plasma glucose profile after 26 weeks of treatment - supportive statistical | 209 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019<br>1.0<br>Final<br>2 of 412 | Novo Nordisk |
|---|---|---|---|---|
| 20: Mean of 9-point self-measure baseline - supportive statistic | d plasma glucose profile after 2<br>al analysis - full analysis set | | _ | 277 |
| 21: Prandial increment after 26 w change from baseline - suppo | eeks of treatment - 9-point self-<br>ortive statistical analysis - full a | | | 287 |
| 22: Fasting insulin after 26 weeks | of treatment - supportive statis | tical analysis - f | full analysis set | 327 |
| 23: Fasting C-peptide after 26 we | eks of treatment - supportive sta | atistical analysis | s - full analysis set | 330 |
| 24: Fasting glucagon after 26 wee | eks of treatment - supportive sta | tistical analysis | - full analysis set | 336 |
| 25: HOMA-B after 26 weeks of tr | reatment - supportive statistical | analysis - full a | nalysis set | 339 |
| 26: HDL cholesterol after 26 wee | ks of treatment - supportive stat | tistical analysis | - full analysis set | 342 |
| 27: LDL cholesterol after 26 week | ks of treatment - supportive stat | istical analysis - | - full analysis set | 348 |
| 28: VLDL cholesterol after 26 we | eks of treatment - supportive st | atistical analysi | s - full analysis set | 354 |
| 29: Triglycerides after 26 weeks of | of treatment - supportive statistic | cal analysis - fu | ll analysis set | 360 |
| 30: Total cholesterol after 26 wee | ks of treatment - supportive stat | tistical analysis | - full analysis set | 366 |
| 31: Free fatty acid after 26 weeks | of treatment - supportive statist | tical analysis - f | ull analysis set | 372 |
| 32: Hypoglycaemic episodes - tre | atment emergent - confirmatory | statistical anal | ysis - full analysis se | t378 |
| 33: Hypoglycaemic episodes - tre - full analysis set | atment emergent - statistical ser | , , | 1 1 | |
| 34: Hypoglycaemic episodes - tre | atment emergent - supportive st | tatistical analysi | s - full analysis set | 389 |
| 35: Nocturnal hypoglycaemic epi-<br>analysis set | sodes - treatment emergent - su | | | 392 |
| 36: Pulse after 26 weeks of treatmanalysis set | nent - change from baseline - su | 1 1 | • | 398 |
| 37: Systolic blood pressure after 2 | | from baseline - | supportive statistical | |
| 38: Diastolic blood pressure after | | from baseline - | - supportive statistica | ıl |

| NN9068 | | Date: | 16 December 2019 1 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 3 of 412 | |

#### **Statistical documentation**

# 1: Actual daily total insulin dose after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=TOTDDAC

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtpn 2 1 2

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 6
Columns in Z 0
Subjects 1
Max Obs per Subject 530

Number of Observations

Number of Observations Read 540 Number of Observations Used 530 Number of Observations Not Used 10

Covariance Parameter Estimates

Cov Parm Estimate Residual 156.79

Fit Statistics

-2 Res Log Likelihood 4173.3 AIC (Smaller is Better) 4175.3 AICC (Smaller is Better) 4175.3 BIC (Smaller is Better) 4179.6

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t| Alpha 9.5426 5.5886 0.0883 0.05 526 1.71 Intercept -5.4917 -4.73 0.05 trtpn 1.1603 526 <.0001 trtpn PREOAD2 Metformin -0.8080 1.1686 526 -0.69 0.4896 0.05 PREOAD2 Metformin + OAD 2.5256 0.6569 526 3.84 0.0001 0.05 HBA1CBL

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 4 of 412 | |

Actual daily total insulin dose after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=TOTDDAC

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn | | 1 2 | -1.4362<br>-7.7712 | 20.5213<br>-3.2123 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | _ | -3.1038 | 1.4877 |
| HBA1CBL | Meclormin ( OAD | | 1.2352 | 3.8160 |

trtpn Treatment contrast, IDegLira - IDeg 0.000422

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 1 | 526 | 22.40 | <.0001 |
| PREOAD2 | 1 | 526 | 0.48 | 0.4896 |
| HBA1CBL | 1 | 526 | 14.78 | 0.0001 |

#### Least Squares Means Estimates

Standard

0.04027

| Effect | Label | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | | | 0.6640<br>0.9504 | | | <.0001<br><.0001 | 0.05<br>0.05 |
| | | Least Squ | ares Means | s Estimates | | | | |
| Effect | Label | Lower | Upper H | Exponentiated | Expon | entiated<br>Lower | Exponentia<br>Up | |
| trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg | 23.3095 2<br>28.2385 3 | | | | 1.328E10<br>1.836E12 | 1.804<br>7.684 | |
| | Least Squares Means Estimate | | | | | | | |
| Effect | Label | | Margins | s Estima | | andard<br>Error | DF t Va | lue |
| trtpn | Treatment contrast, | IDegLira - IDe | g WORK.AI | DATA2 -5.49 | 17 | 1.1603 | 526 -4 | .73 |
| | | Least Sq | uares Mear | ns Estimate | | | | |
| Effect | Label | | Pr > t | t Alpha | Lower | Upper | Exponentia | ted |
| trtpn | Treatment contrast, | IDegLira - IDe | g <.000 | 0.05 - | 7.7712 | -3.2123 | 0.004 | 121 |
| | Leas | t Squares Means | Estimate | | | | | |
| | | | _ | ntiated Exp | | + 3 | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 5 of 412 | |

# 2: HbA1c after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values
TRTPN 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.5548

Fit Statistics

-2 Res Log Likelihood 1635.3 AIC (Smaller is Better) 1637.3 AICC (Smaller is Better) 1637.3 BIC (Smaller is Better) 1641.9

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t| Alpha 0.2879 0.06796 4.5634 715 715 <.0001 0.05 15.85 Intercept TRTPN -0.6283 -9.25 <.0001 0.05 TRTPN -0.03366 0.07869 715 -0.43 0.6690 0.05 TRTPN PREOAD2 Metformin -0.3922 0.05944 715 -6.60 <.0001 0.05 PREOAD2 Metformin + OAD 0.3338 0.03413 715 9.78 <.0001 0.05 BASE

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 6 of 412 | |

HbAlc after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=C64849B

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>TRTPN<br>TRTPN<br>TRTPN | | 1<br>2<br>3 | 3.9982<br>-0.7618<br>-0.1882 | 5.1287<br>-0.4949<br>0.1208 |
| PREOAD2 | Metformin<br>Metformin + OAD | | -0.5089 | -0.2755 |
| BASE | 110010111111111111111111111111111111111 | | 0.2668 | 0.4008 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| TRTPN | 2 | 715 | 60.69 | <.0001 |
| PREOAD2 | 1 | 715 | 43.53 | <.0001 |
| BASE | 1 | 715 | 95.66 | <.0001 |

#### Least Squares Means Estimates

| | | | | Standard | | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
| TRTPN | LSMeans, IDegLira | WORK.ADATA2 | 6.5559 | | 715 | 167.18 | <.0001 | 0.05 |
| TRTPN<br>TRTPN | LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2 | 7.1506<br>7.1842 | | 715<br>715 | 128.29<br>129.40 | <.0001<br><.0001 | 0.05 |
| | | Least Sq | uares Mean | s Estimates | | | | |
| Effect | Label | Lower | Upper | Exponentiated | Expon | entiated<br>Lower | Exponentia<br>Up | ted<br>per |
| TRTPN | LSMeans, IDegLira | 6.4789 | 6.6329 | 703.38 | | 651.26 | 759 | .68 |
| TRTPN | LSMeans, IDeg | 7.0412 | 7.2600 | 1274.85 | | 1142.71 | 1422 | |
| TRTPN | LSMeans, Lira | 7.0752 | 7.2933 | 1318.50 | | 1182.33 | 1470 | .34 |
| | | Least Squ | uares Mean | s Estimates | | | | |
| | | | | | St | andard | | |
| Effect | Label | | Margin | s Estima | te | Error | DF t Va | lue |
| TRTPN | Treatment contrast | . IDegLira - IDe | eg WORK.A | DATA2 -0.59 | 47 0 | .06819 | 715 -8 | 3.72 |
| | | Least Squ | uares Mean | s Estimates | | | | |
| Effect | Label | | Pr > | t Alpha | Lower | Upper | Exponentia | ited |
| TRTPN | Treatment contrast | . IDegLira - IDe | eg <.00 | 01 0.05 - | 0.7286 | -0.4608 | 0.5 | 517 |

| пттссс | дарсі | | 11 / 101 | Атрпа | HOWCI | opper | Баропенстасса |
|---|---|---|---|---|---|---|---|
| TRTPN | Treatment contrast, | IDegLira - IDeg | <.0001 | 0.05 | -0.7286 | -0.4608 | 0.5517 |
| | T | + G | | | | | |

#### Least Squares Means Estimates

| Effect | Label | | | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| TRTPN | Treatment of | contrast, | IDegLira - | - IDeg | 0.4826 | 0.6308 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date: 16 D<br>Version:<br>Status:<br>Page: | ecember 2019 Novo Nordisk 1.0 Final 7 of 412 |
|---|---|---|---|
| HbAlc after 26 weeks of treatment analysis set | ent - change from baseline - | confirmatory statistic | al analysis - full |
| Parameter Code=C64849B | | | |
| The Mixed Procedure | | | |
| | Least Squares Means Estima | tes | |
| Effect Label | Margins | Standard<br>Estimate Error | DF t Value |
| TRTPN Treatment contrast, IDe | egLira - Lira WORK.ADATA2 | -0.6283 0.06796 | 715 -9.25 |
| | Least Squares Means Estima | tes | |
| Effect Label | Pr > t Alp | ha Lower Upper | Exponentiated |
| TRTPN Treatment contrast, IDe | egLira - Lira <.0001 0. | 05 -0.7618 -0.4949 | 0.5335 |
| Least So | quares Means Estimates | | |
| Effect Label | Exponentiated Lower | Exponentiated<br>Upper | |
| TRTPN Treatment contrast, IDe | egLira - Lira 0.4668 | 0.6096 | |

# NN9068 NN9068-4148 Clinical Trial Report Statistical document Date: 16 December 2019 Version: 1.0 Status: Final 

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

TRTPN 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate Residual 66.2773

Fit Statistics

-2 Res Log Likelihood 5060.0 AIC (Smaller is Better) 5062.0 AICC (Smaller is Better) 5066.5 BIC (Smaller is Better) 5066.5

Solution for Fixed Effects

Planned

Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 34.2233 Intercept 2.3673 715 14.46 <.0001 0.05 TRTPN -6.8678 0.7428 715 -9.25 < .0001 0.05 2 0.6690 TRTPN -0.3679 0.8601 715 -0.43 0.05 TRTPN 3 -4.2869 PREOAD2 0.6497 715 -6.60 <.0001 0.05 Metformin Metformin + OAD PREOAD2 BASE 0.3338 0.03413 715 9.78 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 9 of 412 | |

HbAlc after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>TRTPN<br>TRTPN<br>TRTPN | | 1<br>2<br>3 | 29.5757<br>-8.3262<br>-2.0566 | 38.8709<br>-5.4094<br>1.3207 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -5.5625 | -3.0113 |
| BASE | | | 0.2668 | 0.4008 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| TRTPN | 2 | 715 | 60.69 | <.0001 |
| PREOAD2 | 1 | 715 | 43.53 | <.0001 |
| BASE | 1 | 715 | 95.66 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| TRTPN<br>TRTPN<br>TRTPN | LSMeans, I<br>LSMeans, I<br>LSMeans, L | Deg | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2<br>Least Squ | 48.1560<br>54.6559<br>55.0238<br>wares Means | 0.4286<br>0.6092<br>0.6068<br>Estimates | 715<br>715<br>715 | 112.35<br>89.72<br>90.67 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| TRTPN | LSMeans, IDegLira | 47.3145 | 48.9975 | 8.201E20 | 3.535E20 | 1.903E21 |
| TRTPN | LSMeans, IDeg | 53.4599 | 55.8519 | 5.454E23 | 1.649E23 | 1.804E24 |
| TRTPN | LSMeans, Lira | 53.8324 | 56.2152 | 7.88E23 | 2.394E23 | 2.594E24 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| TRTPN | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -6.4999 | 0.7453 | 715 | -8.72 |

#### Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| TRTPN | Treatment contrast, | IDegLira - IDeg | <.0001 | 0.05 | -7.9631 | -5.0367 | 0.001504 |

#### Least Squares Means Estimates

| Effect | Label | | | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| TRTPN | Treatment | contrast, | IDegLira - | IDeg | 0.000348 | 0.006495 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date: 16 D<br>Version:<br>Status:<br>Page: | 1.0 Final 10 of 412 |
|---|---|---|---|
| HbAlc after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set | | | |
| Parameter Code=HBA1CONV | | | |
| The Mixed Procedure | | | |
| Leas | st Squares Means Estimate | es | |
| Effect Label | Margins E | Standard<br>stimate Error | DF t Value |
| TRTPN Treatment contrast, IDegLira | - Lira WORK.ADATA2 | -6.8678 0.7428 | 715 -9.25 |
| Leas | st Squares Means Estimate | es | |
| Effect Label | Pr > t Alpha | a Lower Upper | Exponentiated |
| TRTPN Treatment contrast, IDegLira | - Lira <.0001 0.0 | 5 -8.3262 -5.4094 | 0.001041 |
| Least Squares | Means Estimates | | |
| Effect Label | Exponentiated Lower | Exponentiated<br>Upper | |
| TRTPN Treatment contrast, IDegLira | - Lira 0.000242 | 0.004474 | |


 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

TRTPN 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.5548

Fit Statistics

-2 Res Log Likelihood 1635.3 AIC (Smaller is Better) 1637.3 AICC (Smaller is Better) 1637.3 BIC (Smaller is Better) 1641.9

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 4.5634 0.2879 715 15.85 <.0001 0.05 TRTPN 1 -0.6283 0.06796 715 -9.25 <.0001 0.05 -0.43 0.6690 TRTPN -0.03366 0.07869 715 0.05 TRTPN 3 -0.3922 PREOAD2 0.05944 715 -6.60 <.0001 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.6662 0.03413 715 -19.52 <.0001 0.05
| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 12 of 412 | |

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=C64849B

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>TRTPN<br>TRTPN<br>TRTPN | | 1<br>2<br>3 | 3.9982<br>-0.7618<br>-0.1882 | 5.1287<br>-0.4949<br>0.1208 |
| PREOAD2<br>PREOAD2<br>BASE | Metformin<br>Metformin + OAD | | -0.5089<br>-0.7332 | -0.2755<br>-0.5992 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| TRTPN | 2 | 715 | 60.69 | <.0001 |
| PREOAD2 | 1 | 715 | 43.53 | <.0001 |
| BASE | 1 | 715 | 380.96 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| TRTPN<br>TRTPN<br>TRTPN | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -1.0822 | 0.03921<br>0.05574<br>0.05552 | 715<br>715<br>715 | -42.76<br>-19.42<br>-18.89 | <.0001<br><.0001<br><.0001 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| TRTPN<br>TRTPN<br>TRTPN | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -1.7539<br>-1.1916<br>-1.1575 | -1.5999<br>-0.9728<br>-0.9395 | | | |


 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

TRTPN 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate Residual 66.2773

Fit Statistics

-2 Res Log Likelihood 5060.0
AIC (Smaller is Better) 5062.0
BIC (Smaller is Better) 5066.5

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 34.2233 Intercept 2.3673 715 14.46 <.0001 0.05 TRTPN 1 -6.8678 0.7428 715 -9.25 < .0001 0.05 -0.43 0.6690 TRTPN -0.3679 0.8601 715 0.05 TRTPN 3 -4.2869 PREOAD2 0.6497 715 -6.60 <.0001 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.6662 0.03413 715 -19.52 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 14 of 412 | |

HbAlc after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>TRTPN<br>TRTPN<br>TRTPN | | 1<br>2<br>3 | 29.5757<br>-8.3262<br>-2.0566 | 38.8709<br>-5.4094<br>1.3207 |
| PREOAD2<br>PREOAD2<br>BASE | Metformin<br>Metformin + OAD | | -5.5625<br>-0.7332 | -3.0113<br>-0.5992 |

#### Type 3 Tests of Fixed Effects

| Effect | DF | DF | F Value | Pr > F |
|---------|----|-----|---------|--------|
| TRTPN | 2 | 715 | 60.69 | <.0001 |
| PREOAD2 | | 715 | 43.53 | <.0001 |
| BASE | | 715 | 380.96 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| TRTPN<br>TRTPN<br>TRTPN | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -11.8284 | 0.4286<br>0.6092<br>0.6068 | 715<br>715<br>715 | -42.76<br>-19.42<br>-18.89 | <.0001<br><.0001<br><.0001 |
| | Least Squares Mean | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| TRTPN<br>TRTPN<br>TRTPN | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 -3 | | -17.4868<br>-10.6323<br>-10.2690 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 15 of 412 | |

### 3: HbA1c after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtan 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 674

Number of Observations

Number of Observations Read 674
Number of Observations Used 674
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.4940

Fit Statistics

-2 Res Log Likelihood 1453.8
AIC (Smaller is Better) 1455.8
AICC (Smaller is Better) 1455.8
BIC (Smaller is Better) 1460.3

Solution for Fixed Effects

Actual Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t| Alpha 0.2803 0.06726 4.7125 -0.5903 669 16.81 -8.78 <.0001 0.05 Intercept 669 <.0001 0.05 trtan -0.00164 0.07752 669 -0.02 0.9832 0.05 trtan trtan PREOAD2 Metformin -0.3963 0.05779 669 -6.86 <.0001 0.05 PREOAD2 Metformin + OAD 0.3060 0.03321 669 9.21 <.0001 0.05 BASE

#### NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

HbA1c after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set

Parameter Code=C64849B

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtan<br>trtan<br>trtan | | 1<br>2<br>3 | 4.1621<br>-0.7224<br>-0.1538 | 5.2628<br>-0.4583<br>0.1506 |
| PREOAD2 | Metformin<br>Metformin + OAD | | -0.5097 | -0.2828 |
| BASE | | | 0.2408 | 0.3712 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtan | 2 | 669 | 59.18 | <.0001 |
| PREOAD2 | 1 | 669 | 47.01 | <.0001 |
| BASE | 1 | 669 | 84.90 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Es | stimate | | andard<br>Error | DF | t | Value | Pr : | > t | Alph | a | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| trtan<br>trtan<br>trtan | LSMeans, II<br>LSMeans, II<br>LSMeans, Li | , IDeg WORK.ADATA2 7.0999 | | A2 7.0999 | | .ADATA2 7.0999 | | 7.0999 0.05398 | | 669<br>669 | | 171.78<br>131.54<br>127.78 | < | .0001<br>.0001 | 0.0 | 5 |
| | | | Least | Square | es Mean | s Est | imates | | | | | | | | | |
| Effect | Label | | Lower | Uŗ | per | Expone | entiate | | onen | tiated<br>Lower | Exp | onenti<br>U | ated<br>pper | | | |
| trtan<br>trtan<br>trtan | LSMeans, II<br>LSMeans, II<br>LSMeans, Li | Deg | 6.4368<br>6.9939<br>6.9924 | 7.2 | 5856<br>2059<br>2107 | 672.65<br>1211.88<br>1213.87 | | 8 | | | | 134 | 4.62<br>7.38<br>3.83 | | | |
| | | | Least | Square | es Mean | s Est: | imates | | | | | | | | | |
| Effect | Label | | | | Margin | s | Esti | mate | Stan<br>E | dard<br>rror | DF | t V | alue | | | |
| trtan | Treatment co | ontrast, | IDegLira - | IDeg | WORK.A | DATA2 | -0. | 5887 | 0.0 | 6599 | 669 | - | 8.92 | | | |
| | | | Least | Square | es Mean | s Est: | imates | | | | | | | | | |
| Effect | Label | | | | Pr > | tl i | Alpha | Lowe | r | Upper | Exp | onenti | ated | | | |
| trtan | Treatment co | ontrast, | IDegLira - | IDeg | <.00 | 01 | 0.05 | -0.718 | 3 | -0.4591 | | 0. | 5550 | | | |

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtan | Treatment contrast, | IDegLira - IDeg | <.0001 | 0.05 | -0.7183 | -0.4591 | 0.5550 |

| Effect | Label | | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|
| trtan | Treatment contrast, | IDegLira - IDeg | 0.4876 | 0.6318 |

| NN9068 NN9068-4148 Clinical Trial Report Statistical document | CONFIDENTIAL Date:<br>Version Status<br>Page: | on: 1.0 s: Final | Novo Nordisk |
|---|---|---|---|
| HbA1c after 26 weeks of treatment - chan protocol analysis set | nge from baseline – statist | tical sensitivity analysis - | - per |
| Parameter Code=C64849B | | | |
| The Mixed Procedure | | | |
| Least S | Squares Means Estimates | | |
| Effect Label | Margins Estimat | Standard<br>te Error DF t Va | ılue |
| trtan Treatment contrast, IDegLira - I | ira WORK.ADATA2 -0.590 | 03 0.06726 669 -8 | 3.78 |
| Least S | Squares Means Estimates | | |
| Effect Label | Pr > t Alpha | Lower Upper Exponentia | ited |
| trtan Treatment contrast, IDegLira - I | ira <.0001 0.05 -0 | 0.7224 -0.4583 0.5 | 5541 |
| Least Squares Mea | ans Estimates | | |
| Effect Label | Exponentiated Expo | onentiated<br>Upper | |
| trtan Treatment contrast, IDegLira - I | 0.4856 | 0.6324 | |


 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtan 3 123

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 674

Number of Observations

Number of Observations Read 674 Number of Observations Used 674 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 59.0097

Fit Statistics

-2 Res Log Likelihood 4658.5 AIC (Smaller is Better) 4660.5 AICC (Smaller is Better) 4660.5 BIC (Smaller is Better) 4665.0

Solution for Fixed Effects

Actual Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 35.1977 2.3063 669 15.26 <.0001 0.05 trtan 1 -6.4525 0.7351 669 -8.78 < .0001 0.05 -0.01787 0.9832 trtan 0.8472 669 -0.02 0.05 3 t.rt.an -4.3311 PREOAD2 0.6317 669 -6.86 <.0001 0.05 Metformin Metformin + OAD PREOAD2 BASE 0.3060 0.03321 669 9.21 <.0001 0.05

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtan<br>trtan<br>trtan | | 1<br>2<br>3 | 30.6693<br>-7.8959<br>-1.6814 | 39.7261<br>-5.0090<br>1.6457 |
| PREOAD2 | Metformin<br>Metformin + OAD | Ü | -5.5714 | -3.0908 |
| BASE | 110010111111 1 0110 | | 0.2408 | 0.3712 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtan | 2 | 669 | 59.18 | <.0001 |
| PREOAD2 | 1 | 669 | 47.01 | <.0001 |
| BASE | 1 | 669 | 84.90 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtan<br>trtan<br>trtan | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 47.6677<br>54.1023<br>54.1201 | 0.4143<br>0.5900<br>0.6075 | 669<br>669<br>669 | 115.06<br>91.71<br>89.09 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |
| | | Least Sq | uares Means | Estimates | | | | |
| | | _ | | | Expo | nentiated | Exponentia | ted |

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtan | LSMeans, IDegLira | 46.8542 | 48.4811 | 5.033E20 | 2.231E20 | 1.135E21 |
| trtan | LSMeans, IDeg | 52.9439 | 55.2606 | 3.136E23 | 9.845E22 | 9.986E23 |
| trtan | LSMeans, Lira | 52.9274 | 55.3129 | 3.192E23 | 9.684E22 | 1.052E24 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtan | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -6.4346 | 0.7213 | 669 | -8.92 |

#### Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtan | Treatment contrast, | IDegLira - IDeg | <.0001 | 0.05 | -7.8508 | -5.0183 | 0.001605 |

| Effect | Label | | | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtan | Treatment | contrast, | IDegLira | - IDeg | 0.000389 | 0.006615 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date: 16 D<br>Version:<br>Status:<br>Page: | ecember 2019 Novo Nordisk 1.0 Final 20 of 412 |
|---|---|---|---|
| HbA1c after 26 weeks of treatment protocol analysis set | - change from baseline - s | statistical sensitivit | y analysis – per |
| Parameter Code=HBA1CONV | | | |
| The Mixed Procedure | | | |
| | Least Squares Means Estimat | ces | |
| Effect Label | Margins F | Standard<br>Estimate Error | DF t Value |
| trtan Treatment contrast, IDegL | ira - Lira WORK.ADATA2 | -6.4525 0.7351 | 669 -8.78 |
| | Least Squares Means Estimat | ces | |
| Effect Label | Pr > t Alph | na Lower Upper | Exponentiated |
| trtan Treatment contrast, IDegL | ira - Lira <.0001 0.0 | 05 -7.8959 -5.0090 | 0.001577 |
| Least Squa | res Means Estimates | | |
| Effect Label | Exponentiated<br>Lower | Exponentiated<br>Upper | |
| trtan Treatment contrast, IDegL | ira - Lira 0.000372 | 0.006678 | |


 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtan 3 123

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 674

Number of Observations

Number of Observations Read 674
Number of Observations Used 674
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.4940

Fit Statistics

-2 Res Log Likelihood 1453.8 AIC (Smaller is Better) 1455.8 AICC (Smaller is Better) 1455.8 BIC (Smaller is Better) 1460.3

Solution for Fixed Effects

Actual Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 4.7125 0.2803 669 16.81 <.0001 0.05 trtan 1 -0.5903 0.06726 669 -8.78 <.0001 0.05 -0.00164 -0.02 0.9832 trtan 0.07752 669 0.05 3 t.rt.an -0.3963 PREOAD2 0.05779 669 -6.86 <.0001 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.6940 0.03321 669 -20.90 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 22 of 412 | |

HbA1c after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set

Parameter Code=C64849B

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtan<br>trtan | | 1 2 | 4.1621<br>-0.7224<br>-0.1538 | 5.2628<br>-0.4583<br>0.1506 |
| trtan | | 3 | | |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -0.5097 | -0.2828 |
| BASE | | | -0.7592 | -0.6288 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtan | 2 | 669 | 59.18 | <.0001 |
| PREOAD2 | 1 | 669 | 47.01 | <.0001 |
| BASE | 1 | 669 | 436.75 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtan<br>trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -1.1346 | 0.03790<br>0.05398<br>0.05558 | 669<br>669<br>669 | -45.47<br>-21.02<br>-20.39 | <.0001<br><.0001<br><.0001 |
| | Least Squares Mean | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtan<br>trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -1.7978<br>-1.2406<br>-1.2421 | -1.6489<br>-1.0287<br>-1.0239 | | | |


 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtan 3 123

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 674

Number of Observations

Number of Observations Read 674
Number of Observations Used 674
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 59.0097

Fit Statistics

-2 Res Log Likelihood 4658.5 AIC (Smaller is Better) 4660.5 AICC (Smaller is Better) 4660.5 BIC (Smaller is Better) 4665.0

Solution for Fixed Effects

Actual Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 35.1977 2.3063 669 15.26 <.0001 0.05 trtan 1 -6.4525 0.7351 669 -8.78 <.0001 0.05 -0.01787 -0.02 0.9832 trtan 0.8472 669 0.05 3 t.rt.an -4.3311 PREOAD2 0.6317 669 -6.86 <.0001 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.6940 0.03321 669 -20.90 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 24 of 412 | |

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtan<br>trtan<br>trtan | | 1<br>2<br>3 | 30.6693<br>-7.8959<br>-1.6814 | 39.7261<br>-5.0090<br>1.6457 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -5.5714 | -3.0908 |
| BASE | TICCIOIMIN , OND | | -0.7592 | -0.6288 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---|---|---|---|---|
| trtan<br>PREOAD2 | 2 | 669<br>669 | 59.18<br>47.01 | <.0001<br><.0001 |
| PREUADZ | 1 | 009 | 4 / . 01 | <.0001 |
| BASE | 1 | 669 | 436.75 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtan<br>trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -12.4016 | 0.4143<br>0.5900<br>0.6075 | 669<br>669 | -45.47<br>-21.02<br>-20.39 | <.0001<br><.0001<br><.0001 |
| | Least Squares Means Estimates | | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtan<br>trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 -1 | 19.6496<br>13.5600<br>13.5765 | -18.0227<br>-11.2432<br>-11.1910 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 25 of 412 | |

### 4: HbA1c after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 659

Number of Observations

Number of Observations Read 659 Number of Observations Used 659 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.4598

Fit Statistics

-2 Res Log Likelihood 1374.9
AIC (Smaller is Better) 1376.9
AICC (Smaller is Better) 1376.9
BIC (Smaller is Better) 1381.4

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t| Alpha 0.2736 0.06629 4.8534 17.74 -8.26 <.0001 0.05 654 Intercept trtpn -0.5474 654 <.0001 0.05 0.02449 0.07622 654 0.32 0.7481 0.05 trtpn trtpn PREOAD2 Metformin -0.4131 0.05637 654 -7.33 <.0001 0.05 PREOAD2 Metformin + OAD 0.2840 0.03241 654 8.77 <.0001 0.05 BASE

### NN9068 | Date: 16 December 2019 | Novo Nordisk NN9068-4148 | CONFIDENTIAL | Version: 1.0 | Clinical Trial Report | Status: Final | Statistical document |  |

HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set

Parameter Code=C64849B

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 4.3162<br>-0.6776<br>-0.1252 | 5.3906<br>-0.4173<br>0.1742 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | - | -0.5238 | -0.3025 |
| BASE | | | 0.2204 | 0.3477 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 654 | 56.18 | <.0001 |
| PREOAD2 | 1 | 654 | 53.71 | <.0001 |
| BASE | 1 | 654 | 76.83 | <.0001 |

#### Least Squares Means Estimates

| | | | | Standard | | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2<br>Least Sq | 6.5085<br>7.0805<br>7.0560<br>uares Means | 0.03673<br>0.05252<br>0.05520<br>Estimates | 654<br>654<br>654 | 177.21<br>134.81<br>127.83 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |
| | | | | | F | | Europontio | ± a al |

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | 6.4364 | 6.5807 | 670.84 | 624.16 | 721.01 |
| trtpn | LSMeans, IDeg | 6.9773 | 7.1836 | 1188.52 | 1072.06 | 1317.64 |
| trtpn | LSMeans, Lira | 6.9476 | 7.1644 | 1159.77 | 1040.64 | 1292.54 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -0.5719 | 0.06411 | 654 | -8.92 |

#### Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | <.0001 | 0.05 | -0.6978 | -0.4460 | 0.5644 |

| Effect | Label | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment contras | t, IDegLira - IDe | eg 0.4977 | 0.6402 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date: 16 D<br>Version:<br>Status:<br>Page: | ecember 2019 Novo Nordisk<br>1.0 Final<br>27 of 412 |
|---|---|---|---|
| HbA1c after 26 weeks of treatme<br>completer analysis set | ent - change from baseline - | statistical sensitivit | y analysis - |
| Parameter Code=C64849B | | | |
| The Mixed Procedure | | | |
| | Least Squares Means Estima | tes | |
| Effect Label | Margins | Standard<br>Estimate Error | DF t Value |
| trtpn Treatment contrast, IDe | egLira - Lira WORK.ADATA2 | -0.5474 0.06629 | 654 -8.26 |
| | Least Squares Means Estima | tes | |
| Effect Label | Pr > t Alp | ha Lower Upper | Exponentiated |
| trtpn Treatment contrast, IDe | egLira - Lira <.0001 0. | 05 -0.6776 -0.4173 | 0.5784 |
| Least So | quares Means Estimates | | |
| Effect Label | Exponentiated Lower | Exponentiated<br>Upper | |
| trtpn Treatment contrast, IDe | egLira - Lira 0.5078 | 0.6588 | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis completer analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 659

Number of Observations

Number of Observations Read 659 Number of Observations Used 659 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 54.9347

Fit Statistics

-2 Res Log Likelihood 4507.8 AIC (Smaller is Better) AICC (Smaller is Better) 4509.8 4509.8 BIC (Smaller is Better) 4514.3

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 36.2227 Intercept 2.2522 654 16.08 <.0001 0.05 trtpn 1 -5.9836 0.7246 654 -8.26 <.0001 0.05 0.7481 trtpn 0.2677 0.8331 654 0.32 0.05 3 trtpn PREOAD2 -4.5157 0.6162 654 -7.33 <.0001 0.05 Metformin Metformin + OAD PREOAD2 BASE 0.2840 0.03241 654 8.77 <.0001 0.05

### NN9068 NN9068-4148 Clinical Trial Report Statistical document Date: 16 December 2019 Version: 1.0 Status: Final 

HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 31.8002<br>-7.4064<br>-1.3682 | 40.6451<br>-4.5608<br>1.9036 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | ŭ | -5.7256 | -3.3058 |
| BASE | TICCIOIMITI ( OILD | | 0.2204 | 0.3477 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 654 | 56.18 | <.0001 |
| PREOAD2 | 1 | 654 | 53.71 | <.0001 |
| BASE | 1 | 654 | 76.83 | <.0001 |

#### Least Squares Means Estimates

| | | | | Standard | | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2 | 47.6382<br>53.8895<br>53.6218<br>uares Means | 0.4014<br>0.5741<br>0.6033<br>Estimates | 654<br>654<br>654 | 118.67<br>93.87<br>88.88 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |
| | | | | | Exno | nentiated | Exponentia | ated |

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | 46.8500 | 48.4265 | 4.887E20 | 2.222E20 | 1.075E21 |
| trtpn | LSMeans, IDeg | 52.7623 | 55.0167 | 2.535E23 | 8.211E22 | 7.825E23 |
| trtpn | LSMeans, Lira | 52.4372 | 54.8065 | 1.939E23 | 5.932E22 | 6.341E23 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -6.2513 | 0.7007 | 654 | -8.92 |

#### Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | <.0001 | 0.05 | -7.6272 | -4.8753 | 0.001928 |

| Effect | Label | | | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira · | - IDeg | 0.000487 | 0.007633 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | NFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 Decer | mber 2019 <b>Novo Nordisk</b> 1.0 Final 30 of 412 |
|---|---|---|---|---|
| HbAlc after 26 weeks of treatment - change completer analysis set | from baseline - | statistical se | ensitivity a | nalysis - |
| Parameter Code=HBA1CONV | | | | |
| The Mixed Procedure | | | | |
| Least Squ | ares Means Estima | tes | | |
| Effect Label | Margins | | andard<br>Error | DF t Value |
| trtpn Treatment contrast, IDegLira - Lir | a WORK.ADATA2 | -5.9836 | .7246 6 | 54 -8.26 |
| Least Squ | ares Means Estima | tes | | |
| Effect Label | Pr > t Alp | ha Lower | Upper E | xponentiated |
| trtpn Treatment contrast, IDegLira - Lir | a <.0001 0. | 05 -7.4064 | -4.5608 | 0.002520 |
| Least Squares Means | Estimates | | | |
| Effect Label | Exponentiated Lower | Exponentiat<br>Upp | | |
| trtpn Treatment contrast, IDegLira - Lir | 0.000607 | 0.010 | )45 | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis completer analysis set

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 659

Number of Observations

Number of Observations Read 659 Number of Observations Used 659 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 0.4598

Fit Statistics

-2 Res Log Likelihood 1374.9 AIC (Smaller is Better) AICC (Smaller is Better) 1376.9 1376.9 BIC (Smaller is Better) 1381.4

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 4.8534 0.2736 654 17.74 <.0001 0.05 trtpn 1 -0.5474 0.06629 654 -8.26 <.0001 0.05 0.7481 0.02449 trtpn 0.07622 654 0.32 0.05 3 trtpn PREOAD2 -0.4131 0.05637 654 -7.33 <.0001 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.7160 0.03241 654 -22.09 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 32 of 412 | |

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set

Parameter Code=C64849B

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 4.3162<br>-0.6776<br>-0.1252 | 5.3906<br>-0.4173<br>0.1742 |
| PREOAD2<br>PREOAD2<br>BASE | Metformin<br>Metformin + OAD | | -0.5238<br>-0.7796 | -0.3025<br>-0.6523 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 654 | 56.18 | <.0001 |
| PREOAD2 | 1 | 654 | 53.71 | <.0001 |
| BASE | 1 | 654 | 488.10 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -1.1528 | 0.03673<br>0.05252<br>0.05520 | 654<br>654<br>654 | -46.96<br>-21.95<br>-21.33 | <.0001<br><.0001<br><.0001 |
| | Least Squares Mean | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -1.7968<br>-1.2559<br>-1.2856 | -1.6526<br>-1.0496<br>-1.0689 | | | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis completer analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 659

Number of Observations

Number of Observations Read 659 Number of Observations Used 659 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 54.9347

Fit Statistics

-2 Res Log Likelihood 4507.8 AIC (Smaller is Better) AICC (Smaller is Better) 4509.8 4509.8 BIC (Smaller is Better) 4514.3

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 36.2227 Intercept 2.2522 654 16.08 <.0001 0.05 trtpn 1 -5.9836 0.7246 654 -8.26 <.0001 0.05 0.7481 trtpn 0.2677 0.8331 654 0.32 0.05 3 trtpn PREOAD2 -4.5157 0.6162 654 -7.33 <.0001 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.7160 0.03241 654 -22.09 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 34 of 412 | |

HbA1c after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 31.8002<br>-7.4064<br>-1.3682 | 40.6451<br>-4.5608<br>1.9036 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -5.7256 | -3.3058 |
| BASE | INCCIONNIN , OND | | -0.7796 | -0.6523 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---|---|---|---|---|
| trtpn<br>PREOAD2 | 2 | 654<br>654 | 56.18<br>53.71 | <.0001<br><.0001 |
| BASE | 1 | 654 | 488.10 | <.0001 |

| Effect | Label | | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from<br>Change from<br>Change from | baseline, | IDeg | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -12.5997 | 0.4014<br>0.5741<br>0.6033 | 654<br>654<br>654 | -46.96<br>-21.95<br>-21.33 | <.0001<br><.0001<br><.0001 |
| | | Least Squ | ares Means | Estimates | | | | | |
| Effect | Label | | | Alpha | Lower | Upper | | | |

| Effect | Label | | | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|
| trtpn<br>trtpn | | baseline, | _ | 0.05 | -19.6393<br>-13.7269 | -18.0627<br>-11.4725 |
| trtpn | | baseline, | _ | 0.05 | -14.0521 | -11.6827 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 35 of 412 | |

### 5: HbA1c after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

#### Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Subjuct Effect
Stimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Satterthwaite

### Class Level Information

| Class | Levels | Values |
|---------|--------|---------------------------|
| TRT01PN | 3 | 1 2 3 |
| AVISITN | 6 | 60 100 140 180 220 280 |
| PREOAD2 | 2 | Metformin Metformin + OAD |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 36 of 412 | |

 $\label{thm:main_model} \begin{tabular}{ll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set \end{tabular}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 720



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 37 of 412 | |

 $\label{thm:main_model} \begin{tabular}{ll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set \end{tabular}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure



| NN9068 | | Date: | 16 December 2019 <b>Novo Nordis</b> | sk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 38 of 412 | |

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure



#### Dimensions

| Covariance | Parameters | 21 |
|------------|------------|-----|
| Columns in | X | 37 |
| Columns in | Z | 0 |
| Subjects | | 720 |
| Max Obs pe | r Subject | 6 |

#### Number of Observations

| Number | of | Observations | Read | 4320 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 4041 |
| Number | of | Observations | Not Used | 279 |


HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

#### Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 7781.56844929 | |
| 1 | 3 | 2512.22254080 | 0.00036020 |
| 2 | 1 | 2511.34737835 | 0.00000107 |
| 3 | 1 | 2511.34477278 | 0.00000000 |

Convergence criteria met.

#### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | |
| UN(2,1) | SUBJID | |
| UN(2,2) | SUBJID | |
| UN(3,1) | SUBJID | |
| UN(3,2) | SUBJID | |
| UN(3,3) | SUBJID | |
| UN(4,1) | SUBJID | |
| UN(4,2) | SUBJID | |
| UN(4,3) | SUBJID | |
| UN (4,4) | SUBJID | |
| UN(5,1) | SUBJID | |
| UN(5,2) | SUBJID | |
| UN(5,3) | SUBJID | |
| UN(5,4) | SUBJID | |
| UN(5,5) | SUBJID | |
| UN(6,1) | SUBJID | |
| UN(6,2) | SUBJID | |
| UN(6,3) | SUBJID | |
| UN(6,4) | SUBJID | |
| UN(6,5) | SUBJID | |
| UN(6,6) | SUBJID | |

#### Fit Statistics

| -2 Res Log Likelihood | 2511.3 |
|--------------------------|--------|
| AIC (Smaller is Better) | 2553.3 |
| AICC (Smaller is Better) | 2553.6 |
| BIC (Smaller is Better) | 2649.5 |

### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr | > ChiSq |
|----|------------|----|---------|
| 20 | 5270.22 | | <.0001 |

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---|---|---|---|---|
| TRT01PN (AVISITN) PREOAD2 (AVISITN) BASE (AVISITN) | 12 | 828 | 18.08 | <.0001 |
| | 6 | 668 | 10.71 | <.0001 |
| | 6 | 670 | 308.22 | <.0001 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 40 of 412 | |

 ${\tt HbAlc\ after\ 26\ weeks\ of\ treatment\ -\ change\ from\ baseline\ -\ statistical\ sensitivity\ analysis\ -\ MMRM\ -\ full\ analysis\ set}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| TRT01PN (AVISITN)<br>TRT01PN (AVISITN)<br>TRT01PN (AVISITN) | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ANA_DATA<br>WORK.ANA_DATA<br>WORK.ANA_DATA | 6.5097<br>7.1047<br>7.1015 | 0.03704<br>0.05281<br>0.05446 | 658.2<br>660.9<br>683.2 | 175.76<br>134.54<br>130.40 | <.0001<br><.0001<br><.0001 |
| | Least Squares Mea | ans Estimates | | | | | |
| Effect | Label | Alpha I | Lower | Upper | | | |
| TRT01PN (AVISITN)<br>TRT01PN (AVISITN)<br>TRT01PN (AVISITN) | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | 0.05 7. | .4370<br>.0011<br>.9946 | 6.5825<br>7.2084<br>7.2085 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 41 of 412 | |

 $\begin{tabular}{ll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set \\ \end{tabular}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

#### Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Subject Effect
Subject Effect
Subject Effect
Subject Effect
SubJID
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Satterthwaite

#### Class Level Information

| Class | Levels | Values |
|---------|--------|---------------------------|
| TRT01PN | 3 | 1 2 3 |
| AVISITN | 6 | 60 100 140 180 220 280 |
| PREOAD2 | 2 | Metformin Metformin + OAD |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 42 of 412 | |

 ${\tt HbAlc\ after\ 26\ weeks\ of\ treatment\ -\ change\ from\ baseline\ -\ statistical\ sensitivity\ analysis\ -\ MMRM\ -\ full\ analysis\ set}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

Class Level Information

Class Levels Values
SUBJID 720



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 43 of 412 | |

 $\label{thm:main_model} \begin{tabular}{ll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set \end{tabular}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 44 of 412 | |

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure



#### Dimensions

| Covariance | Parameters | 21 |
|------------|------------|-----|
| Columns in | X | 37 |
| Columns in | Z | 0 |
| Subjects | | 720 |
| Max Obs pe | r Subject | 6 |

### Number of Observations

| Number of | Observations Observations Observations | Used | 4320<br>4041<br>279 |
|---|---|---|---|
| Number of | Observations | Not Usea | 2/9 |

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

#### Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 26994.97025107 | |
| 1 | 3 | 21725.62434258 | 0.00012195 |
| 2 | 1 | 21724.74918014 | 0.00000036 |
| 3 | 1 | 21724.74657456 | 0.00000000 |

Convergence criteria met.

#### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | |
| UN(2,1) | SUBJID | |
| UN(2,2) | SUBJID | |
| UN(3,1) | SUBJID | |
| UN(3,2) | SUBJID | |
| UN(3,3) | SUBJID | |
| UN(4,1) | SUBJID | |
| UN(4,2) | SUBJID | |
| UN(4,3) | SUBJID | |
| UN(4,4) | SUBJID | |
| UN(5,1) | SUBJID | |
| UN(5,2) | SUBJID | |
| UN(5,3) | SUBJID | |
| UN(5,4) | SUBJID | |
| UN(5,5) | SUBJID | |
| UN(6,1) | SUBJID | |
| UN(6,2) | SUBJID | |
| UN(6,3) | SUBJID | |
| UN(6,4) | SUBJID | |
| UN(6,5) | SUBJID | |
| UN(6,6) | SUBJID | |

#### Fit Statistics

| -2 Res Log Likelihood | 21724.7 |
|--------------------------|---------|
| AIC (Smaller is Better) | 21766.7 |
| AICC (Smaller is Better) | 21767.0 |
| BIC (Smaller is Better) | 21862.9 |

### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr | > | ChiSq |
|----|------------|----|---|--------|
| 20 | 5270.22 | | 4 | <.0001 |

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---|---|---|---|---|
| TRT01PN(AVISITN) PREOAD2(AVISITN) BASE(AVISITN) | 12 | 828 | 18.08 | <.0001 |
| | 6 | 668 | 10.71 | <.0001 |
| | 6 | 670 | 308.22 | <.0001 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 46 of 412 | |

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| TRT01PN (AVISITN)<br>TRT01PN (AVISITN)<br>TRT01PN (AVISITN) | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ANA_DATA<br>WORK.ANA_DATA<br>WORK.ANA_DATA | 47.6513<br>54.1549<br>54.1197 | 0.4048<br>0.5772<br>0.5952 | 658.2<br>660.9<br>683.2 | 117.71<br>93.83<br>90.92 | <.0001<br><.0001<br><.0001 |
| Least Squares Means Estimates | | | | | | | |
| Effect | Label | Alpha I | Lower | Upper | | | |
| TRT01PN (AVISITN)<br>TRT01PN (AVISITN)<br>TRT01PN (AVISITN) | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | 0.05 53. | .0216 5 | 18.4462<br>55.2882<br>55.2884 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 47 of 412 | |

 ${\tt HbAlc\ after\ 26\ weeks\ of\ treatment\ -\ change\ from\ baseline\ -\ statistical\ sensitivity\ analysis\ -\ MMRM\ -\ full\ analysis\ set}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

#### Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
SWBK.ANA\_DATA
CHG
Unstructured
SUBJID
REML
None
Method
Model-Based
Satterthwaite

#### Class Level Information

| Class | Levels | Values |
|--------------------|--------|---------------------------------|
| TRT01PN<br>AVISITN | 3 | 1 2 3<br>60 100 140 180 220 280 |
| PREOAD2 | 2 | Metformin Metformin + OAD |
| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 48 of 412 | |

 ${\tt HbAlc\ after\ 26\ weeks\ of\ treatment\ -\ change\ from\ baseline\ -\ statistical\ sensitivity\ analysis\ -\ MMRM\ -\ full\ analysis\ set}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

Class Level Information

Class Levels Values
SUBJID 720

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 49 of 412 | |

 ${\tt HbAlc\ after\ 26\ weeks\ of\ treatment\ -\ change\ from\ baseline\ -\ statistical\ sensitivity\ analysis\ -\ MMRM\ -\ full\ analysis\ set}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure



| NN9068 | | Date: | 16 December 2019 Novo Nor | disk |
|---|---|---|---|---|
| NN9068-4148 | | Version: | 1.0 | |
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 50 of 412 | |

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure



## Dimensions

| Covariance | Parameters | 21 |
|------------|------------|-----|
| Columns in | X | 37 |
| Columns in | Z | 0 |
| Subjects | | 720 |
| Max Obs pe | r Subject | 6 |

## Number of Observations

| Number | of | Observations | Read | 4320 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 4041 |
| Number | of | Observations | Not Used | 279 |


HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

## Iteration History

| Criterion | -2 Res Log Like | Evaluations | Iteration |
|------------|-----------------|-------------|-----------|
| | 7781.56844929 | 1 | 0 |
| 0.00036020 | 2512.22254080 | 3 | 1 |
| 0.00000107 | 2511.34737835 | 1 | 2 |
| 0.00000000 | 2511.34477278 | 1 | 3 |

Convergence criteria met.

## Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | |
| UN(2,1) | SUBJID | |
| UN(2,2) | SUBJID | |
| UN(3,1) | SUBJID | |
| UN(3,2) | SUBJID | |
| UN(3,3) | SUBJID | |
| UN(4,1) | SUBJID | |
| UN(4,2) | SUBJID | |
| UN(4,3) | SUBJID | |
| UN(4,4) | SUBJID | |
| UN(5,1) | SUBJID | |
| UN(5,2) | SUBJID | |
| UN(5,3) | SUBJID | |
| UN(5,4) | SUBJID | |
| UN(5,5) | SUBJID | |
| UN(6,1) | SUBJID | |
| UN(6,2) | SUBJID | |
| UN(6,3) | SUBJID | |
| UN(6,4) | SUBJID | |
| UN(6,5) | SUBJID | |
| UN(6,6) | SUBJID | |

## Fit Statistics

| -2 Res Log Likelihood | 2511.3 |
|--------------------------|--------|
| AIC (Smaller is Better) | 2553.3 |
| AICC (Smaller is Better) | 2553.6 |
| BIC (Smaller is Better) | 2649.5 |

# Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 20 | 5270.22 | <.0001 |

# Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---|---|---|---|---|
| TRT01PN(AVISITN) PREOAD2(AVISITN) BASE(AVISITN) | 12 | 828 | 18.08 | <.0001 |
| | 6 | 668 | 10.71 | <.0001 |
| | 6 | 670 | 83.04 | <.0001 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 52 of 412 | |

 $\label{thm:main_model} \begin{tabular}{ll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set \end{tabular}$ 

Short Topic Code=C64849B Long label=HbA1c (%)

The Mixed Procedure

## Least Squares Means Estimates

| Effect | Label | Margins | | ndard<br>Error DF t Value |
|---|---|---|---|---|
| TRT01PN (AVISITN)<br>TRT01PN (AVISITN)<br>TRT01PN (AVISITN) | | WORK.ANA_DATA<br>WORK.ANA_DATA<br>WORK.ANA_DATA | -1.1325 0. | 03704 658.2 -46.64<br>05281 660.9 -21.45<br>05446 683.2 -20.85 |
| | Least Squares Mean | s Estimates | | |
| Effect | Label | Pr > t | Alpha Low | er Upper |
| TRT01PN (AVISITN) TRT01PN (AVISITN) TRT01PN (AVISITN) | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | <.0001 | 0.05 -1.80<br>0.05 -1.23<br>0.05 -1.24 | -1.0288 |
| | Least Squares M | Means Estimates | | |
| Effect | Label | Margins | Estimat | Standard<br>Error DF |
| TRT01PN (AVISITN) TRT01PN (AVISITN) | Treatment contrast, IDegLira -<br>Treatment contrast, IDegLira - | | | |
| Least Squares Means Estimates | | | | |
| Effect | Label | t Value | Pr > t Alp | na Lower Upper |
| TRT01PN (AVISITN) TRT01PN (AVISITN) | Treatment contrast, IDegLira -<br>Treatment contrast, IDegLira - | | <.0001 0.<br><.0001 0. | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 53 of 412 | |

 ${\tt HbAlc\ after\ 26\ weeks\ of\ treatment\ -\ change\ from\ baseline\ -\ statistical\ sensitivity\ analysis\ -\ MMRM\ -\ full\ analysis\ set}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

## Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
SWBK.ANA\_DATA
CHG
Unstructured
SUBJID
REML
None
Method
Model-Based
Satterthwaite

## Class Level Information

| Class | Levels | Values | |
|---------|--------|------------|-----|
| TRT01PN | 3 | 1 2 3 | |
| AVISITN | 6 | 60 100 140 | 180 |

AVISITN 6 60 100 140 180 220 280 PREOAD2 2 Metformin Metformin + OAD

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 54 of 412 | |

 ${\tt HbAlc\ after\ 26\ weeks\ of\ treatment\ -\ change\ from\ baseline\ -\ statistical\ sensitivity\ analysis\ -\ MMRM\ -\ full\ analysis\ set}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

Class Level Information

Class Levels Values
SUBJID 720



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 55 of 412 | |

 $\label{thm:main_model} \begin{tabular}{ll} HbAlc after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set \end{tabular}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 56 of 412 | |

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure



## Dimensions

| Covariance | Parameters | 21 |
|------------|------------|-----|
| Columns in | X | 37 |
| Columns in | Z | 0 |
| Subjects | | 720 |
| Max Obs pe | r Subject | 6 |

# Number of Observations

| Number of Observations Read 4320<br>Number of Observations Used 4041<br>Number of Observations Not Used 279 | Number | of | Used | 1011 |
|---|---|---|---|---|
|---|---|---|---|---|

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 57 of 412 | |

 ${\tt HbAlc\ after\ 26\ weeks\ of\ treatment\ -\ change\ from\ baseline\ -\ statistical\ sensitivity\ analysis\ -\ MMRM\ -\ full\ analysis\ set}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

## Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 26994.97025107 | |
| 1 | 3 | 21725.62434258 | 0.00012195 |
| 2 | 1 | 21724.74918014 | 0.00000036 |
| 3 | 1 | 21724.74657456 | 0.00000000 |

Convergence criteria met.

## Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|-----------|---------|----------|
| UN(1,1) | SUBJID | |
| UN(2,1) | SUBJID | |
| UN(2,2) | SUBJID | |
| UN(3,1) | SUBJID | |
| UN(3,2) | SUBJID | |
| UN(3,3) | SUBJID | |
| UN(4,1) | SUBJID | |
| UN(4,2) | SUBJID | |
| UN(4,3) | SUBJID | |
| UN(4,4) | SUBJID | |
| - ( - , , | SUBJID | |
| UN(5,2) | SUBJID | |
| UN(5,3) | SUBJID | |
| UN(5,4) | SUBJID | |
| UN(5,5) | SUBJID | |
| UN(6,1) | SUBJID | |
| UN(6,2) | SUBJID | |
| UN(6,3) | SUBJID | |
| UN(6,4) | SUBJID | |
| UN(6,5) | SUBJID | |
| UN(6,6) | SUBJID | |

## Fit Statistics

| -2 Res Log Likelihood | 21724.7 |
|--------------------------|---------|
| AIC (Smaller is Better) | 21766.7 |
| AICC (Smaller is Better) | 21767.0 |
| BIC (Smaller is Better) | 21862.9 |

# Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr | > ChiSq |
|----|------------|----|---------|
| 20 | 5270.22 | | <.0001 |

# Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---|---|---|---|---|
| TRT01PN(AVISITN) PREOAD2(AVISITN) BASE(AVISITN) | 12 | 828 | 18.08 | <.0001 |
| | 6 | 668 | 10.71 | <.0001 |
| | 6 | 670 | 83.04 | <.0001 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 58 of 412 | |

 ${\tt HbAlc\ after\ 26\ weeks\ of\ treatment\ -\ change\ from\ baseline\ -\ statistical\ sensitivity\ analysis\ -\ MMRM\ -\ full\ analysis\ set}$ 

Short Topic Code=HBA1CONV Long label=HbA1c (mmol/mol)

The Mixed Procedure

## Least Squares Means Estimates

| Effect | Label | Margins | Standa<br>Estimate Err | |
|---|---|---|---|---|
| TRT01PN (AVISITN)<br>TRT01PN (AVISITN)<br>TRT01PN (AVISITN) | | WORK.ANA_DATA<br>WORK.ANA_DATA<br>WORK.ANA_DATA | -12.3779 0.5 | |
| | Least Squares Mear | ns Estimates | | |
| Effect | Label | Pr > t | Alpha Lower | Upper |
| TRT01PN (AVISITN) TRT01PN (AVISITN) TRT01PN (AVISITN) | Change from baseline, IDeg | <.0001 | 0.05 -19.6764<br>0.05 -13.5112<br>0.05 -13.5818 | -11.2446 |
| | Least Squares N | Means Estimates | | |
| Effect | Label | Margins | Estimate | Standard<br>Error DF |
| TRT01PN (AVISITN) TRT01PN (AVISITN) | Treatment contrast, IDegLira -<br>Treatment contrast, IDegLira - | | | 0.7053 659.9<br>0.7197 675.3 |
| Least Squares Means Estimates | | | | |
| Effect | Label | t Value | Pr > t Alpha | Lower Upper |
| TRT01PN (AVISITN) TRT01PN (AVISITN) | Treatment contrast, IDegLira -<br>Treatment contrast, IDegLira - | | <.0001 0.05<br><.0001 0.05 | -7.8885 -5.1186<br>-7.8815 -5.0552 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 59 of 412 | |

PARAM ANA SORT=12 Parameter Code=C64849B Label=LSMeans, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME ABS MI2 Number of Imputations WORK 1000

Variance Information (1000 Imputations)

-----Variance-----

Parameter Between Within Total 0.002826 0.003022 238192 Estimate 0.000195

Variance Information (1000 Imputations)

Relative Fraction Increase Missing Relative in Variance Information Efficiency Parameter

0.069246 0.064770 Estimate 0.999935

Parameter Estimates (1000 Imputations)

7.062800

7.156116

95% Confidence Std Error Limits DF Estimate Minimum Maximum Parameter

Estimate 7.103584 0.054969 6.995846 7.211322 238192 Parameter Estimates (1000 Imputations)

t for HO:

Theta0 Parameter=Theta0 Pr > |t| Parameter 129.23 <.0001 Estimate

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=12 Parameter Code=C64849B Label=LSMeans, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

Parameter Between Within Total DF

Estimate 0.000084942 0.001399 0.001484 304281

Variance Information (1000 Imputations)

Relative Fraction Increase Missing Relative Parameter in Variance Information Efficiency

Estimate 0.060781 0.057305 0.999943

Parameter Estimates (1000 Imputations)

 Parameter
 Estimate
 Std Error
 Limits
 DF
 Minimum
 Maximum

 Estimate
 6.548286
 0.038522
 6.472785
 6.623788
 304281
 6.518629
 6.575295

Parameter Estimates (1000 Imputations)

Parameter Theta0 Parameter=Theta0 Pr > |t| Estimate 0 169.99 <.0001

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=12 Parameter Code=C64849B Label=LSMeans, Lira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total

0.002804 0.003230 57506 Estimate 0.000425

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency Estimate 0.151813 0.131833 0.999868

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits

Minimum Maximum 0.056832 6.995953 7.218735 57506 7.045183 7.178137 7.107344 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|

0 125.06 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Page: Statistical document 62 of 412

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=22 Parameter Code=HBA1CONV Label=LSMeans, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total

0.337598 0.360976 238192 Estimate 0.023354

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency 0.064770 0.999935 Estimate 0.069246

Parameter Estimates (1000 Imputations)

95% Confidence

DF Minimum Parameter Estimate Std Error Limits Maximum 0.600812 52.96460 55.31975 238192 53.696405 54.716345 54.142174 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 90.11 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Page: Statistical document 63 of 412

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=22 Parameter Code=HBA1CONV Label=LSMeans, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.167118 0.177276 304281 Estimate 0.010148

Variance Information (1000 Imputations)

Relative

Fraction Missing Relative Increase Parameter in Variance Information Efficiency 0.057305 Estimate 0.060781 0.999943

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum

48.072770 0.421042 47.24754 48.89800 304281 47.748618 48.367977 Estimate

Maximum

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|

0 114.18 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Page: Statistical document 64 of 412

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=22 Parameter Code=HBA1CONV Label=LSMeans, Lira Statement Number=1

The MIANALYZE Procedure

Estimate

Model Information

Data Set WORK.LSME\_ABS\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.334999 0.385856 57506

Estimate 0.050806

Variance Information (1000 Imputations)

Fraction Missing Relative Relative Increase Parameter in Variance Information Efficiency

0.151813

Parameter Estimates (1000 Imputations)

0.131833

DF Minimum Parameter Estimate Std Error Limits Maximum 0.621173 52.96577 55.40078 57506 53.503846 54.957040 54.183273 Estimate

95% Confidence

0.999868

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 87.23 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 65 of 412 | |

PARAM\_ANA\_SORT=12 Parameter Code=C64849B Label=Change from baseline, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2
Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.002826 0.003022 238192 0.000195 Estimate

Variance Information (1000 Imputations)

Relative Fraction Missing Increase

Relative Increase Missing in Variance Information Parameter Efficiency 0.069246 0.064770 0.999935 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits e DF Minimum Estimate Std Error Parameter Maximum Estimate -1.129194 0.054969 -1.23693 -1.02146 238192 -1.169978 -1.076662

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -20.54 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 66 of 412 | |

PARAM\_ANA\_SORT=12 Parameter Code=C64849B Label=Change from baseline, IDegLira Statement Number=1

The MIANALYZE Procedure

Estimate

Model Information

Data Set WORK.LSME\_CHG\_MI2
Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.001399 0.001484 304281 0.000084942 Estimate

Variance Information (1000 Imputations)

Relative Fraction Missing

Increase Missing in Variance Information Relative Parameter Efficiency 0.060781 0.057305 0.999943 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits

nce DF Minimum Estimate Std Error Parameter Maximum Estimate -1.684491 0.038522 -1.75999 -1.60899 304281 -1.714149 -1.657483

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -43.73 <.0001

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 67 of 412 | |

PARAM ANA SORT=12 Parameter Code=C64849B Label=Change from baseline, Lira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2
Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.000425 0.002804 0.003230 57506 Estimate

Variance Information (1000 Imputations)

Relative Fraction Missing

Increase Missing in Variance Information Relative Parameter Efficiency 0.151813 0.131833 0.999868 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits DF Minimum Estimate Std Error Parameter Maximum Estimate -1.125433 0.056832 -1.23682 -1.01404 57506 -1.187595 -1.054641

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter

0 -19.80 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Page: Statistical document 68 of 412

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=12 Parameter Code=C64849B Label=Treatment contrast, IDegLira - IDeg

The MIANALYZE Procedure

Estimate

Model Information

Data Set WORK.LSME\_CHG\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total

0.004230 0.004495 286688 Estimate 0.000265

Variance Information (1000 Imputations)

Relative Fraction Missing Relative Increase Parameter in Variance Information Efficiency

0.059037 Estimate 0.062734 0.999941

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum -0.555298 0.067045 -0.68670 -0.42389 286688 -0.609658 -0.503912

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 -8.28 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 69 of 412 | |

PARAM\_ANA\_SORT=22 Parameter Code=HBA1CONV Label=Change from baseline, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2
Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter 0.023354 0.337598 0.360976 238192 Estimate

Variance Information (1000 Imputations)

Relative

Fraction Missing Relative Increase Increase Missing in Variance Information Parameter Efficiency 0.069246 0.064770 0.999935 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits

e DF Minimum Maximum Estimate Std Error Parameter Estimate -12.342087 0.600812 -13.5197 -11.1645 238192 -12.787856 -11.767916

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -20.54 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 70 of 412 | |

PARAM\_ANA\_SORT=22 Parameter Code=HBA1CONV Label=Change from baseline, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2
Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.010148 0.167118 0.177276 304281 Estimate

Variance Information (1000 Imputations)

Relative Fraction Missing

Increase Missing in Variance Information Relative Parameter Efficiency 0.060781 0.057305 0.999943 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits DF Minimum Maximum Parameter Estimate Std Error Estimate -18.411491 0.421042 -19.2367 -17.5863 304281 -18.735643 -18.116284

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -43.73 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 71 of 412 | |

PARAM\_ANA\_SORT=22 Parameter Code=HBA1CONV Label=Change from baseline, Lira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2
Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.050806 0.334999 0.385856 57506 Estimate

Variance Information (1000 Imputations)

Relative Fraction Missing

Increase Missing
in Variance Information Relative Parameter Efficiency 0.151813 0.131833 0.999868 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits

nce DF Minimum Maximum Std Error Estimate Parameter 0.621173 -13.5185 -11.0835 57506 -12.980415 -11.527221 Estimate -12.300988

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -19.80 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Page: Statistical document 72 of 412

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=22 Parameter Code=HBA1CONV Label=Treatment contrast, IDegLira - IDeg

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.505294 0.536993 286688 Estimate 0.031667

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency 0.059037 Estimate 0.062734 0.999941

Parameter Estimates (1000 Imputations)

95% Confidence

DF Minimum Parameter Estimate Std Error Limits Maximum -6.069404 0.732798 -7.50567 -4.63314 286688 -6.663557 -5.507762 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 -8.28 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=13 Parameter Code=C64849B Label=LSMeans, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.002751 0.002945 229712 Estimate 0.000194

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency 0.070602 0.065955 Estimate 0.999934

Parameter Estimates (1000 Imputations)

95% Confidence

DF Parameter Estimate Std Error Limits Minimum Maximum 0.054266 6.996669 7.209389 229712 7.062298 7.103029 7.155185 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 130.89 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Page: Statistical document 74 of 412

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=13 Parameter Code=C64849B Label=LSMeans, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total

0.000072517 0.001362 0.001434 389972 Estimate

Variance Information (1000 Imputations)

Fraction Missing Relative

Relative Increase Parameter in Variance Information Efficiency 0.050618 0.999949 Estimate 0.053312

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum 0.037871 6.458631 6.607083 389972 6.505273 6.532857 6.557992 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 172.50 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final 75 of 412 Statistical document Page:

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=13 Parameter Code=C64849B Label=LSMeans, Lira Statement Number=1

The MIANALYZE Procedure

Estimate

Model Information

Data Set WORK.LSME\_ABS\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.002729 0.003155 54889 Estimate 0.000425

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency 0.999865 Estimate 0.155948 0.134940

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum 7.107487 0.056170 6.997393 7.217581 54889 7.045149 7.178158

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 126.54 <.0001 Estimate

### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Page: Statistical document 76 of 412

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=23 Parameter Code=HBA1CONV Label=LSMeans, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.328601 0.351801 229712 Estimate 0.023177

Variance Information (1000 Imputations)

Relative

Fraction Missing Relative Increase Parameter in Variance Information Efficiency 0.070602 0.065955 Estimate 0.999934

Parameter Estimates (1000 Imputations)

95% Confidence DF Minimum Parameter Estimate Std Error Limits

0.593128 52.97359 55.29862 229712 53.690920 54.706169 54.136108 Estimate

Maximum

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 91.27 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Page: Statistical document 77 of 412

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=23 Parameter Code=HBA1CONV Label=LSMeans, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Within Total DF Parameter Between 0.162664 0.171336 389972 Estimate 0.008663

Variance Information (1000 Imputations)

Relative

Fraction Missing Relative Increase Parameter in Variance Information Efficiency 0.053312 0.050618 0.999949 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence DF Minimum Parameter Estimate Std Error Limits Maximum 0.413928 47.09284 48.71541 389972 47.602638 48.178854

Parameter Estimates (1000 Imputations)

47.904126

Estimate

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|0 115.73 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final  Statistical document

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=23 Parameter Code=HBA1CONV Label=LSMeans, Lira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total

0.326071 0.376921 54889 Estimate 0.050799

Variance Information (1000 Imputations)

Fraction Missing Relative

54.184834

Estimate

Relative Increase Parameter in Variance Information Efficiency Estimate 0.155948 0.134940 0.999865

Parameter Estimates (1000 Imputations)

95% Confidence DF Minimum Parameter Estimate Std Error Limits Maximum 0.613939 52.98151 55.38816 54889 53.503476 54.957268

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 88.26 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 79 of 412 | |

PARAM\_ANA\_SORT=13 Parameter Code=C64849B Label=Change from baseline, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3
Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.002751 0.002945 229712 0.000194 Estimate

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Increase Missing in Variance Information Parameter Efficiency 0.070602 0.065955 0.999934 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits ce DF Minimum Estimate Std Error Parameter Maximum

Estimate -1.129749 0.054266 -1.23611 -1.02339 229712 -1.170480 -1.077593

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter

0 -20.82 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 80 of 412 | |

PARAM\_ANA\_SORT=13 Parameter Code=C64849B Label=Change from baseline, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3
Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance----Between Within Total DF Parameter

0.001362 0.001434 389972 0.000072517 Estimate

Variance Information (1000 Imputations)

Relative Fraction Missing

Increase Missing Parameter in Variance Information Relative Efficiency 0.053312 0.050618 0.999949 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits DF Minimum Estimate Std Error Parameter Maximum

Estimate -1.699921 0.037871 -1.77415 -1.62570 389972 -1.727504 -1.674786

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -44.89 <.0001 Estimate

| NN9068 | CONFIDENTIAL | Date: | 16 December 2019 Novo Nordis | sk |
|---|---|---|---|---|
| NN9068-4148 | | Version: | 1.0 | |
| Clinical Trial Report | | Status: | Final | |
| Statistical document | | Page: | 81 of 412 | |

PARAM ANA SORT=13 Parameter Code=C64849B Label=Change from baseline, Lira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3
Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.000425 0.002729 0.003155 54889 Estimate

Variance Information (1000 Imputations)

Relative Fraction Missing

Increase Missing in Variance Information Relative Parameter Efficiency 0.155948 0.134940 0.999865 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits DF Minimum Estimate Std Error Parameter Maximum Estimate -1.125291 0.056170 -1.23538 -1.01520 54889 -1.187629 -1.054620

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter

0 -20.03 <.0001 Estimate

### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 82 of 412 Page:

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=13 Parameter Code=C64849B Label=Treatment contrast, IDeqLira - Lira

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.004090 0.004588 84745 Estimate 0.000498

Variance Information (1000 Imputations)

Relative

Fraction Missing Relative Increase Parameter in Variance Information Efficiency 0.108595 Estimate 0.121798 0.999891

Parameter Estimates (1000 Imputations)

95% Confidence DF Minimum Parameter Estimate Std Error Limits

-0.574630 0.067735 -0.70739 -0.44187 84745 -0.643691 -0.509073 Estimate

Maximum

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|

0 -8.48 <.0001 Estimate

| NN9068 | CONFIDENTIAL | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| NN9068-4148 | | Version: | 1.0 | |
| Clinical Trial Report | | Status: | Final | |
| Statistical document | | Page: | 83 of 412 | |

PARAM\_ANA\_SORT=23 Parameter Code=HBA1CONV Label=Change from baseline, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3
Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.023177 0.328601 0.351801 229712 Estimate

Variance Information (1000 Imputations)

Relative Fraction Missing

Increase Missing in Variance Information Relative Parameter Efficiency 0.070602 0.065955 0.999934 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits DF Minimum Maximum Estimate Std Error Parameter Estimate -12.348153 0.593128 -13.5107 -11.1856 229712 -12.793341 -11.778092

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -20.82 <.0001 Estimate
#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=23 Parameter Code=HBA1CONV Label=Change from baseline, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total

0.162664 0.171336 389972 Estimate 0.008663

Variance Information (1000 Imputations)

Fraction Missing Relative

Relative Increase Information Parameter in Variance Efficiency 0.053312 0.050618 0.999949 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence

DF Minimum Parameter Estimate Std Error Limits Maximum -18.580135 0.413928 -19.3914 -17.7688 389972 -18.881623 -18.305407 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|0 -44.89 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIALE | Status: | Final | |
| Statistical document | | Page: | 85 of 412 | |

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM\_ANA\_SORT=23 Parameter Code=HBA1CONV Label=Change from baseline, Lira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3
Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter 0.050799 0.326071 0.376921 54889 Estimate

Variance Information (1000 Imputations)

Relative Fraction Missing

Increase Missing
in Variance Information Relative Parameter Efficiency 0.155948 0.134940 0.999865 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits

nce DF Minimum Maximum Estimate Std Error Parameter Estimate -12.299427 0.613939 -13.5028 -11.0961 54889 -12.980785 -11.526993

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -20.03 <.0001 Estimate

### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

 $\tt HbAlc$  after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

PARAM ANA SORT=23 Parameter Code=HBA1CONV Label=Treatment contrast, IDeqLira - Lira

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total

0.488595 0.548105 84745 Estimate 0.059450

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency 0.108595 Estimate 0.121798 0.999891

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum

-6.280708 0.740341 -7.73177 -4.82965 84745 -7.035540 -5.564170 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|

0 -8.48 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 87 of 412 | |

# 7: HbA1c after 26 weeks of treatment – change from baseline – supportive statistical analysis – full analysis set

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.5548

Fit Statistics

-2 Res Log Likelihood 1635.3 AIC (Smaller is Better) 1637.3 AICC (Smaller is Better) 1637.3 BIC (Smaller is Better) 1641.9

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t| Alpha 0.2879 0.06796 4.5634 715 715 <.0001 0.05 15.85 Intercept trtpn -0.6283 -9.25 <.0001 0.05 -0.03366 0.07869 715 -0.43 0.6690 0.05 trtpn trtpn PREOAD2 Metformin -0.3922 0.05944 715 -6.60 <.0001 0.05 PREOAD2 Metformin + OAD 0.3338 0.03413 715 9.78 <.0001 0.05 BASE


HbAlc after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=C64849B

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 3.9982<br>-0.7618<br>-0.1882 | 5.1287<br>-0.4949<br>0.1208 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -0.5089 | -0.2755 |
| BASE | | | 0.2668 | 0.4008 |

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 715 | 60.69 | <.0001 |
| PREOAD2 | 1 | 715 | 43.53 | <.0001 |
| BASE | 1 | 715 | 95.66 | <.0001 |

### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 6.5559<br>7.1500<br>7.1842 | 0.05574 | 715<br>715<br>715 | 167.18<br>128.29<br>129.40 | | 0.05<br>0.05<br>0.05 |
| | | Least Squ | ares Mean | ns Estimates | | | | |
| Effect | Label | Lower | Upper | Exponentiated | Expor | nentiated<br>Lower | Exponentia<br>Up | ted |
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | | 6.6329<br>7.2600<br>7.2933 | 703.38<br>1274.85<br>1318.50 | | 651.26<br>1142.71<br>1182.33 | 759<br>1422<br>1470 | |
| | | Least Squ | ares Mean | ns Estimates | | | | |
| Effect | Label | | Margi | ns Estima | | andard<br>Error | DF t Va | lue |
| trtpn | Treatment contrast, | IDegLira - IDe | eg WORK. | ADATA2 -0.59 | 947 ( | 0.06819 | 715 -8 | .72 |
| | | Least Squ | uares Mean | ns Estimates | | | | |
| Effect | Label | | Pr > | t Alpha | Lower | Upper | Exponentia | ted |
| trtpn | Treatment contrast, | . IDegLira - IDe | eg <.00 | 0.05 - | -0.7286 | -0.4608 | 0.5 | 517 |

| Effect | Label | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment contrast | , IDegLira - IDeg | 0.4826 | 0.6308 |

| | 4148<br>Trial Report<br>document | | CONF | IDENTIAL | | Date:<br>Version:<br>Status:<br>Page: | 161 | December 2019<br>1.0<br>Fina<br>89 of 412 | 1 |
|---|---|---|---|---|---|---|---|---|---|
| HbA1c as | | of treatr | ment - change f | rom baselin | e – suj | pportive | statistica | l analysis · | - full |
| Paramete | er Code=C64849 | В | | | | | | | |
| The Mixe | ed Procedure | | | | | | | | |
| Least Squares Means Estimates | | | | | | | | | |
| Effect | Label | | | Margins | Est | timate | Standard<br>Error | DF t | /alue |
| trtpn | Treatment con | ntrast, II | DegLira - Lira | WORK.ADATA | .2 –( | 0.6283 | 0.06796 | 715 | -9.25 |
| | | | Least Squar | es Means Es | timate | 3 | | | |
| Effect | Label | | | Pr > t | Alpha | Lowe | er Uppe | r Exponent: | iated |
| trtpn | Treatment con | ntrast, II | DegLira - Lira | <.0001 | 0.05 | -0.761 | .8 -0.494 | 9 0 | .5335 |
| | | Least S | Squares Means E | stimates | | | | | |
| Effect | Label | | | Exponentia<br>Lo | ted<br>wer | Exponent | iated<br>Upper | | |
| trtpn | Treatment con | ntrast, II | DegLira - Lira | 0.4 | 668 | C | .6096 | | |

Nordisk

### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

HbAlc after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 66.2773

Fit Statistics

-2 Res Log Likelihood 5060.0 AIC (Smaller is Better) AICC (Smaller is Better) 5062.0 BIC (Smaller is Better) 5066.5

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 34.2233 Intercept 2.3673 715 14.46 <.0001 0.05 trtpn 1 -6.8678 0.7428 715 -9.25 < .0001 0.05 0.6690 trtpn -0.3679 0.8601 715 -0.43 0.05 3 trtpn PREOAD2 -4.2869 0.6497 715 -6.60 <.0001 0.05 Metformin Metformin + OAD PREOAD2 BASE 0.3338 0.03413 715 9.78 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 91 of 412 | |

HbAlc after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

Effect Label

### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 29.5757<br>-8.3262<br>-2.0566 | 38.8709<br>-5.4094<br>1.3207 |
| PREOAD2 | Metformin<br>Metformin + OAD | | -5.5625 | -3.0113 |
| BASE | IICCICIMIII / OAD | | 0.2668 | 0.4008 |

trtpn Treatment contrast, IDegLira - IDeg 0.000348

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 715 | 60.69 | <.0001 |
| PREOAD2 | 1 | 715 | 43.53 | <.0001 |
| BASE | 1 | 715 | 95.66 | <.0001 |

### Least Squares Means Estimates

| 7.55 | T 1 1 | | | Standard | 5.5 | | 5 | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
| trtpn | LSMeans, IDegLira | WORK.ADATA2 | 48.1560 | 0.4286 | 715 | 112.35 | <.0001 | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | 54.6559 | | | 89.72 | | 0.05 |
| trtpn | LSMeans, Lira | WORK.ADATA2 | 55.0238 | 0.6068 | 715 | 90.67 | <.0001 | 0.05 |
| | | Least Squ | ares Mean | s Estimates | | | | |
| | | | | | Expor | entiated | Exponentia | ated |
| Effect | Label | Lower | Upper | Exponentiated | - | Lower | Uŗ | per |
| trtpn | LSMeans, IDegLira | 47.3145 4 | 8.9975 | 8.201E20 | | 3.535E20 | 1.903 | BE21 |
| trtpn | LSMeans, IDeg | 53.4599 5 | | 5.454E23 | | 1.649E23 | 1.804 | |
| trtpn | LSMeans, Lira | 53.8324 5 | 6.2152 | 7.88E23 | | 2.394E23 | 2.594 | E24 |
| | | Least Squ | ares Mean | s Estimates | | | | |
| | | | | | St | andard | | |
| Effect | Label | | Margin | s Estima | ate | Error | DF t Va | lue |
| trtpn | Treatment contrast | IDegLira - IDe | a WORK.A | DATA2 -6.49 | 999 | 0.7453 | 715 -8 | 3.72 |
| 1 | | | , | | | | | |
| | | Least Squ | ares Mean | s Estimates | | | | |
| Effect | Label | | Pr > | t Alpha | Lower | Upper | Exponentia | ated |
| trtpn | Treatment contrast, | IDegLira - IDe | g <.00 | 01 0.05 | -7.9631 | -5.0367 | 0.001 | 504 |
| | Leas | st Squares Means | Estimate | S | | | | |
| | Loude bytates means betimeees | | | | | | | |

Exponentiated Exponentiated Lower Upper

0.006495

| | 4148<br>Trial Report<br>document | CONFI | DENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 De | ecember 2019<br>1.0<br>Final<br>92 of 412 | Novo I |
|---|---|---|---|---|---|---|---|
| HbA1c as | fter 26 weeks of treat<br>s set | tment - change f | rom baseline - | supportive | statistical | analysis - | full |
| Paramete | er Code=HBA1CONV | | | | | | |
| The Mixe | ed Procedure | | | | | | |
| | | Least Squar | es Means Estim | ates | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF t Va | alue |
| trtpn | Treatment contrast, I | DegLira - Lira | WORK.ADATA2 | -6.8678 | 0.7428 | 715 -9 | 9.25 |
| | | Least Squar | es Means Estim | ates | | | |
| Effect | Label | | Pr > t Al | pha Lowe | er Upper | Exponentia | ated |
| trtpn | Treatment contrast, I | DegLira - Lira | <.0001 0 | .05 -8.326 | 52 -5.4094 | 0.001 | 1041 |
| | Least | Squares Means E | stimates | | | | |
| Effect | Label | | Exponentiated Lower | | iated<br>Upper | | |
| trtpn | Treatment contrast, I | DegLira - Lira | 0.000242 | 0.0 | 004474 | | |

Nordisk

### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

HbAlc after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=C64849B

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 0.5548

Fit Statistics

-2 Res Log Likelihood 1635.3 AIC (Smaller is Better) AICC (Smaller is Better) 1637.3 BIC (Smaller is Better) 1641.9

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 4.5634 0.2879 715 15.85 <.0001 0.05 trtpn 1 -0.6283 0.06796 715 -9.25 <.0001 0.05 -0.03366 -0.43 0.6690 trtpn 0.07869 715 0.05 3 trtpn PREOAD2 -0.3922 0.05944 715 -6.60 <.0001 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.6662 0.03413 715 -19.52 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 94 of 412 | |

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=C64849B

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 3.9982<br>-0.7618<br>-0.1882 | 5.1287<br>-0.4949<br>0.1208 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -0.5089 | -0.2755 |
| BASE | | | -0.7332 | -0.5992 |

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 715 | 60.69 | <.0001 |
| PREOAD2 | 1 | 715 | 43.53 | <.0001 |
| BASE | 1 | 715 | 380.96 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -1.0822 | 0.03921<br>0.05574<br>0.05552 | 715<br>715<br>715 | -42.76<br>-19.42<br>-18.89 | <.0001<br><.0001<br><.0001 |
| | Least Squares Mean | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -1.7539<br>-1.1916<br>-1.1575 | -1.5999<br>-0.9728<br>-0.9395 | | | |

### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

HbAlc after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 66.2773

Fit Statistics

-2 Res Log Likelihood 5060.0 AIC (Smaller is Better) AICC (Smaller is Better) 5062.0 BIC (Smaller is Better) 5066.5

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 34.2233 Intercept 2.3673 715 14.46 <.0001 0.05 trtpn 1 -6.8678 0.7428 715 -9.25 < .0001 0.05 -0.43 0.6690 trtpn -0.3679 0.8601 715 0.05 3 trtpn PREOAD2 -4.2869 0.6497 715 -6.60 <.0001 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.6662 0.03413 715 -19.52 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 96 of 412 | |

 ${\tt HbAlc}$  after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=HBA1CONV

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 29.5757<br>-8.3262<br>-2.0566 | 38.8709<br>-5.4094<br>1.3207 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -5.5625 | -3.0113 |
| BASE | | | -0.7332 | -0.5992 |

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|-----------|---------|------------------|
| trtpn<br>PREOAD2 | 2 | 715 | 60.69 | <.0001<br><.0001 |
| | 1 | 715 | 43.53 | |
| BASE | 1 | 715 | 380.96 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -11.8284 | 0.4286<br>0.6092<br>0.6068 | 715<br>715<br>715 | -42.76<br>-19.42<br>-18.89 | <.0001<br><.0001<br><.0001 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 -1 | L9.1697<br>L3.0244<br>L2.6519 | -17.4868<br>-10.6323<br>-10.2690 | | | |

NN9068 Date: 16 December 2019 Novo Nordisk

NN9068-4148 CONFIDENTIAL
Clinical Trial Report Status: Final
Statistical document 

## 8: Responder for HbA1c treatment target - supportive statistical analysis - full analysis set

Parameter Code=HBA BL65

The GENMOD Procedure

Model Information

Data Set WORK.ADATA2
Distribution Binomial
Link Function Logit

Dependent Variable AVALC Analysis Value (C)

Number of Observations Read 720 Number of Observations Used 720 Number of Events 298 Number of Trials 720

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Response Profile

Ordered Total
Value AVALC Frequency

1 Y 298
2 N 422

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

Effect trtpn PREOAD2 Parameter Prm1 Intercept Prm2 trtpn Prm3 trtpn 2 Prm4 trtpn PREOAD2 PREOAD2 Prm5 Metformin Metformin + OAD Prm6 HBA1CBL Prm7

Criteria For Assessing Goodness Of Fit

Criterion DF Value Value/DF

Log Likelihood -412.3951
Full Log Likelihood -412.3951
AIC (smaller is better) 834.7901
AICC (smaller is better) 834.8741
BIC (smaller is better) 857.6864

Algorithm converged.

Analysis Of Maximum Likelihood Parameter Estimates

| | | | | Standard | Wald 9 | 95% | Wald | |
|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Error | Confidence | e Limits | Chi-Square | Pr > ChiSq |
| | | | | | | | - | - |
| Intercept | | 1 | 3.3360 | 0.8860 | 1.5994 | 5.0726 | 14.18 | 0.0002 |
| trtpn | 1 | 1 | 1.5276 | 0.2163 | 1.1037 | 1.9514 | 49.90 | <.0001 |
| trtpn | 2 | 1 | 0.1533 | 0.2546 | -0.3456 | 0.6522 | 0.36 | 0.5469 |

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Responder for HbAlc treatment target - supportive statistical analysis - full analysis set

Parameter Code=HBA\_BL65

The GENMOD Procedure

### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidence | | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>PREOAD2<br>PREOAD2 | 3 Metformin Metformin + OAD | 0<br>1<br>0 | 0.0000<br>1.1477<br>0.0000 | 0.0000<br>0.1809<br>0.0000 | 0.0000<br>0.7933<br>0.0000 | 0.0000<br>1.5022<br>0.0000 | 40.27 | <.0001 |
| HBA1CBL<br>Scale | | 1 | -0.6000<br>1.0000 | 0.1074 | -0.8105<br>1.0000 | -0.3894<br>1.0000 | 31.19 | <.0001 |

NOTE: The scale parameter was held fixed.

### Least Squares Means Estimates

| Effect | Label | | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans frequency,<br>LSMeans frequency,<br>LSMeans frequency, | IDeg | 0.4980<br>-0.8762<br>-1.0295 | 0.1204<br>0.1800<br>0.1821 | 4.14<br>-4.87<br>-5.65 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |

### Least Squares Means Estimates

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | LSMeans frequency, IDegLira | 0.2621 | 0.7340 | 1.6455 | 1.2997 | 2.0833 |
| trtpn | LSMeans frequency, IDeg | -1.2289 | -0.5235 | 0.4164 | 0.2926 | 0.5925 |
| trtpn | LSMeans frequency, Lira | -1.3864 | -0.6727 | 0.3572 | 0.2500 | 0.5103 |

### Least Squares Means Estimates

| Effect | Label | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Treatment odds ratio, IDegLira / IDeg<br>Treatment odds ratio, IDegLira / Lira | 1.3742<br>1.5276 | 0.2140<br>0.2163 | 6.42<br>7.06 | <.0001<br><.0001 | 0.05<br>0.05 |
| | Least Squares Means | Estimates | | | | |

| Effect | Label | Lower | Upper | Exponentiated |
|--------|-----------------------|--------|--------|---------------|
| trtpn | Treatment odds ratio, | 0.9549 | 1.7936 | 3.9521 |
| trtpn | Treatment odds ratio, | 1.1037 | 1.9514 | 4.6070 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | | io, IDegLira / IDeg | 2.5984 | 6.0111 |
| trtpn | | io, IDegLira / Lira | 3.0154 | 7.0387 |

# NN9068 NN9068-4148 Clinical Trial Report Date: 16 December 2019 Version: 1.0 Status: Final

Page:

99 of 412

Responder for HbAlc treatment target - supportive statistical analysis - full analysis set

Parameter Code=HBA\_BL7

The GENMOD Procedure

Statistical document

Model Information

Data Set WORK.ADATA2
Distribution Binomial
Link Function Logit

Dependent Variable AVALC Analysis Value (C)

Number of Observations Read 720
Number of Observations Used 720
Number of Events 448
Number of Trials 720

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Response Profile

Ordered Total
Value AVALC Frequency

1 Y 448
2 N 272

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

Effect Parameter PREOAD2 trtpn Prm1 Intercept Prm2 trtpn Prm3 trtpn Prm4 trtpn 3 PREOAD2 Prm5 Metformin Metformin + OAD PRECAD2 Prm6 HBA1CBL Prm7

Criteria For Assessing Goodness Of Fit

Criterion DF Value Value/DF
Log Likelihood -402.2667
Full Log Likelihood -402.2667

Algorithm converged.

Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidenc | | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| Intercept | | 1 | 5.2013 | 0.9001 | 3.4371 | 6.9654 | 33.39 | <.0001 |
| trtpn | 1 | 1 | 1.4327 | 0.2089 | 1.0234 | 1.8420 | 47.06 | <.0001 |
| trtpn | 2 | 1 | -0.0143 | 0.2262 | -0.4576 | 0.4291 | 0.00 | 0.9497 |


Responder for HbAlc treatment target - supportive statistical analysis - full analysis set

Parameter Code=HBA\_BL7

The GENMOD Procedure

### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidence | | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>PREOAD2<br>PREOAD2 | 3 Metformin Metformin + OAD | 0<br>1<br>0 | 0.0000<br>1.1167<br>0.0000 | 0.0000<br>0.1969<br>0.0000 | 0.0000<br>0.7307<br>0.0000 | 0.0000<br>1.5026<br>0.0000 | 32.16 | <.0001 |
| HBA1CBL<br>Scale | 1100101111111 7 0115 | 1 | -0.6859<br>1.0000 | 0.1082 | -0.8979<br>1.0000 | -0.4739<br>1.0000 | 40.22 | <.0001 |

NOTE: The scale parameter was held fixed.

### Least Squares Means Estimates

| Effect | Label | | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans frequency, | IDeg | 1.5454 | 0.1465 | 10.55 | <.0001 | 0.05 |
| trtpn | LSMeans frequency, | | 0.09841 | 0.1657 | 0.59 | 0.5526 | 0.05 |
| trtpn | LSMeans frequency, | | 0.1127 | 0.1628 | 0.69 | 0.4889 | 0.05 |

### Least Squares Means Estimates

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | LSMeans frequency, IDegLira | 1.2582 | 1.8325 | 4.6897 | 3.5191 | 6.2497 |
| trtpn | LSMeans frequency, IDeg | -0.2264 | 0.4232 | 1.1034 | 0.7974 | 1.5268 |
| trtpn | LSMeans frequency, Lira | -0.2064 | 0.4317 | 1.1193 | 0.8135 | 1.5399 |

### Least Squares Means Estimates

| Effect | Label | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Treatment odds ratio, IDegLira / IDeg<br>Treatment odds ratio, IDegLira / Lira | 1.4470<br>1.4327 | 0.2100<br>0.2089 | 6.89<br>6.86 | <.0001<br><.0001 | 0.05<br>0.05 |
| | Least Squares Means | Estimates | | | | |

| Effect | Label | Lower | Upper | Exponentiated |
|---|---|---|---|---|
| - | Treatment odds ratio,<br>Treatment odds ratio, | <br>1.0354<br>1.0234 | 1.8585<br>1.8420 | 4.2502<br>4.1900 |

| Effect | Label | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|
| trtpn | Treatment odds ratio, IDegLira / II | | 6.4142 |
| trtpn | Treatment odds ratio, IDegLira / Li | | 6.3095 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 101 of 412 | |

# 9: Responder for HbA1c treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes - supportive statistical analysis - full analysis set

Parameter Code=HB65CHY

The GENMOD Procedure

Model Information

Data Set Distribution WORK.ADATA2 Binomial Link Function Dependent Variable Logit AVALC

Analysis Value (C)

Number of Observations Read Number of Observations Used Number of Events Number of Trials 720 720 284 720

Class Level Information

Levels Class Values 1 2 3

3 1 2 3 2 Metformin Metformin + OAD trtpn PREOAD2

Response Profile

| Ordered | | Total |
|---------|-------|-----------|
| Value | AVALC | Frequency |
| 1 | Y | 284 |
| 2 | N | 436 |

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

| Parameter | Effect | trtpn | PREOAD2 |
|---|---|---|---|
| Prm1<br>Prm2<br>Prm3<br>Prm4<br>Prm5<br>Prm6<br>Prm7 | Intercept<br>trtpn<br>trtpn<br>trtpn<br>PREOAD2<br>PREOAD2<br>HBA1CBL | 1<br>2<br>3 | Metformin<br>Metformin + OAD |

Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|---|---|---|---|
| Log Likelihood<br>Full Log Likelihood<br>AIC (smaller is better)<br>AICC (smaller is better)<br>BIC (smaller is better) | - | -415.4484<br>-415.4484<br>840.8968<br>840.9808<br>863.7930 | |

Algorithm converged.

Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald 95%<br>Confidence Limits | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|
| Intercept<br>trtpn | 1 | _ | | 0.8796<br>0.2161 | 0.9962 4.4443<br>1.0242 1.8713 | | 0.0020<br><.0001 |


Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes – supportive statistical analysis – full analysis set

Parameter Code=HB65CHY

The GENMOD Procedure

### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidenc | | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | 2 | 1 | 0.1498 | 0.2562 | -0.3523<br>0.0000 | 0.6519 | 0.34 | 0.5587 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | 1 | 1.0974 | 0.1785 | 0.7475 | 1.4473 | 37.79 | <.0001 |
| HBA1CBL<br>Scale | | 1 0 | -0.5290<br>1.0000 | 0.1063 | -0.7374<br>1.0000 | -0.3207<br>1.0000 | 24.77 | <.0001 |
| NOTE: The | scale parameter w | as h | eld fixed. | | | | | |
| | | L | east Squar | es Means E | stimates | | | |

| Effect | Label | | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans frequency, | IDeg | 0.3613 | 0.1179 | 3.06 | 0.0022 | 0.05 |
| trtpn | LSMeans frequency, | | -0.9366 | 0.1807 | -5.18 | <.0001 | 0.05 |
| trtpn | LSMeans frequency, | | -1.0864 | 0.1834 | -5.92 | <.0001 | 0.05 |

### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans frequenc<br>LSMeans frequenc<br>LSMeans frequenc | y, IDeg | 0.1302<br>-1.2908<br>-1.4458 | 0.5923<br>-0.5825<br>-0.7270 | 1.4352<br>0.3920<br>0.3374 | 1.1390<br>0.2751<br>0.2356 | 1.8082<br>0.5585<br>0.4833 |

| Effect | Label | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Treatment odds ratio, IDegLira / IDeg<br>Treatment odds ratio, IDegLira / Lira | 1.2979<br>1.4477 | 0.2134<br>0.2161 | 6.08<br>6.70 | <.0001<br><.0001 | 0.05<br>0.05 |
| | Least Squares Means | Estimates | | | | |
| Effect | Label | Lower | Upper | Expone | ntiated | |
| trtpn<br>trtpn | Treatment odds ratio, IDegLira / IDeg<br>Treatment odds ratio, IDegLira / Lira | 0.8796<br>1.0242 | 1.7162<br>1.8712 | | 3.6616<br>4.2533 | |
| | Least Squares Means Es | timates | | | | |

| Effect | Label | Exponentiate Lowe | Exponentiated<br>Upper |
|---|---|---|---|
| trtpn<br>trtpn | Treatment<br>Treatment | 2.409<br>2.784 | 5.5632<br>6.4958 |

### NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes – supportive statistical analysis – full analysis set

Parameter Code=HB7CHY

The GENMOD Procedure

Model Information

Data Set WORK.ADATA2 Distribution Binomial Logit AVALC Link Function

Dependent Variable Analysis Value (C)

Number of Observations Read Number of Observations Used Number of Events Number of Trials 720 720 429 720

Class Level Information

Class Levels Values

trtpn 1 2 3 PREOAD2 Metformin Metformin + OAD

Response Profile

| Ordered | | Total |
|---------|-------|-----------|
| Value | AVALC | Frequency |
| 1 | Y | 429 |
| 2 | N | 291 |

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

| Parameter | Effect | trtpn | PREOAD2 |
|---|---|---|---|
| Prm1<br>Prm2<br>Prm3<br>Prm4<br>Prm5<br>Prm6 | Intercept<br>trtpn<br>trtpn<br>trtpn<br>PREOAD2<br>PREOAD2 | 1<br>2<br>3 | Metformin<br>Metformin + OAD |
| Prm7 | HBA1CBI. | | |

Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|---|---|---|---|
| Log Likelihood Full Log Likelihood AIC (smaller is better) AICC (smaller is better) BIC (smaller is better) | | -422.3970<br>-422.3970<br>854.7939<br>854.8780<br>877.6902 | |

Algorithm converged.

### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | Estimate | Standard<br>Error | | <br>Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|
| Intercept | _ | | | 2.4773 | <br>23.21 | <.0001 |


Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes – supportive statistical analysis – full analysis set

Parameter Code=HB7CHY

The GENMOD Procedure

### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidence | | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn | 2 | 1 | -0.0256<br>0.0000 | 0.2239 | -0.4644<br>0.0000 | 0.4133 | 0.01 | 0.9091 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | 1 | 1.0552 | 0.1883 | 0.6862 | 1.4243 | 31.40 | <.0001 |
| HBA1CBL<br>Scale | | 1 | -0.5676<br>1.0000 | 0.1040 | -0.7714<br>1.0000 | -0.3638<br>1.0000 | 29.80 | <.0001 |

NOTE: The scale parameter was held fixed.

### Least Squares Means Estimates

| Effect | Label | | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans frequency, | IDeg | 1.2949 | 0.1364 | 9.49 | <.0001 | 0.05 |
| trtpn | LSMeans frequency, | | 0.005601 | 0.1631 | 0.03 | 0.9726 | 0.05 |
| trtpn | LSMeans frequency, | | 0.03115 | 0.1606 | 0.19 | 0.8462 | 0.05 |

### Least Squares Means Estimates

| Effect | Label | | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans | frequency, frequency, frequency, | IDeg | 1.0275<br>-0.3142<br>-0.2836 | 1.5623<br>0.3254<br>0.3459 | 3.6507<br>1.0056<br>1.0316 | 2.7941<br>0.7304<br>0.7530 | 4.7700<br>1.3845<br>1.4133 |

## Least Squares Means Estimates

| Effect | Label | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Treatment odds ratio, IDegLira / IDeg<br>Treatment odds ratio, IDegLira / Lira | 1.2893<br>1.2638 | 0.2034<br>0.2022 | 6.34<br>6.25 | <.0001<br><.0001 | 0.05<br>0.05 |
| | Least Squares Means | Estimates | | | | |

# Effect Label Lower Upper Exponentiated trtpn Treatment odds ratio, IDegLira / IDeg 0.8906 1.6881 3.6303 trtpn Treatment odds ratio, IDegLira / Lira 0.8675 1.6600 3.5387

| Effect | Label | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|
| trtpn<br>trtpn | Treatment<br>Treatment | 2.4365<br>2.3810 | 5.4090<br>5.2593 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 105 of 412 | |

## 10: Responder for HbA1c treatment target without weight gain - supportive statistical analysis - full analysis set

Parameter Code=HB65WOWG

The GENMOD Procedure

Model Information

Data Set WORK.ADATA2 Distribution Binomial Logit AVALC Link Function

Analysis Value (C) Dependent Variable

Number of Observations Read Number of Observations Used Number of Events Number of Trials 169 720

Class Level Information

Class Levels Values 1 2 3 trtpn

PREOAD2 2 Metformin Metformin + OAD

Response Profile

Ordered Total AVALC Frequency Value 551

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

Effect trtpn PREOAD2 Parameter Prm1 Intercept Prm2 trtpn Prm3 trtpn 3 trtpn PREOAD2 Prm4 Metformin Prm5 Prm6 PREOAD2 Metformin + OAD Prm7 HBA1CBL Prm8 WGTBL

Criteria For Assessing Goodness Of Fit

Value Criterion Value/DF

Log Likelihood -365.5852 Full Log Likelihood
AIC (smaller is better)
AICC (smaller is better)
BIC (smaller is better) -365.5852 743.1705 743.2883

Algorithm converged.

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 106 of 412 | |

Responder for  $\tt HbAlc$  treatment target without weight gain - supportive statistical analysis - full analysis set

Parameter Code=HB65WOWG

The GENMOD Procedure

### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidenc | 95%<br>ce Limits | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| Intercept | | 1 | 1.8407 | 1.1171 | -0.3489 | 4.0302 | 2.71 | 0.0994 |
| trtpn | 1 | 1 | 0.5428 | 0.2209 | 0.1097 | 0.9758 | 6.04 | 0.0140 |
| trtpn | 2 | 1 | -0.6440 | 0.3007 | -1.2334 | -0.0546 | 4.59 | 0.0322 |
| trtpn | 3 | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 | | |
| PREOAD2 | Metformin | 1 | 0.4953 | 0.1891 | 0.1247 | 0.8660 | 6.86 | 0.0088 |
| PREOAD2 | Metformin + OAD | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 | | |
| HBA1CBL | | 1 | -0.4657 | 0.1184 | -0.6978 | -0.2336 | 15.46 | <.0001 |
| WGTBL | | 1 | 0.0056 | 0.0066 | -0.0072 | 0.0185 | 0.73 | 0.3923 |
| Scale | | 0 | 1.0000 | 0.0000 | 1.0000 | 1.0000 | | |

NOTE: The scale parameter was held fixed.

### Least Squares Means Estimates

| Effect | Label | | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans frequency, | IDeg | -0.7874 | 0.1214 | -6.48 | <.0001 | 0.05 |
| trtpn | LSMeans frequency, | | -1.9742 | 0.2366 | -8.34 | <.0001 | 0.05 |
| trtpn | LSMeans frequency, | | -1.3302 | 0.1898 | -7.01 | <.0001 | 0.05 |

### Least Squares Means Estimates

| Effect | Label | | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans | <pre>frequency, frequency, frequency,</pre> | IDeg | -1.0254<br>-2.4380<br>-1.7021 | -0.5494<br>-1.5104<br>-0.9582 | 0.4550<br>0.1389<br>0.2644 | 0.3586<br>0.08734<br>0.1823 | 0.5773<br>0.2208<br>0.3836 |

### Least Squares Means Estimates

| Effect | Label | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Treatment odds ratio, IDegLira / IDeg<br>Treatment odds ratio, IDegLira / Lira | 1.1867<br>0.5428 | 0.2630<br>0.2209 | 4.51<br>2.46 | <.0001<br>0.0140 | 0.05<br>0.05 |
| | Least Squares Means | Estimates | | | | |
| Effect | Label | Lower | Upper | Exponen | tiated | |
| trtpn<br>trtpn | Treatment odds ratio, IDegLira / IDeg<br>Treatment odds ratio, IDegLira / Lira | 0.6713<br>0.1097 | 1.7021<br>0.9758 | | 3.2764<br>1.7207 | |

| Effect | Label | Exponentiated Lowe: | Exponentiated Upper |
|---|---|---|---|
| trtpn<br>trtpn | Treatment<br>Treatment | 1.956<br>1.116 | 5.4856<br>2.6532 |

### NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

Responder for HbAlc treatment target without weight gain - supportive statistical analysis - full analysis set

Parameter Code=HBA7WOWG

The GENMOD Procedure

Model Information

Data Set WORK.ADATA2 Distribution Link Function Binomial Logit AVALC

Dependent Variable Analysis Value (C)

Number of Observations Read Number of Observations Used Number of Events Number of Trials 720 720 255 720

Class Level Information

Class Levels Values

trtpn 1 2 3 PREOAD2 Metformin Metformin + OAD

Response Profile

| Total | | Ordered |
|-----------|-------|---------|
| Frequency | AVALC | Value |
| 255 | Y | 1 |
| 465 | N | 2. |

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

| Parameter | Effect | trtpn | PREOAD2 |
|---|---|---|---|
| Prm1<br>Prm2<br>Prm3<br>Prm4<br>Prm5<br>Prm6<br>Prm7 | Intercept<br>trtpn<br>trtpn<br>trtpn<br>PREOAD2<br>PREOAD2<br>HBA1CBL<br>WGTBL | 1<br>2<br>3 | Metformin<br>Metformin + OAD |

Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|---|---|---|---|
| Log Likelihood Full Log Likelihood AIC (smaller is better) AICC (smaller is better) BIC (smaller is better) | | -443.5697<br>-443.5697<br>899.1394<br>899.2572<br>926.6149 | |

Algorithm converged.

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 108 of 412 | |

Responder for HbAlc treatment target without weight gain - supportive statistical analysis - full analysis set

Parameter Code=HBA7WOWG

The GENMOD Procedure

### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidence | 95%<br>ce Limits | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| Intercept | | 1 | 2.8025 | 0.9850 | 0.8719 | 4.7331 | 8.09 | 0.0044 |
| trtpn | 1 | 1 | -0.0231 | 0.1881 | -0.3918 | 0.3456 | 0.02 | 0.9024 |
| trtpn | 2 | 1 | -1.0805 | 0.2462 | -1.5630 | -0.5979 | 19.26 | <.0001 |
| trtpn | 3 | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 | | |
| PREOAD2 | Metformin | 1 | 0.2349 | 0.1710 | -0.1003 | 0.5701 | 1.89 | 0.1696 |
| PREOAD2 | Metformin + OAD | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 | | |
| HBA1CBL | | 1 | -0.3991 | 0.1024 | -0.5999 | -0.1983 | 15.18 | <.0001 |
| WGTBL | | 1 | 0.0004 | 0.0059 | -0.0111 | 0.0119 | 0.00 | 0.9458 |
| Scale | | 0 | 1.0000 | 0.0000 | 1.0000 | 1.0000 | | |

NOTE: The scale parameter was held fixed.

### Least Squares Means Estimates

| Effect | Label | | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans frequenc | y, IDeg | -0.3592 | 0.1129 | -3.18 | 0.0015 | 0.05 |
| trtpn | LSMeans frequenc | | -1.4167 | 0.1942 | -7.29 | <.0001 | 0.05 |
| trtpn | LSMeans frequenc | | -0.3362 | 0.1562 | -2.15 | 0.0314 | 0.05 |

### Least Squares Means Estimates

| Effect | Label | | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans | <pre>frequency, frequency, frequency,</pre> | IDeg | -1.7973 | -0.1380<br>-1.0360<br>-0.03007 | 0.6982<br>0.2425<br>0.7145 | 0.5596<br>0.1657<br>0.5261 | 0.8711<br>0.3549<br>0.9704 |

## Least Squares Means Estimates

| Effect | Label | stimate | Standard<br>Error z | : Value Pr | > z | Alpha |
|---|---|---|---|---|---|---|
| trtpn<br>trtpn | | 1.0574 | 0.2213<br>0.1881 | | <.0001<br>0.9024 | 0.05<br>0.05 |
| | Least Squares Means Est | imates | | | | |
| Effect | Label | Lower | Upper | Exponentia | ted | |
| trtpn<br>trtpn | Treatment odds ratio, IDegLira / IDeg<br>Treatment odds ratio, IDegLira / Lira - | 0.6237<br>-0.3918 | 1.4911<br>0.3456 | 2.8 | | |

| Effect | Label | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|
| trtpn<br>trtpn | Treatment<br>Treatment | 1.8658<br>0.6759 | 4.4421<br>1.4129 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 109 of 412 | |

# 11: Responder for HbA1c treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes and weight gain - supportive statistical analysis - full analysis set

Parameter Code=H65WOCHY

The GENMOD Procedure

Model Information

Data Set Distribution WORK.ADATA2 Binomial Link Function Dependent Variable Logit AVALC

Analysis Value (C)

Number of Observations Read Number of Observations Used Number of Events Number of Trials 720 720 160 720

Class Level Information

Levels Class Values 1 2 3

3 1 2 3 2 Metformin Metformin + OAD trtpn PREOAD2

Response Profile

| Ordered | | Total |
|---------|-------|-----------|
| Value | AVALC | Frequency |
| 1 | Y | 160 |
| 2 | N | 560 |

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

| Parameter | Effect | trtpn | PREOAD2 |
|---|---|---|---|
| Prm1<br>Prm2<br>Prm3<br>Prm4<br>Prm5<br>Prm6<br>Prm7 | Intercept<br>trtpn<br>trtpn<br>trtpn<br>PREOAD2<br>PREOAD2<br>HBA1CBL<br>WGTBL | 1<br>2<br>3 | Metformin<br>Metformin + OAD |

Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|---|---|---|---|
| Log Likelihood Full Log Likelihood AIC (smaller is better) AICC (smaller is better) BIC (smaller is better) | | -359.6463<br>-359.6463<br>731.2926<br>731.4104<br>758.7681 | |

Algorithm converged.

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIALE | Status: | Final | |
| Statistical document | | Page: | 110 of 412 | |

Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes and weight gain - supportive statistical analysis - full analysis set

Parameter Code=H65WOCHY

The GENMOD Procedure

trtpn trtpn

### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidence | 95%<br>ce Limits | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| Intercept | | 1 | 1.4599 | 1.1291 | -0.7530 | 3.6729 | 1.67 | 0.1960 |
| trtpn | 1 | 1 | 0.4667 | 0.2232 | 0.0292 | 0.9041 | 4.37 | 0.0366 |
| trtpn | 2 | 1 | -0.6089 | 0.3013 | -1.1994 | -0.0184 | 4.08 | 0.0433 |
| trtpn | 3 | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 | | |
| PREOAD2 | Metformin | 1 | 0.4783 | 0.1912 | 0.1036 | 0.8531 | 6.26 | 0.0124 |
| PREOAD2 | Metformin + OAD | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 | | |
| HBA1CBL | | 1 | -0.4171 | 0.1192 | -0.6508 | -0.1833 | 12.23 | 0.0005 |
| WGTBL | | 1 | 0.0051 | 0.0066 | -0.0079 | 0.0181 | 0.58 | 0.4450 |
| Scale | | 0 | 1.0000 | 0.0000 | 1.0000 | 1.0000 | | |

NOTE: The scale parameter was held fixed.

### Least Squares Means Estimates

| Effect | Label | | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans frequency, | IDeg | -0.8921 | 0.1233 | -7.23 | <.0001 | 0.05 |
| trtpn | LSMeans frequency, | | -1.9677 | 0.2360 | -8.34 | <.0001 | 0.05 |
| trtpn | LSMeans frequency, | | -1.3588 | 0.1911 | -7.11 | <.0001 | 0.05 |

### Least Squares Means Estimates

| Effect | Label | | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans | frequency, frequency, frequency, | IDeg | -2.4303 | -0.6504<br>-1.5050<br>-0.9843 | 0.4098<br>0.1398<br>0.2570 | 0.3218<br>0.08801<br>0.1767 | 0.5218<br>0.2220<br>0.3737 |

## Least Squares Means Estimates

| Effect | Label | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|
| trtpn<br>trtpn | Treatment odds ratio, IDegLira / IDeg<br>Treatment odds ratio, IDegLira / Lira | 1.0755<br>0.4667 | 0.2634<br>0.2232 | 4.08<br>2.09 | <.0001<br>0.0366 | 0.05<br>0.05 |
| | Least Squares Means | Estimates | | | | |
| Effect | Label | Lower | Upper | Exponer | itiated | |

0.5592 0.02919

1.5919 0.9041 2.9315 1.5947

### Least Squares Means Estimates

Treatment odds ratio, IDegLira / IDeg Treatment odds ratio, IDegLira / Lira

| Effect | Label | <u> </u> | Exponentiated<br>Lower | Exponentiated Upper |
|---|---|---|---|---|
| trtpn | Treatment odds ratio, IDeg | | 1.7492 | 4.9129 |
| trtpn | Treatment odds ratio, IDeg | | 1.0296 | 2.4698 |

### NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final 111 of 412 Statistical document Page:

Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes and weight gain - supportive statistical analysis - full analysis set

Parameter Code=HB7WOCHY

The GENMOD Procedure

Model Information

Data Set WORK.ADATA2 Distribution Link Function Binomial Logit AVALC

Dependent Variable Analysis Value (C)

Number of Observations Read Number of Observations Used Number of Events Number of Trials 720 720 241 720

Class Level Information

Class Levels Values

trtpn 1 2 3 PREOAD2 Metformin Metformin + OAD

Response Profile

| Ordered<br>Value | AVALC | Total<br>Frequency |
|------------------|--------|--------------------|
| 1 2 | Y<br>N | 241<br>479 |

PROC GENMOD is modeling the probability that AVALC='Y'.

Parameter Information

| Parameter | Effect | trtpn | PREOAD2 |
|---|---|---|---|
| Prm1<br>Prm2<br>Prm3<br>Prm4<br>Prm5<br>Prm6<br>Prm7<br>Prm8 | Intercept<br>trtpn<br>trtpn<br>trtpn<br>PREOAD2<br>PREOAD2<br>HBA1CBL<br>WGTBL | 1<br>2<br>3 | Metformin<br>Metformin + OAD |

Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|---|---|---|---|
| Log Likelihood Full Log Likelihood AIC (smaller is better) AICC (smaller is better) BIC (smaller is better) | | -438.4315<br>-438.4315<br>888.8631<br>888.9809<br>916.3386 | |

Algorithm converged.

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 112 of 412 | |

Responder for HbAlc treatment target without treatment emergent severe or BG confirmed hypoglycaemic episodes and weight gain - supportive statistical analysis - full analysis set

Parameter Code=HB7WOCHY

The GENMOD Procedure

### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confiden | 95%<br>ce Limits | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| Intercept | | 1 | 2.1921 | 0.9893 | 0.2532 | 4.1311 | 4.91 | 0.0267 |
| trtpn | 1 | 1 | -0.1069 | 0.1890 | -0.4774 | 0.2636 | 0.32 | 0.5717 |
| trtpn | 2 | 1 | -1.0692 | 0.2478 | -1.5549 | -0.5836 | 18.62 | <.0001 |
| trtpn | 3 | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 | | |
| PREOAD2 | Metformin | 1 | 0.2598 | 0.1720 | -0.0773 | 0.5968 | 2.28 | 0.1309 |
| PREOAD2 | Metformin + OAD | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 | | |
| HBA1CBL | | 1 | -0.3417 | 0.1029 | -0.5433 | -0.1401 | 11.03 | 0.0009 |
| WGTBL | | 1 | 0.0016 | 0.0059 | -0.0100 | 0.0131 | 0.07 | 0.7916 |
| Scale | | 0 | 1.0000 | 0.0000 | 1.0000 | 1.0000 | | |

NOTE: The scale parameter was held fixed.

### Least Squares Means Estimates

| Effect | Label | | Estimate | Standard<br>Error | z Value | Pr > z | Alpha |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans frequency,<br>LSMeans frequency,<br>LSMeans frequency, | IDeg | -0.4823<br>-1.4447<br>-0.3754 | 0.1139<br>0.1959<br>0.1564 | -4.23<br>-7.37<br>-2.40 | <.0001<br><.0001<br>0.0164 | 0.05<br>0.05<br>0.05 |

### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans frequency,<br>LSMeans frequency,<br>LSMeans frequency, | IDeg | -1.8286 | -0.2591<br>-1.0607<br>-0.06891 | 0.6173<br>0.2358<br>0.6870 | 0.4938<br>0.1606<br>0.5056 | 0.7718<br>0.3462<br>0.9334 |

### Least Squares Means Estimates

| Effect | Label | Estimate | Standard<br>Error | z Value Pr > z | Alpha |
|---|---|---|---|---|---|
| trtpn<br>trtpn | Treatment odds ratio, IDegLira / IDeg<br>Treatment odds ratio, IDegLira / Lira | 0.9623<br>-0.1069 | 0.2234<br>0.1890 | 4.31 <.0001<br>-0.57 0.5717 | 0.05<br>0.05 |
| | Least Squares Means | Estimates | | | |
| Effect | Label | Lower | Upper | Exponentiated | |
| trtpn<br>trtpn | Treatment odds ratio, IDegLira / IDeg<br>Treatment odds ratio, IDegLira / Lira | 0.5244<br>-0.4774 | 1.4002<br>0.2636 | 2.6177<br>0.8986 | |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | | tio, IDegLira / IDeg | 1.6894 | 4.0562 |
| trtpn | | tio, IDegLira / Lira | 0.6204 | 1.3016 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 113 of 412 | |

# 12: Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=C25208X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate Residual 6.8139

Fit Statistics

-2 Res Log Likelihood 3434.3
AIC (Smaller is Better) 3436.3
AICC (Smaller is Better) 3436.3
BIC (Smaller is Better) 3440.9

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t|Alpha -1.9302 2.5706 0.5566 0.2383 715 715 -3.47 10.79 0.0006 0.05 Intercept trtpn <.0001 0.05 3.6551 0.2756 715 13.26 <.0001 0.05 trtpn trtpn PREOAD2 Metformin 0.6254 0.2084 715 3.00 0.0028 0.05 PREOAD2 Metformin + OAD 0.9906 0.007083 715 139.86 <.0001 0.05 BASE

### NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=C25208X

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | -3.0230<br>2.1028<br>3.1140 | -0.8375<br>3.0384<br>4.1961 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | 0.2162 | 1.0347 |
| BASE | | | 0.9767 | 1.0045 |

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 715 | 95.37 | <.0001 |
| PREOAD2 | 1 | 715 | 9.00 | 0.0028 |
| BASE | 1 | 715 | 19562.2 | <.0001 |

### Least Squares Means Estimates

Standard

| Effect | Label | Margins | Estimate | e Erro | r DF | t Value | Pr > | t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 74.2782<br>75.362<br>71.707 | 7 0.1952 | 2 715 | 540.36<br>386.03<br>368.53 | <. ( | 0001<br>0001<br>0001 | 0.05<br>0.05<br>0.05 |
| | | Least Sq | uares Mean | ns Estimate: | S | | | | |
| Effect | Label | Lower | Upper | Exponentia | | nentiated<br>Lower | Expo | nentiate<br>Uppe | |
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | 74.9794 | 74.5480<br>75.7460<br>72.0896 | 1.814I<br>5.365I<br>1.387I | E32 | 1.385E32<br>3.657E32<br>9.469E30 | | 2.376E3<br>7.871E3<br>2.033E3 | 2 |
| | | Least Sq | uares Mean | ns Estimate: | S | | | | |
| Effect | Label | | Margi | ns Est | timate | Standard<br>Error | DF | t Valu | е |
| trtpn | Treatment contrast, | IDegLira - ID | eg WORK. | ADATA2 - | 1.0845 | 0.2389 | 715 | -4.5 | 4 |
| | | Least Sq | uares Mean | ns Estimate: | s | | | | |

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | <.0001 | 0.05 | -1.5535 | -0.6155 | 0.3381 |

| Effect | Label | | | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira - | - IDeg | 0.2115 | 0.5404 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 115 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=C25208X

The Mixed Procedure

Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | tandard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, IDe | egLira - Lira | WORK.ADATA2 | 2.5706 | 0.2383 | 715 | 10.79 |
| | | Least Square | es Means Estir | nates | | | |
| Effect | Label | | Pr > t Al | lpha Lower | Upper | Expone | ntiated |
| trtpn | Treatment contrast, IDe | egLira - Lira | <.0001 | 2.1028 | 3.0384 | | 13.0733 |
| | Least Squares Means Estimates | | | | | | |
| Effect | Label | | Exponentiated Lower | _ | ated<br>pper | | |

trtpn Treatment contrast, IDegLira - Lira 8.1888 20.8714

Upper

### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=WEIGHTU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 33.1179

Fit Statistics

-2 Res Log Likelihood 4566.4 AIC (Smaller is Better) AICC (Smaller is Better) 4568.4 BIC (Smaller is Better) 4572.9

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error -4.2554 -3.47 Intercept 1.2271 715 0.0006 0.05 trtpn 1 5.6671 0.5253 715 10.79 <.0001 0.05 <.0001 trtpn 8.0581 0.6075 715 13.26 0.05 3 trtpn PREOAD2 1.3789 0.4595 715 3.00 0.0028 0.05 Metformin Metformin + OAD PREOAD2 BASE 0.9906 0.007083 715 139.86 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 117 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=WEIGHTU

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | -6.6645<br>4.6358<br>6.8653 | -1.8463<br>6.6985<br>9.2509 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | 0.4766 | 2.2811 |
| BASE | | | 0.9767 | 1.0045 |

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 715 | 95.37 | <.0001 |
| PREOAD2 | 1 | 715 | 9.00 | 0.0028 |
| BASE | 1 | 715 | 19562.2 | <.0001 |

### Least Squares Means Estimates

| Effect. | Label | Margins | Estimat | Standard<br>e Error | DF | t Value | Day > 1±1 | 71.000 |
|---|---|---|---|---|---|---|---|---|
| FILECT | Label | Margins | ESTIMAT | e Filor | DF | t value | Pr > t | Alpha |
| trtpn | LSMeans, IDegLira | WORK.ADATA2 | 163.7 | 6 0.3030 | 715 | 540.36 | <.0001 | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | 166.1 | | 715 | 386.03 | | |
| trtpn | LSMeans, Lira | WORK.ADATA2 | 158.0 | 9 0.4290 | 715 | 368.53 | <.0001 | 0.05 |
| | | Least Sq | uares Mea | ns Estimates | | | | |
| | | | | | Expor | nentiated | Exponentia | ited |
| Effect | Label | Lower | Upper | Exponentiated | | Lower | Up | per |
| trtpn | LSMeans, IDegLira | 163.16 | 164.35 | 1.312E71 | | 7.238E70 | 2.379 | E71 |
| trtpn | LSMeans, IDeg | 165.30 | 166.99 | 1.434E72 | | 6.158E71 | 3.337 | |
| trtpn | LSMeans, Lira | 157.25 | 158.93 | 4.538E68 | | 1.955E68 | 1.053 | E69 |
| | | Least Sq | uares Mea | ns Estimates | | | | |
| Standard | | | | | | | | |
| Effect | Label | | Margi | ns Estima | | Error | DF t Va | lue |
| | | TD T' TD | | 3.53.53.0 | 0.0 | 0 5067 | 715 | F 4 |
| trtpn | Treatment contrast, | IDegLira - IDe | eg WORK. | ADATA2 -2.39 | 09 | 0.5267 | 715 -4 | .54 |
| Least Squares Means Estimates | | | | | | | | |
| Effect | Label | | Pr > | t Alpha | Lower | Upper | Exponentia | ted |
| trtpn | Treatment contrast, | IDegLira - IDe | eg <.0 | 001 0.05 - | 3.4249 | -1.3570 | 0.09 | 154 |

| Effect | Label | | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 0.03255 | 0.2574 |

| NN9068 | | Date: | 16 December 2019 <b>No</b> | ovo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 118 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=WEIGHTU

The Mixed Procedure

Least Squares Means Estimates

Effect Label Margins Estimate Error DF t Value trtpn Treatment contrast, IDegLira - Lira WORK.ADATA2 5.6671 0.5253 715 10.79

Least Squares Means Estimates

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - Lira <.0001 0.05 4.6358 6.6985 289.21

Least Squares Means Estimates

Effect Label Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - Lira 103.11 Exponentiated 311.17

### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=C25208X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 6.8139

Fit Statistics

-2 Res Log Likelihood 3434.3 AIC (Smaller is Better) AICC (Smaller is Better) 3436.3 BIC (Smaller is Better) 3440.9

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error -3.47 Intercept -1.9302 0.5566 715 0.0006 0.05 trtpn 1 2.5706 0.2383 715 10.79 <.0001 0.05 <.0001 trtpn 3.6551 0.2756 715 13.26 0.05 3 trtpn PREOAD2 0.6254 0.2084 715 3.00 0.0028 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.00938 0.007083 715 -1.32 0.1856 0.05
| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 120 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=C25208X

The Mixed Procedure

## Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | -3.0230<br>2.1028<br>3.1140 | -0.8375<br>3.0384<br>4.1961 |
| PREOAD2<br>PREOAD2<br>BASE | Metformin<br>Metformin + OAD | | 0.2162 | 1.0347 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 715 | 95.37 | <.0001 |
| PREOAD2 | 1 | 715 | 9.00 | 0.0028 |
| BASE | 1 | 715 | 1.76 | 0.1856 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 0.1480<br>1.2325<br>-2.4226 | 0.1375<br>0.1952<br>0.1946 | 715<br>715<br>715 | 1.08<br>6.31<br>-12.45 | 0.2819<br><.0001<br><.0001 |
| | Least Squares Mean | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -0.1219<br>0.8493<br>-2.8046 | 0.4179<br>1.6158<br>-2.0405 | | | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=WEIGHTU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 33.1179

Fit Statistics

-2 Res Log Likelihood 4566.4 AIC (Smaller is Better) AICC (Smaller is Better) 4568.4 BIC (Smaller is Better) 4572.9

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error -4.2554 -3.47 Intercept 1.2271 715 0.0006 0.05 trtpn 1 5.6671 0.5253 715 10.79 <.0001 0.05 trtpn 8.0581 0.6075 715 13.26 < .0001 0.05 3 trtpn PREOAD2 1.3789 0.4595 715 3.00 0.0028 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.00938 0.007083 715 -1.32 0.1856 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 122 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - confirmatory statistical analysis - full analysis set

Parameter Code=WEIGHTU

The Mixed Procedure

## Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | -6.6645<br>4.6358<br>6.8653 | -1.8463<br>6.6985<br>9.2509 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | 0.4766 | 2.2811 |
| BASE | | | -0.02329 | 0.004522 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 715 | 95.37 | <.0001 |
| PREOAD2 | 1 | 715 | 9.00 | 0.0028 |
| BASE | 1 | 715 | 1.76 | 0.1856 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 0.3263<br>2.7173<br>-5.3408 | 0.3030<br>0.4304<br>0.4290 | 715<br>715<br>715 | 1.08<br>6.31<br>-12.45 | 0.2819<br><.0001<br><.0001 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -0.2686<br>1.8723<br>-6.1830 | 0.9213<br>3.5623<br>-4.4986 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 123 of 412 | |

Parameter Code=C25208X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtan 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 674

Number of Observations

Number of Observations Read 674 Number of Observations Used 674 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 7.0840

Fit Statistics

-2 Res Log Likelihood 3241.1 AIC (Smaller is Better) 3243.1 AICC (Smaller is Better) 3243.1 BIC (Smaller is Better) 3247.6

Solution for Fixed Effects

Actual Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t| Alpha -2.1023 2.7218 0.5882 0.2548 669 -3.57 0.0004 0.05 Intercept 669 10.68 <.0001 0.05 trtan 3.8575 0.2933 669 13.15 <.0001 0.05 trtan trtan PREOAD2  ${\tt Metformin}$ 0.6458 0.2192 669 2.95 0.0033 0.05 PREOAD2 Metformin + OAD 0.9910 0.007451 669 132.99 <.0001 0.05 BASE

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 124 of 412 | |

Parameter Code=C25208X

The Mixed Procedure

## Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtan<br>trtan<br>trtan | | 1<br>2<br>3 | -3.2572<br>2.2216<br>3.2817 | -0.9475<br>3.2221<br>4.4334 |
| PREOAD2 | Metformin<br>Metformin + OAD | | 0.2154 | 1.0762 |
| BASE | | | 0.9764 | 1.0056 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtan | 2 | 669 | 92.95 | <.0001 |
| PREOAD2 | 1 | 669 | 8.68 | 0.0033 |
| BASE | 1 | 669 | 17686.7 | <.0001 |

## Least Squares Means Estimates

| | | | | Standard | | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
| trtan<br>trtan<br>trtan | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 74.3557<br>75.4914<br>71.6338 | 0.1436<br>0.2043<br>0.2104 | 669<br>669 | 517.92<br>369.57<br>340.39 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |
| | | Least Sq | uares Means | Estimates | | | | |

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtan | LSMeans, IDegLira | 74.0738 | 74.6376 | 1.96E32 | 1.479E32 | 2.598E32 |
| trtan | LSMeans, IDeg | 75.0903 | 75.8924 | 6.102E32 | 4.086E32 | 9.113E32 |
| trtan | LSMeans, Lira | 71.2206 | 72.0471 | 1.289E31 | 8.526E30 | 1.948E31 |

## Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtan | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -1.1357 | 0.2498 | 669 | -4.55 |

## Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtan | Treatment contrast, | IDegLira - IDeg | <.0001 | 0.05 | -1.6262 | -0.6452 | 0.3212 |

| Effect | Label | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtan | Treatment contrast, | IDegLira - IDeg | 0.1967 | 0.5245 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019<br>1.0<br>Final<br>125 of 412 | |
|---|---|---|---|---|
| Body weight after 26 weeks of | treatment - change from basel | ine - statist | ical sensitivity anal | ysis - |

per protocol analysis set

Parameter Code=C25208X

The Mixed Procedure

Least Squares Means Estimates

Standard Margins Estimate Error DF t Value Effect Label trtan Treatment contrast, IDegLira - Lira WORK.ADATA2 2.7218 0.2548 669 10.68 Least Squares Means Estimates Pr > |t| Alpha Lower Upper Exponentiated Effect Label trtan Treatment contrast, IDegLira - Lira <.0001 0.05 2.2216 3.2221 15.2082 Least Squares Means Estimates

Exponentiated Exponentiated Lower Upper Upper Effect Label trtan Treatment contrast, IDegLira - Lira 9.2217 25.0810


Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set

Parameter Code=WEIGHTU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtan 3 123

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 674

Number of Observations

Number of Observations Read 674 Number of Observations Used 674 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 34.4308

Fit Statistics

-2 Res Log Likelihood 4300.5 AIC (Smaller is Better) 4302.5 AICC (Smaller is Better) 4302.5 BIC (Smaller is Better) 4307.0

Solution for Fixed Effects

Actual Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error -3.57 Intercept -4.6348 1.2967 669 0.0004 0.05 trtan 1 6.0006 0.5617 669 10.68 <.0001 0.05 <.0001 trtan 8.5044 0.6465 669 13.15 0.05 3 t.rt.an 1.4238 PREOAD2 0.4832 669 2.95 0.0033 0.05 Metformin Metformin + OAD PREOAD2 BASE 0.9910 0.007451 669 132.99 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 127 of 412 | |

Parameter Code=WEIGHTU

The Mixed Procedure

## Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtan<br>trtan<br>trtan | | 1<br>2<br>3 | -7.1808<br>4.8977<br>7.2349 | -2.0888<br>7.1035<br>9.7739 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | 0.4750 | 2.3727 |
| BASE | | | 0.9764 | 1.0056 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtan | 2 | 669 | 92.95 | <.0001 |
| PREOAD2 | 1 | 669 | 8.68 | 0.0033 |
| BASE | 1 | 669 | 17686.7 | <.0001 |

## Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>e Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtan<br>trtan<br>trtan | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 163.93<br>166.43<br>157.93 | 3 0.4503 | 669<br>669 | 517.92<br>369.57<br>340.39 | | 0.05<br>0.05<br>0.05 |
| | | Least Sq | uares Mean | ns Estimates | | | | |
| Effect | Label | Lower | Upper | Exponentiated | Expo | nentiated<br>Lower | Exponent: | lated<br>Jpper |
| trtan<br>trtan<br>trtan | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | 163.30<br>165.55<br>157.01 | 164.55<br>167.31<br>158.84 | 1.557E71<br>1.904E72<br>3.857E68 | | 8.363E70<br>7.863E71<br>1.551E68 | 4.60 | 98E71<br>99E72<br>91E68 |
| | | Least Sq | uares Mea | ns Estimates | | | | |
| Effect | Label | | Margi | ns Estima | _ | tandard<br>Error | DF t | /alue |
| trtan | Treatment contrast, | . IDegLira - ID | eg WORK. | ADATA2 -2.50 | 38 | 0.5507 | 669 - | -4.55 |
| | | Least Sq | uares Mean | ns Estimates | | | | |
| Effect | Label | | Pr > | t Alpha | Lower | Upper | Exponent | lated |

trtan Treatment contrast, IDegLira - IDeg <.0001 0.05 -3.5850 -1.4225 0.08178

| Effect | Label | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtan | Treatment contrast, | IDegLira - IDeg | 0.02774 | 0.2411 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019 1.0 Final 128 of 412 | Novo Nordisk |
|---|---|---|---|---|
| Body weight after 26 weeks of t<br>per protocol analysis set | treatment - change from basel. | ine - statistical | sensitivity anal | ysis - |
| Parameter Code=WEIGHTU | | | | |
| The Mixed Procedure | | | | |
| | Least Squares Means Estima | tes | | |
| Effect Label | Margins | Standa<br>Estimate Erre | | lue |
| trtan Treatment contrast, IDe | egLira - Lira WORK.ADATA2 | 6.0006 0.56 | 17 669 10 | .68 |

Least Squares Means Estimates

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtan Treatment contrast, IDegLira - Lira <.0001 0.05 4.8977 7.1035 403.68

Least Squares Means Estimates

Exponentiated Lower Upper trtan Treatment contrast, IDegLira - Lira 133.98 Exponentiated 1216.26


Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set

Parameter Code=C25208X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtan 3 123

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 674

Number of Observations

Number of Observations Read 674
Number of Observations Used 674
Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 7.0840

Fit Statistics

-2 Res Log Likelihood 3241.1 AICC (Smaller is Better) 3243.1 AICC (Smaller is Better) 3243.1 BIC (Smaller is Better) 3247.6

Solution for Fixed Effects

Actual Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error -3.57 Intercept -2.1023 0.5882 669 0.0004 0.05 trtan 1 2.7218 0.2548 669 10.68 < .0001 0.05 <.0001 trtan 3.8575 0.2933 669 13.15 0.05 3 t.rt.an PREOAD2 0.6458 0.2192 669 2.95 0.0033 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.00902 0.007451 669 -1.21 0.2267 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 130 of 412 | |

Parameter Code=C25208X

The Mixed Procedure

## Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtan<br>trtan<br>trtan | | 1<br>2<br>3 | -3.2572<br>2.2216<br>3.2817 | -0.9475<br>3.2221<br>4.4334 |
| PREOAD2 | Metformin<br>Metformin + OAD | | 0.2154 | 1.0762 |
| BASE | | | -0.02365 | 0.005614 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtan | 2 | 669 | 92.95 | <.0001 |
| PREOAD2 | 1 | 669 | 8.68 | 0.0033 |
| BASE | 1 | 669 | 1.46 | 0.2267 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtan<br>trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 1.2989 | 0.1436<br>0.2043<br>0.2104 | 669<br>669<br>669 | 1.14<br>6.36<br>-12.16 | 0.2559<br><.0001<br><.0001 |
| | Least Squares Mear | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtan<br>trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -0.1186<br>0.8979<br>-2.9718 | 0.4451<br>1.7000<br>-2.1454 | | | |


Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - per protocol analysis set

Parameter Code=WEIGHTU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable CHG
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values

trtan 3 123

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 674

Number of Observations

Number of Observations Read 674 Number of Observations Used 674 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 34.4308

Fit Statistics

-2 Res Log Likelihood 4300.5 AIC (Smaller is Better) 4302.5 AICC (Smaller is Better) 4302.5 BIC (Smaller is Better) 4307.0

Solution for Fixed Effects

Actual Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept -4.6348 1.2967 669 -3.57 0.0004 0.05 trtan 1 6.0006 0.5617 669 10.68 <.0001 0.05 <.0001 trtan 8.5044 0.6465 669 13.15 0.05 3 t.rt.an 1.4238 PREOAD2 0.4832 669 2.95 0.0033 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.00902 0.007451 669 -1.21 0.2267 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 132 of 412 | |

Parameter Code=WEIGHTU

The Mixed Procedure

## Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Actual<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtan<br>trtan<br>trtan | | 1<br>2<br>3 | -7.1808<br>4.8977<br>7.2349 | -2.0888<br>7.1035<br>9.7739 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | 0.4750 | 2.3727 |
| BASE | | | -0.02365 | 0.005614 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtan | 2 | 669 | 92.95 | <.0001 |
| PREOAD2 | 1 | 669 | 8.68 | 0.0033 |
| BASE | 1 | 669 | 1.46 | 0.2267 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtan<br>trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 2.8637 | 0.3165<br>0.4503<br>0.4640 | 669<br>669<br>669 | 1.14<br>6.36<br>-12.16 | 0.2559<br><.0001<br><.0001 |
| | Least Squares Mean | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtan<br>trtan<br>trtan | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -0.2616<br>1.9794<br>-6.5517 | 0.9814<br>3.7479<br>-4.7297 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 133 of 412 | |

Parameter Code=C25208X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 659

Number of Observations

Number of Observations Read 659 Number of Observations Used 659 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 7.1903

Fit Statistics

-2 Res Log Likelihood 3178.8
AIC (Smaller is Better) 3180.8
AICC (Smaller is Better) 3180.8
BIC (Smaller is Better) 3185.3

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t| Alpha -2.0338 0.5997 0.2623 -3.39 10.27 0.0007 0.05 654 Intercept trtpn 2.6948 654 <.0001 0.05 3.8227 0.3012 654 12.69 <.0001 0.05 trtpn trtpn PREOAD2  ${\tt Metformin}$ 0.6288 0.2232 654 2.82 0.0050 0.05 PREOAD2 Metformin + OAD 0.9907 0.007605 654 130.26 <.0001 0.05 BASE

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 134 of 412 | |

Parameter Code=C25208X

The Mixed Procedure

## Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | -3.2114<br>2.1797<br>3.2313 | -0.8561<br>3.2099<br>4.4141 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | 0.1905 | 1.0670 |
| BASE | | | 0.9757 | 1.0056 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 654 | 85.96 | <.0001 |
| PREOAD2 | 1 | 654 | 7.94 | 0.0050 |
| BASE | 1 | 654 | 16968.0 | <.0001 |

## Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > | t Alpha | ì |
|---|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 74.3137<br>75.4416<br>71.6190 | 0.2076 | 654<br>654<br>654 | 511.41<br>363.33<br>328.11 | <.00<br><.00<br><.00 | 01 0.05 | 5 |
| Least Squares Means Estimates | | | | | | | | | |
| Effect | Label | Lower | Upper | Exponentiated | Expo | nentiated<br>Lower | Expone | ntiated<br>Upper | |
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | 75.0339 | 74.5991<br>75.8493<br>72.0476 | 1.88E32<br>5.806E32<br>1.27E31 | | 1.413E32<br>3.862E32<br>8.271E30 | | 2.5E32<br>.729E32<br>.949E31 | |
| | | Least Sq | uares Mear | ns Estimates | | | | | |
| Effect | Label | | Margin | ns Estimat | | tandard<br>Error | DF | t Value | |
| trtpn | Treatment contrast | , IDegLira - ID | eg WORK. | ADATA2 -1.123 | 79 | 0.2536 | 654 | -4.45 | |
| | | Ioast So | ularos Moar | ne Fetimatos | | | | | |

## Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | <.0001 | 0.05 | -1.6258 | -0.6299 | 0.3237 |

| Effect | Label | | | | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira | - ID | eg | 0.1968 | 0.5326 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 201<br>1<br>Fin<br>135 of 4 | 0<br>al |
|---|---|---|---|---|
| Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set | | | | |
| Parameter Code=C25208X | | | | |
| The Mixed Procedure | | | | |
| Least Squares Means Estimates | | | | |
| Effect Label | Margins | | ndard<br>Error DF t | Value |
| trtpn Treatment contrast, II | DegLira - Lira WORK.ADATA2 | 2.6948 0 | .2623 654 | 10.27 |
| Least Squares Means Estimates | | | | |
| Effect Label | Pr > t | Alpha Lower | Upper Exponent | iated |
| trtpn Treatment contrast, II | DegLira - Lira <.0001 | 0.05 2.1797 | 3.2099 1 | 1.8025 |
| Least Squares Means Estimates | | | | |

Effect Label Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - Lira 8.8438 Exponentiated Upper

#### NN9068 16 December 2019 Date: Novo Nordisk NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis completer analysis set

Parameter Code=WEIGHTU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 659

Number of Observations

Number of Observations Read 659 Number of Observations Used 659 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 34.9472

Fit Statistics

-2 Res Log Likelihood 4214.4 AIC (Smaller is Better) AICC (Smaller is Better) 4216.4 BIC (Smaller is Better) 4220.9

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect treatment2 01 (N) Estimate DF t Value Pr > |t| Alpha Error -4.4837 -3.39 Intercept 1.3222 654 0.0007 0.05 trtpn 1 5.9410 0.5783 654 10.27 <.0001 0.05 <.0001 trtpn 8.4275 0.6640 654 12.69 0.05 3 trtpn PREOAD2 1.3862 0.4920 654 2.82 0.0050 0.05 Metformin Metformin + OAD PREOAD2 BASE 0.9907 0.007605 654 130.26 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 137 of 412 | |

Parameter Code=WEIGHTU

The Mixed Procedure

## Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn<br>PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | 1<br>2<br>3 | -7.0800<br>4.8055<br>7.1237<br>0.4201 | -1.8874<br>7.0766<br>9.7313<br>2.3524 |
| BASE | | | 0.9757 | 1.0056 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 654 | 85.96 | <.0001 |
| PREOAD2 | 1 | 654 | 7.94 | 0.0050 |
| BASE | 1 | 654 | 16968.0 | <.0001 |

## Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans,<br>LSMeans,<br>LSMeans, | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 163.83<br>166.32<br>157.89 | 0.3204<br>0.4578<br>0.4812<br>Estimates | 654<br>654<br>654 | 511.41<br>363.33<br>328.11 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | 163.20 | 164.46 | 1.419E71 | 7.567E70 | 2.663E71 |
| trtpn | LSMeans, IDeg | 165.42 | 167.22 | 1.706E72 | 6.944E71 | 4.191E72 |
| trtpn | LSMeans, Lira | 156.95 | 158.84 | 3.732E68 | 1.451E68 | 9.601E68 |

## Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Error | DF | t Value | |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -2.4865 | 0.5591 | 654 | -4.45 |

## Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | <.0001 | 0.05 | -3.5843 | -1.3887 | 0.08320 |

| Effect | Label | | | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira - | IDeg | 0.02776 | 0.2494 |

| | -4148<br>Trial Report<br>I document | CONF | IDENTIAL | Date:<br>Version<br>Status<br>Page: | on:<br>s: | 16 Dec | cember 2<br>I<br>138 of | 1.0<br>Final | Novo Nordisk |
|---|---|---|---|---|---|---|---|---|---|
| | Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - completer analysis set | | | | | | | | |
| Paramet | er Code=WEIGHTU | | | | | | | | |
| The Mix | ed Procedure | | | | | | | | |
| | | Least Squar | res Means Esti | imates | | | | | |
| Effect | Label | | Margins | Estimat | Standa<br>te Err | | DF | t Valı | ie |
| trtpn | Treatment contrast, | IDegLira - Lira | WORK.ADATA2 | 5.941 | 10 0.57 | 83 | 654 | 10.2 | 27 |
| Least Squares Means Estimates | | | | | | | | | |
| Effect | Label | | Pr > t A | Alpha | Lower | Upper | Expone | entiate | ed |
| trtpn | Treatment contrast, | IDegLira - Lira | <.0001 | 0.05 | 1.8055 7 | .0766 | | 380.3 | 32 |
| | Least Squares Means Estimates | | | | | | | | |

Exponentiated Exponentiated Lower Upper

trtpn Treatment contrast, IDegLira - Lira 122.18 1183.89

Effect Label

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis completer analysis set

Parameter Code=C25208X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 659

Number of Observations

Number of Observations Read 659 Number of Observations Used 659 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 7.1903

Fit Statistics

-2 Res Log Likelihood 3178.8 AIC (Smaller is Better) AICC (Smaller is Better) 3180.8 BIC (Smaller is Better) 3185.3

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect treatment2 01 (N) Estimate DF t Value Pr > |t| Alpha Error -3.39 Intercept -2.0338 0.5997 654 0.0007 0.05 trtpn 1 2.6948 0.2623 654 10.27 <.0001 0.05 12.69 <.0001 trtpn 3.8227 0.3012 654 0.05 3 trtpn PREOAD2 0.6288 0.2232 654 2.82 0.0050 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.00935 0.007605 654 -1.23 0.2194 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 140 of 412 | |

Parameter Code=C25208X

The Mixed Procedure

## Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | -3.2114<br>2.1797<br>3.2313 | -0.8561<br>3.2099<br>4.4141 |
| PREOAD2 | Metformin<br>Metformin + OAD | - | 0.1905 | 1.0670 |
| BASE | 1100101111111 / 0112 | | -0.02428 | 0.005584 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 654 | 85.96 | <.0001 |
| PREOAD2 | 1 | 654 | 7.94 | 0.0050 |
| BASE | 1 | 654 | 1.51 | 0.2194 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLin<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2 WORK.ADATA2 WORK.ADATA2 | 1.3028 | 0.1453<br>0.2076<br>0.2183 | 654<br>654<br>654 | 1.20<br>6.27<br>-11.54 | 0.2292<br><.0001<br><.0001 |
| | Least Squares Mea | ns Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLin<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -0.1104<br>0.8951<br>-2.9485 | 0.4602<br>1.7105<br>-2.0913 | | | |

#### NN9068 16 December 2019 Date: Novo Nordisk NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis completer analysis set

Parameter Code=WEIGHTU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 659

Number of Observations

Number of Observations Read 659 Number of Observations Used 659 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 34.9472

Fit Statistics

-2 Res Log Likelihood 4214.4 AIC (Smaller is Better) AICC (Smaller is Better) 4216.4 BIC (Smaller is Better) 4220.9

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect treatment2 01 (N) Estimate DF t Value Pr > |t| Alpha Error -4.4837 Intercept 1.3222 654 -3.39 0.0007 0.05 trtpn 1 5.9410 0.5783 654 10.27 <.0001 0.05 12.69 <.0001 trtpn 8.4275 0.6640 654 0.05 3 trtpn PREOAD2 0.05 1.3862 0.4920 654 2.82 0.0050 Metformin Metformin + OAD PREOAD2 BASE -0.00935 0.007605 654 -1.23 0.2194 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 142 of 412 | |

Parameter Code=WEIGHTU

The Mixed Procedure

## Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn<br>preoad2 | Metformin | 1<br>2<br>3 | -7.0800<br>4.8055<br>7.1237 | -1.8874<br>7.0766<br>9.7313 |
| PREOAD2<br>BASE | Metformin + OAD | | -0.02428 | 0.005584 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 654 | 85.96 | <.0001 |
| PREOAD2 | 1 | 654 | 7.94 | 0.0050 |
| BASE | 1 | 654 | 1.51 | 0.2194 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 2.8721 | 0.3204<br>0.4578<br>0.4812 | 654<br>654<br>654 | 1.20<br>6.27<br>-11.54 | 0.2292<br><.0001<br><.0001 |
| | Least Squares Mean | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -0.2435<br>1.9733<br>-6.5003 | 1.0146<br>3.7710<br>-4.6105 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 143 of 412 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

### Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Subject Effect
Stimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
Satterthwaite

## Class Level Information

| Class | Levels | Values |
|---------|--------|---------------------------|
| TRT01PN | 3 | 1 2 3 |
| avisitn | 6 | 60 100 140 180 220 280 |
| PREOAD2 | 2 | Metformin Metformin + OAD |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 144 of 412 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 720



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 145 of 412 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 146 of 412 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure



## Dimensions

| Covariance | Parameters | 21 |
|------------|------------|-----|
| Columns in | X | 37 |
| Columns in | Z | 0 |
| Subjects | | 720 |
| Max Obs pe | r Subject | 6 |

## Number of Observations

| Number | of | Observations | Read | 4320 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 4046 |
| Number | of | Observations | Not Used | 274 |


Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

## Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 17548.36814718 | 0.00000775 |
| 1 | 2 | 13253.73696060 | |
| 2 | 1 | 13253.71397046 | |

Convergence criteria met.

## Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|---|---|---|
| UN(1,1)<br>UN(2,1)<br>UN(2,2)<br>UN(3,1)<br>UN(3,2)<br>UN(3,3)<br>UN(4,1)<br>UN(4,2)<br>UN(4,3)<br>UN(4,4)<br>UN(5,1) | SUBJID | Estimate |
| UN (5,3)<br>UN (5,4)<br>UN (5,5)<br>UN (6,1)<br>UN (6,2)<br>UN (6,3)<br>UN (6,4) | SUBJID | |

## Fit Statistics

| -2 Res Log Likelihood | 13253.7 |
|--------------------------|---------|
| AIC (Smaller is Better) | 13295.7 |
| AICC (Smaller is Better) | 13295.9 |
| BIC (Smaller is Better) | 13391.9 |

## Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|-----|------------|------------|
| 2.0 | 4294.65 | < .0001 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---|---|---|---|---|
| TRT01PN(avisitn) PREOAD2(avisitn) BASE(avisitn) | 12 | 814 | 20.33 | <.0001 |
| | 6 | 674 | 2.75 | 0.0120 |
| | 6 | 676 | 12856.3 | <.0001 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 148 of 412 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| TRT01PN(avisitn) TRT01PN(avisitn) TRT01PN(avisitn) | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ANA_DATA<br>WORK.ANA_DATA<br>WORK.ANA_DATA | 74.3474<br>75.4830<br>71.6194 | 0.1440<br>0.2052<br>0.2118 | 672.4<br>675.4<br>698.6 | 516.20<br>367.88<br>338.12 | <.0001<br><.0001<br><.0001 |
| | Least Squares Mea | ans Estimates | | | | | |
| Effect | Label | Alpha I | lower | Upper | | | |
| TRT01PN(avisitn) TRT01PN(avisitn) TRT01PN(avisitn) | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | 0.05 75. | .0801 7 | 74.6302<br>75.8858<br>72.0353 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 149 of 412 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

## Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
SVAL
WORK.ANA\_DATA
AVAL
Unstructured
SUBJID
REML
None
Method
Model-Based
Satterthwaite

## Class Level Information

| Class | Levels | Values |
|--------------------|--------|---------------------------------|
| TRT01PN<br>avisitn | 3<br>6 | 1 2 3<br>60 100 140 180 220 280 |
| PREOAD2 | 2 | Metformin Metformin + OAD |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 150 of 412 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

Class Level Information

Class Levels Values
SUBJID 720



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 151 of 412 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 152 of 412 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure



## Dimensions

| Covariance | Parameters | 21 |
|------------|------------|-----|
| Columns in | X | 37 |
| Columns in | Z | 0 |
| Subjects | | 720 |
| Max Obs pe | r Subject | 6 |

## Number of Observations

| Number of Observat<br>Number of Observat<br>Number of Observat | tions Used 4046 |
|---|---|
|---|---|


Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

## Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 23907.60340805 | |
| 1 | 2 | 19612.97222150 | 0.00000372 |
| 2 | 1 | 19612.94923134 | 0.00000000 |

Convergence criteria met.

## Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|---|---|---|
| UN(1,1)<br>UN(2,1)<br>UN(2,2)<br>UN(3,1)<br>UN(3,2)<br>UN(3,3)<br>UN(4,1)<br>UN(4,2)<br>UN(4,3)<br>UN(4,4)<br>UN(5,1)<br>UN(5,2) | Subject SUBJID | Estimate |
| UN(6,4)<br>UN(6,5)<br>UN(6,6) | SUBJID<br>SUBJID<br>SUBJID | |

## Fit Statistics

| -2 Res Log Likelihood | 19612.9 |
|--------------------------|---------|
| AIC (Smaller is Better) | 19654.9 |
| AICC (Smaller is Better) | 19655.2 |
| BIC (Smaller is Better) | 19751.1 |

## Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|-----|------------|------------|
| 2.0 | 4294.65 | < .0001 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|-------------------|-----------|-----------|---------|--------|
| TRT01PN(avisitn) | 12 | 814 | 20.33 | <.0001 |
| PREOAD2 (avisitn) | 6 | 674 | 2.75 | 0.0120 |
| BASE(avisitn) | 6 | 676 | 12856.3 | <.0001 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 154 of 412 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| TRT01PN(avisitn) TRT01PN(avisitn) TRT01PN(avisitn) | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ANA_DATA<br>WORK.ANA_DATA<br>WORK.ANA_DATA | 163.91<br>166.41<br>157.89 | 0.3175<br>0.4524<br>0.4670 | 672.4<br>675.4<br>698.6 | 516.20<br>367.88<br>338.12 | <.0001<br><.0001<br><.0001 |
| Least Squares Means Estimates | | | | | | | |
| Effect | Label | Alpha I | Lower | Upper | | | |
| TRT01PN(avisitn) TRT01PN(avisitn) TRT01PN(avisitn) | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | 0.05 16 | 55.52 | 164.53<br>167.30<br>158.81 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 155 of 412 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

## Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
SWBK.ANA\_DATA
CHG
Unstructured
SUBJID
REML
None
Method
Model-Based
Satterthwaite

## Class Level Information

| Class | Levels | Values |
|--------------------|--------|---------------------------------|
| TRT01PN<br>avisitn | 3<br>6 | 1 2 3<br>60 100 140 180 220 280 |
| PREOAD2 | 2 | Metformin Metformin + OAD |
| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 156 of 412 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 720



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 157 of 412 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 158 of 412 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure



## Dimensions

| Covariance | Parameters | 21 |
|-------------|------------|-----|
| Columns in | X | 37 |
| Columns in | Z | 0 |
| Subjects | | 720 |
| Max Obs per | : Subject | 6 |

## Number of Observations

| Number | of | Observations | Read | 4320 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 4046 |
| Number | of | Observations | Not Used | 274 |


Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

## Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 17548.36814717 | |
| 1 | 2 | 13253.73696060 | 0.00000775 |
| 2 | 1 | 13253.71397046 | 0.00000000 |

Convergence criteria met.

### Covariance Parameter Estimates

| a 5 | 0.1. | |
|------------------|---------|----------|
| Cov Parm | Subject | Estimate |
| UN(1,1) | SUBJID | |
| UN(2,1) | SUBJID | |
| UN(2,2) | SUBJID | |
| UN(3,1) | SUBJID | |
| UN(3,2) | SUBJID | |
| UN(3,3) | SUBJID | |
| UN(4,1) | SUBJID | |
| UN(4,2) | SUBJID | |
| UN(4,3) | SUBJID | |
| UN(4,4) | SUBJID | |
| ( - <b>/</b> - / | SUBJID | |
| UN(5,2) | SUBJID | |
| UN(5,3) | SUBJID | |
| UN(5,4) | SUBJID | |
| UN(5,5) | SUBJID | |
| UN(6,1) | SUBJID | |
| UN(6,2) | SUBJID | |
| UN(6,3) | SUBJID | |
| UN(6,4) | SUBJID | |
| UN(6,5) | SUBJID | |
| UN(6,6) | SUBJID | |

## Fit Statistics

| -2 Res Log Likelihood | 13253.7 |
|--------------------------|---------|
| AIC (Smaller is Better) | 13295.7 |
| AICC (Smaller is Better) | 13295.9 |
| BIC (Smaller is Better) | 13391.9 |

## Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|-----|------------|------------|
| 2.0 | 4294.65 | < .0001 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|-------------------|-----------|-----------|---------|--------|
| TRT01PN(avisitn) | 12 | 814 | 20.33 | <.0001 |
| PREOAD2 (avisitn) | 6 | 674 | 2.75 | 0.0120 |
| BASE(avisitn) | 6 | 676 | 6.16 | <.0001 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 160 of 412 | |

Short Topic Code=C25208X Long label=Body weight (kg)

The Mixed Procedure

## Least Squares Means Estimates

| | • | | | | | |
|---|---|---|---|---|---|---|
| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value |
| TRT01PN(avisitn) TRT01PN(avisitn) TRT01PN(avisitn) | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ANA_DATA<br>WORK.ANA_DATA<br>WORK.ANA_DATA | 1.2938 | 0.2052 | | 1.10<br>6.31<br>-12.13 |
| | Least Squares Mean | s Estimates | | | | |
| Effect | Label | Pr > t A | Alpha | Lower | Upper | |
| TRT01PN(avisitn) TRT01PN(avisitn) TRT01PN(avisitn) | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | <.0001 | 0.05 | -0.1246<br>0.8909<br>-2.9857 | 0.4410<br>1.6967<br>-2.1539 | |
| | Least Squares M | Means Estimates | | | | |
| Effect | Label | Manaina | Fat | | andard<br>Error | DF |
| EIIeCt | Label | Margins | EST | imate | Error | DF |
| TRT01PN(avisitn) TRT01PN(avisitn) | Treatment contrast, IDegLira - Treatment contrast, IDegLira - | | | | 0.2508<br>0.2562 | 674.4<br>690.4 |
| Least Squares Means Estimates | | | | | | |
| Effect | Label | t Value | Pr > t | Alpha | Lower | Upper |
| TRT01PN(avisitn) TRT01PN(avisitn) | Treatment contrast, IDegLira -<br>Treatment contrast, IDegLira - | | <.0001<br><.0001 | 0.05<br>0.05 | -1.6281<br>2.2250 | -0.6431<br>3.2310 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 161 of 412 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

## Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
SWBK.ANA\_DATA
CHG
Unstructured
SUBJID
REML
None
Method
Model-Based
Satterthwaite

### Class Level Information

| Class | Levels | Values |
|--------------------|--------|---------------------------------|
| TRT01PN<br>avisitn | 3 | 1 2 3<br>60 100 140 180 220 280 |
| PREOAD2 | 2 | Metformin Metformin + OAD |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| NN9068-4148 | | Version: | 1.0 | |
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 162 of 412 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

Class Level Information

Class Levels Values
SUBJID 720



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| NN9068-4148 | | Version: | 1.0 | |
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 163 of 412 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure



| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 164 of 412 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure



## Dimensions

| Covariance | Parameters | 21 |
|-------------|------------|-----|
| Columns in | X | 37 |
| Columns in | Z | 0 |
| Subjects | | 720 |
| Max Obs per | Subject | 6 |

## Number of Observations

| Number | of | Observations | Read | 4320 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 4046 |
| Number | of | Observations | Not Used | 274 |

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 CONFIDENTIAL Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - MMRM - full analysis set

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

## Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|----------------------------------|------------|
| 0 | 1 2 | 23907.60340805<br>19612.97222148 | 0.00000372 |
| 2 | 1 | 19612.94923134 | 0.00000000 |

Convergence criteria met.

### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|---|---|---|
| Cov Parm UN(1,1) UN(2,1) UN(2,2) UN(3,1) UN(3,2) UN(3,3) UN(4,1) UN(4,2) UN(4,3) UN(4,4) UN(5,1) UN(5,2) UN(5,4) UN(5,5) UN(6,1) UN(6,2) | Subject SUBJID | Estimate |
| UN (6, 3)<br>UN (6, 4)<br>UN (6, 5)<br>UN (6, 6) | SUBJID<br>SUBJID<br>SUBJID<br>SUBJID | |

## Fit Statistics

| -2 Res Log Likelihood | 19612.9 |
|--------------------------|---------|
| AIC (Smaller is Better) | 19654.9 |
| AICC (Smaller is Better) | 19655.2 |
| BIC (Smaller is Better) | 19751.1 |

## Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 20 | 4294.65 | <.0001 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|-----------|---------|--------|
| TRT01PN(avisitn) | 12 | 814 | 20.33 | <.0001 |
| PREOAD2(avisitn) | 6 | 674 | 2.75 | 0.0120 |
| BASE(avisitn) | 6 | 676 | 6.16 | <.0001 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 166 of 412 | |

Short Topic Code=WEIGHTU Long label=Body weight (lb)

The Mixed Procedure

## Least Squares Means Estimates

| Effect | Label | Margins | Stand<br>Estimate Er | lard<br>ror DF t Value |
|---|---|---|---|---|
| TRT01PN (avisitn) TRT01PN (avisitn) TRT01PN (avisitn) | Change from baseline, IDeg | WORK.ANA_DATA<br>WORK.ANA_DATA<br>WORK.ANA_DATA | 2.8523 0.4 | 175 672.4 1.10<br>524 675.4 6.31<br>670 698.6 -12.13 |
| | Least Squares Mean | s Estimates | | |
| Effect | Label | Pr > t A | Alpha Lower | Upper |
| TRT01PN(avisitn) TRT01PN(avisitn) TRT01PN(avisitn) | | <.0001 | 0.05 -0.2747<br>0.05 1.9641<br>0.05 -6.5822 | 3.7405 |
| | Least Squares M | Means Estimates | | |
| Effect | Label | Margins | Estimate | Standard<br>Error DF |
| TRT01PN(avisitn) TRT01PN(avisitn) | | | | 0.5530 674.4<br>0.5648 690.4 |
| | Least Squares | Means Estimates | 5 | |
| Effect | Label | t Value | Pr > t Alpha | Lower Upper |
| TRT01PN(avisitn) TRT01PN(avisitn) | | | <.0001 0.05<br><.0001 0.05 | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 167 of 412 | |

## 16: Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis conditional multiple imputation - full analysis set

param ana sort=12 Parameter Code=C25208X Label=LSMeans, IDeg Statement Number=1

The MIANALYZE Procedure

Estimate

Model Information

Data Set WORK.LSME ABS MI2 Number of Imputations WORK 1000

Variance Information (1000 Imputations)

-----Variance-----

Parameter Within Total 0.040243 0.042294 424717 Estimate 0.002049

Variance Information (1000 Imputations)

Relative Fraction Increase Missing Relative in Variance Information Efficiency Parameter

0.048503 Estimate 0.050971 0.999951

Parameter Estimates (1000 Imputations)

95% Confidence Std Error Limits DF Estimate Minimum Parameter Maximum

0.205654 75.02980 75.83595 424717

75.291050

75.598927

Parameter Estimates (1000 Imputations)

t for HO:

75.432878

Theta0 Parameter=Theta0 Pr > |t| Parameter 366.79 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Page: Statistical document 168 of 412

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=12 Parameter Code=C25208X Label=LSMeans, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total 0.020855 531569 Estimate 0.000903 0.019951

Variance Information (1000 Imputations)

Relative

Fraction Missing Relative Increase Parameter in Variance Information Efficiency 0.043355 0.999957 Estimate 0.045316

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum 74.335940 0.144413 74.05290 74.61899 531569 74.250861 74.416588 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 514.74 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final  Statistical document

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=12 Parameter Code=C25208X Label=LSMeans, Lira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.045238 73847 Estimate 0.005256 0.039976

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency Estimate 0.131619 0.116334 0.999884

Parameter Estimates (1000 Imputations)

95% Confidence

DF Parameter Estimate Std Error Limits Minimum Maximum 71.554362 0.212692 71.13749 71.97124 73847 71.264993 71.786081 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 336.42 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 170 of 412 Statistical document Page:

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=22 Parameter Code=WEIGHTU Label=LSMeans, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total

0.195593 0.205563 424717 Estimate 0.009960

Variance Information (1000 Imputations)

Fraction Missing Relative

Relative Increase Parameter in Variance Information Efficiency 0.048503 Estimate 0.050971 0.999951

Parameter Estimates (1000 Imputations)

95% Confidence Parameter Estimate Std Error Limits

DF Minimum Maximum 0.453390 165.4124 167.1897 424717 165.988353 166.667105 166.301030 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|0 366.79 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=22 Parameter Code=WEIGHTU Label=LSMeans, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total

0.096969 0.101364 531569 Estimate 0.004390

Variance Information (1000 Imputations)

Fraction Missing Relative

163.882696

Estimate

Relative Increase Parameter in Variance Information Efficiency 0.999957 Estimate 0.045316 0.043355

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum 0.318376 163.2587 164.5067 531569 163.695128 164.060492

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|0 514.74 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Page: Statistical document 172 of 412

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=22 Parameter Code=WEIGHTU Label=LSMeans, Lira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.219873 73847 Estimate 0.025548 0.194299

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency Estimate 0.131619 0.116334 0.999884

Parameter Estimates (1000 Imputations)

95% Confidence Parameter Estimate Std Error Limits

DF Minimum Maximum 0.468906 156.8313 158.6694 73847 157.112416 158.261218 157.750364 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|

0 <.0001 336.42 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Page: Statistical document 173 of 412

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=12 Parameter Code=C25208X Label=Change from baseline, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total

0.040243 0.042294 424717 Estimate 0.002049

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency 0.048503 Estimate 0.050971 0.999951

Parameter Estimates (1000 Imputations)

95% Confidence

DF Parameter Estimate Std Error Limits Minimum Maximum 0.205654 0.899663 1.705816 424717 1.160912 1.302740 1.468788 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|

0 6.33 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 174 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=12 Parameter Code=C25208X Label=Change from baseline, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total

0.019951 0.020855 531569 Estimate 0.000903

Variance Information (1000 Imputations)

Relative Fraction Missing

0.205802

Estimate

Relative Increase Increase Missing in Variance Information Parameter Efficiency 0.045316 0.043355 0.999957 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum 0.144413 -0.07724 0.488847 531569 0.120722

0.286449

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 1.43 0.1541 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 175 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=12 Parameter Code=C25208X Label=Change from baseline, Lira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.039976 0.045238 73847 Estimate 0.005256

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Increase Missing in Variance Information Parameter Efficiency 0.131619 0.999884 Estimate 0.116334

Parameter Estimates (1000 Imputations)

95% Confidence

DF Minimum Std Error Parameter Estimate Limits Maximum -2.575777 0.212692 -2.99265 -2.15890 73847 -2.865146 Estimate -2.344058

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter

0 -12.11 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Page: Statistical document 176 of 412

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=12 Parameter Code=C25208X Label=Treatment contrast, IDegLira - IDeg

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total

0.060258 0.063074 501172 Estimate 0.002813

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency 0.999955 Estimate 0.046733 0.044651

Parameter Estimates (1000 Imputations)

95% Confidence

DF Parameter Estimate Std Error Limits Minimum Maximum -1.096938 0.251145 -1.58917 -0.60470 501172 -1.276007 -0.942857 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 -4.37 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final  Statistical document

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=22 Parameter Code=WEIGHTU Label=Change from baseline, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total

0.195593 0.205563 424717 Estimate 0.009960

Variance Information (1000 Imputations)

Relative Fraction Missing Increase

2.872049

Estimate

Relative Parameter in Variance Information Efficiency 0.048503 Estimate 0.050971 0.999951

Parameter Estimates (1000 Imputations)

0.453390 1.983418 3.760680 424717

2.559372

3.238123

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|0 6.33 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 178 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=22 Parameter Code=WEIGHTU Label=Change from baseline, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.096969 0.101364 531569 Estimate 0.004390

Variance Information (1000 Imputations)

Relative Fraction Missing Relative Increase Increase Missing in Variance Information Parameter Efficiency 0.045316 0.043355 0.999957 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence DF Std Error Parameter Estimate Limits Minimum Maximum 0.453715 0.318376 -0.17029 1.077723 531569 0.266147 0.631511 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 1.43 0.1541 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 179 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=22 Parameter Code=WEIGHTU Label=Change from baseline, Lira Statement Number=1

The MIANALYZE Procedure

Estimate

Model Information

Data Set WORK.LSME\_CHG\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance----Between Within Total DF Parameter

0.116334

0.194299 0.219873 73847 Estimate 0.025548

Variance Information (1000 Imputations)

Relative Fraction Missing Relative Increase Increase Missing in Variance Information Parameter Efficiency 0.131619

Parameter Estimates (1000 Imputations)

0.999884

95% Confidence Limits DF Minimum Std Error Parameter Estimate Maximum -5.678617 0.468906 -6.59767 -4.75956 73847 -6.316565 -5.167763 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -12.11 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final  Statistical document

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=22 Parameter Code=WEIGHTU Label=Treatment contrast, IDegLira - IDeg

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total

0.306562 501172 Estimate 0.013673 0.292875

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency 0.999955 Estimate 0.046733 0.044651

Parameter Estimates (1000 Imputations)

95% Confidence

DF Parameter Estimate Std Error Limits Minimum Maximum 0.553680 -3.50353 -1.33314 501172 -2.813114 -2.078643 -2.418334 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 -4.37 <.0001 Estimate

## NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=13 Parameter Code=C25208X Label=LSMeans, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

Parameter Between Within Total DF

Estimate 0.002050 0.040747 0.042799 434662

Variance Information (1000 Imputations)

Relative Fraction Increase Missing Relative Parameter in Variance Information Efficiency

Estimate 0.050355 0.047945 0.999952

Parameter Estimates (1000 Imputations)

 
 Parameter
 Estimate
 Std Error
 95% Confidence Limits
 DF
 Minimum
 Maximum

 Estimate
 75.434346
 0.206879
 75.02887
 75.83982
 434662
 75.292957
 75.599366

Parameter Estimates (1000 Imputations)

Parameter Theta0 Parameter=Theta0 Pr > |t| Estimate 0 364.63 <.0001

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Page: Statistical document 182 of 412

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=13 Parameter Code=C25208X Label=LSMeans, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total

0.021187 461469 Estimate 0.000985 0.020201

Variance Information (1000 Imputations)

Fraction Missing Relative

Relative Increase Parameter in Variance Information Efficiency Estimate 0.048798 0.046532 0.999953

Parameter Estimates (1000 Imputations)

95% Confidence

DF Parameter Estimate Std Error Limits Minimum Maximum 74.184327 0.145558 73.89904 74.46962 461469 74.065477 74.270842 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 509.66 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Page: Statistical document 183 of 412

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=13 Parameter Code=C25208X Label=LSMeans, Lira Statement Number=1

The MIANALYZE Procedure

Estimate

Model Information

Data Set WORK.LSME\_ABS\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.045745 75344 Estimate 0.005262 0.040478

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency 0.999885 Estimate 0.130133 0.115172

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum 71.554942 0.213881 71.13574 71.97415 75344 71.265539 71.787147

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 334.56 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=23 Parameter Code=WEIGHTU Label=LSMeans, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total

0.208018 434662 Estimate 0.009963 0.198046

Variance Information (1000 Imputations)

Fraction Missing Relative

Relative Increase Parameter in Variance Information Efficiency 0.047945 0.999952 Estimate 0.050355

Parameter Estimates (1000 Imputations)

95% Confidence

DF Minimum Parameter Estimate Std Error Limits Maximum 0.456090 165.4103 167.1982 434662 165.992557 166.668072 166.304265 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|0 364.63 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=23 Parameter Code=WEIGHTU Label=LSMeans, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total

0.102976 461469 Estimate 0.004786 0.098185

Variance Information (1000 Imputations)

Fraction Missing Relative

Relative Increase Parameter in Variance Information Efficiency Estimate 0.048798 0.046532 0.999953

Parameter Estimates (1000 Imputations)

95% Confidence

DF Minimum Parameter Estimate Std Error Limits Maximum 0.320899 162.9195 164.1774 461469 163.286426 163.739178 163.548445 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|0 509.66 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Page: Statistical document 186 of 412

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=23 Parameter Code=WEIGHTU Label=LSMeans, Lira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_ABS\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total 0.222337 75344 Estimate 0.025576 0.196735

Variance Information (1000 Imputations)

Fraction Missing Relative

Relative Increase Parameter in Variance Information Efficiency 0.999885 Estimate 0.130133 0.115172

Parameter Estimates (1000 Imputations)

95% Confidence

DF Minimum Parameter Estimate Std Error Limits Maximum 0.471526 156.8275 158.6758 75344 157.113619 158.263568 157.751645 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t| 0 334.56 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final  Statistical document

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=13 Parameter Code=C25208X Label=Change from baseline, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total

0.040747 0.042799 434662 Estimate 0.002050

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency 0.047945 0.999952 Estimate 0.050355

Parameter Estimates (1000 Imputations)

95% Confidence Estimate Std Error Limits

DF Parameter Minimum Maximum 0.206879 0.898730 1.709683 434662 1.162818 1.304207 1.469227 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|

0 6.30 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 188 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=13 Parameter Code=C25208X Label=Change from baseline, IDegLira Statement Number=1

The MIANALYZE Procedure

Estimate

Model Information

Data Set WORK.LSME\_CHG\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between DF Parameter Within Total

0.020201 0.021187 461469 Estimate 0.000985

Variance Information (1000 Imputations)

Relative Fraction Missing Increase

0.054188

Relative in Variance Information Parameter Efficiency 0.048798 0.046532 0.999953 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence DF Minimum Parameter Estimate Std Error Limits Maximum 0.145558 -0.23110 0.339476 461469 -0.064662

0.140703

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 0.37 0.7097 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 189 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=13 Parameter Code=C25208X Label=Change from baseline, Lira Statement Number=1

The MIANALYZE Procedure

Estimate

Model Information

Data Set WORK.LSME\_CHG\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.040478 0.045745 75344 Estimate 0.005262

Variance Information (1000 Imputations)

Fraction Missing Relative Relative Increase Increase Missing in Variance Information Parameter Efficiency 0.130133 0.115172 0.999885

Parameter Estimates (1000 Imputations)

95% Confidence Limits ce DF Minimum Std Error Parameter Estimate

-2.575196 0.213881 -2.99440 -2.15599 75344 -2.864600 -2.342992 Estimate

Maximum

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -12.04 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Page: Statistical document 190 of 412

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=13 Parameter Code=C25208X Label=Treatment contrast, IDegLira - Lira

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total

0.066917 115773 Estimate 0.006210 0.060701

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency 0.092908 0.999907 Estimate 0.102405

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits

Minimum Maximum 0.258683 2.122370 3.136398 115773 2.405082 2.629384 2.939673 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|0 10.16 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Page: Statistical document 191 of 412

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=23 Parameter Code=WEIGHTU Label=Change from baseline, IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total

0.208018 434662 Estimate 0.009963 0.198046

Variance Information (1000 Imputations)

Relative Fraction Missing

2.875284

Estimate

Relative Increase Parameter in Variance Information Efficiency 0.047945 0.999952 Estimate 0.050355

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum 0.456090 1.981361 3.769207 434662 2.563576 3.239091

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|0 6.30 <.0001 Estimate
| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 192 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=23 Parameter Code=WEIGHTU Label=Change from baseline, IDegLira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3 Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.098185 0.102976 461469 Estimate 0.004786

Variance Information (1000 Imputations)

Relative Fraction Missing Increase

Relative Increase Missing in Variance Information Parameter Efficiency 0.048798 0.046532 0.999953 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Limits

DF Minimum Std Error Parameter Estimate Maximum 0.320899 -0.50949 0.748417 461469 -0.142555 0.310196 Estimate 0.119464

Parameter Estimates (1000 Imputations)

t for HO:

Theta0 Parameter=Theta0 Pr > |t| Parameter 0 0.37 0.7097 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 193 of 412 | |

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=23 Parameter Code=WEIGHTU Label=Change from baseline, Lira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter 0.196735 0.222337 75344 Estimate 0.025576

Variance Information (1000 Imputations)

Relative

Fraction Missing Relative Increase Increase Missing in Variance Information Parameter Efficiency 0.130133 0.115172 0.999885 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Timits DF Minimum Std Error Parameter Estimate Maximum -5.677336 0.471526 -6.60153 -4.75315 75344 -6.315363 -5.165413 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 -12.04 <.0001 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final  Statistical document

Body weight after 26 weeks of treatment - change from baseline - statistical sensitivity analysis - conditional multiple imputation - full analysis set

param\_ana\_sort=23 Parameter Code=WEIGHTU Label=Treatment contrast, IDegLira - Lira

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME\_CHG\_MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----DF Parameter Between Within Total

0.295027 0.325239 115773 Estimate 0.030182

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Parameter in Variance Information Efficiency 0.092908 0.999907 Estimate 0.102405

Parameter Estimates (1000 Imputations)

95% Confidence

DF Parameter Estimate Std Error Limits Minimum Maximum 0.570298 4.679026 6.914575 115773 5.302299 6.480870 5.796800 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|

0 10.16 <.0001 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 195 of 412 | |

# 17: Waist circumference after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=MEANWAIC

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 717

Number of Observations

Number of Observations Read 720 Number of Observations Used 717 Number of Observations Not Used 3

Covariance Parameter Estimates

Cov Parm Estimate
Residual 12.8901

Fit Statistics

-2 Res Log Likelihood 3873.2
AIC (Smaller is Better) 3875.2
AICC (Smaller is Better) 3875.3
BIC (Smaller is Better) 3879.8

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t| Alpha 4.4327 712 712 3.40 0.0007 0.05 1.3030 Intercept trtpn 2.4135 0.3281 7.36 <.0001 0.05 3.8648 0.3795 712 10.18 <.0001 0.05 trtpn trtpn PREOAD2 Metformin 0.6340 0.2863 712 2.21 0.0271 0.05 PREOAD2 Metformin + OAD 0.9234 0.01353 712 68.27 <.0001 0.05 BASE

#### NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Waist circumference after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=MEANWAIC

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.8746<br>1.7693<br>3.1197 | 6.9908<br>3.0578<br>4.6099 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | 0.07184 | 1.1961 |
| BASE | | | 0.8968 | 0.9499 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 712 | 53.53 | <.0001 |
| PREOAD2 | 1 | 712 | 4.90 | 0.0271 |
| BASE | 1 | 712 | 4660.89 | <.0001 |

#### Least Squares Means Estimates

Standard

| Effect | Label | Margins | Estimat | e E | rror | DF | t Value | Pr > | t | Alpha |
|---|---|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 94.603<br>96.054<br>92.190 | 9 0. | 1896<br>2692<br>2677 | 712<br>712<br>712 | 498.98<br>356.83<br>344.41 | <.( | 0001<br>0001<br>0001 | 0.05<br>0.05<br>0.05 |
| | | Least Sq | uares Mea | ns Estim | ates | | | | | |
| Effect | Label | Lower | Upper | Exponen | tiated | Expo | nentiated<br>Lower | Expor | nentiat<br>Upp | |
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | 95.5264 | 94.9758<br>96.5834<br>92.7156 | 5. | 218E41<br>201E41<br>091E40 | | 8.398E40<br>3.066E41<br>6.448E39 | | 1.768E<br>8.823E<br>1.844E | 41 |
| | | Least Sq | uares Mea | ns Estim | ates | | | | | |
| Effect | Label | | Margi | ns | Estimat | | tandard<br>Error | DF | t Val | ue |
| trtpn | Treatment contrast | , IDegLira - ID | eg WORK. | ADATA2 | -1.451 | 3 | 0.3294 | 712 | -4. | 41 |
| | | Least Sq | uares Mea | ns Estim | ates | | | | | |

| Effect | Label | | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - I | Deg | <.0001 | 0.05 | -2.0980 | -0.8046 | 0.2343 |

### Least Squares Means Estimates

| Effect | Label | | | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira | - IDe | g 0.1227 | 0.4473 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019<br>1.0<br>Final<br>197 of 412 |
|---|---|---|---|
|---|---|---|---|

Waist circumference after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=MEANWAIC

The Mixed Procedure

Least Squares Means Estimates

| Effect | Label | | Margins | Estir | | andard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - Lira | WORK.ADATA | 2 2. | 4135 | 0.3281 | 712 | 7.36 |
| | | Least Squar | es Means Es | timates | | | | |
| Effect | Label | | Pr > t | Alpha | Lower | Upper | Expon | entiated |
| trtpn | Treatment contrast, | IDegLira - Lira | <.0001 | 0.05 | 1.7693 | 3.0578 | | 11.1735 |
| | Leas | t Squares Means E | stimates | | | | | |
| | | | Exponentia | ted E: | xponentia | ted | | |

| Effect | Label | | | | Lower | Upper |
|--------|-----------|-----------|----------|--------|--------|---------|
| trtpn | Treatment | contrast, | IDegLira | - Lira | 5.8669 | 21.2799 |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 198 of 412 Statistical document Page:

Waist circumference after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=MEANWAIC

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 717

Number of Observations

Number of Observations Read 720 Number of Observations Used 717 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 12.8901

Fit Statistics

-2 Res Log Likelihood 3873.2 AIC (Smaller is Better) AICC (Smaller is Better) 3875.3 BIC (Smaller is Better) 3879.8

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 4.4327 1.3030 712 3.40 0.0007 0.05 trtpn 1 2.4135 0.3281 712 7.36 <.0001 0.05 10.18 <.0001 trtpn 3.8648 0.3795 712 0.05 3 trtpn PREOAD2 0.6340 0.2863 712 2.21 0.0271 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.07661 0.01353 712 -5.66 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 199 of 412 | |

Waist circumference after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=MEANWAIC

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.8746<br>1.7693<br>3.1197 | 6.9908<br>3.0578<br>4.6099 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | 0.07184 | 1.1961 |
| BASE | | | -0.1032 | -0.05005 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|------------|---------------|------------------|
| trtpn<br>PREOAD2 | 2 | 712<br>712 | 53.53<br>4.90 | <.0001<br>0.0271 |
| BASE | 1 | 712 | 32.08 | <.0001 |

## Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 1.2408 | 0.1896<br>0.2692<br>0.2677 | 712<br>712<br>712 | -1.11<br>4.61<br>-9.80 | 0.2674<br><.0001<br><.0001 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -0.5827<br>0.7123<br>-3.1495 | 0.1618<br>1.7693<br>-2.0985 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 200 of 412 | |

# 18: Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=C105585P

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used 2

Covariance Parameter Estimates

Cov Parm Estimate
Residual 2.7090

Fit Statistics

-2 Res Log Likelihood 2763.3
AIC (Smaller is Better) 2765.3
AICC (Smaller is Better) 2765.3
BIC (Smaller is Better) 2769.9

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t| Alpha 6.7293 -1.8662 0.3170 0.1503 713 713 21.23 -12.42 <.0001 0.05 Intercept trtpn <.0001 0.05 -1.4011 0.1742 713 -8.04 <.0001 0.05 trtpn trtpn PREOAD2 Metformin -0.3263 0.1311 713 -2.49 0.0130 0.05 PREOAD2 Metformin + OAD 0.1393 0.03019 713 4.61 <.0001 0.05 BASE

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=C105585P

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 6.1069<br>-2.1612<br>-1.7431 | 7.3516<br>-1.5712<br>-1.0591 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | 3 | -0.5837 | -0.06898 |
| BASE | 110010111111111111111111111111111111111 | | 0.08005 | 0.1986 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 713 | 77.73 | <.0001 |
| PREOAD2 | 1 | 713 | 6.20 | 0.0130 |
| BASE | 1 | 713 | 21.29 | <.0001 |

#### Least Squares Means Estimates

| 766 | T 1 1 | | | Standard | | 3 | 5 2 111 | 7.1.1 |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
| trtpn | LSMeans, IDegLira | WORK.ADATA2 | 6.1008 | 0.08676 | 713 | 70.32 | <.0001 | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | 6.5659 | 0.1235 | 713 | 53.17 | <.0001 | 0.05 |
| trtpn | LSMeans, Lira | WORK.ADATA2 | 7.9670 | 0.1227 | 713 | 64.92 | <.0001 | 0.05 |
| | | Least Sq | uares Means | s Estimates | | | | |
| Effect | Lahel | Lower | Unner F | Exponentiated | Expo | nentiated | Exponentia | ted |

| Effect | Label | | Lower | Upper | Exponentiated | Lower | Upper |
|--------|----------|---|--------|--------|---------------|---------|---------|
| trtpn | LSMeans, | _ | 5.9305 | 6.2712 | 446.22 | 376.34 | 529.09 |
| trtpn | LSMeans, | | 6.3235 | 6.8084 | 710.47 | 557.51 | 905.40 |
| trtpn | LSMeans, | | 7.7261 | 8.2080 | 2884.34 | 2266.80 | 3670.11 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -0.4651 | 0.1510 | 713 | -3.08 |

### Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 0.0021 | 0.05 | -0.7615 | -0.1687 | 0.6281 |

### Least Squares Means Estimates

| Effect | Label | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment contrast | , IDegLira - IDeg | 0.4670 | 0.8447 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019<br>1.0<br>Final<br>202 of 412 | |
|---|---|---|---|---|
| Fasting plasma glucose after 26 | weeks of treatment - change | from baselin | e - supportive statis | tical |

analysis - full analysis set

Parameter Code=C105585P

The Mixed Procedure

Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF t Value |
|---|---|---|---|---|---|
| trtpn | Treatment contrast, IDegLira - Lira | work.ADATA2 | -1.8662 | 0.1503 | 713 -12.42 |
| | Least Squa | ares Means Est | imates | | |
| Effect | Label | Pr > t 2 | Alpha Low | er Upper | Exponentiated |
| trtpn | Treatment contrast, IDegLira - Lira | <.0001 | 0.05 -2.16 | 12 -1.5712 | 0.1547 |
| | Least Squares Means | Estimates | | | |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - Lira | 0.1152 | 0.2078 |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 203 of 412 Statistical document Page:

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=FPGU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 879.68

Fit Statistics

-2 Res Log Likelihood 6892.3 AIC (Smaller is Better) AICC (Smaller is Better) 6894.3 6894.3 BIC (Smaller is Better) 6898.9

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect treatment2 01 (N) Estimate DF t Value Pr > |t| Alpha Error 21.23 Intercept 121.26 5.7125 713 < .0001 0.05 trtpn 1 -33.6294 2.7077 713 -12.42 <.0001 0.05 trtpn -25.2482 3.1389 713 -8.04 < .0001 0.05 3 trtpn PREOAD2 -5.8804 2.3620 713 -2.49 0.0130 0.05 Metformin PREOAD2 Metformin + OAD BASE 0.1393 0.03019 713 4.61 <.0001 0.05

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=FPGU

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 110.05<br>-38.9455<br>-31.4108 | 132.48<br>-28.3134<br>-19.0856 |
| PREOAD2 | Metformin<br>Metformin + OAD | | -10.5177 | -1.2431 |
| BASE | THE CTOTALLIT . OTHE | | 0.08005 | 0.1986 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 713 | 77.73 | <.0001 |
| PREOAD2 | 1 | 713 | 6.20 | 0.0130 |
| BASE | 1 | 713 | 21.29 | <.0001 |

#### Least Squares Means Estimates

| | | | | Standard | | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2 WORK.ADATA2 WORK.ADATA2 Least Squ | 109.94<br>118.32<br>143.57 | 1.5634<br>2.2253<br>2.2113<br>Estimates | 713<br>713<br>713 | 70.32<br>53.17<br>64.92 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |
| | | - | | | Evno | nontiatod | Evnonontia | +00 |

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | 106.87 | 113.01 | 5.558E47 | 2.582E46 | 1.197E49 |
| trtpn | LSMeans, | | 113.95 | 122.69 | 2.426E51 | 3.072E49 | 1.916E53 |
| trtpn | LSMeans, | | 139.22 | 147.91 | 2.239E62 | 2.914E60 | 1.72E64 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -8.3812 | 2.7204 | 713 | -3.08 |

### Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 0.0021 | 0.05 | -13.7223 | -3.0402 | 0.000229 |

### Least Squares Means Estimates

| Effect | Label | | | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira | - IDeg | 1.098E-6 | 0.04782 |

| NN9068 | | Date: | 16 December 2019 Nov | o Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 205 of 412 | |

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=FPGU

The Mixed Procedure

Least Squares Means Estimates

Effect Label Margins Estimate Standard Error DF t Value trtpn Treatment contrast, IDegLira - Lira WORK.ADATA2 -33.6294 2.7077 713 -12.42

Least Squares Means Estimates

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - Lira < .0001 0.05 -38.9455 -28.3134 2.48E-15

Least Squares Means Estimates

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - Lira 1.22E-17 5.05E-13

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=C105585P

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 2.7090

Fit Statistics

-2 Res Log Likelihood 2763.3 AIC (Smaller is Better) AICC (Smaller is Better) 2765.3 2765.3 BIC (Smaller is Better) 2769.9

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 21.23 Intercept 6.7293 0.3170 713 < .0001 0.05 trtpn 1 -1.8662 0.1503 713 -12.42 < .0001 0.05 trtpn -1.4011 0.1742 713 -8.04 < .0001 0.05 3 trtpn PREOAD2 -0.3263 0.1311 713 -2.49 0.0130 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.8607 0.03019 713 -28.50 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 207 of 412 | |

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=C105585P

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 6.1069<br>-2.1612<br>-1.7431 | 7.3516<br>-1.5712<br>-1.0591 |
| PREOAD2<br>PREOAD2<br>BASE | Metformin<br>Metformin + OAD | Ü | -0.5837<br>-0.9199 | -0.06898<br>-0.8014 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 713 | 77.73 | <.0001 |
| PREOAD2 | 1 | 713 | 6.20 | 0.0130 |
| BASE | 1 | 713 | 812.50 | <.0001 |

## Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | | 0.08676<br>0.1235<br>0.1227 | 713<br>713<br>713 | -40.87<br>-24.95<br>-13.69 | <.0001<br><.0001<br><.0001 |
| | Least Squares Mean: | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 - | -3.7164<br>-3.3235<br>-1.9208 | -3.3758<br>-2.8386<br>-1.4390 | | | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=FPGU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 879.68

Fit Statistics

-2 Res Log Likelihood 6892.3 AIC (Smaller is Better) AICC (Smaller is Better) 6894.3 6894.3 BIC (Smaller is Better) 6898.9

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 21.23 Intercept 121.26 5.7125 713 <.0001 0.05 trtpn 1 -33.6294 2.7077 713 -12.42 <.0001 0.05 <.0001 trtpn -25.2482 3.1389 713 -8.04 0.05 3 trtpn PREOAD2 -5.8804 2.3620 713 -2.49 0.0130 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.8607 0.03019 713 -28.50 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 209 of 412 | |

Fasting plasma glucose after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=FPGU

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 110.05<br>-38.9455<br>-31.4108 | 132.48<br>-28.3134<br>-19.0856 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -10.5177 | -1.2431 |
| BASE | IICCIOIMIII I OIID | | -0.9199 | -0.8014 |

Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|---------|
| trtpn | 2 | 713 | 77.73 | <.0001 |
| PREOAD2 | 1 | 713 | 6.20 | 0.0130 |
| BASE | 1 | 71.3 | 812.50 | < .0001 |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -55.5197 | 1.5634<br>2.2253<br>2.2113 | 713<br>713<br>713 | -40.87<br>-24.95<br>-13.69 | <.0001<br><.0001<br><.0001 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 -5 | 56.9703<br>59.8887<br>34.6130 | -60.8317<br>-51.1508<br>-25.9300 | | | |

# 19: 9-point self-measured plasma glucose profile after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C105585Y

The Mixed Procedure

Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
WORK.ANA\_DATA
AVAL
Compound Symmetry
USUBJID
REML
Profile
Kenward-Roger
Kenward-Roger

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 210 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

Class Level Information

Class Levels Values USUBJID 720 NN9068-4148/

NN9068-4148/

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 211 of 412 | |

Parameter Code=C105585Y

```
NN9068-4148/
NN9068-4146/

NN9068-4148/

NN9068-4148/

NN9068-4148/

NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 212 of 412 | |

Parameter Code=C105585Y

```
NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 213 of 412 | |

Parameter Code=C105585Y

```
NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 214 of 412 | |

Parameter Code=C105585Y

```
NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 215 of 412 | |

Parameter Code=C105585Y

```
NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 216 of 412 | |

Parameter Code=C105585Y

```
NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 217 of 412 | |

Parameter Code=C105585Y

```
NN9068-4148/

NN9068-4148/
  NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 218 of 412 | |

Parameter Code=C105585Y

```
NN9068-4148/

NN9068-4148/
  NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 219 of 412 | |

Parameter Code=C105585Y

```
NN9068-4148/

NN9068-4148/
  NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 220 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

```
NN9068-4148/

NN9068-4148/

NN9068-4148/

NN9068-4148/

NN9068-4148/

NN9068-4148/

NN9068-4148/

NN9068-4148/
     NN9068-4148/
    1 2 3
1 2 3 4 5 6 7 8 9
    Metformin Metformin + OAD
```

#### Dimensions

3

TRTPN ATPTN

PREOAD2

| Covariance | Parameters | 2 |
|------------|------------|-----|
| Columns in | | 49 |
| Columns in | Z | 0 |
| Subjects | | 720 |
| Max Obs pe | r Subject | 9 |


9-point self-measured plasma glucose profile after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C105585Y

The Mixed Procedure

Number of Observations

Number of Observations Read 6480 Number of Observations Used 6401 Number of Observations Not Used 79

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 28226.72908143
1 2 26184.01976519 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Standard Value Subject Estimate Alpha Cov Parm Error Pr Z Lower Upper <.0001 0.05 1.7835 2.2688 USUBJID 2.0262 0.1238 16.37 Residual 2.7716 0.05215 53.15 <.0001 0.05 2.6721 2.8767

Asymptotic Covariance Matrix of Estimates

Row Cov Parm CovP1 CovP2

1 CS 0.01533 -0.00031
2 Residual -0.00031 0.002720

Fit Statistics

-2 Res Log Likelihood 26184.0 AIC (Smaller is Better) 26188.0 BIC (Smaller is Better) 26187.2

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1 2042.71 <.0001

Solution for Fixed Effects

Planned Treatment Pre Trial anti-Diabetic for Analysis Period Standard Timepoint 01 (N) (N) Effect Estimate DF t Value Pr > |t| treatment2 Error Intercept 7.1788 0.1737 2673 41.34 <.0001 0.2005 TRTPN 1 -1.6069 2664 -8.02 <.0001 TRTPN -1.4114 0.2316 2655 -6.09 <.0001 2 3 1 TRTPN 0 0.05534 TRTPN (ATPTN) 0.1385 5650 0.40 0.6895 1 TRTPN (ATPTN) 2 1 0.1714 0.1858 5649 0.3565 0.92 TRTPN (ATPTN) 3 0.03570 0.1866 0.19 0.8483 5650 TRTPN (ATPTN) 2 3.7916 0.1387 5650 <.0001 TRTPN (ATPTN) 4.4526 0.1868 5654 23.83 <.0001

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 222 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | | 3 | 2 | 3.4643 | 0.1873 | 5652 | 18.50 | <.0001 |
| TRTPN (ATPTN) | | 1 | 3 | 1.1290 | 0.1391 | 5652 | 8.12 | <.0001 |
| TRTPN (ATPTN) | | 2 | 3 | 1.6932 | 0.1867 | 5654 | 9.07 | <.0001 |
| TRTPN (ATPTN) | | 3 | 3 | 0.9288 | 0.1866 | 5651 | 4.98 | <.0001 |
| TRTPN (ATPTN) | | 1 | 4 | 3.6173 | 0.1390 | 5651 | 26.03 | <.0001 |
| TRTPN (ATPTN) | | 2 | 4 | 4.7494 | 0.1869 | 5655 | 25.41 | <.0001 |
| TRTPN (ATPTN) | | 2 3 | 4 | 2.8978 | 0.1868 | 5651 | 15.51 | <.0001 |
| TRTPN (ATPTN) | | | 5 | 1.2618 | 0.1387 | 5652 | 9.10 | <.0001 |
| TRTPN (ATPTN) | | 1<br>2<br>3 | 5 | 1.9783 | 0.1860 | 5652 | 10.63 | <.0001 |
| TRTPN (ATPTN) | | 3 | 5 | 0.9111 | 0.1866 | 5651 | 4.88 | <.0001 |
| TRTPN (ATPTN) | | 1 2 | 6 | 4.0292 | 0.1390 | 5653 | 28.99 | <.0001 |
| TRTPN (ATPTN) | | 2 | 6 | 4.8940 | 0.1861 | 5652 | 26.30 | <.0001 |
| TRTPN (ATPTN) | | 3 | 6 | 2.9201 | 0.1867 | 5651 | 15.64 | <.0001 |
| TRTPN (ATPTN) | | | 7 | 2.7960 | 0.1392 | 5654 | 20.08 | <.0001 |
| TRTPN (ATPTN) | | 1<br>2 | 7 | 3.4588 | 0.1873 | 5655 | 18.47 | <.0001 |
| TRTPN (ATPTN) | | 3 | 7 | 1.8831 | 0.1871 | 5652 | 10.07 | <.0001 |
| TRTPN (ATPTN) | | | 8 | 0.2813 | 0.1397 | 5654 | 2.01 | 0.0440 |
| TRTPN (ATPTN) | | 1 2 | 8 | 0.6376 | 0.1880 | 5657 | 3.39 | 0.0007 |
| TRTPN (ATPTN) | | 3 | 8 | 0.1064 | 0.1877 | 5653 | 0.57 | 0.5710 |
| TRTPN (ATPTN) | | 1 | 9 | 0 | | | | |
| TRTPN (ATPTN) | | 2 | 9 | 0 | | | | |
| TRTPN (ATPTN) | | 3 | 9 | 0 | | | | |
| PREOAD2 (ATPTN) | Metformin | | 1 | -0.1375 | 0.1743 | 2641 | -0.79 | 0.4302 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 1 | 0 | | | | |
| PREOAD2 (ATPTN) | Metformin | | 2 | -0.7606 | 0.1750 | 2671 | -4.35 | < .0001 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 2 | 0 | | | | |
| PREOAD2 (ATPTN) | Metformin | | 3 | -0.5825 | 0.1749 | 2665 | -3.33 | 0.0009 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 3 | 0 | | | | |
| PREOAD2 (ATPTN) | Metformin | | 4 | -0.4914 | 0.1752 | 2678 | -2.80 | 0.0051 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 4 | 0 | | | | |
| PREOAD2 (ATPTN) | Metformin | | 5 | -0.6473 | 0.1749 | 2664 | -3.70 | 0.0002 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 5 | 0 | | | | |
| PREOAD2 (ATPTN) | Metformin | | 6 | -0.7595 | 0.1751 | 2675 | -4.34 | <.0001 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 6 | 0 | | | | |
| PREOAD2 (ATPTN) | Metformin | | 7 | -0.7914 | 0.1758 | 2705 | -4.50 | <.0001 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 7 | 0 | 0 4555 | 0.000 | 0.00 | 0 0 1 0 5 |
| PREOAD2 (ATPTN) | Metformin | | 8 | -0.3572 | 0.1766 | 2738 | -2.02 | 0.0432 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 8 | 0 | 0 45 | 0646 | | 0 0 4 4 5 |
| PREOAD2 (ATPTN) | Metformin | | 9 | -0.2029 | 0.1744 | 2648 | -1.16 | 0.2449 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 9 | 0 | | | | |

Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|-----------------|-----------|-----------|---------|--------|
| TRTPN | 2 | 716 | 39.78 | <.0001 |
| TRTPN (ATPTN) | 16 | 5652 | 8.63 | <.0001 |
| PREOAD2 (ATPTN) | 9 | 5392 | 5.07 | <.0001 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 223 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | WORK.ANA DATA | 5.5825 | 0.1153 | 2641 | 48.42 | <.0001 |
| TRTPN (ATPTN) | 2 | 1 | WORK.ANA DATA | 5.8941 | 0.1637 | 2641 | 36.00 | <.0001 |
| TRTPN (ATPTN) | 3 | 1 | WORK.ANA DATA | 7.1698 | 0.1633 | 2641 | 43.92 | <.0001 |
| TRTPN (ATPTN) | 1 | 2 | WORK.ANA DATA | 9.1163 | 0.1155 | 2655 | 78.92 | <.0001 |
| TRTPN (ATPTN) | 2 | 2 | WORK.ANA DATA | 9.9728 | 0.1650 | 2697 | 60.45 | < .0001 |
| TRTPN (ATPTN) | 3 | 2 | WORK.ANA DATA | 10.3959 | 0.1638 | 2669 | 63.45 | < .0001 |
| TRTPN (ATPTN) | 1 | 3 | WORK.ANA DATA | 6.5115 | 0.1158 | 2676 | 56.22 | < .0001 |
| TRTPN (ATPTN) | 2 | 3 | WORK.ANA DATA | 7.2713 | 0.1647 | 2683 | 44.15 | < .0001 |
| TRTPN (ATPTN) | 3 | 3 | WORK.ANA_DATA | 7.9183 | 0.1633 | 2641 | 48.50 | <.0001 |
| TRTPN (ATPTN) | 1 | 4 | WORK.ANA_DATA | 9.0295 | 0.1157 | 2669 | 78.03 | <.0001 |
| TRTPN (ATPTN) | 2 | 4 | WORK.ANA DATA | 10.3571 | 0.1650 | 2697 | 62.77 | <.0001 |
| TRTPN (ATPTN) | 3 | 4 | WORK.ANA DATA | 9.9170 | 0.1636 | 2655 | 60.63 | < .0001 |
| TRTPN (ATPTN) | 1 | 5 | WORK.ANA_DATA | 6.6233 | 0.1156 | 2662 | 57.29 | <.0001 |
| TRTPN (ATPTN) | 2 | 5 | WORK.ANA_DATA | 7.5353 | 0.1641 | 2654 | 45.93 | <.0001 |
| TRTPN (ATPTN) | 3 | 5 | WORK.ANA_DATA | 7.8796 | 0.1633 | 2641 | 48.26 | <.0001 |
| TRTPN (ATPTN) | 1 | 6 | WORK.ANA_DATA | 9.3542 | 0.1159 | 2683 | 80.69 | <.0001 |
| TRTPN (ATPTN) | 2 | 6 | WORK.ANA_DATA | 10.4145 | 0.1641 | 2654 | 63.48 | <.0001 |
| TRTPN (ATPTN) | 3 | 6 | WORK.ANA_DATA | 9.8521 | 0.1633 | 2641 | 60.35 | <.0001 |
| TRTPN (ATPTN) | 1 | 7 | WORK.ANA_DATA | 8.1106 | 0.1163 | 2704 | 69.77 | <.0001 |
| TRTPN (ATPTN) | 2 | 7 | WORK.ANA_DATA | 8.9690 | 0.1653 | 2712 | 54.26 | <.0001 |
| TRTPN (ATPTN) | 3 | 7 | WORK.ANA_DATA | 8.8047 | 0.1636 | 2655 | 53.83 | <.0001 |
| TRTPN (ATPTN) | 1 | 8 | WORK.ANA_DATA | 5.7371 | 0.1167 | 2733 | 49.17 | <.0001 |
| TRTPN (ATPTN) | 2 | 8 | WORK.ANA_DATA | 6.2889 | 0.1659 | 2741 | 37.90 | <.0001 |
| TRTPN (ATPTN) | 3 | 8 | WORK.ANA_DATA | 7.1691 | 0.1644 | 2697 | 43.60 | <.0001 |
| TRTPN (ATPTN) | 1 | 9 | WORK.ANA_DATA | 5.5059 | 0.1155 | 2655 | 47.67 | <.0001 |
| TRTPN (ATPTN) | 2 | 9 | WORK.ANA_DATA | 5.7015 | 0.1637 | 2641 | 34.82 | <.0001 |
| TRTPN (ATPTN) | 3 | 9 | WORK.ANA_DATA | 7.1129 | 0.1638 | 2669 | 43.41 | <.0001 |

Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Alpha | Lower | Upper |
|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | 0.05 | 5.3565 | 5.8086 |
| TRTPN (ATPTN) | 2 | 1 | 0.05 | 5.5730 | 6.2151 |
| TRTPN (ATPTN) | 3 | 1<br>2<br>2<br>2<br>3<br>3<br>3<br>4 | 0.05 | 6.8497 | 7.4900 |
| TRTPN (ATPTN) | 1 | 2 | 0.05 | 8.8898 | 9.3428 |
| TRTPN (ATPTN) | 2 | 2 | 0.05 | 9.6493 | 10.2963 |
| TRTPN (ATPTN) | 3 | 2 | 0.05 | 10.0746 | 10.7172 |
| TRTPN (ATPTN) | 1 | 3 | 0.05 | 6.2844 | 6.7387 |
| TRTPN (ATPTN) | 2 | 3 | 0.05 | 6.9483 | 7.5942 |
| TRTPN (ATPTN) | 3 | 3 | 0.05 | 7.5982 | 8.2384 |
| TRTPN (ATPTN) | 1 | | 0.05 | 8.8026 | 9.2564 |
| TRTPN (ATPTN) | 2 | 4 | 0.05 | 10.0335 | 10.6806 |
| TRTPN (ATPTN) | 3 | 4 | 0.05 | 9.5962 | 10.2377 |
| TRTPN (ATPTN) | 1 | 5 | 0.05 | 6.3966 | 6.8500 |
| TRTPN (ATPTN) | 2 | 5<br>5<br>6 | 0.05 | 7.2136 | 7.8571 |
| TRTPN (ATPTN) | 3 | 5 | 0.05 | 7.5594 | 8.1997 |
| TRTPN (ATPTN) | 1 | | 0.05 | 9.1269 | 9.5815 |
| TRTPN (ATPTN) | 2 | 6 | 0.05 | 10.0928 | 10.7362 |
| TRTPN (ATPTN) | 3 | 6 | 0.05 | 9.5320 | 10.1722 |
| TRTPN (ATPTN) | 1 | 7 | 0.05 | 7.8827 | 8.3386 |
| TRTPN (ATPTN) | 2 | 7 | 0.05 | 8.6449 | 9.2931 |
| TRTPN (ATPTN) | 3 | 7 | 0.05 | 8.4840 | 9.1254 |
| TRTPN (ATPTN) | 1 | 8 | 0.05 | 5.5083 | 5.9660 |
| TRTPN (ATPTN) | 2 | 8 | 0.05 | 5.9636 | 6.6142 |

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

9-point self-measured plasma glucose profile after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C105585Y

The Mixed Procedure

#### Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Alpha | Lower | Upper |
|---|---|---|---|---|---|
| TRTPN (ATPTN) | 3 | 8 | 0.05 | 6.8466 | 7.4915 |
| TRTPN (ATPTN) | 1 | 9 | 0.05 | 5.2795 | 5.7324 |
| TRTPN (ATPTN) | 2 | 9 | 0.05 | 5.3804 | 6.0225 |
| TRTPN (ATPTN) | 3 | 9 | 0.05 | 6.7916 | 7.4342 |

#### Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | 2 | 1 | WORK.ANA DATA | -0.3115 | 0.2002 | 2641 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 1 | WORK.ANA DATA | -1.5873 | 0.1999 | 2641 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 2 | WORK.ANA DATA | -3.5338 | 0.1241 | 5652 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 2 | WORK.ANA DATA | -4.3903 | 0.2013 | 2679 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 2 | WORK.ANA DATA | -4.8133 | 0.2003 | 2660 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 3 | WORK.ANA DATA | -0.9290 | 0.1244 | 5653 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 3 | WORK.ANA DATA | -1.6887 | 0.2010 | 2669 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 3 | WORK.ANA_DATA | -2.3358 | 0.1999 | 2641 |

## Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | 2 | 1 | -1.56 | 0.1199 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 1 | -7.94 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 2 | -28.47 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 2 | -21.81 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 2 | -24.03 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 3 | -7.47 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 3 | -8.40 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 3 | -11.69 | <.0001 | 0.05 |

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1<br>1<br>1<br>1<br>1<br>1 | 1<br>1<br>1<br>1<br>1<br>1 | 2<br>3<br>1<br>2<br>3<br>1<br>2 | 1<br>1<br>2<br>2<br>2<br>2<br>3<br>3 | -0.7042<br>-1.9792<br>-3.7771<br>-4.7850<br>-5.2062<br>-1.1729<br>-2.0829 | 0.08110<br>-1.1954<br>-3.2904<br>-3.9956<br>-4.4205<br>-0.6851<br>-1.2945 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 3 | -2.7277 | -1.9439 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 225 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

| | | DILL | CICHCCD OI | beabe bquar | CD IICUIID | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
| TRTPN (ATPTN) | 1 | 1 | 1 | 4 | WORK.ANA DATA | -3.4470 | 0.1243 | 5653 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 4 | WORK.ANA DATA | -4.7745 | 0.2013 | 2679 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 4 | WORK.ANA DATA | -4.3344 | 0.2013 | 2650 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 5 | WORK.ANA DATA | -1.0408 | 0.1242 | 5652 |
| TRTPN (ATPTN) | ī | 1 | 2 | 5 | WORK.ANA DATA | -1.9528 | 0.2005 | 2650 |
| TRTPN (ATPTN) | 1 | ī | 3 | 5 | WORK.ANA DATA | -2.2970 | 0.1999 | 2641 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 6 | WORK.ANA DATA | -3.7717 | 0.1245 | 5653 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 6 | WORK.ANA DATA | -4.8320 | 0.2005 | 2650 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 6 | WORK.ANA DATA | -4.2696 | 0.1999 | 2641 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 7 | WORK.ANA DATA | -2.5281 | 0.1248 | 5654 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 7 | WORK.ANA DATA | -3.3864 | 0.2015 | 2688 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 7 | WORK.ANA DATA | -3.2222 | 0.2001 | 2650 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 8 | WORK.ANA DATA | -0.1546 | 0.1252 | 5656 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 8 | WORK.ANA DATA | -0.7064 | 0.2020 | 2708 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 8 | WORK.ANA_DATA | -1.5866 | 0.2008 | 2679 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 9 | WORK.ANA_DATA | 0.07658 | 0.1241 | 5650 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 9 | WORK.ANA_DATA | -0.1189 | 0.2002 | 2641 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 9 | WORK.ANA_DATA | -1.5304 | 0.2003 | 2660 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 1 | WORK.ANA_DATA | -1.2758 | 0.2312 | 2641 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 2 | WORK.ANA_DATA | -3.2222 | 0.2004 | 2645 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 2 | WORK.ANA_DATA | -4.0788 | 0.1772 | 5656 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 2 | WORK.ANA_DATA | -4.5018 | 0.2316 | 2655 |
| TRTPN (ATPTN) | 2 | 1 | 1 2 | 3 | WORK.ANA_DATA | -0.6175 | 0.2006<br>0.1769 | 2652<br>5656 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 1 | 3 | 3 | WORK.ANA_DATA<br>WORK.ANA DATA | -1.3772<br>-2.0242 | 0.1769 | 2641 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 4 | WORK.ANA DATA | -3.1354 | 0.2005 | 2650 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 4 | WORK.ANA DATA | -4.4630 | 0.1772 | 5656 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 4 | WORK.ANA DATA | -4.0229 | 0.2314 | 2648 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 5 | WORK.ANA DATA | -0.7292 | 0.2004 | 2648 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 5 | WORK.ANA DATA | -1.6413 | 0.1763 | 5653 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 5 | WORK.ANA DATA | -1.9855 | 0.2312 | 2641 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 6 | WORK.ANA DATA | -3.4602 | 0.2006 | 2655 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 6 | WORK.ANA DATA | -4.5205 | 0.1763 | 5653 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 6 | WORK.ANA DATA | -3.9580 | 0.2312 | 2641 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 7 | WORK.ANA DATA | -2.2166 | 0.2008 | 2662 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 7 | WORK.ANA_DATA | -3.0749 | 0.1774 | 5656 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 7 | WORK.ANA_DATA | -2.9106 | 0.2314 | 2648 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 8 | WORK.ANA_DATA | 0.1569 | 0.2011 | 2672 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 8 | WORK.ANA_DATA | -0.3948 | 0.1780 | 5658 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 8<br>9 | WORK.ANA_DATA | -1.2750 | 0.2320 | 2669 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 9 | WORK.ANA_DATA | 0.3881 | 0.2004<br>0.1760 | 2646<br>5649 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 1 | 3 | 9 | WORK.ANA_DATA<br>WORK.ANA DATA | -1.2188 | 0.2316 | 2655 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 2 | WORK.ANA DATA | -1.9465 | 0.2000 | 2646 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 2 | WORK.ANA DATA | -2.8030 | 0.2321 | 2669 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 2 | WORK.ANA DATA | -3.2260 | 0.1760 | 5650 |
| TRTPN (ATPTN) | 3 | ī | 1 | 3 | WORK.ANA DATA | 0.6583 | 0.2002 | 2653 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 3 | WORK.ANA DATA | -0.1014 | 0.2319 | 2662 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 3 | WORK.ANA DATA | -0.7485 | 0.1755 | 5649 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 4 | WORK.ANA DATA | -1.8597 | 0.2001 | 2650 |
| TRTPN (ATPTN) | 3 | ī | 2 | 4 | WORK.ANA DATA | -3.1872 | 0.2321 | 2669 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 4 | WORK.ANA_DATA | -2.7471 | 0.1758 | 5650 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 5 | WORK.ANA DATA | 0.5465 | 0.2001 | 2648 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 5 | WORK.ANA_DATA | -0.3655 | 0.2315 | 2648 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 5 | WORK.ANA_DATA | -0.7097 | 0.1755 | 5649 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 6 | WORK.ANA_DATA | -2.1844 | 0.2002 | 2655 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 6 | WORK.ANA_DATA | -3.2447 | 0.2315 | 2648 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 6 | WORK.ANA_DATA | -2.6823 | 0.1755 | 5649 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 7 | WORK.ANA_DATA | -0.9408 | 0.2004 | 2662 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 226 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

| | | DILIEIGN | es or heast | . squares me | alis | | |
|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
| TRTPN (ATPTN) | 1 | 1 | 1 | 4 | -27.73 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 4 | -23.72 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 4 | -21.66 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 5 | -8.38 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 5 | -9.74 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 5 | -11.49 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 6 | -30.29 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 6 | -24.10 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 6 | -21.36 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 7 | -20.25 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 7 | -16.80 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 7 | -16.10 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 1 2 | 8 | -1.23 | 0.2170 | 0.05 |
| TRTPN (ATPTN) | 1 | 1<br>1 | 3 | 8 | -3.50 | 0.0005 | 0.05<br>0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 1 | 1 | 9 | -7.90<br>0.62 | <.0001<br>0.5372 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 9 | -0.59 | 0.5526 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 9 | -7.64 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 1 | -5.52 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 2 | -16.08 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 2 | -23.02 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 2 | -19.44 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 3 | -3.08 | 0.0021 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 3 | -7.79 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 3 | -8.75 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 4 | -15.64 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 4 | -25.19 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 4 | -17.38 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 5 | -3.64 | 0.0003 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 5 | -9.31 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1<br>1 | 3 | 5<br>6 | -8.59 | <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 1 | 2 | 6 | -17.25<br>-25.64 | <.0001<br><.0001 | 0.05<br>0.05 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 6 | -17.12 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 7 | -11.04 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 7 | -17.33 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 7 | -12.58 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 8 | 0.78 | 0.4351 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 2 3 | 8 | -2.22 | 0.0266 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 8 | -5.49 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 9 | 1.94 | 0.0528 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 9 | 1.09 | 0.2738 | 0.05 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 9 | -5.26 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 2 | -9.73 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 2 | -12.08 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 2 | -18.33 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 1<br>1 | 1 | 3 | 3.29 | 0.0010 | 0.05<br>0.05 |
| TRTPN (ATPTN)<br>TRTPN (ATPTN) | 3 | 1 | 2 3 | 3 | -0.44<br>-4.27 | 0.6619<br><.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 4 | -9.29 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 4 | -13.73 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 4 | -15.63 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 5 | 2.73 | 0.0063 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 5 | -1.58 | 0.1144 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 5 | -4.04 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 6 | -10.91 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 6 | -14.02 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 6 | -15.28 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 7 | -4.69 | <.0001 | 0.05 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 227 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | 1 | 4 | -3.6907 | -3.2032 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 4 | -5.1692 | -4.3798 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 4 | -4.7268 | -3.9421 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 5 | -1.2843 | -0.7972 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 5 | -2.3460 | -1.5596 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 5 | -2.6889 | -1.9051 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 6 | -4.0158 | -3.5276 |
| TRTPN (ATPTN) | 1 | 1<br>1 | 2 3 | 6<br>6 | -5.2252 | -4.4388<br>-3.8777 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 1 | 1 | 7 | -4.6615<br>-2.7728 | -2.2834 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 7 | -3.7816 | -2.9913 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 7 | -3.6145 | -2.8298 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 8 | -0.4001 | 0.09088 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 8 | -1.1025 | -0.3102 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 8 | -1.9804 | -1.1928 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 9 | -0.1667 | 0.3199 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 9 | -0.5116 | 0.2737 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 9 | -1.9232 | -1.1375 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 1 | -1.7291 | -0.8224 |
| TRTPN (ATPTN) | 2 2 | 1 | 1 | 2 | -3.6151 | -2.8293 |
| TRTPN (ATPTN) | 2 | 1<br>1 | 2 3 | 2 2 | -4.4261<br>-4.9560 | -3.7315<br>-4.0476 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 1 | 1 | 3 | -1.0107 | -0.2242 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 3 | -1.7239 | -1.0304 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 3 | -2.4776 | -1.5708 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 4 | -3.5286 | -2.7423 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 4 | -4.8103 | -4.1157 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 4 | -4.4767 | -3.5691 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 5 | -1.1223 | -0.3362 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 5 | -1.9869 | -1.2957 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 5 | -2.4389 | -1.5321 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 6 | -3.8535 | -3.0668 |
| TRTPN (ATPTN) | 2 | 1 | 2 3 | 6 | -4.8661 | -4.1748 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 1<br>1 | 1 | 6<br>7 | -4.4114<br>-2.6103 | -3.5047<br>-1.8228 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 7 | -3.4227 | -2.7271 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 7 | -3.3644 | -2.4568 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 8 | -0.2373 | 0.5512 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 8 | -0.7438 | -0.04583 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 8 | -1.7300 | -0.8200 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 9 | -0.00476 | 0.7810 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 9 | -0.1524 | 0.5376 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 9 | -1.6730 | -0.7646 |
| TRTPN (ATPTN) | 3 | 1<br>1 | 1 2 | 2 | -2.3386 | -1.5543 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 2 | -3.2581<br>-3.5711 | -2.3479<br>-2.8810 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 1 | 1 | 3 | 0.2658 | 1.0508 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 3 | -0.5562 | 0.3533 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 3 | -1.0925 | -0.4044 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 4 | -2.2521 | -1.4673 |
| TRTPN (ATPTN) | 3 | ī | 2 | 4 | -3.6424 | -2.7321 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 4 | -3.0917 | -2.4026 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 5 | 0.1542 | 0.9388 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 5<br>5 | -0.8194 | 0.08834 |
| TRTPN (ATPTN) | 3 | 1 | 3 | | -1.0538 | -0.3657 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 6 | -2.5770 | -1.7918 |
| TRTPN (ATPTN) | 3 | 1 | 2 3 | 6 | -3.6986 | -2.7908 |
| TRTPN (ATPTN) | 3 | 1 | 3<br>1 | 6<br>7 | -3.0263<br>-1.3338 | -2.3383<br>-0.5478 |
| TRTPN (ATPTN) | J | ± | ± | 1 | -I.JJJ0 | -0.34/0 |
| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 228 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

| | | DILL | CICHCCD OI | nearc bquar | CD HCGHD | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
| TRTPN (ATPTN) | 3 | 1 | 2 | 7 | WORK.ANA DATA | -1.7991 | 0.2323 | 2676 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 7 | WORK.ANA DATA | -1.6349 | 0.1758 | 5650 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 8 | WORK.ANA DATA | 1.4327 | 0.2007 | 2672 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 8 | WORK.ANA DATA | 0.8809 | 0.2328 | 2691 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 8 | WORK.ANA DATA | 0.000731 | 0.1766 | 5651 |
| TRTPN (ATPTN) | 3 | ī | 1 | 9 | WORK.ANA DATA | 1.6639 | 0.2000 | 2646 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 9 | WORK.ANA DATA | 1.4684 | 0.2312 | 2641 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 9 | WORK, ANA DATA | 0.05695 | 0.1760 | 5650 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 2 | WORK.ANA DATA | -0.8566 | 0.2014 | 2683 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 2 | WORK.ANA DATA | -1.2796 | 0.2005 | 2664 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 3 | WORK.ANA DATA | 2.6048 | 0.1246 | 5650 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 3 | WORK.ANA DATA | 1.8450 | 0.2012 | 2673 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 3 | WORK.ANA DATA | 1.1980 | 0.2000 | 2646 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 4 | WORK.ANA DATA | 0.08679 | 0.1245 | 5650 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 4 | WORK.ANA_DATA | -1.2408 | 0.2014 | 2683 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 4 | WORK.ANA_DATA | -0.8007 | 0.2002 | 2655 |
| TRTPN (ATPTN) | 1 | 2 2 | 1 | 5 | WORK.ANA_DATA | 2.4930 | 0.1244 | 5651 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 5 | WORK.ANA_DATA | 1.5809 | 0.2007 | 2654 |
| TRTPN (ATPTN) | 1 | 2 2 | 3 | 5 | WORK.ANA_DATA | 1.2367 | 0.2000 | 2646 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 6 | WORK.ANA_DATA | -0.2379 | 0.1247 | 5652 |
| TRTPN (ATPTN) | 1 | 2 2 | 2 | 6 | WORK.ANA_DATA | -1.2982 | 0.2007 | 2654 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 6<br>7 | WORK.ANA_DATA | -0.7358 | 0.2000 | 2646 |
| TRTPN (ATPTN) | 1 | 2 2 | 1 2 | 7 | WORK.ANA_DATA | 1.0056<br>0.1473 | 0.1250<br>0.2017 | 5653<br>2693 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 2 | 3 | 7 | WORK.ANA_DATA<br>WORK.ANA DATA | 0.1473 | 0.2017 | 2655 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 8 | WORK.ANA DATA | 3.3791 | 0.1254 | 5653 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 8 | WORK.ANA DATA | 2.8274 | 0.2022 | 2712 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 8 | WORK.ANA DATA | 1.9472 | 0.2010 | 2683 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 9 | WORK.ANA DATA | 3.6103 | 0.1243 | 5651 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 9 | WORK.ANA DATA | 3.4148 | 0.2004 | 2645 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 9 | WORK.ANA DATA | 2.0034 | 0.2005 | 2664 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 2 | WORK.ANA DATA | -0.4230 | 0.2325 | 2683 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 3 | WORK.ANA DATA | 3.4613 | 0.2016 | 2690 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 3 | WORK.ANA_DATA | 2.7016 | 0.1778 | 5652 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 3 | WORK.ANA DATA | 2.0546 | 0.2321 | 2669 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 4 | WORK.ANA_DATA | 0.9433 | 0.2015 | 2688 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 4 | WORK.ANA_DATA | -0.3842 | 0.1781 | 5652 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 4 | WORK.ANA_DATA | 0.05589 | 0.2323 | 2676 |
| TRTPN (ATPTN) | 2 | 2 2 | 1 | 5 | WORK.ANA_DATA | 3.3495 | 0.2015 | 2685 |
| TRTPN (ATPTN) | 2 | | 2 | 5 | WORK.ANA_DATA | 2.4375 | 0.1773 | 5651<br>2669 |
| TRTPN (ATPTN) | 2 | 2 2 | 1 | 5<br>6 | WORK.ANA_DATA<br>WORK.ANA DATA | 2.0933<br>0.6186 | 0.2321 | 2692 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 2 | 2 | 6 | WORK.ANA DATA | -0.4417 | 0.1773 | 5651 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 6 | WORK.ANA DATA | 0.1207 | 0.2321 | 2669 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 7 | WORK.ANA DATA | 1.8622 | 0.2018 | 2699 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 7 | WORK.ANA DATA | 1.0039 | 0.1784 | 5653 |
| TRTPN (ATPTN) | 2 | 2 2 | 3 | 7 | WORK.ANA DATA | 1.1682 | 0.2323 | 2676 |
| TRTPN (ATPTN) | 2 | 2 | ĺ | 8 | WORK.ANA DATA | 4.2357 | 0.2021 | 2709 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 8 | WORK.ANA DATA | 3.6840 | 0.1790 | 5654 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 8 | WORK.ANA DATA | 2.8037 | 0.2329 | 2697 |
| TRTPN (ATPTN) | 2 | 2 2 | 1 | 9 | WORK.ANA DATA | 4.4669 | 0.2014 | 2683 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 9 | WORK.ANA_DATA | 4.2714 | 0.1772 | 5656 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 9 | WORK.ANA DATA | 2.8600 | 0.2325 | 2683 |
| TRTPN (ATPTN) | 3 | 2 2 | 1 | 3 | WORK.ANA_DATA | 3.8843 | 0.2007 | 2671 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 3 | WORK.ANA_DATA | 3.1246 | 0.2323 | 2676 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 3 | WORK.ANA_DATA | 2.4776 | 0.1760 | 5650 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 4 | WORK.ANA_DATA | 1.3664 | 0.2006 | 2669 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 4 | WORK.ANA_DATA | 0.03882 | 0.2325 | 2683 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 4 | WORK.ANA_DATA | 0.4789 | 0.1763 | 5651 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 229 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

| | | DILIEIGUC | es or heast | oquares Me | allo | | |
|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
| TRTPN (ATPTN) | 3 3 3 3 3 3 3 1 1 1 1 1 1 1 1 1 1 1 1 1 | 1<br>2<br>2 | 2 3 1 2 2 3 1 1 2 3 3 | 7 | -7.74 -9.30 7.14 3.78 0.00 8.32 6.35 0.32 -4.25 -6.38 20.91 9.17 5.99 0.70 -6.16 -4.00 20.04 7.88 6.18 -1.91 -6.47 -3.68 8.05 0.73 1.56 26.96 13.99 9.69 29.05 17.04 9.99 -1.82 17.17 15.19 8.85 4.68 | <pre>&lt;.0001 &lt;.0001 &lt;.0001 0.0002 0.9967 &lt;.0001 0.7463 &lt;.0001 &lt;.00</pre> | 0.05 |
| TRTPN (ATPTN) | 2<br>2 | 2<br>2 | 1<br>2<br>3<br>3<br>3<br>3 | 4<br>4<br>4<br>5<br>5<br>5<br>5<br>6<br>6<br>6<br>6<br>7<br>7<br>7<br>8<br>8<br>8<br>9<br>9<br>9<br>9<br>3<br>3<br>3<br>3<br>4 | 4.68 -2.16 0.24 16.63 13.75 9.02 3.07 -2.49 0.52 9.23 5.63 5.03 20.96 20.58 12.04 22.18 24.11 12.30 19.36 13.45 14.07 6.81 0.17 2.72 | <.0001 0.0310 0.8099 <.0001 <.0001 <.0001 0.0022 0.0128 0.6030 <.0001 0.0001 | 0.05 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 230 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

| | D.1 | riterences c | or neast sat | iales Means | | |
|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
| TRTPN (ATPTN) | 3 | 1 | 2 | 7 | -2.2547 | -1.3436 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 7 | -1.9794 | -1.2903 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 8 | 1.0392 | 1.8262 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 8 | 0.4245 | 1.3374 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 8 | -0.3454 | 0.3469 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 9 | 1.2717 | 2.0560 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 1 | 2 3 | 9 | 1.0150<br>-0.2881 | 1.9217<br>0.4020 |
| TRIPN (AIPIN) | 3<br>1 | 2 | 2 | 2 | -1.2515 | -0.4616 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 2 | -1.6727 | -0.8865 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 3 | 2.3606 | 2.8489 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 3 | 1.4506 | 2.2395 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 3 | 0.8058 | 1.5902 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 4 | -0.1572 | 0.3308 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 4 | -1.6357 | -0.8458 |
| TRTPN (ATPTN) | 1 | 2 2 | 3<br>1 | 4<br>5 | -1.1933 | -0.4080<br>2.7368 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1<br>1 | 2 | 2 | 5 | 2.2491<br>1.1875 | 1.9744 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 5 | 0.8446 | 1.6289 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 6 | -0.4824 | 0.006482 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 6 | -1.6917 | -0.9048 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 6 | -1.1280 | -0.3437 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 7 | 0.7606 | 1.2507 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 7 | -0.2481 | 0.5427 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 7 | -0.08103 | 0.7042 |
| TRTPN (ATPTN) | 1 | 2 2 | 1 2 | 8 | 3.1334 | 3.6249 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1<br>1 | 2 | 3 | 8 | 2.4310<br>1.5531 | 3.2238<br>2.3412 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 9 | 3.3667 | 3.8540 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 9 | 3.0219 | 3.8077 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 9 | 1.6103 | 2.3965 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 2 | -0.8790 | 0.03292 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 3 | 3.0660 | 3.8566 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 3 | 2.3530 | 3.0502 |
| TRTPN (ATPTN) | 2 | 2 2 | 3<br>1 | 3 | 1.5994 | 2.5097 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 2 | 2 | 4 | 0.5482<br>-0.7334 | 1.3385<br>-0.03505 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 4 | -0.3996 | 0.5114 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 5 | 2.9545 | 3.7446 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 5 | 2.0899 | 2.7851 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 5 | 1.6381 | 2.5484 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 6 | 0.2232 | 1.0140 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 6 | -0.7893 | -0.09404 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 6 | -0.3344 | 0.5759 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 2 2 | 1 2 | 7<br>7 | 1.4664<br>0.6541 | 2.2580<br>1.3536 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 7 | 0.7126 | 1.6237 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 8 | 3.8395 | 4.6319 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 8 | 3.3331 | 4.0348 |
| TRTPN (ATPTN) | 2 | | 3 | 8 | 2.3470 | 3.2605 |
| TRTPN (ATPTN) | 2 | 2 2 | 1 | 9 | 4.0720 | 4.8618 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 9 | 3.9241 | 4.6187 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 9 | 2.4040 | 3.3159 |
| TRTPN (ATPTN) | 3 | 2 2 | 1 2 | 3 | 3.4909 | 4.2778 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 2 | 3 | 3 | 2.6691<br>2.1325 | 3.5801<br>2.8227 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 4 | 0.9730 | 1.7597 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 4 | -0.4171 | 0.4948 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 4 | 0.1333 | 0.8245 |
| ,, | | | | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 231 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

| | | DILL | CICHCCD OI | nearc bquar | CD HCGHD | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
| TRTPN (ATPTN) | 3 | 2 | 1 | 5 | WORK.ANA DATA | 3.7726 | 0.2005 | 2667 |
| | 3 | 2 | 2 | 5 | WORK.ANA DATA | 2.8605 | 0.2319 | 2662 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 2 | 3 | 5 | WORK.ANA DATA | 2.5163 | 0.1760 | 5650 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 6 | WORK.ANA DATA | 1.0416 | 0.2007 | 2674 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 6 | WORK.ANA DATA | -0.01865 | 0.2319 | 2662 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 6 | WORK.ANA DATA | 0.5438 | 0.1760 | 5650 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 7 | WORK.ANA DATA | 2.2852 | 0.2009 | 2681 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 7 | WORK.ANA DATA | 1.4269 | 0.2327 | 2690 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 7 | WORK.ANA DATA | 1.5912 | 0.1763 | 5651 |
| TRTPN (ATPTN) | 3 | 2 2 | 1 | 8 | WORK.ANA DATA | 4.6587 | 0.2012 | 2690 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 8 | WORK, ANA DATA | 4.1070 | 0.2332 | 2705 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 8 | WORK.ANA DATA | 3.2268 | 0.1771 | 5652 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 9 | WORK.ANA DATA | 4.8899 | 0.2005 | 2664 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 9 | WORK.ANA DATA | 4.6944 | 0.2316 | 2655 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 9 | WORK.ANA DATA | 3.2830 | 0.1766 | 5651 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 3 | WORK.ANA DATA | -0.7597 | 0.2013 | 2680 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 3 | WORK.ANA DATA | -1.4068 | 0.2002 | 2653 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 4 | WORK.ANA DATA | -2.5180 | 0.1247 | 5650 |
| TRTPN (ATPTN) | 1 | 3 | 2 3 | 4 | WORK.ANA DATA | -3.8455 | 0.2016 | 2690 |
| TRTPN (ATPTN) | 1 | 3 | | 4 | WORK.ANA_DATA | -3.4054 | 0.2004 | 2662 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 5 | WORK.ANA_DATA | -0.1118 | 0.1247 | 5651 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 5 | WORK.ANA_DATA | -1.0238 | 0.2008 | 2661 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 5 | WORK.ANA_DATA | -1.3680 | 0.2002 | 2653 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 6 | WORK.ANA_DATA | -2.8427 | 0.1250 | 5653 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 6 | WORK.ANA_DATA | -3.9030 | 0.2008 | 2661 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 6 | WORK.ANA_DATA | -3.3406 | 0.2002 | 2653 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 7 | WORK.ANA_DATA | -1.5991 | 0.1252 | 5653 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 7 | WORK.ANA_DATA | -2.4574 | 0.2018 | 2700 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 7 | WORK.ANA_DATA | -2.2932 | 0.2004 | 2662 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 8 | WORK.ANA_DATA | 0.7744 | 0.1256 | 5653 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 8 | WORK.ANA_DATA | 0.2226 | 0.2023 | 2719<br>2690 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 9 | WORK.ANA_DATA<br>WORK.ANA DATA | -0.6576<br>1.0056 | 0.2011<br>0.1246 | 2690<br>5653 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 3 | 2 | 9 | WORK.ANA DATA | 0.8101 | 0.2006 | 2652 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 9 | WORK.ANA DATA | -0.6013 | 0.2007 | 2671 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 3 | WORK.ANA DATA | -0.6470 | 0.2319 | 2662 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 4 | WORK.ANA DATA | -1.7582 | 0.2013 | 2678 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 4 | WORK.ANA DATA | -3.0858 | 0.1778 | 5650 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 4 | WORK.ANA DATA | -2.6457 | 0.2321 | 2669 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 5 | WORK.ANA DATA | 0.6480 | 0.2012 | 2676 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 5 | WORK.ANA DATA | -0.2641 | 0.1771 | 5651 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 5 | WORK.ANA DATA | -0.6083 | 0.2319 | 2662 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 6 | WORK.ANA DATA | -2.0830 | 0.2014 | 2683 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 6 | WORK.ANA DATA | -3.1433 | 0.1771 | 5651 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 6 | WORK.ANA DATA | -2.5809 | 0.2319 | 2662 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 7 | WORK.ANA DATA | -0.8394 | 0.2016 | 2690 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 7 | WORK.ANA_DATA | -1.6977 | 0.1781 | 5652 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 7 | WORK.ANA_DATA | -1.5334 | 0.2321 | 2669 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 8 | WORK.ANA_DATA | 1.5341 | 0.2018 | 2699 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 8 | WORK.ANA_DATA | 0.9824 | 0.1786 | 5651 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 8 | WORK.ANA_DATA | 0.1022 | 0.2327 | 2690 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 9 | WORK.ANA_DATA | 1.7653 | 0.2012 | 2673 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 9 | WORK.ANA_DATA | 1.5698 | 0.1769 | 5656 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 9 | WORK.ANA_DATA | 0.1584 | 0.2323 | 2676 |
| TRTPN (ATPTN) | 3 | ى<br>د | 1 | 4 | WORK.ANA_DATA | -1.1112 | 0.2001 | 2650 |
| TRTPN (ATPTN) | 3 | 3 | 2 | 4 | WORK.ANA_DATA | -2.4388 | 0.2321 | 2669 |
| TRTPN (ATPTN) | 3 | 3 | 1 | 4<br>5 | WORK.ANA_DATA | -1.9987<br>1.2950 | 0.1758<br>0.2001 | 5650<br>2648 |
| TRTPN (ATPTN)<br>TRTPN (ATPTN) | 3 | 3 | 2 | 5 | WORK.ANA_DATA<br>WORK.ANA DATA | 0.3829 | 0.2315 | 2648 |
| TIVIEIN (WILIN) | J | J | 4 | J | MOIVIV. ANA DATA | 0.3029 | 0.2313 | 2010 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 232 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

| | | DILIEIGUC | es or heast | oquares Me | allo | | |
|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
| TRTPN (ATPTN) | 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 1 1 1 1 1 | 2<br>2 | 1 2 3 3 1 2 2 3 3 1 2 2 3 3 1 | 5556666777788889999334444555566667777888899934445555 | 18.81 12.34 14.29 5.19 -0.08 3.09 11.38 6.13 9.03 23.16 17.61 18.22 24.39 20.27 18.59 -3.77 -7.03 -20.19 -19.08 -16.99 -0.90 -5.10 -6.83 -22.75 -19.43 -16.69 -12.77 -12.18 -11.44 6.16 1.10 -3.27 8.07 4.04 -3.00 -2.79 -8.74 -17.36 -11.40 3.22 -1.49 -2.62 | <pre>&lt;.0001 &lt;.0001 &lt;.0001 &lt;.0001 &lt;.0001 0.9359 0.0020 &lt;.0001 &lt;.00</pre> | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 2<br>2<br>2<br>2<br>2 | 3<br>3<br>3<br>3 | 1<br>2<br>3<br>1<br>2 | 6<br>6<br>7<br>7 | -10.34<br>-17.75<br>-11.13<br>-4.16<br>-9.53 | <.0001<br><.0001<br><.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05<br>0.05<br>0.05 |
| TRTPN (ATPTN) | 2<br>3<br>3<br>3<br>3<br>3 | 3<br>3 | 3<br>1<br>2<br>3<br>1<br>2<br>3<br>1<br>1<br>2<br>3<br>1<br>2<br>3<br>1<br>2<br>2<br>3<br>1<br>2<br>2<br>3 | 7<br>8<br>8<br>8<br>9<br>9<br>9<br>9<br>4<br>4<br>4<br>4<br>5<br>5<br>5 | -6.61<br>7.60<br>5.50<br>0.44<br>8.78<br>8.87<br>0.68<br>-5.55<br>-10.51<br>-11.37<br>6.47 | <.0001<br><.0001<br><.0001<br>0.6607<br><.0001<br><.0001<br>0.4955<br><.0001<br><.0001<br><.0001 | 0.05 |
| TT/TT 14 (WTE TIA) | J | J | - | J | 1.00 | 0.0002 | 0.00 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 233 of 412 | |

Parameter Code=C105585Y

Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
|---|---|---|---|---|---|---|
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 2 2 | 1 2 | 5<br>5 | 3.3794<br>2.4059 | 4.1658<br>3.3152 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 2 | 3<br>1 | 5<br>6 | 2.1712<br>0.6481 | 2.8614<br>1.4352 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 6 | -0.4733 | 0.4360 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 6 | 0.1987 | 0.8889 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 7 | 1.8913 | 2.6792 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 7 | 0.9705 | 1.8833 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 7 | 1.2456 | 1.9368 |
| TRTPN (ATPTN) | 3 | 2 | 1 2 | 8 | 4.2643<br>3.6498 | 5.0532<br>4.5642 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 2 | 3 | 8 | 2.8795 | 3.5740 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 9 | 4.4968 | 5.2830 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 9 | 4.2402 | 5.1486 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 9 | 2.9368 | 3.6292 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 3 | -1.1545 | -0.3649 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 3 | 3<br>1 | 3<br>4 | -1.7993<br>-2.7625 | -1.0142<br>-2.2734 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 4 | -4.2408 | -3.4502 |
| TRTPN (ATPTN) | ī | 3 | 3 | 4 | -3.7984 | -3.0124 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 5 | -0.3562 | 0.1326 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 5 | -1.4176 | -0.6300 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 5 | -1.7606 | -0.9755 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 3 | 1 2 | 6<br>6 | -3.0877<br>-4.2968 | -2.5977<br>-3.5092 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 6 | -3.7331 | -2.9481 |
| TRTPN (ATPTN) | ī | 3 | 1 | 7 | -1.8446 | -1.3536 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 7 | -2.8532 | -2.0617 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 7 | -2.6861 | -1.9002 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 8 | 0.5281 | 1.0207 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 3 | 2 3 | 8 | -0.1741<br>-1.0520 | 0.6194<br>-0.2632 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 9 | 0.7613 | 1.2498 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 9 | 0.4168 | 1.2033 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 9 | -0.9948 | -0.2079 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 3 | -1.1017 | -0.1923 |
| TRTPN (ATPTN) | 2 | 3 | 1 2 | 4 | -2.1529 | -1.3636<br>-2.7373 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 3 | 3 | 4 | -3.4343<br>-3.1008 | -2.1906 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 5 | 0.2534 | 1.0425 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 5 | -0.6112 | 0.08300 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 5 | -1.0630 | -0.1536 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 6 | -2.4779 | -1.6881 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 3 | 2 | 6<br>6 | -3.4904<br>-3.0356 | -2.7962<br>-2.1261 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 7 | -1.2347 | -0.4441 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 7 | -2.0469 | -1.3486 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 7 | -1.9886 | -1.0783 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 8 | 1.1383 | 1.9299 |
| TRTPN (ATPTN) | 2 2 | 3 | 2 3 | 8 | 0.6322 | 1.3325 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 3 | 1 | 9 | -0.3542<br>1.3709 | 0.5585<br>2.1597 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 9 | 1.2230 | 1.9165 |
| TRTPN (ATPTN) | 2 | 3 | 3<br>1 | 9 | -0.2972 | 0.6139 |
| TRTPN (ATPTN) | 3 | 3 | | 4 | -1.5036 | -0.7188 |
| TRTPN (ATPTN) | 3 | 3 | 2 | 4 | -2.8939 | -1.9836 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 3 | 3 | 4<br>5 | -2.3432<br>0.9027 | -1.6541<br>1.6873 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 3 | 2 | 5 | -0.07093 | 0.8368 |
| (/ | ~ | ~ | _ | - | 0.0.00 | 0.0000 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 234 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 3 | 3 | 3 | 5 | WORK.ANA DATA | 0.03871 | 0.1755 | 5649 |
| TRTPN (ATPTN) | 3 | 3 | 1 | 6 | WORK.ANA_DATA | -1.4359 | 0.2002 | 2655 |
| TRTPN (ATPTN) | 3 | 3 | 2 | 6 | WORK.ANA_DATA | -2.4962 | 0.2315 | 2648 |
| TRTPN (ATPTN) | 3 | 3 | 3 | 6 | WORK.ANA_DATA | -1.9338 | 0.1755 | 5649 |
| TRTPN (ATPTN) | 3 | 3 | 1 2 | 7<br>7 | WORK.ANA_DATA | -0.1924 | 0.2004 | 2662 |
| TRTPN (ATPTN) | 3 | 3 | 3 | 7 | WORK.ANA_DATA<br>WORK.ANA DATA | -1.0507<br>-0.8864 | 0.2323<br>0.1758 | 2676 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 3 | 1 | 8 | WORK.ANA DATA | 2.1811 | 0.1738 | 5650<br>2672 |
| TRTPN (ATPTN) | 3 | 3 | 2 | 8 | WORK.ANA DATA | 1.6294 | 0.2328 | 2691 |
| TRTPN (ATPTN) | 3 | 3 | 3 | 8 | WORK.ANA DATA | 0.7492 | 0.1766 | 5651 |
| TRTPN (ATPTN) | 3 | 3 | 1 | 9 | WORK.ANA DATA | 2.4123 | 0.2000 | 2646 |
| TRTPN (ATPTN) | 3 | 3 | 2 | 9 | WORK.ANA_DATA | 2.2168 | 0.2312 | 2641 |
| TRTPN (ATPTN) | 3 | 3 | 3 | 9 | WORK.ANA_DATA | 0.8054 | 0.1760 | 5650 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 4 | WORK.ANA_DATA | -1.3276 | 0.2015 | 2688 |
| TRTPN (ATPTN) | 1 | 4 | 3 | 4<br>5 | WORK.ANA_DATA | -0.8875<br>2.4062 | 0.2004<br>0.1246 | 2659<br>5652 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 4 | 2 | 5 | WORK.ANA_DATA<br>WORK.ANA DATA | 1.4941 | 0.2008 | 2659 |
| TRTPN (ATPTN) | 1 | 4 | 3 | 5 | WORK.ANA DATA | 1.1499 | 0.2001 | 2650 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 6 | WORK.ANA DATA | -0.3247 | 0.1249 | 5652 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 6 | WORK.ANA_DATA | -1.3850 | 0.2008 | 2659 |
| TRTPN (ATPTN) | 1 | 4 | 3 | 6 | WORK.ANA_DATA | -0.8226 | 0.2001 | 2650 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 7 | WORK.ANA_DATA | 0.9189 | 0.1252 | 5654 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 7<br>7 | WORK.ANA_DATA | 0.06053 | 0.2018 | 2697 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 4 | 3 | 8 | WORK.ANA_DATA<br>WORK.ANA DATA | 0.2248<br>3.2924 | 0.2004<br>0.1255 | 2660<br>5653 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 8 | WORK.ANA DATA | 2.7406 | 0.2023 | 2717 |
| TRTPN (ATPTN) | 1 | 4 | 3 | 8 | WORK.ANA DATA | 1.8604 | 0.2011 | 2688 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 9 | WORK.ANA DATA | 3.5235 | 0.1245 | 5652 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 9 | WORK.ANA_DATA | 3.3280 | 0.2005 | 2650 |
| TRTPN (ATPTN) | 1 | 4 | 3 | 9 | WORK.ANA_DATA | 1.9166 | 0.2006 | 2669 |
| TRTPN (ATPTN) | 2 | 4 | 3 | 4 | WORK.ANA_DATA | 0.4401 | 0.2323 | 2676 |
| TRTPN (ATPTN) | 2 | 4 | 1 2 | 5<br>5 | WORK.ANA_DATA | 3.7338 | 0.2015 | 2685 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 4 | 3 | 5 | WORK.ANA_DATA<br>WORK.ANA DATA | 2.8217<br>2.4775 | 0.1773<br>0.2321 | 5652<br>2669 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 6 | WORK.ANA DATA | 1.0028 | 0.2017 | 2692 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 6 | | -0.05746 | 0.1773 | 5652 |
| TRTPN (ATPTN) | 2 | 4 | 3 | 6 | WORK.ANA DATA | 0.5049 | 0.2321 | 2669 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 7 | WORK.ANA_DATA | 2.2464 | 0.2018 | 2699 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 7 | WORK.ANA_DATA | 1.3881 | 0.1784 | 5653 |
| TRTPN (ATPTN) | 2 | 4 | 3 | 7<br>8 | WORK.ANA_DATA | 1.5524 | 0.2323 | 2676 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 4 | 1 2 | 8 | WORK.ANA_DATA<br>WORK.ANA DATA | 4.6199<br>4.0682 | 0.2021<br>0.1789 | 2709<br>5652 |
| TRTPN (ATPTN) | 2 | 4 | 3 | 8 | WORK.ANA DATA | 3.1880 | 0.2329 | 2697 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 9 | WORK.ANA DATA | 4.8511 | 0.2014 | 2683 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 9 | WORK.ANA DATA | 4.6556 | 0.1772 | 5656 |
| TRTPN (ATPTN) | 2 | 4 | 3 | 9 | WORK.ANA_DATA | 3.2442 | 0.2325 | 2683 |
| TRTPN (ATPTN) | 3 | 4 | 1 | 5 | WORK.ANA_DATA | 3.2936 | 0.2003 | 2657 |
| TRTPN (ATPTN) | 3 | 4 | 2 | 5 | WORK.ANA_DATA | 2.3816 | 0.2317 | 2655 |
| TRTPN (ATPTN) | 3 | 4 | 1 | 5<br>6 | WORK.ANA_DATA<br>WORK.ANA DATA | 2.0374<br>0.5627 | 0.1758<br>0.2005 | 5650<br>2664 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 4 | 2 | 6 | WORK.ANA DATA | -0.4976 | 0.2005 | 2655 |
| TRTPN (ATPTN) | 3 | 4 | 3 | 6 | WORK.ANA DATA | 0.06484 | 0.1758 | 5650 |
| TRTPN (ATPTN) | 3 | 4 | 1 | 7 | WORK.ANA DATA | 1.8063 | 0.2007 | 2671 |
| TRTPN (ATPTN) | 3 | 4 | 2 | 7 | WORK.ANA_DATA | 0.9480 | 0.2325 | 2683 |
| TRTPN (ATPTN) | 3 | 4 | 3 | 7 | WORK.ANA_DATA | 1.1123 | 0.1760 | 5650 |
| TRTPN (ATPTN) | 3 | 4 | 1 | 8 | WORK.ANA_DATA | 4.1798 | 0.2009 | 2681 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 4 | 2 | 8 | WORK.ANA_DATA<br>WORK.ANA DATA | 3.6281<br>2.7479 | 0.2330<br>0.1769 | 2698<br>5652 |
| TRIPN (AIPIN) | 3 | 4 | 1 | 9 | WORK.ANA_DATA | 4.4110 | 0.2002 | 2655 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 235 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

| | | DILIEIGUC | es or heast | squares Me | allo | | |
|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
| TRTPN (ATPTN) | 3 3 3 3 3 3 3 3 3 3 3 3 3 1 1 1 1 1 1 1 | 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 | 3 1 2 | 5666677778888999944555566667777888899994555566667 | 0.22<br>-7.17<br>-10.78<br>-11.02<br>-0.96<br>-4.52<br>-5.04<br>10.87<br>7.00<br>4.24<br>12.06<br>9.59<br>4.58<br>-6.59<br>-4.43<br>19.31<br>7.44<br>5.75<br>-2.60<br>-6.90<br>-4.11<br>7.34<br>0.30<br>1.12<br>26.23<br>13.55<br>9.25<br>28.30<br>16.60<br>9.59<br>1.89<br>18.53<br>15.91<br>10.67<br>4.97<br>-0.32<br>2.18<br>11.13 | 0.8254 <.0001 | 0.05 |
| TRTPN (ATPTN) | 2<br>3<br>3 | 4<br>4 | 2<br>3<br>1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>3 | 7<br>7<br>8<br>8<br>8<br>9<br>9<br>9<br>9<br>5<br>5<br>5<br>5<br>6<br>6<br>6<br>6<br>7<br>7<br>7<br>8<br>8<br>8<br>9<br>9 | 7.78 6.68 22.86 22.74 13.69 24.09 26.28 13.95 16.44 10.28 11.59 2.81 -2.15 0.37 9.00 4.08 6.32 20.80 15.57 15.54 22.03 | <.0001 | 0.05 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 236 of 412 | |

Parameter Code=C105585Y

Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
|---|---|---|---|---|---|---|
| Effect TRTPN (ATPTN) | for<br>Period | Timepoint | for<br>Period | Timepoint (N) 5 6 6 6 7 7 7 8 8 8 9 9 4 4 5 5 5 6 6 6 7 7 7 8 8 8 9 9 9 4 5 5 5 6 6 6 7 7 7 8 8 8 8 9 9 9 9 9 9 9 9 9 9 9 | Lower -0.3053 -1.8286 -2.9501 -2.2778 -0.5854 -1.5062 -1.2310 1.7876 1.1730 0.4030 2.0202 1.7634 0.4603 -1.7227 -1.2803 2.1620 1.1005 0.7575 -0.5695 -1.7787 -1.2150 0.6735 -0.3351 -0.1681 3.0463 2.3440 1.4661 3.2795 2.9349 1.5233 -0.01544 3.3387 2.4741 2.0223 0.6074 -0.4051 0.04980 1.8506 1.0384 1.0968 4.2237 3.7175 2.7312 4.4562 4.3083 2.7882 | Upper 0.3827 -1.0433 -2.0424 -1.5898 0.2006 -0.5951 -0.5419 2.5746 2.0858 1.0954 2.8045 2.6702 1.1505 -0.9324 -0.4946 2.6504 1.8878 1.5423 -0.07997 -0.9913 -0.4302 1.1642 0.4562 0.6177 3.5384 3.1373 2.2547 3.7676 3.7212 2.3100 0.8957 4.1288 3.1694 2.9326 1.3982 0.2902 0.9601 2.6422 1.7378 2.0079 5.0162 4.4189 3.6447 5.2460 5.0029 |
| TRTPN (ATPTN) | 2<br>3 | 4<br>4 | 1<br>2<br>3<br>1<br>1<br>2<br>3<br>1<br>1<br>1<br>2<br>3<br>1<br>1<br>2<br>3<br>1<br>1<br>1<br>1 | 5<br>5<br>5<br>6<br>6<br>6<br>7<br>7<br>7<br>8<br>8<br>8<br>8<br>9 | 2.9009<br>1.9273<br>1.6928<br>0.1696<br>-0.9518<br>-0.2797<br>1.4128<br>0.4920<br>0.7672<br>3.7858<br>3.1712<br>2.4011<br>4.0184 | 3.6864<br>2.8359<br>2.3819<br>0.9558<br>-0.04331<br>0.4094<br>2.1998<br>1.4573<br>4.5733<br>4.5734<br>4.0849<br>3.0946<br>4.8036 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 237 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

| | | DILL | CICHCCD OI | nearc bquar | es means | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
| TRTPN (ATPTN) | 3 | 4 | 2 | 9 | WORK.ANA DATA | 4.2155 | 0.2314 | 2648 |
| TRTPN (ATPTN) | 3 | 4 | 3 | 9 | WORK.ANA DATA | 2.8041 | 0.1763 | 5651 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 5 | WORK.ANA DATA | -0.9120 | 0.2007 | 2657 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 5 | WORK.ANA DATA | -1.2563 | 0.2001 | 2648 |
| TRTPN (ATPTN) | ī | 5 | 1 | 6 | WORK.ANA DATA | -2.7309 | 0.1247 | 5651 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 6 | WORK.ANA DATA | -3.7912 | 0.2007 | 2657 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 6 | WORK.ANA DATA | -3.2288 | 0.2001 | 2648 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 7 | WORK.ANA DATA | -1.4873 | 0.1250 | 5651 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 7 | WORK.ANA DATA | -2.3457 | 0.2017 | 2695 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 7 | WORK.ANA DATA | -2.1814 | 0.2003 | 2657 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 8 | WORK.ANA DATA | 0.8862 | 0.1254 | 5653 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 8 | WORK.ANA DATA | 0.3344 | 0.2022 | 2715 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 8 | WORK.ANA DATA | -0.5458 | 0.2010 | 2685 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 9 | WORK.ANA DATA | 1.1174 | 0.1244 | 5654 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 9 | WORK.ANA_DATA | 0.9218 | 0.2004 | 2648 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 9 | WORK.ANA_DATA | -0.4896 | 0.2005 | 2667 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 5 | WORK.ANA_DATA | -0.3442 | 0.2315 | 2648 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 6 | WORK.ANA_DATA | -1.8189 | 0.2009 | 2664 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 6 | WORK.ANA_DATA | -2.8792 | 0.1765 | 5649 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 6 | WORK.ANA_DATA | -2.3168 | 0.2315 | 2648 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 7<br>7 | WORK.ANA_DATA | -0.5753 | 0.2011 | 2671 |
| TRTPN (ATPTN) | 2 | 5<br>5 | 2 | 7 | WORK.ANA_DATA | -1.4336 | 0.1776 | 5652 |
| TRTPN (ATPTN) | 2 | 5<br>5 | 3 | 8 | WORK.ANA_DATA | -1.2693<br>1.7982 | 0.2317<br>0.2013 | 2655<br>2681 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 5 | 2 | 8 | WORK.ANA_DATA<br>WORK.ANA DATA | 1.2465 | 0.2013 | 5654 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 8 | WORK.ANA DATA | 0.3663 | 0.2323 | 2676 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 9 | WORK.ANA DATA | 2.0294 | 0.2006 | 2655 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 9 | WORK.ANA DATA | 1.8339 | 0.1763 | 5653 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 9 | WORK.ANA DATA | 0.4225 | 0.2319 | 2662 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 6 | WORK.ANA DATA | -1.4747 | 0.2002 | 2655 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 6 | WORK.ANA DATA | -2.5349 | 0.2315 | 2648 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 6 | WORK.ANA DATA | -1.9725 | 0.1755 | 5649 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 7 | WORK.ANA DATA | -0.2311 | 0.2004 | 2662 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 7 | WORK.ANA_DATA | -1.0894 | 0.2323 | 2676 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 7 | WORK.ANA DATA | -0.9251 | 0.1758 | 5650 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 8 | WORK.ANA_DATA | 2.1424 | 0.2007 | 2672 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 8 | WORK.ANA_DATA | 1.5907 | 0.2328 | 2691 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 8 | WORK.ANA_DATA | 0.7105 | 0.1766 | 5651 |
| TRTPN (ATPTN) | 3 | 5<br>5 | 1 2 | 9 | WORK.ANA_DATA | 2.3736 | 0.2000 | 2646 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 9 | WORK.ANA_DATA | 2.1781 | 0.2312 | 2641<br>5650 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 6 | WORK.ANA_DATA<br>WORK.ANA DATA | 0.7667<br>-1.0603 | 0.1760<br>0.2009 | 2664 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 6 | 3 | 6 | WORK.ANA DATA | -0.4979 | 0.2003 | 2655 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 7 | WORK.ANA DATA | 1.2436 | 0.1253 | 5653 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 7 | WORK.ANA DATA | 0.3853 | 0.2019 | 2702 |
| TRTPN (ATPTN) | ī | 6 | 3 | 7 | WORK.ANA DATA | 0.5495 | 0.2005 | 2664 |
| TRTPN (ATPTN) | 1 | 6 | ĺ | 8 | WORK.ANA DATA | 3.6171 | 0.1257 | 5654 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 8 | WORK.ANA DATA | 3.0653 | 0.2024 | 2722 |
| TRTPN (ATPTN) | 1 | 6 | 3 | 8 | WORK.ANA DATA | 2.1851 | 0.2012 | 2692 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 9 | WORK.ANA DATA | 3.8483 | 0.1247 | 5654 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 9 | WORK.ANA_DATA | 3.6528 | 0.2006 | 2655 |
| TRTPN (ATPTN) | 1 | 6 | 3 | 9 | WORK.ANA_DATA | 2.2413 | 0.2007 | 2674 |
| TRTPN (ATPTN) | 2 | 6 | 3 | 6 | WORK.ANA_DATA | 0.5624 | 0.2315 | 2648 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 7 | WORK.ANA_DATA | 2.3039 | 0.2011 | 2671 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 7 | WORK.ANA_DATA | 1.4456 | 0.1776 | 5652 |
| TRTPN (ATPTN) | 2 | 6 | 3 | 7 | WORK.ANA_DATA | 1.6098 | 0.2317 | 2655 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 8 | WORK.ANA_DATA | 4.6774 | 0.2013 | 2681 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 8 | WORK.ANA_DATA | 4.1256 | 0.1782 | 5654 |
| TRTPN (ATPTN) | 2 | 6 | 3 | 8 | WORK.ANA_DATA | 3.2454 | 0.2323 | 2676 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 238 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

| | | DILIEIGUC | es or heast | oquares me | alio | | |
|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
| TRTPN (ATPTN) | 3 3 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | 4 4 5 5 5 5 5 5 5 5 5 5 5 5 5 5 5 5 5 5 | 2 3 1 2 3 1 2 3 3 1 2 3 3 1 2 3 3 1 2 3 3 1 2 3 3 1 2 2 | 9955666677778888999566667777888899996666777888 | 18.22<br>15.90<br>-4.54<br>-6.28<br>-21.89<br>-18.89<br>-16.14<br>-11.90<br>-11.63<br>-10.89<br>7.06<br>1.65<br>-2.72<br>8.98<br>4.60<br>-2.44<br>-1.49<br>-9.05<br>-16.31<br>-10.01<br>-2.86<br>-8.07<br>-5.48<br>8.93<br>6.99<br>1.58<br>10.11<br>10.40<br>1.82<br>-7.36<br>-10.95<br>-11.24<br>-1.15<br>-4.69<br>-5.26<br>10.68<br>6.83 | <pre>&lt;.0001 &lt;.0001 &lt;.00</pre> | 0.05 |
| TRTPN (ATPTN) | 3<br>3<br>3<br>3<br>1<br>2<br>2<br>2<br>2 | 555566666666666666666666666666666666666 | 3<br>1<br>2<br>3<br>2<br>3<br>1<br>2<br>3<br>1<br>2<br>3<br>1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>3 | 8<br>9<br>9<br>9<br>9<br>6<br>6<br>7<br>7<br>7<br>8<br>8<br>8<br>9<br>9<br>9<br>9<br>6<br>6<br>7<br>7<br>7<br>7<br>8<br>8<br>8<br>8<br>9 | 4.02<br>11.87<br>9.42<br>4.36<br>-5.28<br>-2.49<br>9.92<br>1.91<br>2.74<br>28.77<br>15.14<br>10.86<br>30.86<br>18.21<br>11.17<br>2.43<br>11.46<br>8.14<br>6.95<br>23.23<br>23.15<br>13.97 | <.0001 <.0001 <.0001 <.0001 <.0001 <.0001 0.0130 <.0001 0.0565 0.0062 <.0001 | 0.05 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 239 of 412 | |

Parameter Code=C105585Y

Differences of Least Squares Means

| | | .IICICIICCO C | or neare by | arco neano | | |
|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
| TRTPN (ATPTN) | 3 | 4 | 2 | 9 | 3.7617 | 4.6693 |
| TRTPN (ATPTN) | 3 | 4 | 3 | 9 | 2.4584 | 3.1497 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 5 | -1.3056 | -0.5185 |
| | 1 | 5 | 3 | 5 | -1.6486 | -0.8640 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 5 | 1 | 6 | -2.9755 | -2.4864 |
| | | 5 | 2 | | -4.1848 | -3.3976 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 6 | | |
| TRTPN (ATPTN) | | | | 6 | -3.6211 | -2.8365 |
| TRTPN (ATPTN) | 1 | 5<br>5 | 1 2 | 7<br>7 | -1.7324 | -1.2422 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 7 | -2.7412 | -1.9501 |
| TRTPN (ATPTN) | 1 | | | | -2.5741 | -1.7886 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 8 | 0.6403 | 1.1321 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 8 | -0.06211 | 0.7309 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 8 | -0.9400 | -0.1516 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 9 | 0.8734 | 1.3613 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 9 | 0.5288 | 1.3149 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 9 | -0.8828 | -0.09636 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 5 | -0.7981 | 0.1096 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 6 | -2.2128 | -1.4250 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 6 | -3.2251 | -2.5332 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 6 | -2.7706 | -1.8629 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 7 | -0.9696 | -0.1810 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 7 | -1.7818 | -1.0854 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 7 | -1.7236 | -0.8151 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 8 | 1.4034 | 2.1930 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 8 | 0.8971 | 1.5958 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 8 | -0.08924 | 0.8217 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 9 | 1.6360 | 2.4228 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 9 | 1.4883 | 2.1795 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 9 | -0.03220 | 0.8771 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 6 | -1.8673 | -1.0820 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 6 | -2.9888 | -2.0811 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 6 | -2.3166 | -1.6285 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 7 | -0.6241 | 0.1619 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 7 | -1.5449 | -0.6338 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 7 | -1.2697 | -0.5806 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 8 | 1.7489 | 2.5359 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 8 | 1.1343 | 2.0471 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 8 | 0.3643 | 1.0567 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 9 | 1.9815 | 2.7658 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 9 | 1.7247 | 2.6315 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 9 | 0.4216 | 1.1118 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 6 | -1.4542 | -0.6664 |
| TRTPN (ATPTN) | 1 | 6 | 3 | 6 | -0.8905 | -0.1053 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 7 | 0.9979 | 1.4893 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 7 | -0.01062 | 0.7811 |
| TRTPN (ATPTN) | 1 | 6 | 3 | 7 | 0.1564 | 0.9426 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 8 | 3.3706 | 3.8635 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 8 | 2.6685 | 3.4622 |
| TRTPN (ATPTN) | 1 | 6 | 3 | 8 | 1.7906 | 2.5797 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 9 | 3.6038 | 4.0928 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 9 | 3.2594 | 4.0461 |
| TRTPN (ATPTN) | 1 | 6 | 3 | 9 | 1.8478 | 2.6349 |
| TRTPN (ATPTN) | 2 | 6 | 3 | 6 | 0.1085 | 1.0163 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 7 | 1.9096 | 2.6982 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 7 | 1.0974 | 1.7937 |
| TRTPN (ATPTN) | 2 | 6 | 3 | 7 | 1.1556 | 2.0641 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 8 | 4.2826 | 5.0722 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 8 | 3.7763 | 4.4750 |
| , , | 2 | 6 | 3 | 8 | 2.7899 | 3.7009 |
| TRTPN (ATPTN) | ∠ | U | J | U | 2.1099 | 5.7009 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 240 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

# Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 2 | 6 | 1 | 9 | WORK.ANA DATA | 4.9086 | 0.2006 | 2655 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 9 | WORK.ANA DATA | 4.7131 | 0.1763 | 5653 |
| TRTPN (ATPTN) | 2 | 6 | 3 | 9 | WORK.ANA DATA | 3.3016 | 0.2319 | 2662 |
| TRTPN (ATPTN) | 3 | 6 | 1 | 7 | WORK.ANA DATA | 1.7415 | 0.2004 | 2662 |
| TRTPN (ATPTN) | 3 | 6 | 2 | 7 | WORK.ANA DATA | 0.8831 | 0.2323 | 2676 |
| TRTPN (ATPTN) | 3 | 6 | 3 | 7 | WORK.ANA DATA | 1.0474 | 0.2323 | 5650 |
| TRTPN (ATPTN) | 3 | 6 | 1 | 8 | WORK.ANA DATA | 4.1150 | 0.2007 | 2672 |
| TRTPN (ATPTN) | 3 | 6 | 2 | 8 | WORK.ANA DATA | 3.5632 | 0.2328 | 2691 |
| TRTPN (ATPTN) | 3 | 6 | 3 | 8 | WORK.ANA DATA | 2.6830 | 0.2326 | 5651 |
| TRTPN (ATPTN) | 3 | 6 | 1 | 9 | WORK.ANA DATA | 4.3462 | 0.2000 | 2646 |
| TRTPN (ATPTN) | 3 | 6 | 2 | 9 | WORK.ANA DATA | 4.1506 | 0.2312 | 2641 |
| TRTPN (ATPTN) | 3 | 6 | 3 | 9 | WORK.ANA DATA | 2.7392 | 0.2312 | 5650 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 7 | WORK.ANA DATA | -0.8583 | 0.2021 | 2709 |
| TRTPN (ATPTN) | 1 | 7 | 3 | 7 | WORK.ANA DATA | -0.6940 | 0.2021 | 2671 |
| TRTPN (ATPTN) | 1 | 7 | 1 | 8 | WORK.ANA DATA | 2.3735 | 0.1260 | 5654 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 8 | WORK.ANA DATA | 1.8218 | 0.2026 | 2729 |
| TRTPN (ATPTN) | 1 | 7 | 3 | 8 | WORK.ANA DATA | 0.9415 | 0.2014 | 2700 |
| TRTPN (ATPTN) | 1 | 7 | 1 | 9 | WORK.ANA DATA | 2.6047 | 0.1250 | 5655 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 9 | WORK.ANA DATA | 2.4092 | 0.2008 | 2662 |
| TRTPN (ATPTN) | 1 | 7 | 3 | 9 | WORK.ANA DATA | 0.9978 | 0.2009 | 2681 |
| TRTPN (ATPTN) | 2 | 7 | 3 | 7 | WORK.ANA DATA | 0.1643 | 0.2325 | 2683 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 8 | WORK.ANA DATA | 3.2318 | 0.2023 | 2719 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 8 | WORK.ANA DATA | 2.6801 | 0.1792 | 5654 |
| TRTPN (ATPTN) | 2 | 7 | 3 | 8 | WORK.ANA DATA | 1.7999 | 0.2332 | 2704 |
| TRTPN (ATPTN) | 2 | 7 | ĭ | 9 | WORK.ANA DATA | 3.4630 | 0.2016 | 2693 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 9 | WORK.ANA DATA | 3.2675 | 0.1774 | 5656 |
| TRTPN (ATPTN) | 2 | 7 | 3 | 9 | WORK.ANA DATA | 1.8561 | 0.2327 | 2690 |
| TRTPN (ATPTN) | 3 | 7 | 1 | 8 | WORK.ANA DATA | 3.0675 | 0.2009 | 2681 |
| TRTPN (ATPTN) | 3 | 7 | 2 | 8 | WORK.ANA DATA | 2.5158 | 0.2330 | 2698 |
| TRTPN (ATPTN) | 3 | 7 | 3 | 8 | WORK.ANA DATA | 1.6356 | 0.1769 | 5652 |
| TRTPN (ATPTN) | 3 | 7 | ĺ | 9 | WORK.ANA DATA | 3.2987 | 0.2002 | 2655 |
| TRTPN (ATPTN) | 3 | 7 | 2 | 9 | WORK.ANA DATA | 3.1032 | 0.2314 | 2648 |
| TRTPN (ATPTN) | 3 | 7 | 3 | 9 | WORK.ANA DATA | 1.6918 | 0.1763 | 5651 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 8 | WORK.ANA DATA | -0.5517 | 0.2028 | 2738 |
| TRTPN (ATPTN) | 1 | 8 | 3 | 8 | WORK.ANA DATA | -1.4320 | 0.2016 | 2709 |
| TRTPN (ATPTN) | 1 | 8 | ĺ | 9 | WORK.ANA DATA | 0.2312 | 0.1254 | 5655 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 9 | WORK.ANA DATA | 0.03568 | 0.2011 | 2672 |
| TRTPN (ATPTN) | 1 | 8 | 3 | 9 | WORK.ANA DATA | -1.3757 | 0.2012 | 2690 |
| TRTPN (ATPTN) | 2 | 8 | 3 | 8 | WORK.ANA DATA | -0.8802 | 0.2336 | 2719 |
| TRTPN (ATPTN) | 2 | 8 | 1 | 9 | WORK.ANA DATA | 0.7829 | 0.2022 | 2712 |
| TRTPN (ATPTN) | 2 | 8 | 2 | 9 | WORK.ANA DATA | 0.5874 | 0.1780 | 5658 |
| TRTPN (ATPTN) | 2 | 8 | 3 | 9 | WORK.ANA DATA | -0.8240 | 0.2332 | 2705 |
| TRTPN (ATPTN) | 3 | 8 | 1 | 9 | WORK.ANA DATA | 1.6631 | 0.2010 | 2683 |
| TRTPN (ATPTN) | 3 | 8 | 2 | 9 | WORK.ANA DATA | 1.4676 | 0.2320 | 2669 |
| TRTPN (ATPTN) | 3 | 8 | 3 | 9 | WORK.ANA DATA | 0.05621 | 0.1771 | 5652 |
| TRTPN (ATPTN) | 1 | 9 | 2 | 9 | WORK.ANA DATA | -0.1955 | 0.2004 | 2646 |
| TRTPN (ATPTN) | 1 | 9 | 3 | 9 | WORK.ANA DATA | -1.6069 | 0.2005 | 2664 |
| TRTPN (ATPTN) | 2 | 9 | 3 | 9 | WORK.ANA DATA | -1.4114 | 0.2316 | 2655 |
| | | | | | _ | | | |

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 01 (N)<br>2 | 6 | 01 (N)<br>1 | 9 | 24.46 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 9 | 26.73 | <.0001 | 0.05 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 241 of 412 | |

Parameter Code=C105585Y

The Mixed Procedure

## Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| Effect TRTPN (ATPTN) | | _ | 01 (N) 3 1 2 3 1 1 2 3 1 2 3 3 1 2 3 3 3 1 2 3 3 3 1 2 3 3 3 1 2 3 3 3 1 2 3 3 3 1 2 3 3 3 3 | - | t Value 14.24 8.69 3.80 5.96 20.51 15.31 15.19 21.73 17.95 15.56 -4.25 -3.46 18.84 8.99 4.68 20.84 12.00 4.97 0.71 15.97 14.95 7.72 17.17 18.41 7.98 15.27 10.80 9.25 16.48 | Pr > t <.0001 | Alpha 0.05 0.05 0.05 0.05 0.05 0.05 0.05 0. |
| TRTPN (ATPTN) | 3<br>3<br>1<br>1<br>1<br>1<br>1<br>2<br>2<br>2<br>2<br>2<br>2<br>3<br>3<br>3<br>3<br>1<br>1<br>1<br>2 | 7 7 7 8 8 8 8 8 8 8 8 8 8 8 8 8 8 8 8 8 | 2<br>3<br>2<br>3<br>1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>3 | 998899998999999999999999999 | 13.41<br>9.60<br>-2.72<br>-7.10<br>1.84<br>0.18<br>-6.84<br>-3.77<br>3.87<br>3.30<br>-3.53<br>8.28<br>6.32<br>0.32<br>-0.98<br>-8.02<br>-6.09 | <pre>&lt;.0001 &lt;.0001 &lt;.0001 0.0066 &lt;.0001 0.0653 0.8592 &lt;.0001 0.0002 0.0001 0.0010 0.0010 0.0010 0.0010 &lt;.0001 &lt;.00</pre> | 0.05 |

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
|---|---|---|---|---|---|---|
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 2<br>2<br>2<br>3 | 6<br>6<br>6 | 1<br>2<br>3<br>1 | 9<br>9<br>9<br>7 | 4.5151<br>4.3674<br>2.8470<br>1.3485 | 5.3020<br>5.0587<br>3.7563<br>2.1345 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 242 of 412 | |

Parameter Code=C105585Y

Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 3 | 6 | 2 | 7 | 0.4276 | 1.3387 |
| TRTPN (ATPTN) | 3 | 6 | 3 | 7 | 0.7029 | 1.3920 |
| TRTPN (ATPTN) | 3 | 6 | 1 | 8 | 3.7215 | 4.5085 |
| TRTPN (ATPTN) | 3 | 6 | 2 | 8 | 3.1068 | 4.0197 |
| TRTPN (ATPTN) | 3 | 6 | 3 | 8 | 2.3368 | 3.0292 |
| TRTPN (ATPTN) | 3 | 6 | 1 | 9 | 3.9540 | 4.7383 |
| TRTPN (ATPTN) | 3 | 6 | 2 | 9 | 3.6973 | 4.6040 |
| TRTPN (ATPTN) | 3 | 6 | 3 | 9 | 2.3941 | 3.0843 |
| TRTPN (ATPTN) | ĺ | 7 | 2 | 7 | -1.2546 | -0.4621 |
| TRTPN (ATPTN) | 1 | 7 | 3 | 7 | -1.0875 | -0.3006 |
| TRTPN (ATPTN) | 1 | 7 | 1 | 8 | 2.1265 | 2.6205 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 8 | 1.4245 | 2.2190 |
| TRTPN (ATPTN) | 1 | 7 | 3 | 8 | 0.5467 | 1.3364 |
| TRTPN (ATPTN) | 1 | 7 | 1 | 9 | 2.3596 | 2.8498 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 9 | 2.0154 | 2.8029 |
| TRTPN (ATPTN) | 1 | 7 | 3 | 9 | 0.6038 | 1.3917 |
| TRTPN (ATPTN) | 2 | 7 | 3 | 7 | -0.2917 | 0.6202 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 8 | 2.8351 | 3.6286 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 8 | 2.3287 | 3.0315 |
| TRTPN (ATPTN) | 2 | 7 | 3 | 8 | 1.3427 | 2.2571 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 9 | 3.0676 | 3.8584 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 9 | 2.9197 | 3.6154 |
| TRTPN (ATPTN) | 2 | 7 | 3 | 9 | 1.3997 | 2.3125 |
| TRTPN (ATPTN) | 3 | 7 | 1 | 8 | 2.6736 | 3.4615 |
| TRTPN (ATPTN) | 3 | 7 | 2 | 8 | 2.0590 | 2.9726 |
| TRTPN (ATPTN) | 3 | 7 | 3 | 8 | 1.2889 | 1.9823 |
| TRTPN (ATPTN) | 3 | 7 | 1 | 9 | 2.9061 | 3.6914 |
| TRTPN (ATPTN) | 3 | 7 | 2 | 9 | 2.6494 | 3.5570 |
| TRTPN (ATPTN) | 3 | 7 | 3 | 9 | 1.3462 | 2.0374 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 8 | -0.9495 | -0.1540 |
| TRTPN (ATPTN) | 1 | 8 | 3 | 8 | -1.8273 | -1.0366 |
| TRTPN (ATPTN) | 1 | 8 | 1 | 9 | -0.01462 | 0.4770 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 9 | -0.3586 | 0.4299 |
| TRTPN (ATPTN) | 1 | 8 | 3 | 9 | -1.7702 | -0.9813 |
| TRTPN (ATPTN) | 2 | 8 | 3 | 8 | -1.3383 | -0.4222 |
| TRTPN (ATPTN) | 2 | 8 | 2 | 9 | 0.3865 | 1.1793 |
| TRTPN (ATPTN) | | | | | 0.2384 | 0.9364 |
| TRTPN (ATPTN) | 2 | 8 | 3 | 9 | -1.2812 | -0.3668 |
| TRTPN (ATPTN) | 3 | 8 | 2 | 9 | 1.2691 | 2.0572<br>1.9226 |
| TRTPN (ATPTN) | 3 | 8 | 3 | 9 | 1.0126<br>-0.2910 | |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 9 | 2 | 9 | -0.2910 | 0.4035<br>0.1974 |
| TRIPN (AIPIN) | 1 | 9 | 3 | 9 | -2.0000 | -1.2139 |
| | 2 | 9 | 3 | 9 | -1.8656 | -0.9572 |
| TRTPN (ATPTN) | ۷ | J | J | J | T.0000 | 0.3312 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 243 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

Model Information

Data Set
Dependent Variable
Covariance Structure
Subject Effect
Estimation Method
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method
WORK.ANA\_DATA
AVAL
Compound Symmetry
USUBJID
REML
Profile
Kenward-Roger
Kenward-Roger

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 244 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

Class Level Information

Class Levels Values USUBJID 720 NN9068-4148/ NN9068-4146/ NN9068-4148/

NN9068-4148/

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 245 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

NN9068-4148/

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 246 of 412 | |

Parameter Code=SMPGCOL

```
NN9068-4148/

NN9068-4148/
    NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 247 of 412 | |

Parameter Code=SMPGCOL

```
NN9068-4148/

NN9068-4148/
    NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 248 of 412 | |

Parameter Code=SMPGCOL

```
NN9068-4148/

NN9068-4148/
    NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 249 of 412 | |

Parameter Code=SMPGCOL

```
NN9068-4148/

NN9068-4148/
    NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 250 of 412 | |

Parameter Code=SMPGCOL

```
NN9068-4148/

NN9068-4148/
    NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 251 of 412 | |

Parameter Code=SMPGCOL

```
NN9068-4148/

NN9068-4148/
    NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 252 of 412 | |

Parameter Code=SMPGCOL

```
NN9068-4148/

NN9068-4148/
    NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 253 of 412 | |

Parameter Code=SMPGCOL

```
NN9068-4148/

NN9068-4148/
    NN9068-4148/
```

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 254 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

```
NN9068-4148/
  1 2 3
1 2 3 4 5 6 7 8 9
  Metformin Metformin + OAD
```

#### Dimensions

3

TRTPN ATPTN

PREOAD2

| Covariance | Parameters | 2 |
|------------|------------|-----|
| Columns in | X | 49 |
| Columns in | Z | 0 |
| Subjects | | 720 |
| Max Obs pe | r Subject | 9 |


9-point self-measured plasma glucose profile after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=SMPGCOL

The Mixed Procedure

Number of Observations

Number of Observations Read 6480 Number of Observations Used 6401 Number of Observations Not Used 79

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 65035.29815169
1 2 62992.58883544 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate | Standard<br>Error | Z<br>Value | Pr Z | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| CS<br>Residual | USUBJID | 657.94<br>899.99 | 40.2013<br>16.9343 | 16.37<br>53.15 | <.0001<br><.0001 | 0.05 | 579.15<br>867.70 | 736.73<br>934.12 |

Asymptotic Covariance Matrix of Estimates

| Row | Cov Parm | CovP1 | CovP2 |
|-----|----------|----------|----------|
| 1 | CS | 1616.14 | -32.4580 |
| 2 | Residual | -32.4580 | 286.77 |

Fit Statistics

-2 Res Log Likelihood 62992.6 AIC (Smaller is Better) 62996.6 AICC (Smaller is Better) 62996.6 BIC (Smaller is Better) 63005.7

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1 2042.71 <.0001

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| Intercept | | | | 129.36 | 3.1296 | 2673 | 41.34 | <.0001 |
| TRTPN | | 1 | | -28.9569 | 3.6123 | 2664 | -8.02 | <.0001 |
| TRTPN | | 2 | | -25.4338 | 4.1740 | 2655 | -6.09 | <.0001 |
| TRTPN | | 3 | | 0 | | | | |
| TRTPN (ATPTN) | | 1 | 1 | 0.9972 | 2.4959 | 5650 | 0.40 | 0.6895 |
| TRTPN (ATPTN) | | 2 | 1 | 3.0880 | 3.3486 | 5649 | 0.92 | 0.3565 |
| TRTPN (ATPTN) | | 3 | 1 | 0.6433 | 3.3621 | 5650 | 0.19 | 0.8483 |
| TRTPN (ATPTN) | | 1 | 2 | 68.3246 | 2.4993 | 5650 | 27.34 | <.0001 |
| TRTPN (ATPTN) | | 2 | 2 | 80.2365 | 3.3670 | 5654 | 23.83 | <.0001 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 256 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

## Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | | 3 | 2 | 62.4258 | 3.3750 | 5652 | 18.50 | <.0001 |
| TRTPN (ATPTN) | | 1 | 3 | 20.3438 | 2.5061 | 5652 | 8.12 | <.0001 |
| TRTPN (ATPTN) | | 2 | 3 | 30.5109 | 3.3645 | 5654 | 9.07 | <.0001 |
| TRTPN (ATPTN) | | 3 | 3 | 16.7365 | 3.3632 | 5651 | 4.98 | <.0001 |
| TRTPN (ATPTN) | | 1 | 4 | 65.1838 | 2.5044 | 5651 | 26.03 | <.0001 |
| TRTPN (ATPTN) | | 2 | 4 | 85.5833 | 3.3675 | 5655 | 25.41 | <.0001 |
| TRTPN (ATPTN) | | 3 | 4 | 52.2188 | 3.3660 | 5651 | 15.51 | <.0001 |
| TRTPN (ATPTN) | | 1 | 5 | 22.7376 | 2.4997 | 5652 | 9.10 | <.0001 |
| TRTPN (ATPTN) | | 2 | 5 | 35.6495 | 3.3524 | 5652 | 10.63 | <.0001 |
| TRTPN (ATPTN) | | 3 | 5 | 16.4187 | 3.3632 | 5651 | 4.88 | <.0001 |
| TRTPN (ATPTN) | | 1 | 6 | 72.6059 | 2.5049 | 5653 | 28.99 | <.0001 |
| TRTPN (ATPTN) | | 2 | 6 | 88.1892 | 3.3528 | 5652 | 26.30 | <.0001 |
| TRTPN (ATPTN) | | 3 | 6 | 52.6208 | 3.3636 | 5651 | 15.64 | <.0001 |
| TRTPN (ATPTN) | | | 7 | 50.3831 | 2.5089 | 5654 | 20.08 | <.0001 |
| TRTPN (ATPTN) | | 1 2 | 7 | 62.3271 | 3.3743 | 5655 | 18.47 | <.0001 |
| TRTPN (ATPTN) | | 3 | 7 | 33.9330 | 3.3706 | 5652 | 10.07 | <.0001 |
| TRTPN (ATPTN) | | 1 | 8 | 5.0699 | 2.5172 | 5654 | 2.01 | 0.0440 |
| TRTPN (ATPTN) | | 2 | 8 | 11.4891 | 3.3879 | 5657 | 3.39 | 0.0007 |
| TRTPN (ATPTN) | | 2 | 8 | 1.9167 | 3.3824 | 5653 | 0.57 | 0.5710 |
| TRTPN (ATPTN) | | 1 | 9 | 1.5107 | 3.3024 | 3033 | 0.57 | 0.3710 |
| TRTPN (ATPTN) | | 2 | 9 | 0 | | | | |
| TRTPN (ATPTN) | | 3 | 9 | 0 | | | | |
| PREOAD2 (ATPTN) | Metformin | 9 | 1 | -2.4780 | 3.1407 | 2641 | -0.79 | 0.4302 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 1 | -2.4700 | 3.1407 | 2041 | -0.79 | 0.4302 |
| PREOAD2 (ATPTN) | Metformin | | 2 | -13.7059 | 3.1541 | 2671 | -4.35 | <.0001 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 2 | 13.7033 | 3.1341 | 2011 | 4.55 | V.0001 |
| PREOAD2 (ATPTN) | Metformin | | 3 | -10.4963 | 3.1518 | 2665 | -3.33 | 0.0009 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 3 | 10.4505 | 3.1310 | 2005 | 3.33 | 0.0003 |
| PREOAD2 (ATPTN) | Metformin | | 3<br>4 | -8.8544 | 3.1571 | 2678 | -2.80 | 0.0051 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 4 | 0.00.09 | 3.13/1 | 2070 | -2.00 | 0.0031 |
| PREOAD2 (ATPTN) | Metformin | | 5 | -11.6645 | 3.1514 | 2664 | -3.70 | 0.0002 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 5 | 0 | 3.1314 | 2004 | -3.70 | 0.0002 |
| PREOAD2 (ATPTN) | Metformin | | 6 | -13.6864 | 3.1557 | 2675 | -4.34 | <.0001 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 6 | 0 | 3.1337 | 2013 | 4.54 | V.0001 |
| PREOAD2 (ATPTN) | Metformin | | 7 | -14.2607 | 3.1682 | 2705 | -4.50 | <.0001 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 7 | -14.2607 | 3.1002 | 2/03 | -4.30 | <.UUU1 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 8 | -6.4367 | 3.1817 | 2738 | -2.02 | 0.0432 |
| PREOAD2 (ATPIN) | Metformin + OAD | | 8 | -0.4307 | J. 101/ | 2150 | -2.02 | 0.0432 |
| PREOADZ (ATPTN) PREOADZ (ATPTN) | Metformin + OAD | | 0 | -3.6559 | 3.1435 | 2648 | -1.16 | 0.2449 |
| PREOAD2 (ATPTN) | Metformin + OAD | | 9 | -3.6339 | 3.1433 | 2040 | -1.10 | 0.2449 |
| INTOADS (AITIN) | FICCIOIMIII OAD | | , | 0 | | | | |

Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|-----------------|-----------|-----------|---------|---------|
| TRTPN | 2 | 716 | 39.78 | <.0001 |
| TRTPN (ATPTN) | 16 | 5652 | 8.63 | <.0001 |
| PRECAD2 (ATPTN) | 9 | 5392 | 5.07 | < .0001 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 257 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | WORK.ANA DATA | 100.60 | 2.0774 | 2641 | 48.42 | <.0001 |
| TRTPN (ATPTN) | 2 | 1 | WORK.ANA DATA | 106.21 | 2.9502 | 2641 | 36.00 | <.0001 |
| TRTPN (ATPTN) | 3 | 1 | WORK.ANA DATA | 129.20 | 2.9420 | 2641 | 43.92 | <.0001 |
| TRTPN (ATPTN) | 1 | 2 | WORK.ANA DATA | 164.28 | 2.0815 | 2655 | 78.92 | <.0001 |
| TRTPN (ATPTN) | 2 | 2 | WORK.ANA DATA | 179.71 | 2.9730 | 2697 | 60.45 | < .0001 |
| TRTPN (ATPTN) | 3 | 2 | WORK.ANA DATA | 187.33 | 2.9526 | 2669 | 63.45 | < .0001 |
| TRTPN (ATPTN) | 1 | 3 | WORK.ANA DATA | 117.34 | 2.0873 | 2676 | 56.22 | <.0001 |
| TRTPN (ATPTN) | 2 | 3 | WORK.ANA DATA | 131.03 | 2.9677 | 2683 | 44.15 | <.0001 |
| TRTPN (ATPTN) | 3 | 3 | WORK.ANA DATA | 142.69 | 2.9420 | 2641 | 48.50 | <.0001 |
| TRTPN (ATPTN) | 1 | 4 | WORK.ANA DATA | 162.71 | 2.0854 | 2669 | 78.03 | <.0001 |
| TRTPN (ATPTN) | 2 | 4 | WORK.ANA DATA | 186.63 | 2.9732 | 2697 | 62.77 | <.0001 |
| TRTPN (ATPTN) | 3 | 4 | WORK.ANA DATA | 178.70 | 2.9472 | 2655 | 60.63 | <.0001 |
| TRTPN (ATPTN) | 1 | 5 | WORK.ANA DATA | 119.35 | 2.0834 | 2662 | 57.29 | <.0001 |
| TRTPN (ATPTN) | 2 | 5 | WORK.ANA DATA | 135.79 | 2.9565 | 2654 | 45.93 | <.0001 |
| TRTPN (ATPTN) | 3 | 5 | WORK.ANA DATA | 141.99 | 2.9420 | 2641 | 48.26 | <.0001 |
| TRTPN (ATPTN) | 1 | 6 | WORK.ANA DATA | 168.56 | 2.0890 | 2683 | 80.69 | < .0001 |
| TRTPN (ATPTN) | 2 | 6 | WORK.ANA DATA | 187.67 | 2.9565 | 2654 | 63.48 | < .0001 |
| TRTPN (ATPTN) | 3 | 6 | WORK.ANA DATA | 177.54 | 2.9420 | 2641 | 60.35 | < .0001 |
| TRTPN (ATPTN) | 1 | 7 | WORK.ANA DATA | 146.15 | 2.0948 | 2704 | 69.77 | < .0001 |
| TRTPN (ATPTN) | 2 | 7 | WORK.ANA DATA | 161.62 | 2.9785 | 2712 | 54.26 | < .0001 |
| TRTPN (ATPTN) | 3 | 7 | WORK.ANA DATA | 158.66 | 2.9472 | 2655 | 53.83 | < .0001 |
| TRTPN (ATPTN) | 1 | 8 | WORK.ANA DATA | 103.38 | 2.1028 | 2733 | 49.17 | < .0001 |
| TRTPN (ATPTN) | 2 | 8 | WORK.ANA DATA | 113.33 | 2.9898 | 2741 | 37.90 | <.0001 |
| TRTPN (ATPTN) | 3 | 8 | WORK.ANA DATA | 129.19 | 2.9633 | 2697 | 43.60 | < .0001 |
| TRTPN (ATPTN) | 1 | 9 | WORK.ANA_DATA | 99.2172 | 2.0813 | 2655 | 47.67 | < .0001 |
| TRTPN (ATPTN) | 2 | 9<br>9 | WORK.ANA DATA | 102.74 | 2.9502 | 2641 | 34.82 | < .0001 |
| TRTPN (ATPTN) | 3 | 9 | WORK.ANA DATA | 128.17 | 2.9526 | 2669 | 43.41 | <.0001 |

Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Alpha | Lower | Upper |
|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>3 | 1<br>1<br>1<br>2<br>2<br>2<br>2<br>3<br>3<br>3<br>4<br>4<br>4<br>4<br>5<br>5<br>5<br>6<br>6<br>6<br>6<br>7<br>7<br>7<br>7<br>7<br>8 | 0.05 | 96.5237<br>100.43<br>123.43<br>160.19<br>173.88<br>181.54<br>113.24<br>125.21<br>136.92<br>158.62<br>180.80<br>172.92<br>115.27<br>129.99<br>136.22<br>164.47<br>181.87<br>171.77<br>142.05<br>155.78<br>152.88<br>99.2601 | 104.67<br>112.00<br>134.97<br>168.36<br>185.54<br>193.12<br>121.43<br>136.85<br>148.46<br>166.80<br>192.46<br>184.48<br>123.44<br>147.76<br>172.66<br>193.47<br>150.26<br>167.46 |
| TRTPN (ATPTN) | 2 | 8 | 0.05 | 107.46 | 119.19 |

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

9-point self-measured plasma glucose profile after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=SMPGCOL

The Mixed Procedure

## Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Alpha | Lower | Upper |
|---|---|---|---|---|---|
| TRTPN (ATPTN)<br>TRTPN (ATPTN) | 3 | 8 | 0.05 | 123.38<br>95.1361 | 135.00<br>103.30 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 9<br>9 | 0.05<br>0.05 | 96.9553<br>122.38 | 108.53<br>133.96 |

## Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | 2 | 1 | WORK.ANA DATA | -5.6140 | 3.6083 | 2641 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 1 | WORK.ANA DATA | -28.6031 | 3.6015 | 2641 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 2 | WORK.ANA DATA | -63.6784 | 2.2368 | 5652 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 2 | WORK.ANA DATA | -79.1134 | 3.6269 | 2679 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 2 | WORK.ANA DATA | -86.7365 | 3.6102 | 2660 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 3 | WORK.ANA DATA | -16.7407 | 2.2422 | 5653 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 3 | WORK.ANA DATA | -30.4309 | 3.6225 | 2669 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 3 | WORK.ANA_DATA | -42.0903 | 3.6015 | 2641 |

# Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | 2 | 1 | -1.56 | 0.1199 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 1 | -7.94 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 2 | -28.47 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 2 | -21.81 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 2 | -24.03 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 3 | -7.47 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 3 | -8.40 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 3 | -11.69 | <.0001 | 0.05 |

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1<br>1<br>1<br>1<br>1 | 1<br>1<br>1<br>1<br>1 | 2<br>3<br>1<br>2<br>3<br>1<br>2 | 1<br>1<br>2<br>2<br>2<br>3<br>3 | -12.6893<br>-35.6651<br>-68.0634<br>-86.2253<br>-93.8155<br>-21.1361<br>-37.5342 | 1.4614<br>-21.5411<br>-59.2934<br>-72.0016<br>-79.6575<br>-12.3452<br>-23.3276 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 3 | -49.1524 | -35.0283 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 259 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 1 | 1 | 1 | 4 | WORK.ANA DATA | -62.1143 | 2.2404 | 5653 |
| TRTPN (ATPTN) | 1 | i | 2 | 4 | WORK.ANA DATA | -86.0370 | 3.6271 | 2679 |
| | | 1 | 3 | 4 | | | | |
| TRTPN (ATPTN) | 1<br>1 | 1 | 1 | 5 | WORK.ANA_DATA | -78.1063 | 3.6058 | 2650<br>5652 |
| TRTPN (ATPTN) | | | | | WORK.ANA_DATA | -18.7548 | 2.2386 | |
| TRTPN (ATPTN) | 1 | 1 | 2 | 5 | WORK.ANA_DATA | -35.1898 | 3.6134 | 2650 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 5 | WORK.ANA_DATA | -41.3928 | 3.6015 | 2641 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 6 | WORK.ANA_DATA | -67.9660 | 2.2438 | 5653 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 6 | WORK.ANA_DATA | -87.0725 | 3.6134 | 2650 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 6<br>7 | WORK.ANA_DATA | -76.9379 | 3.6015 | 2641 |
| TRTPN (ATPTN) | 1 | | 2 | 7 | WORK.ANA_DATA | -45.5566 | 2.2492 | 5654 |
| TRTPN (ATPTN) | 1 | 1 | | 7 | WORK.ANA_DATA | -61.0237 | 3.6314 | 2688 |
| TRTPN (ATPTN) | 1 | 1 | 3<br>1 | 8 | WORK.ANA_DATA<br>WORK.ANA DATA | -58.0633<br>-2.7861 | 3.6058<br>2.2566 | 2650<br>5656 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 8 | WORK.ANA DATA | -12.7285 | | 2708 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 1 | 3 | 8 | WORK.ANA DATA | -28.5899 | 3.6407<br>3.6189 | 2679 |
| TRTPN (ATPTN) | 1 | 1 | 1 | 9 | WORK.ANA DATA | 1.3800 | 2.2365 | 5650 |
| TRTPN (ATPTN) | 1 | 1 | 2 | 9 | WORK.ANA DATA | -2.1432 | 3.6083 | 2641 |
| TRTPN (ATPTN) | 1 | 1 | 3 | 9 | WORK.ANA DATA | -27.5769 | 3.6102 | 2660 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 1 | WORK.ANA DATA | -22.9891 | 4.1665 | 2641 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 2 | WORK.ANA DATA | -58.0644 | 3.6107 | 2645 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 2 | WORK.ANA DATA | -73.4995 | 3.1924 | 5656 |
| TRTPN (ATPTN) | 2 | ī | 3 | 2 2 | WORK.ANA DATA | -81.1225 | 4.1739 | 2655 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 3 | WORK, ANA DATA | -11.1267 | 3.6140 | 2652 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 3 | WORK.ANA DATA | -24.8169 | 3.1874 | 5656 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 3 | WORK.ANA DATA | -36.4764 | 4.1664 | 2641 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 4 | WORK.ANA DATA | -56.5004 | 3.6129 | 2650 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 4 | WORK.ANA DATA | -80.4230 | 3.1925 | 5656 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 4 | WORK.ANA DATA | -72.4923 | 4.1702 | 2648 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 5 | WORK.ANA DATA | -13.1408 | 3.6118 | 2648 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 5 | WORK.ANA DATA | -29.5759 | 3.1770 | 5653 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 5 | WORK.ANA_DATA | -35.7788 | 4.1664 | 2641 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 6 | WORK.ANA_DATA | -62.3520 | 3.6150 | 2655 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 6 | WORK.ANA_DATA | -81.4585 | 3.1770 | 5653 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 6 | WORK.ANA_DATA | -71.3239 | 4.1664 | 2641 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 7 | WORK.ANA_DATA | -39.9426 | 3.6183 | 2662 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 7 | WORK.ANA_DATA | -55.4097 | 3.1974 | 5656 |
| TRTPN (ATPTN) | 2 | 1 | 3 | 7 | WORK.ANA_DATA | -52.4494 | 4.1702 | 2648 |
| TRTPN (ATPTN) | 2 | 1 | 1 | 8 | WORK.ANA_DATA | 2.8278 | 3.6229 | 2672 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 8 | WORK.ANA_DATA | -7.1146 | 3.2079 | 5658 |
| TRTPN (ATPTN) | 2 | 1 | 3<br>1 | 8<br>9 | WORK.ANA_DATA | -22.9760 | 4.1815 | 2669 |
| TRTPN (ATPTN) | 2 | 1 | 2 | 9 | WORK.ANA_DATA | 6.9940 | 3.6105 | 2646 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 1 | 3 | 9 | WORK.ANA_DATA<br>WORK.ANA DATA | 3.4708<br>-21.9630 | 3.1711<br>4.1739 | 5649<br>2655 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 2 | WORK.ANA DATA | -35.0753 | 3.6039 | 2646 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 2 | WORK.ANA DATA | -50.5103 | 4.1826 | 2669 |
| TRTPN (ATPTN) | 3 | i | 3 | 2 | WORK.ANA DATA | -58.1334 | 3.1721 | 5650 |
| TRTPN (ATPTN) | 3 | ī | 1 | 3 | WORK.ANA DATA | 11.8625 | 3.6072 | 2653 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 3 | WORK.ANA DATA | -1.8278 | 4.1788 | 2662 |
| TRTPN (ATPTN) | 3 | ī | 3 | 3 | WORK.ANA DATA | -13.4872 | 3.1623 | 5649 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 4 | WORK.ANA DATA | -33.5112 | 3.6061 | 2650 |
| TRTPN (ATPTN) | 3 | ī | 2 | 4 | WORK.ANA DATA | -57.4339 | 4.1827 | 2669 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 4 | WORK.ANA DATA | -49.5032 | 3.1671 | 5650 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 5 | WORK.ANA DATA | 9.8483 | 3.6050 | 2648 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 5 | WORK.ANA DATA | -6.5867 | 4.1709 | 2648 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 5 | WORK.ANA_DATA | -12.7897 | 3.1623 | 5649 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 6 | WORK.ANA_DATA | -39.3629 | 3.6082 | 2655 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 6 | WORK.ANA_DATA | -58.4694 | 4.1709 | 2648 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 6 | WORK.ANA_DATA | -48.3347 | 3.1623 | 5649 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 7 | WORK.ANA_DATA | -16.9535 | 3.6116 | 2662 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 260 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | | | | | -27.73 -23.72 -21.66 -8.38 -9.74 -11.49 -30.29 -24.10 -21.36 -20.25 -16.80 -16.10 -1.23 -3.50 -7.90 0.62 -0.59 -7.64 -5.52 -16.08 -23.02 -19.44 -3.08 -7.79 -8.75 -15.64 -25.19 -17.38 -3.64 -9.31 -8.59 -17.25 -25.64 -17.12 -11.04 -17.33 -12.58 0.78 -2.22 -5.49 1.94 1.09 -5.26 -9.73 -12.08 -18.33 -2.22 -5.49 1.94 -1.09 -5.26 -9.73 -12.08 -18.33 -12.58 -15.63 -15.63 -15.63 | Pr > t <.0001 | Alpha 0.05 0.05 0.05 0.05 0.05 0.05 0.05 0. |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 3<br>3<br>3<br>3 | 1<br>1<br>1<br>1 | 2<br>3<br>1<br>2<br>3 | 5<br>5<br>6<br>6 | -1.58<br>-4.04<br>-10.91<br>-14.02<br>-15.28 | 0.1144<br><.0001<br><.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05<br>0.05<br>0.05 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 7 | -4.69 | <.0001 | 0.05 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 261 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| Differences of heast squares means | | | | | | |
|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
| TRTPN (ATPTN) | 1<br>1 | 1<br>1 | 1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>3 | 4<br>4<br>4<br>4<br>5<br>5<br>5<br>5<br>6<br>6<br>6<br>6<br>7<br>7<br>7<br>8<br>8<br>8<br>8<br>9<br>9<br>9<br>9<br>1<br>2<br>2<br>2<br>2<br>2<br>2<br>3<br>3<br>3<br>4 | -66.5063<br>-93.1492<br>-85.1767<br>-23.1432<br>-42.2752<br>-48.4548<br>-72.3647<br>-94.1579<br>-83.9999<br>-49.9658<br>-68.1443<br>-65.1338<br>-7.2099<br>-19.8673<br>-35.6861<br>-3.0045<br>-9.2185<br>-34.6559<br>-31.1590<br>-65.1444<br>-79.7577<br>-89.3070<br>-18.2132<br>-31.0654<br>-44.6462<br>-63.5847<br>-86.6816<br>-80.6694 | -57.7224 -78.9249 -71.0359 -14.3663 -28.1044 -34.3307 -63.5673 -79.9871 -69.8758 -41.1473 -53.9031 -50.9929 1.6376 -5.5898 -21.4938 5.7645 4.9322 -20.4980 -14.8193 -50.9844 -67.2412 -72.9380 -4.0402 -18.5684 -28.3065 -49.4161 -74.1645 -64.3152 |
| TRTPN (ATPTN) | 2<br>2 | 1<br>1 | 3<br>1<br>2<br>3<br>3<br>2<br>3<br>3<br>2<br>3<br>3<br>2<br>3<br>3<br>2<br>3<br>2 | <sup>4</sup> 5 5 5 6 6 6 6 7 7 7 8 8 8 8 9 9 9 9 | -80.6694<br>-20.2230<br>-35.8040<br>-43.9487<br>-69.4405<br>-87.6867<br>-79.4937<br>-47.0376<br>-61.6779<br>-60.6265<br>-4.2762<br>-13.4034<br>-31.1753<br>-0.08570<br>-2.7459<br>-30.1475 | -64.3152<br>-6.0587<br>-23.3477<br>-27.6090<br>-55.2636<br>-75.2304<br>-63.1541<br>-32.8476<br>-49.1415<br>-44.2723<br>9.9319<br>-0.8258<br>-14.7766<br>14.0736<br>9.6875<br>-13.7785 |
| TRTPN (ATPTN) | 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 | 1<br>1 | 1<br>2<br>3<br>1<br>1<br>1<br>2<br>3<br>1<br>1<br>1<br>2<br>3<br>1<br>1<br>1<br>1 | 2<br>2<br>2<br>3<br>3<br>3<br>4<br>4<br>4<br>4<br>5<br>5<br>5<br>6<br>6<br>6<br>6<br>7 | -42.1420<br>-58.7118<br>-64.3520<br>4.7892<br>-10.0218<br>-19.6865<br>-40.5823<br>-65.6356<br>-55.7120<br>2.7795<br>-14.7653<br>-18.9889<br>-46.4381<br>-66.6479<br>-54.5340<br>-24.0353 | -28.0085<br>-42.3088<br>-51.9148<br>18.9357<br>6.3663<br>-7.2880<br>-26.4402<br>-49.2322<br>-43.2944<br>16.9172<br>1.5918<br>-6.5904<br>-32.2877<br>-50.2908<br>-42.1355<br>-9.8717 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 262 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| | | DILL | CICHCCD OI | nearc bquar | es neams | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
| TRTPN (ATPTN) | 3 | 1 | 2 | 7 | WORK.ANA DATA | -32.4206 | 4.1865 | 2676 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 7 | WORK.ANA DATA | -29.4602 | 3.1672 | 5650 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 8 | WORK.ANA DATA | 25.8170 | 3.6162 | 2672 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 8 | WORK.ANA DATA | 15.8746 | 4.1945 | 2691 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 8 | WORK.ANA DATA | 0.01317 | 3.1821 | 5651 |
| TRTPN (ATPTN) | 3 | 1 | 1 | 9 | WORK.ANA DATA | 29.9831 | 3.6037 | 2646 |
| TRTPN (ATPTN) | 3 | 1 | 2 | 9 | WORK.ANA DATA | 26.4599 | 4.1664 | 2641 |
| TRTPN (ATPTN) | 3 | 1 | 3 | 9 | WORK.ANA DATA | 1.0262 | 3.1721 | 5650 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 2 | WORK.ANA DATA | -15.4350 | 3.6293 | 2683 |
| TRTPN (ATPTN) | 1 | 2 2 | 3 | 2 | WORK.ANA DATA | -23.0581 | 3.6125 | 2664 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 3 | WORK.ANA DATA | 46.9377 | 2.2445 | 5650 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 3 | WORK.ANA DATA | 33.2475 | 3.6249 | 2673 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 3 | WORK.ANA DATA | 21.5880 | 3.6039 | 2646 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 4 | WORK.ANA DATA | 1.5640 | 2.2427 | 5650 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 4 | WORK.ANA DATA | -22.3586 | 3.6294 | 2683 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 4 | WORK.ANA DATA | -14.4279 | 3.6082 | 2655 |
| TRTPN (ATPTN) | 1 | 2 2 | 1 | 5 | WORK.ANA DATA | 44.9236 | 2.2415 | 5651 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 5 | WORK.ANA DATA | 28.4885 | 3.6158 | 2654 |
| TRTPN (ATPTN) | 1 | 2 2 | 3 | 5 | WORK.ANA DATA | 22.2856 | 3.6039 | 2646 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 6 | WORK.ANA_DATA | -4.2876 | 2.2467 | 5652 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 6 | WORK.ANA_DATA | -23.3941 | 3.6158 | 2654 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 6 | WORK.ANA_DATA | -13.2595 | 3.6039 | 2646 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 7 | WORK.ANA_DATA | 18.1218 | 2.2521 | 5653 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 7 | WORK.ANA_DATA | 2.6547 | 3.6338 | 2693 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 7 | WORK.ANA_DATA | 5.6150 | 3.6082 | 2655 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 8 | WORK.ANA_DATA | 60.8922 | 2.2589 | 5653 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 8 | WORK.ANA_DATA | 50.9498 | 3.6430 | 2712 |
| TRTPN (ATPTN) | 1 | 2 | 3 | 8 | WORK.ANA_DATA | 35.0884 | 3.6213 | 2683 |
| TRTPN (ATPTN) | 1 | 2 | 1 | 9 | WORK.ANA_DATA | 65.0584 | 2.2398 | 5651 |
| TRTPN (ATPTN) | 1 | 2 | 2 | 9 | WORK.ANA_DATA | 61.5352 | 3.6107 | 2645 |
| TRTPN (ATPTN) | 1 2 | 2 2 | 3 | 9 | WORK.ANA_DATA | 36.1014 | 3.6125 | 2664 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 2 | WORK.ANA_DATA | -7.6231<br>62.3728 | 4.1902<br>3.6326 | 2683<br>2690 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 3 | WORK.ANA_DATA | 48.6825 | 3.2044 | 5652 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 2 | 3 | 3 | WORK.ANA_DATA<br>WORK.ANA DATA | 37.0231 | 4.1826 | 2669 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 4 | WORK.ANA DATA | 16.9991 | 3.6315 | 2688 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 4 | WORK.ANA DATA | -6.9236 | 3.2096 | 5652 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 4 | WORK.ANA DATA | 1.0071 | 4.1863 | 2676 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 5 | WORK.ANA DATA | 60.3586 | 3.6304 | 2685 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 5 | WORK.ANA DATA | 43.9236 | 3.1955 | 5651 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 5 | WORK.ANA DATA | 37.7206 | 4.1826 | 2669 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 6 | WORK.ANA DATA | 11.1474 | 3.6336 | 2692 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 6 | WORK.ANA DATA | -7.9591 | 3.1955 | 5651 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 6 | WORK.ANA DATA | 2.1756 | 4.1826 | 2669 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 7 | WORK.ANA DATA | 33.5568 | 3.6369 | 2699 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 7 | WORK.ANA DATA | 18.0897 | 3.2148 | 5653 |
| TRTPN (ATPTN) | 2 | 2 2 | 3 | 7 | WORK.ANA_DATA | 21.0501 | 4.1863 | 2676 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 8 | WORK.ANA_DATA | 76.3273 | 3.6415 | 2709 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 8 | WORK.ANA_DATA | 66.3849 | 3.2250 | 5654 |
| TRTPN (ATPTN) | 2 | 2 2 | 3 | 8 | WORK.ANA_DATA | 50.5235 | 4.1976 | 2697 |
| TRTPN (ATPTN) | 2 | 2 | 1 | 9 | WORK.ANA_DATA | 80.4934 | 3.6291 | 2683 |
| TRTPN (ATPTN) | 2 | 2 | 2 | 9 | WORK.ANA_DATA | 76.9702 | 3.1924 | 5656 |
| TRTPN (ATPTN) | 2 | 2 | 3 | 9 | WORK.ANA_DATA | 51.5365 | 4.1901 | 2683 |
| TRTPN (ATPTN) | 3 | 2 2 | 1 | 3 | WORK.ANA_DATA | 69.9958 | 3.6158 | 2671 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 3 | WORK.ANA_DATA | 56.3056 | 4.1863 | 2676 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 3 | WORK.ANA_DATA | 44.6462 | 3.1721 | 5650 |
| TRTPN (ATPTN) | 3 | 2 2 | 2 | 4 | WORK.ANA_DATA | 24.6221<br>0.6995 | 3.6147<br>4.1902 | 2669<br>2683 |
| TRTPN (ATPTN)<br>TRTPN (ATPTN) | 3 | 2 | 3 | 4 | WORK.ANA_DATA<br>WORK.ANA DATA | 8.6302 | 3.1770 | 2683<br>5651 |
| TIVIEIN (WILIN) | J | 4 | J | 7 | MOIVIL' AINA DATA | 0.0302 | J.1// | JUJI |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 263 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | | | | | TValue -7.74 -9.30 -7.14 3.78 0.00 8.32 6.35 0.32 -4.25 -6.38 20.91 9.17 5.99 0.70 -6.16 -4.00 20.04 7.88 6.18 -1.91 -6.47 -3.68 8.05 0.73 1.56 26.96 13.99 9.69 29.05 17.04 9.99 -1.82 17.17 15.19 8.85 4.68 -2.16 0.24 16.63 13.75 9.02 3.07 -2.49 0.52 9.23 5.63 5.03 20.96 20.58 12.04 22.18 24.11 12.30 | Pr > t <.0001 <.0001 <.0001 <.0001 0.0002 0.9967 <.0001 | Alpha 0.05 0.05 0.05 0.05 0.05 0.05 0.05 0. |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 3<br>3<br>3<br>3<br>3<br>3 | 2<br>2<br>2<br>2<br>2<br>2 | 1<br>2<br>3<br>1<br>2 | 3<br>3<br>3<br>4<br>4<br>4 | 19.36<br>13.45<br>14.07<br>6.81<br>0.17<br>2.72 | <.0001<br><.0001<br><.0001<br><.0001<br><.0001<br>0.8674<br>0.0066 | 0.05<br>0.05<br>0.05<br>0.05<br>0.05<br>0.05 |
| TIVILIA (WILIN) | J | ۷ | 5 | 4 | 2.12 | 0.0000 | 0.03 |
| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 264 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| | D-1 | IICICIICCO O | I Deade bqu | arco neano | | |
|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
| TRTPN (ATPTN) | 01 (N) 3 3 3 3 3 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | (N) 1 1 1 1 1 1 1 1 1 1 2 2 2 2 2 2 2 2 2 2 | | (N) 77788889999223334444555566667777888899992333444455556666777788889999 | -40.6297 -35.6691 18.7262 7.6498 -6.2249 22.9167 18.2901 -5.1924 -22.5516 -30.1418 42.5376 26.1395 14.5213 -2.8325 -29.4754 -21.5030 421.3985 15.2188 -8.6921 -30.4842 -20.3262 13.7068 -4.4706 -1.4601 56.4639 43.8065 27.9876 60.6675 54.4552 29.178 -15.8394 55.2498 42.4006 28.8216 9.8783 -13.2156 -7.2016 53.2400 37.6592 29.5191 4.0225 -14.2235 -6.0259 26.4254 11.7875 12.8413 69.1869 60.0627 42.2926 73.3773 70.7120 43.3204 | -24.2115 -23.2514 32.9078 24.0994 6.2513 37.0495 34.6298 7.2447 -8.3185 -15.9745 51.3378 40.3554 28.6548 5.9606 -15.2419 -7.3528 49.3178 35.5786 29.3523 0.1168 -16.3041 -6.1928 22.5368 29.7799 12.6902 65.3206 58.0322 69.4493 68.6152 43.1851 0.5932 69.4493 68.6152 43.1851 0.5932 69.4957 54.9645 44.1198 -0.6316 9.2158 67.4773 50.1880 45.2246 24.1198 -0.6316 9.2158 67.4773 50.1880 45.2246 24.1198 -0.6316 9.2158 67.4773 50.1880 45.2246 24.1198 -0.6316 9.2158 67.4773 50.1880 45.2246 24.1198 -0.6316 9.2158 67.4773 50.1880 45.2246 24.1798 -0.6316 9.2158 67.4773 50.1880 45.2246 58.7544 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 2 2 | 2 | 3 | 62.9057<br>48.0969 | 77.0860<br>64.5143 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 3 | 38.4276 | 50.8647 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 4 | 17.5342 | 31.7101 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 4 | -7.5169 | 8.9158 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 4 | 2.4021 | 14.8583 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 265 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| | | DILL | CICHCCD OI | nearc bquar | es means | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
| TRTPN (ATPTN) | 3 | 2 | 1 | 5 | WORK.ANA DATA | 67.9817 | 3.6136 | 2667 |
| | 3 | 2 | 2 | 5 | | 51.5467 | 4.1784 | 2662 |
| TRTPN (ATPTN) | | 2 | 3 | 5 | WORK.ANA_DATA | | | 5650 |
| TRTPN (ATPTN) | 3 | | 1 | | WORK.ANA_DATA | 45.3437 | 3.1721 | |
| TRTPN (ATPTN) | 3 | 2 | 2 | 6<br>6 | WORK.ANA_DATA | 18.7705 | 3.6169<br>4.1784 | 2674<br>2662 |
| TRTPN (ATPTN) | | 2 | | | WORK.ANA_DATA | -0.3360 | | |
| TRTPN (ATPTN) | 3 | 2 | 3 | 6 | WORK.ANA_DATA | 9.7986 | 3.1721 | 5650 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 7 | WORK.ANA_DATA | 41.1799 | 3.6202 | 2681 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 7<br>7 | WORK.ANA DATA | 25.7128 | 4.1939 | 2690 |
| TRTPN (ATPTN) | 3 | 2 2 | | | WORK.ANA_DATA | 28.6731 | 3.1770 | 5651 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 8 | WORK.ANA_DATA | 83.9504 | 3.6248 | 2690 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 8 | WORK.ANA_DATA | 74.0080 | 4.2020 | 2705 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 8 | WORK.ANA_DATA | 58.1466 | 3.1919 | 5652 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 9 | WORK.ANA_DATA | 88.1165 | 3.6124 | 2664 |
| TRTPN (ATPTN) | 3 | 2 2 | 2 | 9 | WORK.ANA_DATA | 84.5933 | 4.1739 | 2655 |
| TRTPN (ATPTN) | | 3 | 2 | | WORK.ANA_DATA | 59.1595 | 3.1820 | 5651 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 3 | WORK.ANA_DATA | -13.6902 | 3.6283 | 2680 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 4 | WORK.ANA_DATA | -25.3497<br>-45.3737 | 3.6072<br>2.2477 | 2653<br>5650 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 3 | 2 | 4 | WORK.ANA_DATA | -69.2964 | 3.6327 | 2690 |
| TRTPN (ATPTN) | 1 | 3 | 2 3 | 4 | WORK.ANA_DATA | -61.3656 | 3.6115 | 2662 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 5 | WORK.ANA_DATA<br>WORK.ANA DATA | -2.0141 | 2.2463 | 5651 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 5 | WORK.ANA DATA | -18.4492 | 3.6191 | 2661 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 5 | WORK.ANA DATA | -24.6521 | 3.6072 | 2653 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 6 | WORK.ANA DATA | -51.2254 | 2.2521 | 5653 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 6 | WORK.ANA DATA | -70.3318 | 3.6191 | 2661 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 6 | WORK.ANA DATA | -60.1972 | 3.6072 | 2653 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 7 | WORK.ANA DATA | -28.8159 | 2.2569 | 5653 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 7 | WORK.ANA DATA | -44.2830 | 3.6371 | 2700 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 7 | WORK.ANA DATA | -41.3227 | 3.6115 | 2662 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 8 | WORK.ANA DATA | 13.9545 | 2.2637 | 5653 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 8 | WORK.ANA DATA | 4.0121 | 3.6463 | 2719 |
| TRTPN (ATPTN) | ī | 3 | 3 | 8 | WORK.ANA DATA | -11.8493 | 3.6246 | 2690 |
| TRTPN (ATPTN) | ī | 3 | 1 | 9 | WORK.ANA DATA | 18.1207 | 2.2451 | 5653 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 9 | WORK.ANA DATA | 14.5975 | 3.6140 | 2652 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 9 | WORK.ANA DATA | -10.8363 | 3.6158 | 2671 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 3 | WORK.ANA DATA | -11.6594 | 4.1788 | 2662 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 4 | WORK.ANA DATA | -31.6834 | 3.6271 | 2678 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 4 | WORK.ANA DATA | -55.6061 | 3.2032 | 5650 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 4 | WORK.ANA DATA | -47.6754 | 4.1825 | 2669 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 5 | WORK.ANA DATA | 11.6761 | 3.6260 | 2676 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 5 | WORK.ANA DATA | -4.7589 | 3.1905 | 5651 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 5 | WORK.ANA DATA | -10.9619 | 4.1788 | 2662 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 6 | WORK.ANA_DATA | -37.5351 | 3.6292 | 2683 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 6 | WORK.ANA_DATA | -56.6416 | 3.1905 | 5651 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 6 | WORK.ANA DATA | -46.5070 | 4.1788 | 2662 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 7 | WORK.ANA_DATA | -15.1257 | 3.6326 | 2690 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 7 | WORK.ANA_DATA | -30.5928 | 3.2095 | 5652 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 7 | WORK.ANA_DATA | -27.6324 | 4.1825 | 2669 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 8 | WORK.ANA_DATA | 27.6448 | 3.6371 | 2699 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 8 | WORK.ANA_DATA | 17.7024 | 3.2186 | 5651 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 8 | WORK.ANA_DATA | 1.8410 | 4.1938 | 2690 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 9 | WORK.ANA_DATA | 31.8109 | 3.6248 | 2673 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 9 | WORK.ANA_DATA | 28.2877 | 3.1874 | 5656 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 9 | WORK.ANA_DATA | 2.8540 | 4.1863 | 2676 |
| TRTPN (ATPTN) | 3 | 3 | 1 | 4 | WORK.ANA_DATA | -20.0240 | 3.6061 | 2650 |
| TRTPN (ATPTN) | 3 | 3 | 2 | 4 | WORK.ANA_DATA | -43.9467 | 4.1827 | 2669 |
| TRTPN (ATPTN) | 3 | 3 | 3 | 4 | WORK.ANA_DATA | -36.0160 | 3.1671 | 5650 |
| TRTPN (ATPTN) | 3 | 3 | 1 | 5 | WORK.ANA_DATA | 23.3356 | 3.6050 | 2648 |
| TRTPN (ATPTN) | 3 | 3 | 2 | 5 | WORK.ANA_DATA | 6.9005 | 4.1709 | 2648 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 266 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| | | DILIEIGUC | es or heast | oquares Me | allo | | |
|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
| TRTPN (ATPTN) | 3 3 3 3 3 3 3 3 3 3 3 3 3 3 1 1 1 1 1 1 | 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 | 1<br>2<br>3<br>3<br>1<br>2<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>3<br>3<br>3 | 555666677778888999933444455556666777788889999344445 | 18.81 12.34 14.29 5.19 -0.08 3.09 11.38 6.13 9.03 23.16 17.61 18.22 24.39 20.27 18.59 -3.77 -7.03 -20.19 -19.08 -16.99 -0.90 -5.10 -6.83 -22.75 -19.43 -16.69 -12.77 -12.18 -11.44 6.16 1.10 -3.27 8.07 4.04 -3.00 -2.79 -8.74 -17.36 -11.40 3.22 | <.0001 <.0001 <.0001 <.0001 0.9359 0.0020 <.0001 | 0.05 |
| TRTPN (ATPTN) | 2<br>2 | 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 | 2<br>3<br>1<br>2<br>2<br>3<br>3<br>1<br>2<br>2<br>3<br>3<br>1<br>2<br>2<br>3<br>3<br>1<br>2<br>2<br>3<br>3<br>1<br>2<br>2<br>3<br>3<br>3<br>1<br>2<br>3<br>1<br>2<br>2<br>3<br>2<br>3 | 5<br>5<br>6<br>6<br>6<br>7<br>7<br>7<br>8<br>8<br>8<br>8<br>9<br>9<br>9<br>4<br>4<br>4<br>4<br>5<br>5<br>5<br>5 | -1.49 -2.62 -10.34 -17.75 -11.13 -4.16 -9.53 -6.61 7.60 5.50 0.44 8.78 8.87 0.68 -5.55 -10.51 -11.37 6.47 1.65 | 0.1359<br>0.0088<br><.0001<br>0.6607<br><.0001<br><.0001<br><.0001<br><.0001<br><.0001<br><.0001<br><.0001 | 0.05 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 267 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

Differences of Least Squares Means

| | | .IICICIICCO C | or neare by | arco neano | | |
|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
| TRTPN (ATPTN) | 3 | 2 | 1 | 5 | 60.8959 | 75.0675 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 5 | 43.3535 | 59.7399 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 5 | 39.1251 | 51.5623 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 6 | 11.6784 | 25.8626 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 6 | -8.5292 | 7.8572 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 6 | 3.5801 | 16.0172 |
| TRTPN (ATPTN) | 3 | 2 | ĺ | 7 | 34.0812 | 48.2786 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 7 | 17.4891 | 33.9365 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 7 | 22.4450 | 34.9013 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 8 | 76.8427 | 91.0580 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 8 | 65.7686 | 82.2473 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 8 | 51.8892 | 64.4039 |
| TRTPN (ATPTN) | 3 | 2 | 1 | 9 | 81.0332 | 95.1998 |
| TRTPN (ATPTN) | 3 | 2 | 2 | 9 | 76.4088 | 92.7778 |
| TRTPN (ATPTN) | 3 | 2 | 3 | 9 | 52.9217 | 65.3974 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 3 | -20.8047 | -6.5758 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 3 | -32.4229 | -18.2765 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 4 | -49.7800 | -40.9674 |
| TRTPN (ATPTN) | 1 | 3 | 2 3 | 4 | -76.4196 | -62.1731 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 4<br>5 | -68.4472<br>-6.4178 | -54.2840 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 3 | 2 | 5 | -25.5457 | 2.3896<br>-11.3526 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 5 | -31.7254 | -17.5789 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 6 | -55.6402 | -46.8105 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 6 | -77.4284 | -63.2353 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 6 | -67.2704 | -53.1240 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 7 | -33.2404 | -24.3914 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 7 | -51.4147 | -37.1513 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 7 | -48.4043 | -34.2411 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 8 | 9.5168 | 18.3923 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 8 | -3.1377 | 11.1619 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 8 | -18.9565 | -4.7420 |
| TRTPN (ATPTN) | 1 | 3 | 1 | 9 | 13.7193 | 22.5220 |
| TRTPN (ATPTN) | 1 | 3 | 2 | 9 | 7.5110 | 21.6840 |
| TRTPN (ATPTN) | 1 | 3 | 3 | 9 | -17.9264 | -3.7462 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 3 | -19.8535 | -3.4653 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 4 | -38.7957 | -24.5712 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 4 | -61.8856 | -49.3266 |
| TRTPN (ATPTN) | 2 2 | 3 | 3<br>1 | 4<br>5 | -55.8767 | -39.4741 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 3 | 2 | 5 | 4.5661<br>-11.0136 | 18.7862<br>1.4957 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 5 | -19.1560 | -2.7678 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 6 | -44.6515 | -30.4187 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 6 | -62.8963 | -50.3869 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 6 | -54.7010 | -38.3129 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 7 | -22.2486 | -8.0028 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 7 | -36.8847 | -24.3009 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 7 | -35.8338 | -19.4311 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 8 | 20.5129 | 34.7766 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 8 | 11.3927 | 24.0120 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 8 | -6.3825 | 10.0644 |
| TRTPN (ATPTN) | 2 | 3 | 1 | 9 | 24.7033 | 38.9185 |
| TRTPN (ATPTN) | 2 | 3 | 2 | 9 | 22.0392 | 34.5362 |
| TRTPN (ATPTN) | 2 | 3 | 3 | 9 | -5.3547 | 11.0626 |
| TRTPN (ATPTN) | 3 | 3 | 1 | 4 | -27.0951 | -12.9530 |
| TRTPN (ATPTN) | 3 | 3 | 2 | 4 | -52.1484 | -35.7450 |
| TRTPN (ATPTN) | 3 | 3 | 3<br>1 | 4<br>5 | -42.2248 | -29.8071 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 3 | 2 | 5<br>5 | 16.2667<br>-1.2781 | 30.4044<br>15.0791 |
| TMIEN (MIEIN) | J | J | ۷ | J | -1.2/01 | 10.0/91 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 268 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| | | DILL | erences or | neast squar | es means | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
| TRTPN (ATPTN) | 3 | 3 | 3 | 5 | WORK.ANA DATA | 0.6975 | 3.1623 | 5649 |
| TRTPN (ATPTN) | 3 | 3 | 1 | 6 | WORK.ANA DATA | -25.8757 | 3.6082 | 2655 |
| TRTPN (ATPTN) | 3 | 3 | 2 | 6 | WORK.ANA DATA | -44.9822 | 4.1709 | 2648 |
| TRTPN (ATPTN) | 3 | 3 | 3 | 6 | WORK.ANA DATA | -34.8475 | 3.1623 | 5649 |
| TRTPN (ATPTN) | 3 | 3 | 1 | 7 | WORK.ANA DATA | -3.4662 | 3.6116 | 2662 |
| TRTPN (ATPTN) | 3 | 3 | 2 | 7 | WORK.ANA DATA | -18.9334 | 4.1865 | 2676 |
| TRTPN (ATPTN) | 3 | 3 | 3 | 7 | WORK.ANA DATA | -15.9730 | 3.1672 | 5650 |
| TRTPN (ATPTN) | 3 | 3 | 1 | 8 | WORK.ANA DATA | 39.3042 | 3.6162 | 2672 |
| TRTPN (ATPTN) | 3 | 3 | 2 | 8 | WORK.ANA DATA | 29.3618 | 4.1945 | 2691 |
| TRTPN (ATPTN) | 3 | 3 | 3 | 8 | WORK.ANA DATA | 13.5004 | 3.1821 | 5651 |
| TRTPN (ATPTN) | 3 | 3 | 1 | 9 | WORK.ANA DATA | 43.4703 | 3.6037 | 2646 |
| TRTPN (ATPTN) | 3 | 3 | 2 | 9 | WORK.ANA DATA | 39.9472 | 4.1664 | 2641 |
| TRTPN (ATPTN) | 3 | 3 | 3 | 9 | WORK.ANA_DATA | 14.5134 | 3.1721 | 5650 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 4 | WORK.ANA_DATA | -23.9227 | 3.6317 | 2688 |
| TRTPN (ATPTN) | 1 | 4 | 3 | 4 | WORK.ANA_DATA | -15.9919 | 3.6104 | 2659 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 5 | WORK.ANA_DATA | 43.3596 | 2.2451 | 5652 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 5 | WORK.ANA_DATA | 26.9245 | 3.6180 | 2659 |
| TRTPN (ATPTN) | 1 | 4 | 3 | 5 | WORK.ANA_DATA | 20.7216 | 3.6061 | 2650 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 6 | WORK.ANA_DATA | -5.8517 | 2.2498 | 5652 |
| TRTPN (ATPTN) | 1 | 4 | 2 3 | 6<br>6 | WORK.ANA_DATA | -24.9581 | 3.6180 | 2659 |
| TRTPN (ATPTN) | 1 | 4<br>4 | 1 | 7 | WORK.ANA_DATA<br>WORK.ANA DATA | -14.8235<br>16.5578 | 3.6061<br>2.2557 | 2650<br>5654 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 4 | 2 | 7 | WORK.ANA DATA | 1.0907 | 3.6359 | 2697 |
| TRTPN (ATPTN) | 1 | 4 | 3 | 7 | WORK.ANA DATA | 4.0510 | 3.6104 | 2660 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 8 | WORK.ANA DATA | 59.3282 | 2.2620 | 5653 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 8 | WORK.ANA DATA | 49.3858 | 3.6452 | 2717 |
| TRTPN (ATPTN) | 1 | 4 | 3 | 8 | WORK.ANA DATA | 33.5244 | 3.6235 | 2688 |
| TRTPN (ATPTN) | 1 | 4 | 1 | 9 | WORK.ANA DATA | 63.4943 | 2.2434 | 5652 |
| TRTPN (ATPTN) | 1 | 4 | 2 | 9 | WORK.ANA DATA | 59.9712 | 3.6129 | 2650 |
| TRTPN (ATPTN) | 1 | 4 | 3 | 9 | WORK.ANA DATA | 34.5374 | 3.6147 | 2669 |
| TRTPN (ATPTN) | 2 | 4 | 3 | 4 | WORK.ANA DATA | 7.9307 | 4.1864 | 2676 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 5 | WORK.ANA_DATA | 67.2822 | 3.6305 | 2685 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 5 | WORK.ANA_DATA | 50.8472 | 3.1957 | 5652 |
| TRTPN (ATPTN) | 2 | 4 | 3 | 5 | WORK.ANA_DATA | 44.6442 | 4.1827 | 2669 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 6 | WORK.ANA_DATA | 18.0710 | 3.6337 | 2692 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 6 | WORK.ANA_DATA | -1.0355 | 3.1957 | 5652 |
| TRTPN (ATPTN) | 2 | 4 | 3 | 6 | WORK.ANA_DATA | 9.0992 | 4.1827 | 2669 |
| TRTPN (ATPTN) | 2 | 4 | 1 2 | 7<br>7 | WORK.ANA_DATA | 40.4804 | 3.6371 | 2699 |
| TRTPN (ATPTN)<br>TRTPN (ATPTN) | 2 | 4 | 3 | 7 | WORK.ANA DATA<br>WORK.ANA DATA | 25.0133<br>27.9737 | 3.2146<br>4.1864 | 5653<br>2676 |
| TRTPN (ATPTN) | 2 | 4 | 1 | 8 | WORK.ANA DATA | 83.2509 | 3.6417 | 2709 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 8 | WORK.ANA DATA | 73.3085 | 3.2237 | 5652 |
| TRTPN (ATPTN) | 2 | 4 | 3 | 8 | WORK.ANA DATA | 57.4471 | 4.1977 | 2697 |
| TRTPN (ATPTN) | 2 | 4 | ĺ | 9 | WORK.ANA DATA | 87.4170 | 3.6293 | 2683 |
| TRTPN (ATPTN) | 2 | 4 | 2 | 9 | WORK.ANA DATA | 83.8938 | 3.1925 | 5656 |
| TRTPN (ATPTN) | 2 | 4 | 3 | 9 | WORK.ANA DATA | 58.4601 | 4.1902 | 2683 |
| TRTPN (ATPTN) | 3 | 4 | 1 | 5 | WORK.ANA DATA | 59.3515 | 3.6093 | 2657 |
| TRTPN (ATPTN) | 3 | 4 | 2 | 5 | WORK.ANA DATA | 42.9165 | 4.1746 | 2655 |
| TRTPN (ATPTN) | 3 | 4 | 3 | 5 | WORK.ANA_DATA | 36.7135 | 3.1671 | 5650 |
| TRTPN (ATPTN) | 3 | 4 | 1 | 6 | WORK.ANA_DATA | 10.1403 | 3.6125 | 2664 |
| TRTPN (ATPTN) | 3 | 4 | 2 | 6 | WORK.ANA_DATA | -8.9662 | 4.1746 | 2655 |
| TRTPN (ATPTN) | 3 | 4 | 3 | 6 | WORK.ANA_DATA | 1.1684 | 3.1671 | 5650 |
| TRTPN (ATPTN) | 3 | 4 | 1 | 7 | WORK.ANA_DATA | 32.5497 | 3.6159 | 2671 |
| TRTPN (ATPTN) | 3 | 4 | 2 | 7 | WORK.ANA_DATA | 17.0826 | 4.1902 | 2683 |
| TRTPN (ATPTN) | 3 | 4 | 3 | 7 | WORK.ANA_DATA | 20.0429 | 3.1720 | 5650 |
| TRTPN (ATPTN) | 3 | 4 | 1 | 8 | WORK.ANA_DATA | 75.3202 | 3.6205 | 2681 |
| TRTPN (ATPTN) | 3 | 4 | 2 3 | 8 | WORK.ANA_DATA | 65.3778 | 4.1982 | 2698 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 4 | 3<br>1 | 9 | WORK.ANA_DATA<br>WORK.ANA DATA | 49.5164<br>79.4863 | 3.1870<br>3.6080 | 5652<br>2655 |
| TUTEN (WILIN) | 3 | 4 | _ | J | WORK.ANA_DATA | 12.4003 | 3.0000 | 2000 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 269 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | | | | | t Value 0.22 -7.17 -10.78 -11.02 -0.96 -4.52 -5.04 10.87 7.00 4.24 12.06 9.59 -4.43 19.31 7.44 5.75 -2.60 -6.90 -4.11 7.34 0.30 1.12 26.23 13.55 9.25 28.30 16.60 9.55 1.89 18.53 15.91 10.67 4.97 -0.32 2.18 11.13 7.78 6.68 22.84 13.69 24.09 26.28 13.95 16.44 10.28 11.59 2.81 -2.15 0.37 9.00 | Pr > t 0.8254 <.0001 | Alpha 0.05 0.05 0.05 0.05 0.05 0.05 0.05 0. |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 3<br>3<br>3<br>3<br>3 | 4<br>4<br>4<br>4 | 2<br>3<br>1<br>2<br>3 | 7<br>7<br>8<br>8<br>8 | 4.08<br>6.32<br>20.80<br>15.57<br>15.54 | <.0001<br><.0001<br><.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05<br>0.05<br>0.05 |
| TRTPN (ATPTN) | 3 | 4 | 1 | 9 | 22.03 | <.0001 | 0.05 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 270 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| | DI. | rierences o | I neast squ | ares means | | |
|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
| TRTPN (ATPTN) | 3<br>1<br>1<br>1<br>1<br>1<br>1 | (N) 3 3 3 3 3 3 3 3 3 3 4 4 4 4 4 4 4 4 4 | 01 (N) 3 1 2 3 1 1 2 3 1 | (N) 56666777888899944555566667777888899945555666677778888999 | -5.5017 -32.9509 -53.1607 -41.0468 -10.5480 -27.1424 -22.1819 32.2134 21.1370 7.2623 36.4039 31.7773 8.2948 -31.0438 -33.0714 38.9584 19.8302 13.6505 -10.2622 -32.0525 -21.8945 12.1358 -6.0389 -3.0285 54.8938 42.2382 26.4193 59.0965 52.8869 27.4494 -0.2782 60.1633 44.5824 36.4425 10.9458 -7.3002 0.8974 33.3487 18.7114 19.7647 76.1102 66.9888 49.2166 080.3006 77.6353 | 6.8968 -18.8005 -36.8036 -28.6483 3.6156 -10.7243 -9.7642 46.3950 37.5866 19.7385 50.5367 48.1170 20.7319 -16.8015 -8.9125 47.7607 34.0189 27.7926 -1.4411 -17.8638 -7.7525 20.9797 8.2202 11.1305 63.7626 56.5334 40.6295 67.8922 67.8925 41.6254 16.1396 74.4011 57.1119 52.8460 25.1962 57.2293 17.3009 47.6122 31.3153 36.1827 90.3916 79.6281 65.6782 94.5335 90.1524 |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 2 3 3 3 3 3 | 4<br>4<br>4<br>4<br>4 | 3<br>1<br>2<br>3<br>1<br>2 | 9<br>5<br>5<br>5<br>6<br>6 | 50.2438<br>52.2743<br>34.7307<br>30.5047<br>3.0567<br>-17.1520 | 66.6764<br>66.4288<br>51.1023<br>42.9223<br>17.2239<br>-0.7804 |
| TRTPN (ATPTN) | 3<br>3<br>3<br>3<br>3<br>3<br>3<br>3 | 4<br>4<br>4<br>4<br>4<br>4<br>4 | 3<br>1<br>2<br>3<br>1<br>2<br>3<br>1 | 6<br>7<br>7<br>8<br>8<br>8 | -5.0404<br>25.4596<br>8.8663<br>13.8245<br>68.2210<br>57.1457<br>43.2687<br>72.4115 | 7.3773 39.6399 25.2989 26.2614 82.4193 73.6098 55.7640 86.5611 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 271 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 3 | 4 | 2 | 9 | WORK.ANA DATA | 75.9631 | 4.1702 | 2648 |
| TRTPN (ATPTN) | 3 | 4 | 3 | 9 | WORK.ANA DATA | 50.5293 | 3.1770 | 5651 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 5 | WORK.ANA DATA | -16.4351 | 3.6169 | 2657 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 5 | WORK.ANA_DATA | -22.6380 | 3.6050 | 2648 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 6 | WORK.ANA_DATA | -49.2112 | 2.2480 | 5651 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 6 | WORK.ANA_DATA | -68.3177 | 3.6169 | 2657 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 6 | WORK.ANA_DATA | -58.1831 | 3.6050 | 2648 |
| TRTPN (ATPTN) | 1<br>1 | 5<br>5 | 1 2 | 7<br>7 | WORK.ANA_DATA<br>WORK.ANA DATA | -26.8018<br>-42.2689 | 2.2529<br>3.6348 | 5651<br>2695 |
| TRTPN (ATPTN)<br>TRTPN (ATPTN) | 1 | 5 | 3 | 7 | WORK.ANA_DATA | -39.3086 | 3.6093 | 2657 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 8 | WORK.ANA DATA | 15.9686 | 2.2603 | 5653 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 8 | WORK.ANA DATA | 6.0262 | 3.6441 | 2715 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 8 | WORK.ANA DATA | -9.8352 | 3.6224 | 2685 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 9 | WORK.ANA DATA | 20.1348 | 2.2422 | 5654 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 9 | WORK.ANA_DATA | 16.6116 | 3.6118 | 2648 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 9 | WORK.ANA_DATA | -8.8222 | 3.6136 | 2667 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 5 | WORK.ANA_DATA | -6.2030 | 4.1709 | 2648 |
| TRTPN (ATPTN) | 2 | 5<br>5 | 1 2 | 6 | WORK.ANA_DATA | -32.7762 | 3.6201 | 2664 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 5 | 3 | 6<br>6 | WORK.ANA_DATA<br>WORK.ANA DATA | -51.8827<br>-41.7480 | 3.1802<br>4.1709 | 5649<br>2648 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 7 | WORK.ANA DATA | -10.3667 | 3.6235 | 2671 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 7 | WORK.ANA DATA | -25.8338 | 3.2006 | 5652 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 7 | WORK.ANA DATA | -22.8735 | 4.1746 | 2655 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 8 | WORK.ANA_DATA | 32.4037 | 3.6280 | 2681 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 8 | WORK.ANA_DATA | 22.4613 | 3.2111 | 5654 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 8 | WORK.ANA_DATA | 6.5999 | 4.1860 | 2676 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 9 | WORK.ANA_DATA | 36.5698 | 3.6156 | 2655 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 5<br>5 | 2 | 9 | WORK.ANA_DATA<br>WORK.ANA DATA | 33.0467<br>7.6129 | 3.1770<br>4.1784 | 5653<br>2662 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 6 | WORK.ANA DATA | -26.5732 | 3.6082 | 2655 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 6 | WORK.ANA DATA | -45.6797 | 4.1709 | 2648 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 6 | WORK.ANA DATA | -35.5451 | 3.1623 | 5649 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 7 | WORK.ANA_DATA | -4.1638 | 3.6116 | 2662 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 7 | WORK.ANA_DATA | -19.6309 | 4.1865 | 2676 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 7 | WORK.ANA_DATA | -16.6706 | 3.1672 | 5650 |
| TRTPN (ATPTN) | 3 | 5<br>5 | 1 2 | 8 | WORK.ANA_DATA<br>WORK.ANA_DATA | 38.6067<br>28.6643 | 3.6162<br>4.1945 | 2672<br>2691 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 5 | 3 | 8 | WORK.ANA_DATA | 12.8029 | 3.1821 | 5651 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 9 | WORK.ANA DATA | 42.7728 | 3.6037 | 2646 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 9 | WORK.ANA DATA | 39.2496 | 4.1664 | 2641 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 9 | WORK.ANA DATA | 13.8158 | 3.1721 | 5650 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 6 | WORK.ANA DATA | -19.1065 | 3.6201 | 2664 |
| TRTPN (ATPTN) | 1 | 6 | 3 | 6 | WORK.ANA_DATA | -8.9718 | 3.6082 | 2655 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 7 | WORK.ANA_DATA | 22.4094 | 2.2586 | 5653 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 7 | WORK.ANA_DATA | 6.9423 | 3.6381 | 2702 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 6<br>6 | 3 | 7<br>8 | WORK.ANA_DATA<br>WORK.ANA DATA | 9.9027<br>65.1799 | 3.6125<br>2.2655 | 2664<br>5654 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 8 | WORK.ANA_DATA | 55.2375 | 3.6473 | 2722 |
| TRTPN (ATPTN) | 1 | 6 | 3 | 8 | WORK.ANA DATA | 39.3761 | 3.6256 | 2692 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 9 | WORK.ANA DATA | 69.3460 | 2.2474 | 5654 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 9 | WORK.ANA_DATA | 65.8228 | 3.6150 | 2655 |
| TRTPN (ATPTN) | 1 | 6 | 3 | 9 | WORK.ANA_DATA | 40.3891 | 3.6169 | 2674 |
| TRTPN (ATPTN) | 2 | 6 | 3 | 6 | WORK.ANA_DATA | 10.1346 | 4.1709 | 2648 |
| TRTPN (ATPTN) | 2 2 | 6<br>6 | 1 2 | 7<br>7 | WORK.ANA_DATA | 41.5159<br>26.0488 | 3.6235<br>3.2006 | 2671<br>5652 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 6 | 3 | 7 | WORK.ANA_DATA<br>WORK.ANA DATA | 29.0091 | 4.1746 | 2655 |
| TRIPN (AIPIN) | 2 | 6 | 1 | 8 | WORK.ANA_DATA | 84.2864 | 3.6280 | 2681 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 8 | WORK.ANA DATA | 74.3439 | 3.2111 | 5654 |
| TRTPN (ATPTN) | 2 | 6 | 3 | 8 | WORK.ANA_DATA | 58.4826 | 4.1860 | 2676 |
| | | | | | _ | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 272 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| | | DILLETENC | es or heast | squares Me | allo | | |
|---|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
| TRTPN (ATPTN) | 3 | 4 | 2 | 9 | 18.22 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 4 | 3 | 9 | 15.90 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 5 | -4.54 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 5 | -6.28 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 6 | -21.89 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 6 | -18.89 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5<br>5 | 3<br>1 | 6<br>7 | -16.14<br>-11.90 | <.0001<br><.0001 | 0.05<br>0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 5 | 2 | 7 | -11.63 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 7 | -10.89 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 8 | 7.06 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 8 | 1.65 | 0.0983 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 3 | 8 | -2.72 | 0.0067 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 1 | 9 | 8.98 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5 | 2 | 9 | 4.60 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 5<br>5 | 3 | 9<br>5 | -2.44<br>-1.49 | 0.0147 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 5 | 1 | 6 | -1.49<br>-9.05 | 0.1371<br><.0001 | 0.05<br>0.05 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 6 | -16.31 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 6 | -10.01 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 7 | -2.86 | 0.0043 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 7 | -8.07 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 7 | -5.48 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 1 | 8 | 8.93 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 5<br>5 | 2 | 8 | 6.99 | <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 5 | 1 | 9 | 1.58<br>10.11 | 0.1150<br><.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 2 | 9 | 10.40 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 5 | 3 | 9 | 1.82 | 0.0686 | 0.05 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 6 | -7.36 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 6 | -10.95 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 6 | -11.24 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 7 | -1.15 | 0.2491 | 0.05 |
| TRTPN (ATPTN) | 3 | 5<br>5 | 2 3 | 7<br>7 | -4.69<br>-5.26 | <.0001<br><.0001 | 0.05<br>0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 5 | 1 | 8 | 10.68 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 8 | 6.83 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 8 | 4.02 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 5 | 1 | 9 | 11.87 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 5 | 2 | 9 | 9.42 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 5 | 3 | 9 | 4.36 | <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 1 | 6<br>6 | 2 3 | 6<br>6 | -5.28<br>-2.49 | <.0001<br>0.0130 | 0.05<br>0.05 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 7 | 9.92 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 7 | 1.91 | 0.0565 | 0.05 |
| TRTPN (ATPTN) | 1 | 6 | 3 | 7 | 2.74 | 0.0062 | 0.05 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 8 | 28.77 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 6 | 2 | 8 | 15.14 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 6 | 3 | 8 | 10.86 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 6 | 1 | 9 | 30.86 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 6<br>6 | 2 3 | 9 | 18.21 | <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 6 | 3 | 6 | 11.17<br>2.43 | <.0001<br>0.0152 | 0.05<br>0.05 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 7 | 11.46 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 7 | 8.14 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 3 | 7 | 6.95 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 1 | 8 | 23.23 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 8 | 23.15 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 3 | 8 | 13.97 | <.0001 | 0.05 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 273 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

| | DI. | TICICIICCD O | I Leade bqu | arco neamo | | |
|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
| TRTPN (ATPTN) | 01 (N) 3 3 1 1 1 1 1 1 1 1 1 1 1 2 2 2 2 2 2 | (N) 4 4 5 5 5 5 5 5 5 5 5 5 5 5 5 5 5 5 5 | 01 (N) 2 3 2 3 1 2 | (N) 9955666777888899956667778888999966677788889999666777 | 67.7860 44.3012 -23.5272 -29.7069 -53.6182 -75.4099 -65.2520 -31.2183 -49.3963 -46.3859 11.5377 -1.1192 -16.9381 15.7393 9.5295 -15.9080 -14.3816 -39.8747 -58.1170 -49.9266 -17.4718 -32.1082 -31.0594 25.2897 16.1663 -1.6081 29.4801 26.8185 -0.5803 -33.6484 -53.8583 -41.7443 -53.8583 -41.7446 -27.8400 -22.8794 31.5159 20.4394 6.5648 35.7064 31.5159 20.4394 6.5648 35.7064 31.5798 7.5973 -26.2050 -16.0471 17.9818 -0.1913 | 84.1402<br>56.7575<br>-9.3429<br>-15.5691<br>-44.8043<br>-61.2255<br>-51.1142<br>-22.3853<br>-35.1415<br>-32.2313<br>20.3996<br>13.1717<br>-2.7322<br>24.5303<br>23.6937<br>-1.7364<br>1.9757<br>-25.6777<br>-45.6483<br>-33.5695<br>-14.6877<br>39.5177<br>28.7562<br>14.8079<br>43.6596<br>39.2748<br>15.8061<br>-19.4980<br>-37.5011<br>-29.3458<br>29.3458 |
| TRTPN (ATPTN) | 1<br>1<br>1<br>1<br>1<br>1<br>1<br>2 | 6<br>6<br>6<br>6<br>6<br>6<br>6<br>6 | 3<br>1<br>2<br>3<br>1<br>2<br>3<br>3 | 7<br>8<br>8<br>9<br>9<br>9 | 2.8190<br>60.7386<br>48.0857<br>32.2668<br>64.9403<br>58.7344<br>33.2969<br>1.9560 | 16.9863<br>69.6212<br>62.3892<br>46.4853<br>73.7517<br>72.9113<br>47.4812<br>18.3133 |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 2<br>2<br>2<br>2<br>2<br>2 | 6<br>6<br>6<br>6<br>6 | 1<br>2<br>3<br>1<br>2<br>3 | 7<br>7<br>7<br>8<br>8 | 34.4109<br>19.7744<br>20.8233<br>77.1723<br>68.0490<br>50.2745 | 48.6210<br>32.3232<br>37.1950<br>91.4004<br>80.6389<br>66.6906 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 274 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

#### Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Margins | Estimate | Standard<br>Error | DF |
|---|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 2 | 6 | 1 | 9 | WORK.ANA DATA | 88.4525 | 3.6156 | 2655 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 9 | WORK.ANA DATA | 84.9293 | 3.1770 | 5653 |
| TRTPN (ATPTN) | 2 | 6 | 3 | 9 | WORK.ANA DATA | 59.4955 | 4.1784 | 2662 |
| TRTPN (ATPTN) | 3 | 6 | 1 | 7 | WORK.ANA DATA | 31.3813 | 3.6116 | 2662 |
| TRTPN (ATPTN) | 3 | 6 | 2 | 7 | WORK.ANA DATA | 15.9142 | 4.1865 | 2676 |
| TRTPN (ATPTN) | 3 | 6 | 3 | 7 | WORK.ANA DATA | 18.8745 | 3.1672 | 5650 |
| TRTPN (ATPTN) | 3 | 6 | 1 | 8 | WORK.ANA DATA | 74.1517 | 3.6162 | 2672 |
| TRTPN (ATPTN) | 3 | 6 | 2 | 8 | WORK.ANA DATA | 64.2093 | 4.1945 | 2691 |
| TRTPN (ATPTN) | 3 | 6 | 3 | 8 | WORK.ANA DATA | 48.3479 | 3.1821 | 5651 |
| TRTPN (ATPTN) | 3 | 6 | 1 | 9 | WORK.ANA DATA | 78.3179 | 3.6037 | 2646 |
| | 3 | 6 | 2 | 9 | WORK.ANA DATA | 74.7947 | 4.1664 | 2641 |
| TRTPN (ATPTN) | 3 | 6 | 3 | 9 | WORK.ANA DATA | 49.3609 | 3.1721 | 5650 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 7 | WORK.ANA DATA | -15.4671 | 3.6413 | 2709 |
| TRTPN (ATPTN) | 1 | 7 | 3 | 7 | WORK.ANA DATA | -13.4671 | 3.6159 | 2671 |
| TRTPN (ATPTN) | 1 | 7 | 1 | 8 | _ | 42.7704 | 2.2704 | 5654 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 8 | WORK.ANA_DATA<br>WORK.ANA DATA | 32.8280 | 3.6506 | 2729 |
| TRTPN (ATPTN) | 1 | 7 | 3 | 8 | _ | 16.9666 | 3.6290 | 2729 |
| TRTPN (ATPTN) | 1 | 7 | 1 | 9 | WORK.ANA_DATA<br>WORK.ANA DATA | 46.9366 | 2.2528 | 5655 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 9 | _ | | | 2662 |
| TRTPN (ATPTN) | | 7 | 3 | 9 | WORK.ANA_DATA | 43.4134 | 3.6183 | 2681 |
| TRTPN (ATPTN) | 1 | 7 | 3 | 7 | WORK.ANA_DATA<br>WORK.ANA DATA | 17.9796<br>2.9603 | 3.6202<br>4.1903 | 2683 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 8 | _ | | | 2719 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 8 | WORK.ANA_DATA | 58.2375 | 3.6460<br>3.2300 | 5654 |
| TRTPN (ATPTN) | | | | | WORK.ANA_DATA | 48.2951 | | |
| TRTPN (ATPTN) | 2 | 7<br>7 | 3<br>1 | 8<br>9 | WORK.ANA_DATA | 32.4337 | 4.2015 | 2704<br>2693 |
| TRTPN (ATPTN) | | 7 | | | WORK.ANA_DATA | 62.4037 | 3.6336 | |
| TRTPN (ATPTN) | 2 | 7 | 2 | 9 | WORK.ANA_DATA | 58.8805 | 3.1974 | 5656 |
| TRTPN (ATPTN) | 2 | 7 | 3 | 9 | WORK.ANA_DATA | 33.4467 | 4.1939 | 2690 |
| TRTPN (ATPTN) | 3 | 7 | 1 2 | 8 | WORK.ANA_DATA | 55.2772 | 3.6205 | 2681 |
| TRTPN (ATPTN) | 3 | 7 | | 8 | WORK.ANA_DATA | 45.3348 | 4.1982 | 2698 |
| TRTPN (ATPTN) | 3 | | 3 | 8 | WORK.ANA_DATA | 29.4734 | 3.1870 | 5652 |
| TRTPN (ATPTN) | 3 | 7<br>7 | 1 | 9 | WORK.ANA_DATA | 59.4433 | 3.6080 | 2655 |
| TRTPN (ATPTN) | | | 2 | - | WORK.ANA_DATA | 55.9202 | 4.1702 | 2648 |
| TRTPN (ATPTN) | 3 | 7<br>8 | 3 | 9 | WORK.ANA_DATA | 30.4864 | 3.1770 | 5651 |
| TRTPN (ATPTN) | 1 | | 2 | 8 | WORK.ANA_DATA | -9.9424 | 3.6551 | 2738 |
| TRTPN (ATPTN) | 1 | 8 | 3 | 8 | WORK.ANA_DATA | -25.8038 | 3.6335 | 2709 |
| TRTPN (ATPTN) | 1 | 8 | 1 | 9 | WORK.ANA_DATA | 4.1661 | 2.2595 | 5655 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 9 | WORK.ANA_DATA | 0.6430 | 3.6229 | 2672 |
| TRTPN (ATPTN) | 1 | 8 | 3 | 9 | WORK.ANA_DATA | -24.7908 | 3.6248 | 2690 |
| TRTPN (ATPTN) | 2 | 8 | 3 | 8 | WORK.ANA_DATA | -15.8614 | 4.2095 | 2719 |
| TRTPN (ATPTN) | 2 | 8 | 1 | 9 | WORK.ANA_DATA | 14.1085 | 3.6428 | 2712 |
| TRTPN (ATPTN) | 2 | 8 | 2 | 9 | WORK.ANA_DATA | 10.5854 | 3.2079 | 5658 |
| TRTPN (ATPTN) | 2 | 8 | 3 | 9 | WORK.ANA_DATA | -14.8484 | 4.2020 | 2705 |
| TRTPN (ATPTN) | 3 | 8 | 1 | 9 | WORK.ANA_DATA | 29.9699 | 3.6211 | 2683 |
| TRTPN (ATPTN) | 3 | 8 | 2 | 9 | WORK.ANA_DATA | 26.4468 | 4.1815 | 2669 |
| TRTPN (ATPTN) | 3 | 8 | 3 | 9 | WORK.ANA_DATA | 1.0130 | 3.1919 | 5652 |
| TRTPN (ATPTN) | 1 | 9 | 2 | 9 | WORK.ANA_DATA | -3.5232 | 3.6105 | 2646 |
| TRTPN (ATPTN) | 1 | 9 | 3 | 9 | WORK.ANA_DATA | -28.9569 | 3.6123 | 2664 |
| TRTPN (ATPTN) | 2 | 9 | 3 | 9 | WORK.ANA_DATA | -25.4338 | 4.1740 | 2655 |

| | Planned<br>Treatment<br>for<br>Period | Analysis<br>Timepoint | Planned<br>Treatment<br>for<br>Period | Analysis<br>Timepoint | | | |
|---|---|---|---|---|---|---|---|
| Effect | 01 (N) | (N) | 01 (N) | (N) | t Value | Pr > t | Alpha |
| TRTPN (ATPTN) | 2 | 6 | 1 | 9 | 24.46 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 6 | 2 | 9 | 26.73 | <.0001 | 0.05 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 275 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

#### Differences of Least Squares Means

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|
| TRTPN (ATPTN) | 2 | 6 | 3 | 9 | 14.24 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 6 | 1 | 7 | 8.69 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 6 | 2 | 7 | 3.80 | 0.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 6 | 3 | 7 | 5.96 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 6 | 1 | 8 | 20.51 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 6 | 2 | 8 | 15.31 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 6 | 3 | 8 | 15.19 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 6 | 1 | 9 | 21.73 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 6 | 2 | 9 | 17.95 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 6 | 3 | 9 | 15.56 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 7 | -4.25 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 7 | 3 | 7 | -3.46 | 0.0006 | 0.05 |
| TRTPN (ATPTN) | 1 | 7 | 1 | 8 | 18.84 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 7 | 2 | 8 | 8.99 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 7 | 3 | 8 | 4.68 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 7 | 1 | 9 | 20.84 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 7<br>7 | 2 | 9 | 12.00<br>4.97 | <.0001<br><.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 2 | 7 | 3 | 7 | 0.71 | 0.4800 | 0.05 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 8 | 15.97 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 8 | 14.95 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 7 | 3 | 8 | 7.72 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 7 | 1 | 9 | 17.17 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 7 | 2 | 9 | 18.41 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 7 | 3 | 9 | 7.98 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 7 | 1 | 8 | 15.27 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 7 | 2 | 8 | 10.80 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 7 | 3 | 8 | 9.25 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 7 | 1 | 9 | 16.48 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 7 | 2 | 9 | 13.41 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 3 | 7 | 3 | 9 | 9.60 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 8 | -2.72 | 0.0066 | 0.05 |
| TRTPN (ATPTN) | 1 | 8 | 3 | 8 | -7.10 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 1 | 8 | 1 | 9 | 1.84 | 0.0653 | 0.05 |
| TRTPN (ATPTN) | 1 | 8 | 2 | 9 | 0.18 | 0.8592 | 0.05 |
| TRTPN (ATPTN) | 1 | 8 | 3 | 9 | -6.84 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 8 | 3 | 8 | -3.77 | 0.0002 | 0.05 |
| TRTPN (ATPTN) | 2 | 8 | 1 | 9 | 3.87 | 0.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 8 | 2 | 9 | 3.30 | 0.0010 | 0.05 |
| TRTPN (ATPTN) | 2 | 8 | | 9 | -3.53 | 0.0004 | 0.05 |
| TRTPN (ATPTN) | 3 | 8 | 1 2 | 9<br>9 | 8.28<br>6.32 | <.0001 | 0.05 |
| TRTPN (ATPTN) TRTPN (ATPTN) | 3 | 8 | 3 | 9 | 0.32 | <.0001<br>0.7510 | 0.05 |
| TRTPN (ATPIN) | 1 | 9 | 2 | 9 | -0.98 | 0.7310 | 0.05 |
| TRTPN (ATPTN) | 1 | 9 | 3 | 9 | -8.02 | <.0001 | 0.05 |
| TRTPN (ATPTN) | 2 | 9 | 3 | 9 | -6.09 | <.0001 | 0.05 |
| TT/TT 14 (111T T T14) | _ | _ | _ | _ | 0.00 | · • • • • • | 0.00 |

| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint | Lower | Upper |
|---|---|---|---|---|---|---|
| HIICCC | 01 (11) | (14) | 01 (11) | (14) | HOWCI | opper |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 2<br>2<br>2<br>3 | 6<br>6<br>6 | 1<br>2<br>3<br>1 | 9<br>9<br>9<br>7 | 81.3628<br>78.7012<br>51.3024<br>24.2995 | 95.5422<br>91.1575<br>67.6887<br>38.4631 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 276 of 412 | |

Parameter Code=SMPGCOL

The Mixed Procedure

Differences of Least Squares Means

| Differences of Least Squares Means | | | | | | |
|---|---|---|---|---|---|---|
| Effect | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Analysis<br>Timepoint<br>(N) | Lower | Upper |
| TRTPN (ATPTN) | 3 3 3 3 3 3 3 1 1 1 1 1 1 1 1 2 2 2 2 2 | 666666667777777777777777777778888888888 | 2 3 1 1 2 3 3 1 3 3 1 3 3 1 3 3 1 3 3 1 3 3 3 1 3 3 3 1 3 3 3 3 1 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 | 7788899977888899978888999988999989999999 | 7.7051 12.6657 67.0609 55.9845 42.1098 71.2515 66.6248 43.1423 -22.6072 -19.5970 38.3195 25.6698 9.8508 42.5203 36.3184 10.8809 -5.2561 51.0884 41.9630 24.1953 55.2788 52.6123 25.2231 48.1780 37.1027 23.2257 52.3685 47.7431 24.2582 -17.1095 -32.9286 -0.2635 -6.4611 -31.8985 -24.1155 6.9655 4.2966 -23.0878 22.8695 18.2474 -5.2444 | 24.1233<br>25.0834<br>81.2425<br>72.4341<br>54.5860<br>85.3842<br>82.9645<br>55.5795<br>-8.3270<br>-5.4165<br>47.2214<br>39.9863<br>24.0824<br>51.3529<br>50.5084<br>25.0783<br>11.1768<br>65.3867<br>54.6272<br>40.6722<br>40.6722<br>40.6722<br>69.5286<br>65.1487<br>41.6704<br>62.3764<br>53.5669<br>35.7211<br>66.5182<br>64.0973<br>36.7146<br>-2.7753<br>-18.6790<br>8.5957<br>7.7470<br>-17.6832<br>-7.6073<br>21.2516<br>16.8742<br>-6.6090<br>37.0704<br>34.6461<br>7.2704 |
| TRTPN (ATPTN) TRTPN (ATPTN) TRTPN (ATPTN) | 1<br>1<br>2 | 9<br>9<br>9 | 2<br>3<br>3 | 9<br>9<br>9 | -10.6029<br>-36.0402<br>-33.6184 | 3.5566<br>-21.8737<br>-17.2492 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 277 of 412 | |

# 20: Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PSMPGM

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 708

Number of Observations

Number of Observations Read 720 Number of Observations Used 708 Number of Observations Not Used 12

Covariance Parameter Estimates

Cov Parm Estimate
Residual 2.2712

Fit Statistics

-2 Res Log Likelihood 2600.9
AIC (Smaller is Better) 2602.9
AICC (Smaller is Better) 2602.9
BIC (Smaller is Better) 2607.4

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t| Alpha 6.4453 0.3205 703 20.11 <.0001 0.05 Intercept trtpn -1.1247 0.1394 703 -8.07 <.0001 0.05 -0.3415 0.1610 703 -2.12 0.0342 0.05 trtpn trtpn PREOAD2 Metformin -0.5115 0.1210 703 -4.23 <.0001 0.05 PREOAD2 Metformin + OAD 0.2153 0.02875 703 7.49 <.0001 0.05 BASE


Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PSMPGM

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 5.8160<br>-1.3983<br>-0.6575 | 7.0746<br>-0.8511<br>-0.02547 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | - | -0.7490 | -0.2740 |
| BASE | THE CITE THE PARTY OF THE PARTY | | 0.1589 | 0.2718 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 703 | 37.60 | <.0001 |
| PREOAD2 | 1 | 703 | 17.88 | <.0001 |
| BASE | 1 | 703 | 56.10 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans,<br>LSMeans,<br>LSMeans, | IDeg | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2<br>Least Squ | 7.3919<br>8.1751<br>8.5166 | 0.07976<br>0.1133<br>0.1143<br>Estimates | 703<br>703<br>703 | 92.68<br>72.15<br>74.52 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |
| | | | | | | Expor | nentiated | Exponentia | ted |

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | 7.2353 | 7.5485 | 1622.74 | 1387.52 | 1897.83 |
| trtpn | LSMeans, | | 7.9526 | 8.3975 | 3551.30 | 2843.02 | 4436.05 |
| trtpn | LSMeans, | | 8.2922 | 8.7410 | 4996.93 | 3992.62 | 6253.87 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -0.7832 | 0.1386 | 703 | -5.65 |

#### Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | <.0001 | 0.05 | -1.0552 | -0.5112 | 0.4569 |

| Effect | Label | | | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira | - IDeg | 0.3481 | 0.5998 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019<br>1.0<br>Final<br>279 of 412 |
|---|---|---|---|
|---|---|---|---|

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PSMPGM

The Mixed Procedure

Least Squares Means Estimates

Effect Label Margins Estimate Error DF t Value trtpn Treatment contrast, IDegLira - Lira WORK.ADATA2 -1.1247 0.1394 703 -8.07

Least Squares Means Estimates

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - Lira <.0001 0.05 -1.3983 -0.8511 0.3247

Least Squares Means Estimates

Effect Label Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - Lira 0.2470 0.4270

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9SMPGMU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3 trtpn PREOAD2

Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 708

Number of Observations

Number of Observations Read 720 Number of Observations Used 708 Number of Observations Not Used 12

Covariance Parameter Estimates

Estimate Cov Parm Residual 737.49

Fit Statistics

-2 Res Log Likelihood 6672.1 AIC (Smaller is Better) AICC (Smaller is Better) 6674.1 6674.1 BIC (Smaller is Better) 6678.6

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 703 20.11 Intercept 116.14 5.7760 < .0001 0.05 trtpn 1 -20.2673 2.5114 703 -8.07 <.0001 0.05 0.0342 trtpn -6.1540 2.9007 703 -2.120.05 3 trtpn PREOAD2 -9.2178 2.1799 703 -4.23 <.0001 0.05 Metformin PREOAD2 Metformin + OAD 0.2153 BASE 0.02875 703 7.49 <.0001 0.05

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9SMPGMU

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 104.80<br>-25.1980<br>-11.8490 | 127.48<br>-15.3365<br>-0.4590 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -13.4977 | -4.9379 |
| BASE | | | 0.1589 | 0.2718 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 703 | 37.60 | <.0001 |
| PREOAD2 | 1 | 703 | 17.88 | <.0001 |
| BASE | 1 | 703 | 56.10 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2<br>Least Sq | 133.20<br>147.31<br>153.47<br>uares Mean | 2.0417 | 703<br>703<br>703 | 92.68<br>72.15<br>74.52 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |
| Effect | Label | Lower | Upper | Exponentiated | Expo | nentiated<br>Lower | Exponentia<br>Up | ted<br>per |

| Effect | Label | Lower | Upper | Exponentiated | Lower | Upper |
|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | 130.38 | 136.02 | 7.058E57 | 4.199E56 | 1.186E59 |
| trtpn | LSMeans, IDeg | 143.31 | 151.32 | 9.506E63 | 1.726E62 | 5.234E65 |
| trtpn | LSMeans, Lira | 149.43 | 157.51 | 4.473E66 | 7.846E64 | 2.55E68 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -14.1133 | 2.4968 | 703 | -5.65 |

#### Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | <.0001 | 0.05 | -19.0154 | -9.2112 | 7.425E-7 |

| Effect | Label | | | | | Exponentiate<br>Lowe | | Exponentiated Upper |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira | _ | IDeg | 5.517E- | 9 | 0.000100 |

| NN9068 | | Date: | 16 December 2019 Novo Nor | disk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 282 of 412 | |

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9SMPGMU

The Mixed Procedure

Least Squares Means Estimates

Effect Label Margins Estimate Standard Error DF t Value trtpn Treatment contrast, IDegLira - Lira WORK.ADATA2 -20.2673 2.5114 703 -8.07

Least Squares Means Estimates

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - Lira < .0001 0.05 -25.1980 -15.3365 1.578E-9

Least Squares Means Estimates

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - Lira 1.14E-11 2.185E-7

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 283 of 412 Statistical document Page:

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PSMPGM

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3 trtpn PREOAD2

Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 708

Number of Observations

Number of Observations Read 720 Number of Observations Used 708 Number of Observations Not Used 12

Covariance Parameter Estimates

Cov Parm Estimate Residual 2.2712

Fit Statistics

-2 Res Log Likelihood 2600.9 AIC (Smaller is Better) AICC (Smaller is Better) 2602.9 2602.9 BIC (Smaller is Better) 2607.4

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 20.11 Intercept 6.4453 0.3205 703 <.0001 0.05 trtpn 1 -1.1247 0.1394 703 -8.07 <.0001 0.05 0.0342 trtpn -0.3415 0.1610 703 -2.120.05 3 trtpn PREOAD2 -0.5115 0.1210 703 -4.23 <.0001 0.05 Metformin PREOAD2 Metformin + OAD BASE -0.7847 0.02875 703 -27.29 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 284 of 412 | |

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PSMPGM

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | w.6 | 1<br>2<br>3 | 5.8160<br>-1.3983<br>-0.6575 | 7.0746<br>-0.8511<br>-0.02547 |
| PREOAD2<br>PREOAD2<br>BASE | Metformin<br>Metformin + OAD | | -0.7490<br>-0.8411 | -0.2740<br>-0.7282 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 703 | 37.60 | <.0001 |
| PREOAD2 | 1 | 703 | 17.88 | <.0001 |
| BASE | 1 | 703 | 744.98 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -2.2158 | 0.07976<br>0.1133<br>0.1143 | 703<br>703<br>703 | -37.60<br>-19.56<br>-16.40 | <.0001<br><.0001<br><.0001 |
| | Least Squares Mean | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -3.1556<br>-2.4383<br>-2.0987 | -2.8425<br>-1.9934<br>-1.6500 | | | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9SMPGMU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 708

Number of Observations

Number of Observations Read 720 Number of Observations Used 708 Number of Observations Not Used 12

Covariance Parameter Estimates

Estimate Cov Parm Residual 737.49

Fit Statistics

-2 Res Log Likelihood 6672.1 AIC (Smaller is Better) AICC (Smaller is Better) 6674.1 6674.1 BIC (Smaller is Better) 6678.6

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 703 20.11 <.0001 Intercept 116.14 5.7760 0.05 trtpn 1 -20.2673 2.5114 703 -8.07 <.0001 0.05 0.0342 trtpn -6.1540 2.9007 703 -2.120.05 3 trtpn PREOAD2 -9.2178 2.1799 703 -4.23 <.0001 0.05 Metformin PREOAD2 Metformin + OAD BASE -0.7847 0.02875 703 -27.29 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 286 of 412 | |

Mean of 9-point self-measured plasma glucose profile after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9SMPGMU

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 104.80<br>-25.1980<br>-11.8490 | 127.48<br>-15.3365<br>-0.4590 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -13.4977 | -4.9379 |
| BASE | 1100101111111 1 0110 | | -0.8411 | -0.7282 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|------------|----------------|--------|
| trtpn<br>PREOAD2 | 2 | 703<br>703 | 37.60<br>17.88 | <.0001 |
| | 1 | | | <.0001 |
| BASE | 1 | 703 | 744.98 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -54.0429<br>-39.9296<br>-33.7756 | 1.4373<br>2.0417<br>2.0594 | 703<br>703<br>703 | -37.60<br>-19.56<br>-16.40 | <.0001<br><.0001<br><.0001 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 -4 | 56.8648<br>13.9381<br>37.8188 | -51.2210<br>-35.9210<br>-29.7323 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 287 of 412 | |

# 21: Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGIBU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 709

Number of Observations

Number of Observations Read 718
Number of Observations Used 709
Number of Observations Not Used 9

Covariance Parameter Estimates

Cov Parm Estimate
Residual 1902.47

Fit Statistics

-2 Res Log Likelihood 7349.6
AIC (Smaller is Better) 7351.6
AICC (Smaller is Better) 7351.6
BIC (Smaller is Better) 7356.1

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t|Alpha 50.3800 4.2937 704 11.73 <.0001 0.05 Intercept trtpn 5.6651 4.0320 704 1.41 0.1604 0.05 14.1118 4.6635 704 3.03 0.0026 0.05 trtpn trtpn PREOAD2 Metformin -10.8133 3.5012 704 -3.09 0.0021 0.05 PREOAD2 Metformin + OAD 0.1397 0.02911 704 4.80 <.0001 0.05 BASE

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGIBU

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 41.9500<br>-2.2510<br>4.9558 | 58.8101<br>13.5813<br>23.2678 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -17.6874 | -3.9393 |
| BASE | | | 0.08260 | 0.1969 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 704 | 4.67 | 0.0096 |
| PREOAD2 | 1 | 704 | 9.54 | 0.0021 |
| BASE | 1 | 704 | 23.05 | <.0001 |

#### Least Squares Means Estimates

| | | | | Standar | d | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | Margins | Estimate | e Erro | r DF | t Value | Pr > t | Alpha |
| trtpn | LSMeans, IDegLira | WORK.ADATA2 | 63.9851 | | | 27.77 | | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | 72.4317 | | | 22.02 | | 0.05 |
| trtpn | LSMeans, Lira | WORK.ADATA2 | 58.3200 | 3.307 | 3 704 | 17.63 | <.0001 | 0.05 |
| | | Least Sq | uares Mear | ns Estimate | S | | | |
| | | | | | Expo | nentiated | Exponenti | ated |
| Effect | Label | Lower | Upper | Exponentia | ted | Lower | U | pper |
| trtpn | LSMeans, IDegLira | | 68.5081 | 6.143 | | 6.669E25 | 5.65 | |
| trtpn | LSMeans, IDeg | | 78.8910 | 2.862 | | 4.482E28 | 1.82 | |
| trtpn | LSMeans, Lira | 51.8266 | 64.8133 | 2.128 | E25 | 3.221E22 | 1.40 | 6E28 |
| | | Toost Co | wana Maar | oo Potimoto | _ | | | |
| | | Least sq | uares mear | ns Estimate | :S | | | |
| | | | | | S | tandard | | |
| Effect | Label | | Margir | ns Es | timate | Error | DF t V | alue |
| trtpn | Treatment contrast | , IDegLira - ID | eg WORK. | ADATA2 - | 8.4466 | 4.0189 | 704 - | 2.10 |
| - | | | - | | | | | |
| Least Squares Means Estimates | | | | | | | | |
| Effect | Label | | Pr > | t Alpha | Lower | Upper | Exponenti | ated |

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 0.0359 | 0.05 | -16.3372 | -0.5561 | 0.000215 |

| Effect | Label | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 8.033E-8 | 0.5734 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019<br>1.0<br>Final<br>289 of 412 | |
|---|---|---|---|---|
| Prandial increment after 26 we | eks of treatment - 9-point se | lf-measured p | lasma glucose profile | · - |

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGIBU

The Mixed Procedure

| Effect | Label | Margins | Estimate | Standard<br>Error | DF t Value |
|---|---|---|---|---|---|
| trtpn | Treatment contrast, IDegLira - Lira | WORK.ADATA2 | 5.6651 | 4.0320 | 704 1.41 |
| | Least Squares Means Estimates | | | | |
| Effect | Label | Pr > t A | lpha Low | er Upper | Exponentiated |
| trtpn | Treatment contrast, IDegLira - Lira | 0.1604 | 0.05 -2.25 | 10 13.5813 | 288.63 |
| Least Squares Means Estimates | | | | | |

| Effect | Label | | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|
| trtpn | Treatment cont | trast, IDegLira | - Lira | 0.1053 | 791207 |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGIEU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 707

Number of Observations

Number of Observations Read 718 Number of Observations Used 707 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 2035.95

Fit Statistics

-2 Res Log Likelihood 7376.4 AIC (Smaller is Better) AICC (Smaller is Better) 7378.4 7378.4 BIC (Smaller is Better) 7382.9

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 7.38 Intercept 28.2369 3.8281 702 <.0001 0.05 trtpn 1 13.7323 4.1645 702 3.30 0.0010 0.05 trtpn 15.3706 4.7970 702 3.20 0.0014 0.05 3 trtpn PREOAD2 -2.5249 3.6263 702 -0.70 0.4865 0.05 Metformin PREOAD2 Metformin + OAD BASE 0.1860 0.03057 702 6.08 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIALE | Status: | Final | |
| Statistical document | | Page: | 291 of 412 | |

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGIEU

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 20.7210<br>5.5560<br>5.9524 | 35.7529<br>21.9086<br>24.7888 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -9.6446 | 4.5948 |
| BASE | | | 0.1259 | 0.2460 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 702 | 6.70 | 0.0013 |
| PREOAD2 | 1 | 702 | 0.48 | 0.4865 |
| BASE | 1 | 702 | 37.00 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimat | Standard<br>e Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 49.651<br>51.289<br>35.919 | 9 3.3822 | 702<br>702<br>702 | 20.67<br>15.16<br>10.56 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |
| | | Least Sq | uares Mea | ns Estimates | | | | |
| Effect | Label | Lower | Upper | Exponentiated | Expor | nentiated<br>Lower | Exponentia<br>Up | ted |
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | 44.6494 | 54.3671<br>57.9303<br>42.5979 | 3.659E21<br>1.883E22<br>3.977E15 | | 3.277E19<br>2.46E19<br>5.001E12 | 4.087<br>1.442<br>3.162 | E25 |
| | | Least Sq | uares Mea | ns Estimates | | | | |
| Effect | Label | | Margi | ns Estima | | andard<br>Error | DF t Va | lue |
| trtpn | Treatment contrast | , IDegLira - ID | eg WORK. | ADATA2 -1.63 | 383 | 4.1484 | 702 -0 | .39 |
| Least Squares Means Estimates | | | | | | | | |
| Effect | Label | | Pr > | t Alpha | Lower | Upper | Exponentia | ted |
| trtpn | Treatment contrast | , IDegLira - ID | eg 0.6 | 930 0.05 - | -9.7830 | 6.5065 | 0.1 | 943 |

| Effect | Label | | | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment co | ontrast, | IDegLira - | IDeg | 0.000056 | 669.48 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019<br>1.0<br>Final<br>292 of 412 | |
|---|---|---|---|---|
| Prandial increment after 26 we | eks of treatment - 9-point se | | olasma glucose profile | . – |

change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGIEU

The Mixed Procedure

Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF t Value |
|---|---|---|---|---|---|
| trtpn | Treatment contrast, IDegLira - Lir | a WORK.ADATA2 | 13.7323 | 4.1645 | 702 3.30 |
| | Least Squares Means Estimates | | | | |
| Effect | Label | Pr > t A | lpha Lowe | er Upper | Exponentiated |
| trtpn | Treatment contrast, IDegLira - Lir | a 0.0010 | 0.05 5.556 | 21.9086 | 920162 |
| Least Squares Means Estimates | | | | | |

Exponentiated Exponentiated Lower Upper Effect Label trtpn Treatment contrast, IDegLira - Lira 258.79 3.2717E9

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGILU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 708

Number of Observations

Number of Observations Read 718 Number of Observations Used 708 Number of Observations Not Used 10

Covariance Parameter Estimates

Cov Parm Estimate Residual 2006.21

Fit Statistics

-2 Res Log Likelihood 7376.7 AIC (Smaller is Better) AICC (Smaller is Better) 7378.7 7378.7 BIC (Smaller is Better) 7383.2

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 703 Intercept 31.7807 3.6382 8.74 < .0001 0.05 trtpn 1 6.7797 4.1349 703 1.64 0.1015 0.05 0.0005 trtpn 16.6127 4.7770 703 3.48 0.05 3 trtpn PREOAD2 1.7065 3.5950 703 0.47 0.6352 0.05 Metformin PREOAD2 Metformin + OAD BASE 0.1446 0.02759 703 5.24 <.0001 0.05

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGILU

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 24.6377<br>-1.3385<br>7.2337 | 38.9237<br>14.8979<br>25.9916 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -5.3517 | 8.7648 |
| BASE | | | 0.09041 | 0.1987 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 703 | 6.15 | 0.0022 |
| PREOAD2 | 1 | 703 | 0.23 | 0.6352 |
| BASE | 1 | 703 | 27.46 | <.0001 |

#### Least Squares Means Estimates

| | | | | Standard | | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 44.9642<br>54.7972<br>38.1846 | 2.3828<br>3.3775<br>3.3702 | 703<br>703<br>703 | 18.87<br>16.22<br>11.33 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |
| | | Least So | uares Means | Estimates | | | | |

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | 40.2859 | 49.6426 | 3.371E19 | 3.133E17 | 3.627E21 |
| trtpn | LSMeans, IDeg | 48.1661 | 61.4284 | 6.283E23 | 8.284E20 | 4.765E26 |
| trtpn | LSMeans, Lira | 31.5677 | 44.8015 | 3.831E16 | 5.125E13 | 2.864E19 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -9.8330 | 4.1312 | 703 | -2.38 |

#### Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 0.0176 | 0.05 | -17.9439 | -1.7221 | 0.000054 |

| Effect | Label | | | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment c | contrast, | IDegLira | - IDeo | 1.611E-8 | 0.1787 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019<br>1.0<br>Final<br>295 of 412 | Novo Nordisk |
|---|---|---|---|---|
| Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set | | | | |
| Parameter Code=P9PGILU | | | | |
| The Mixed Procedure | | | | |
| Least Squares Means Estimates | | | | |
| Effect Label | Margins I | | dard<br>rror DF t Va | ılue |

| Effect | Label | Margins | Estimate | Error | DF t Value |
|---|---|---|---|---|---|
| trtpn | Treatment contrast, IDegLira - Lira | WORK.ADATA2 | 6.7797 | 4.1349 | 703 1.64 |
| Least Squares Means Estimates | | | | | |
| Effect | Label | Pr > t A | lpha Lowe | r Upper | Exponentiated |
| trtpn | Treatment contrast, IDegLira - Lira | 0.1015 | 0.05 -1.338 | 5 14.8979 | 879.78 |
| | Least Squares Means F | Estimates | | | |

| Effect | Label | | | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira | - Lira | 0.2622 | 2951642 |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 296 of 412 Statistical document Page:

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGINC

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 2.6091

Fit Statistics

-2 Res Log Likelihood 2736.5 AIC (Smaller is Better) AICC (Smaller is Better) 2738.5 2738.5 BIC (Smaller is Better) 2743.1

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 2.0022 0.1527 713 13.12 <.0001 0.05 2.99 trtpn 1 0.4424 0.1479 713 0.0029 0.05 trtpn 0.8538 0.1710 713 < .0001 0.05 3 trtpn PREOAD2 -0.2348 0.1288 713 -1.82 0.0688 0.05 Metformin PREOAD2 Metformin + OAD BASE 0.1750 0.02899 713 6.04 <.0001 0.05

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGINC

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.7025<br>0.1521<br>0.5180 | 2.3019<br>0.7327<br>1.1895 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | ŭ | -0.4876 | 0.01811 |
| BASE | 1100101111111 . 0115 | | 0.1181 | 0.2319 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 713 | 12.47 | <.0001 |
| PREOAD2 | 1 | 713 | 3.32 | 0.0688 |
| BASE | 1 | 713 | 36.43 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2<br>Least Squ | 2.9129<br>3.3242<br>2.4705<br>wares Means | 0.08514<br>0.1208<br>0.1209<br>Estimates | 713<br>713<br>713 | 34.21<br>27.52<br>20.44 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | 2.7457 | 3.0800 | 18.4094 | 15.5757 | 21.7585 |
| trtpn | LSMeans, IDeg | 3.0871 | 3.5614 | 27.7781 | 21.9128 | 35.2134 |
| trtpn | LSMeans, Lira | 2.2332 | 2.7077 | 11.8280 | 9.3295 | 14.9955 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -0.4114 | 0.1478 | 713 | -2.78 |

#### Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 0.0055 | 0.05 | -0.7015 | -0.1213 | 0.6627 |

| Effect | Label | | | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira - | - IDeg | 0.4958 | 0.8858 |

| | 4148<br>Frial Report<br>I document | CONF | IDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 De | 1.0<br>Final<br>298 of 412 | Novo Nordisk |
|---|---|---|---|---|---|---|---|
| Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set | | | | | | | |
| Parameter Code=P9PGINC | | | | | | | |
| The Mixed Procedure | | | | | | | |
| Least Squares Means Estimates | | | | | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF t Va | lue |
| trtpn | Treatment contrast, ID | DegLira - Lira | WORK.ADATA2 | 0.4424 | 0.1479 | 713 2 | .99 |
| Least Squares Means Estimates | | | | | | | |
| Effect | Label | | Pr > t Al | lpha Lowe: | r Upper | Exponentia | ted |
| trtpn | Treatment contrast, ID | DegLira - Lira | 0.0029 | 0.152 | 1 0.7327 | 1.5 | 564 |

Exponentiated Exponentiated Lower Upper

Least Squares Means Estimates

trtpn Treatment contrast, IDegLira - Lira 1.1643 2.0807

Effect Label

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGINCB

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 709

Number of Observations

Number of Observations Read 718 Number of Observations Used 709 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 5.8588

Fit Statistics

-2 Res Log Likelihood 3272.6 AIC (Smaller is Better) AICC (Smaller is Better) 3274.6 3274.6 BIC (Smaller is Better) 3279.2

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 2.7958 0.2383 704 11.73 <.0001 0.05 trtpn 1 0.3144 0.2238 704 1.41 0.1604 0.05 trtpn 0.7831 0.2588 704 3.03 0.0026 0.05 3 trtpn PREOAD2 -0.6001 0.1943 704 -3.09 0.0021 0.05 Metformin PREOAD2 Metformin + OAD BASE 0.1397 0.02911 704 4.80 <.0001 0.05
| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 300 of 412 | |

Parameter Code=P9PGINCB

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 2.3280<br>-0.1249<br>0.2750 | 3.2636<br>0.7537<br>1.2912 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -0.9815 | -0.2186 |
| BASE | | | 0.08260 | 0.1969 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 704 | 4.67 | 0.0096 |
| PREOAD2 | 1 | 704 | 9.54 | 0.0021 |
| BASE | 1 | 704 | 23.05 | <.0001 |

# Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2<br>Least Squ | 3.5508<br>4.0195<br>3.2364<br>uares Means | 0.1278<br>0.1826<br>0.1835<br>Estimates | 704<br>704<br>704 | 27.77<br>22.02<br>17.63 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | LSMeans, | 3.2998 | 3.8018 | 34.8406 | 27.1067 | 44.7809 |
| trtpn | LSMeans, | 3.6611 | 4.3780 | 55.6743 | 38.9029 | 79.6761 |
| trtpn | LSMeans, | 2.8761 | 3.5967 | 25.4420 | 17.7442 | 36.4793 |

## Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -0.4687 | 0.2230 | 704 | -2.10 |

# Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 0.0359 | 0.05 | -0.9066 | -0.03086 | 0.6258 |

| Effect | Label | | | | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira - | IDeg | 0.4039 | 0.9696 |

| | 4148<br>Γrial Report<br>I document | CONF | IDENTIAL | V | ersion:<br>tatus:<br>age: | 16 De | 1.<br>Fina<br>301 of 41 | 0 |
|---|---|---|---|---|---|---|---|---|
| | Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set | | | | | | | |
| Paramet | Parameter Code=P9PGINCB | | | | | | | |
| The Mix | The Mixed Procedure | | | | | | | |
| | Least Squares Means Estimates | | | | | | | |
| Effect | Label | | Margins | Esti | St<br>imate | andard<br>Error | DF t | Value |
| trtpn | Treatment contrast, IDe | egLira - Lira | WORK.ADATA2 | 0. | .3144 | 0.2238 | 704 | 1.41 |
| | Least Squares Means Estimates | | | | | | | |
| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponent | iated |
| trtpn | Treatment contrast, IDe | egLira - Lira | 0.1604 | 0.05 | -0.1249 | 0.7537 | 1 | .3694 |
| | Least So | quares Means E | stimates | | | | | |

trtpn Treatment contrast, IDegLira - Lira 0.8826 2.1248

Effect Label

Exponentiated Exponentiated Lower Upper

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGINCE

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

1 7 Covariance Parameters Columns in X Columns in Z 0 Subjects Max Obs per Subject 707

Number of Observations

Number of Observations Read 718 Number of Observations Used 707 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 6.2699

Fit Statistics

-2 Res Log Likelihood AIC (Smaller is Better) AICC (Smaller is Better) 3313.0 BIC (Smaller is Better) 3317.5

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 7.38 Intercept 1.5670 0.2124 702 < .0001 0.05 trtpn 1 0.7621 0.2311 702 3.30 0.0010 0.05 trtpn 0.8530 0.2662 702 3.20 0.0014 0.05 3 trtpn PREOAD2 -0.1401 0.2012 702 -0.70 0.4865 0.05 Metformin PREOAD2 Metformin + OAD BASE 0.1860 0.03057 702 6.08 <.0001 0.05

# NN9068 | Date: 16 December 2019 | Novo Nordisk NN9068-4148 | CONFIDENTIAL | Version: 1.0 | Clinical Trial Report | Status: Final |  |

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGINCE

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.1499<br>0.3083<br>0.3303 | 1.9841<br>1.2158<br>1.3756 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | Ü | -0.5352 | 0.2550 |
| BASE | TICCIOIMITI ( OIID | | 0.1259 | 0.2460 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 702 | 6.70 | 0.0013 |
| PREOAD2 | 1 | 702 | 0.48 | 0.4865 |
| BASE | 1 | 702 | 37.00 | <.0001 |

# Least Squares Means Estimates

Standard

| Effect | Label | Margins | Estimat | e Error | DF | t Value | Pr > | t Al | pha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | WORK.ADATA2 | 2.755 | 4 0.1333 | 702 | 20.67 | <.00 | | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | 2.846 | 3 0.1877 | 702 | 15.16 | < .00 | 001 0 | 0.05 |
| trtpn | LSMeans, Lira | WORK.ADATA2 | 1.993 | 3 0.1888 | 702 | 10.56 | <.00 | | 0.05 |
| | | Least So | quares Mea | ns Estimates | | | | | |
| | | | | | Expor | nentiated | Expone | entiated | |
| Effect | Label | Lower | Upper | Exponentiated | - | Lower | - | Upper | |
| trtpn | LSMeans, IDegLira | 2.4937 | 3.0170 | 15.7267 | | 12.1057 | | 20.4308 | |
| trtpn | LSMeans, IDeg | 2.4778 | 3.2148 | 17.2235 | | 11.9146 | | 24.8978 | |
| trtpn | LSMeans, Lira | 1.6227 | 2.3639 | 7.3397 | | 5.0666 | | 10.6326 | |
| crepn | Horicano, Hira | 1.0227 | 2.3033 | 7.3337 | | 3.0000 | | 10.0020 | |
| | | Least So | quares Mea | ns Estimates | | | | | |
| | | | | | St | andard | | | |
| Effect | Label | | Margi | ns Estima | te | Error | DF | t Value | |
| trtpn | Treatment contrast | , IDeqLira - ID | Dea WORK. | ADATA2 -0.090 | 91 | 0.2302 | 702 | -0.39 | |
| 1 | | | , | | | | | | |

# Least Squares Means Estimates

| Effect | Label | Pr > t | Alpha | Lower | Upper | Exponentiated | |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 0.6930 | 0.05 | -0.5429 | 0.3611 | 0.9131 |

| Effect | Label | | | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment o | contrast, | IDegLira - | IDeg | 0.5811 | 1.4349 |

| | -4148<br>Γrial Report<br>I document | CONF | <u>IDENTIAL</u> | Date:<br>Version:<br>Status:<br>Page: | 16 De | 1.0<br>Final<br>304 of 412 | Novo Nordisk |
|---|---|---|---|---|---|---|---|
| | Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set | | | | | | |
| Parameter Code=P9PGINCE | | | | | | | |
| The Mix | The Mixed Procedure | | | | | | |
| | Least Squares Means Estimates | | | | | | |
| Effect | Label | | Margins | Estimate S | tandard<br>Error | DF t Va | lue |
| trtpn | Treatment contrast, ID | DegLira - Lira | WORK.ADATA2 | 0.7621 | 0.2311 | 702 3 | .30 |
| Least Squares Means Estimates | | | | | | | |
| Effect | Label | | Pr > t Alp | ha Lower | Upper | Exponentia | ited |
| trtpn | Treatment contrast, ID | DegLira - Lira | 0.0010 0 | 0.3083 | 1.2158 | 2.1 | 427 |

Exponentiated Exponentiated Lower Upper

Least Squares Means Estimates

trtpn Treatment contrast, IDegLira - Lira 1.3611 3.3730

Effect Label

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGINCL

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 708

Number of Observations

Number of Observations Read 718 Number of Observations Used 708 Number of Observations Not Used 10

Covariance Parameter Estimates

Cov Parm Estimate Residual 6.1783

Fit Statistics

-2 Res Log Likelihood 3305.5 AIC (Smaller is Better) AICC (Smaller is Better) 3307.5 3307.5 BIC (Smaller is Better) 3312.0

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 703 Intercept 1.7636 0.2019 8.74 <.0001 0.05 trtpn 1 0.3762 0.2295 703 1.64 0.1015 0.05 trtpn 0.9219 0.2651 703 3.48 0.0005 0.05 3 trtpn PREOAD2 0.09470 0.1995 703 0.47 0.6352 0.05 Metformin PREOAD2 Metformin + OAD BASE 0.1446 0.02759 703 5.24 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 306 of 412 | |

Parameter Code=P9PGINCL

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.3672<br>-0.07428<br>0.4014 | 2.1600<br>0.8267<br>1.4424 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -0.2970 | 0.4864 |
| BASE | TICCIOIMITI ( OIID | | 0.09041 | 0.1987 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 703 | 6.15 | 0.0022 |
| PREOAD2 | 1 | 703 | 0.23 | 0.6352 |
| BASE | 1 | 703 | 27.46 | <.0001 |

# Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2<br>Least Sq | 2.4952<br>3.0409<br>2.1190<br>guares Mean | 9 0.1874 | 703<br>703<br>703 | 18.87<br>16.22<br>11.33 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |
| Effect | Label | Lower | Upper | Exponentiated | Expor | nentiated<br>Lower | Exponentia<br>Up | ted<br>pper |
| t.rt.pn | LSMeans. IDeαLira | 2.2356 | 2.7549 | 12.1247 | | 9.3523 | 15.7 | 188 |

| Effect | Label | | Lower | Upper | Exponentiated | Lower | Upper |
|--------|----------|---|--------|--------|---------------|---------|---------|
| trtpn | LSMeans, | _ | 2.2356 | 2.7549 | 12.1247 | 9.3523 | 15.7188 |
| trtpn | LSMeans, | | 2.6729 | 3.4089 | 20.9243 | 14.4822 | 30.2320 |
| trtpn | LSMeans, | | 1.7518 | 2.4862 | 8.3229 | 5.7650 | 12.0156 |

## Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -0.5457 | 0.2293 | 703 | -2.38 |

# Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 0.0176 | 0.05 | -0.9958 | -0.09557 | 0.5795 |

| Effect | Label | | | | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira · | - IDeg | 0.3694 | 0.9089 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019<br>1.0<br>Final<br>307 of 412 |
|---|---|---|---|

Parameter Code=P9PGINCL

The Mixed Procedure

| Effect | Label | Margins | Estimate | Standard<br>Error | DF t Value |
|---|---|---|---|---|---|
| trtpn | Treatment contrast, IDegLira - Lira | WORK.ADATA2 | 0.3762 | 0.2295 | 703 1.64 |
| | Least Squar | es Means Estin | nates | | |
| Effect | Label | Pr > t Al | pha Lowe | r Upper | Exponentiated |
| trtpn | Treatment contrast, IDegLira - Lira | 0.1015 | 0.05 -0.0742 | 8 0.8267 | 1.4568 |
| | Least Squares Means E | stimates | | | |
| | | Exponentiated | l Exponent | iated | |

| Effect | Label | | | | Exponentiated<br>Lower | ± |
|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira - | - Lira | 0.9284 | 2.2859 |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGIU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable AVAL Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 847.22

Fit Statistics

-2 Res Log Likelihood 6865.6 AIC (Smaller is Better) AICC (Smaller is Better) 6867.6 6867.6 BIC (Smaller is Better) 6872.1

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 36.0789 2.7508 713 13.12 < .0001 0.05 trtpn 1 7.9719 2.6645 713 2.99 0.0029 0.05 4.99 15.3852 trtpn 3.0818 713 < .0001 0.05 3 trtpn PREOAD2 -4.2304 2.3209 713 -1.82 0.0688 0.05 Metformin PREOAD2 Metformin + OAD BASE 0.1750 0.02899 713 6.04 <.0001 0.05


Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGIU

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 30.6782<br>2.7408<br>9.3347 | 41.4796<br>13.2031<br>21.4356 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -8.7870 | 0.3263 |
| BASE | 110010111111111111111111111111111111111 | | 0.1181 | 0.2319 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 713 | 12.47 | <.0001 |
| PREOAD2 | 1 | 713 | 3.32 | 0.0688 |
| BASE | 1 | 713 | 36.43 | <.0001 |

# Least Squares Means Estimates

| | | | | Standard | | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | Margins | Estimate | Error | DF | t Value | Pr > t | Alpha |
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 52.4897<br>59.9030<br>44.5178 | 1.5341<br>2.1769<br>2.1779 | 713<br>713<br>713 | 34.21<br>27.52<br>20.44 | <.0001<br><.0001<br><.0001 | 0.05<br>0.05<br>0.05 |
| | | Least So | uares Means | Estimates | | | | |

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | 49.4777 | 55.5017 | 6.252E22 | 3.075E21 | 1.271E24 |
| trtpn | LSMeans, IDeg | 55.6290 | 64.1769 | 1.036E26 | 1.443E24 | 7.442E27 |
| trtpn | LSMeans, Lira | 40.2420 | 48.7936 | 2.157E19 | 2.998E17 | 1.552E21 |

## Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Error | DF | t Value |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | WORK.ADATA2 | -7.4132 | 2.6629 | 713 | -2.78 |

# Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 0.0055 | 0.05 | -12.6413 | -2.1852 | 0.000603 |

| Effect | Label | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 3.236E-6 | 0.1125 |

| | 4148<br>Frial Report<br>I document | CONFI | <del>DENTIAL</del> | | rsion:<br>tus: | 16 De | 1.0<br>Final<br>310 of 412 | Novo Nordisk |
|---|---|---|---|---|---|---|---|---|
| | Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set | | | | | | | |
| Paramet | er Code=P9PGIU | | | | | | | |
| The Mix | ed Procedure | | | | | | | |
| | | Least Squar | es Means Est | imates | | | | |
| Effect | Label | | Margins | Estin | | andard<br>Error | DF t V | alue |
| trtpn | Treatment contrast, IDe | egLira - Lira | WORK.ADATA2 | 7.9 | 719 | 2.6645 | 713 | 2.99 |
| | Least Squares Means Estimates | | | | | | | |
| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponenti | ated |
| trtpn | Treatment contrast, IDe | egLira - Lira | 0.0029 | 0.05 | 2.7408 | 13.2031 | 289 | 3.47 |
| | Least Squares Means Estimates | | | | | | | |

Exponentiated Exponentiated Lower Upper

trtpn Treatment contrast, IDegLira - Lira 15.4998 542016

Effect Label

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGIBU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 709

Number of Observations

Number of Observations Read 718 Number of Observations Used 709 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 1902.47

Fit Statistics

-2 Res Log Likelihood 7349.6 AIC (Smaller is Better) AICC (Smaller is Better) 7351.6 BIC (Smaller is Better) 7356.1

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 704 Intercept 50.3800 4.2937 11.73 < .0001 0.05 trtpn 1 5.6651 4.0320 704 1.41 0.1604 0.05 trtpn 14.1118 4.6635 704 3.03 0.0026 0.05 3 trtpn PREOAD2 -10.8133 3.5012 704 -3.09 0.0021 0.05 Metformin PREOAD2 Metformin + OAD BASE -0.8603 0.02911 704 -29.56 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 312 of 412 | |

Parameter Code=P9PGIBU

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 41.9500<br>-2.2510<br>4.9558 | 58.8101<br>13.5813<br>23.2678 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -17.6874 | -3.9393 |
| BASE | | | -0.9174 | -0.8031 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|------------|---------|------------------|
| trtpn<br>PREOAD2 | 2 | 704<br>704 | 4.67 | 0.0096<br>0.0021 |
| BASE | 1 | 704 | 873.62 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -9.4894 | 2.3037<br>3.2899<br>3.3073 | 704<br>704<br>704 | -7.79<br>-2.88<br>-7.14 | <.0001<br>0.0040<br><.0001 |
| | Least Squares Mean | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 -1 | 22.4590<br>15.9486<br>30.0945 | -13.4130<br>-3.0301<br>-17.1078 | | | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 313 of 412 Statistical document Page:

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGIEU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 707

Number of Observations

Number of Observations Read 718 Number of Observations Used 707 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 2035.95

Fit Statistics

-2 Res Log Likelihood 7376.4 AIC (Smaller is Better) AICC (Smaller is Better) 7378.4 7378.4 BIC (Smaller is Better) 7382.9

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 7.38 Intercept 28.2369 3.8281 702 < .0001 0.05 trtpn 1 13.7323 4.1645 702 3.30 0.0010 0.05 trtpn 15.3706 4.7970 702 3.20 0.0014 0.05 3 trtpn PREOAD2 -2.5249 3.6263 702 -0.70 0.4865 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.8140 0.03057 702 -26.62 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 314 of 412 | |

Parameter Code=P9PGIEU

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 20.7210<br>5.5560<br>5.9524 | 35.7529<br>21.9086<br>24.7888 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -9.6446 | 4.5948 |
| BASE | IICCICIMIII I OIID | | -0.8741 | -0.7540 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|------------|--------------|------------------|
| trtpn<br>PREOAD2 | 2<br>1 | 702<br>702 | 6.70<br>0.48 | 0.0013<br>0.4865 |
| BASE | 1 | 702 | 708.88 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLir<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 5.5644 | 2.4018<br>3.3822<br>3.4016 | 702<br>702<br>702 | 1.63<br>1.65<br>-2.88 | 0.1026<br>0.1004<br>0.0041 |
| | Least Squares Mea | ns Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLir<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -0.7894<br>-1.0761<br>16.4847 | 8.6417<br>12.2049<br>-3.1275 | | | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGILU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 708

Number of Observations

Number of Observations Read 718 Number of Observations Used 708 Number of Observations Not Used 10

Covariance Parameter Estimates

Cov Parm Estimate Residual 2006.21

Fit Statistics

-2 Res Log Likelihood 7376.7 AIC (Smaller is Better) AICC (Smaller is Better) 7378.7 7378.7 BIC (Smaller is Better) 7383.2

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 703 Intercept 31.7807 3.6382 8.74 <.0001 0.05 trtpn 1 6.7797 4.1349 703 1.64 0.1015 0.05 trtpn 16.6127 4.7770 703 3.48 0.0005 0.05 3 trtpn PREOAD2 1.7065 3.5950 703 0.47 0.6352 0.05 Metformin PREOAD2 Metformin + OAD BASE -0.8554 0.02759 703 -31.01 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 316 of 412 | |

Parameter Code=P9PGILU

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 24.6377<br>-1.3385<br>7.2337 | 38.9237<br>14.8979<br>25.9916 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -5.3517 | 8.7648 |
| BASE | IIOOIOIMIII , OIID | | -0.9096 | -0.8013 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 703 | 6.15 | 0.0022 |
| PREOAD2 | 1 | 703 | 0.23 | 0.6352 |
| BASE | 1 | 703 | 961.45 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 4.5032<br>14.3362<br>-2.2764 | 2.3828<br>3.3775<br>3.3702 | 703<br>703<br>703 | 1.89<br>4.24<br>-0.68 | 0.0592<br><.0001<br>0.4996 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -0.1751<br>7.7051<br>-8.8933 | 9.1816<br>20.9674<br>4.3405 | | | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGINC

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 2.6091

Fit Statistics

-2 Res Log Likelihood 2736.5 AIC (Smaller is Better) AICC (Smaller is Better) 2738.5 2738.5 BIC (Smaller is Better) 2743.1

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 2.0022 0.1527 713 13.12 <.0001 0.05 2.99 trtpn 1 0.4424 0.1479 713 0.0029 0.05 trtpn 0.8538 0.1710 713 < .0001 0.05 3 trtpn PREOAD2 -0.2348 0.1288 713 -1.82 0.0688 0.05 Metformin PREOAD2 Metformin + OAD BASE -0.8250 0.02899 713 -28.46 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 318 of 412 | |

Parameter Code=P9PGINC

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.7025<br>0.1521<br>0.5180 | 2.3019<br>0.7327<br>1.1895 |
| PREOAD2<br>PREOAD2<br>BASE | Metformin<br>Metformin + OAD | | -0.4876<br>-0.8819 | 0.01811 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|------------|---------------|------------------|
| trtpn<br>PREOAD2 | 2 | 713<br>713 | 12.47<br>3.32 | <.0001<br>0.0688 |
| BASE | 1 | 713 | 809.82 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLi<br>Change from baseline, IDeg<br>Change from baseline, Lira | ra WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 0.2127 | 0.08514<br>0.1208<br>0.1209 | 713<br>713<br>713 | -2.33<br>1.76<br>-5.30 | 0.0199<br>0.0787<br><.0001 |
| | Least Squares Me | ans Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLi<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 - | -0.3658<br>0.02447<br>-0.8784 | -0.03153<br>0.4499<br>-0.4038 | | | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGINCB

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 709

Number of Observations

Number of Observations Read 718 Number of Observations Used 709 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 5.8588

Fit Statistics

-2 Res Log Likelihood 3272.6 AIC (Smaller is Better) AICC (Smaller is Better) 3274.6 3274.6 BIC (Smaller is Better) 3279.2

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 2.7958 0.2383 704 11.73 <.0001 0.05 trtpn 1 0.3144 0.2238 704 1.41 0.1604 0.05 3.03 trtpn 0.7831 0.2588 704 0.0026 0.05 3 trtpn PREOAD2 -0.6001 0.1943 704 -3.09 0.0021 0.05 Metformin PREOAD2 Metformin + OAD BASE -0.8603 0.02911 704 -29.56 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 320 of 412 | |

Parameter Code=P9PGINCB

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 2.3280<br>-0.1249<br>0.2750 | 3.2636<br>0.7537<br>1.2912 |
| PREOAD2<br>PREOAD2<br>BASE | Metformin<br>Metformin + OAD | | -0.9815<br>-0.9174 | -0.2186<br>-0.8031 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|------------|---------|------------------|
| trtpn<br>PREOAD2 | 2 | 704<br>704 | 4.67 | 0.0096<br>0.0021 |
| BASE | 1 | 704 | 873.62 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -0.5266 | 0.1278<br>0.1826<br>0.1835 | 704<br>704<br>704 | -7.79<br>-2.88<br>-7.14 | <.0001<br>0.0040<br><.0001 |
| | Least Squares Mean | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -1.2463<br>-0.8851<br>-1.6701 | -0.7443<br>-0.1682<br>-0.9494 | | | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGINCE

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 707

Number of Observations

Number of Observations Read 718 Number of Observations Used 707 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 6.2699

Fit Statistics

-2 Res Log Likelihood AIC (Smaller is Better) AICC (Smaller is Better) 3313.0 BIC (Smaller is Better) 3317.5

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 7.38 Intercept 1.5670 0.2124 702 <.0001 0.05 trtpn 1 0.7621 0.2311 702 3.30 0.0010 0.05 trtpn 0.8530 0.2662 702 3.20 0.0014 0.05 3 trtpn PREOAD2 -0.1401 0.2012 702 -0.70 0.4865 0.05 Metformin PREOAD2 Metformin + OAD BASE -0.8140 0.03057 702 -26.62 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 322 of 412 | |

Parameter Code=P9PGINCE

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.1499<br>0.3083<br>0.3303 | 1.9841<br>1.2158<br>1.3756 |
| PREOAD2 | Metformin<br>Metformin + OAD | | -0.5352 | 0.2550 |
| BASE | | | -0.8741 | -0.7540 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|------------|--------------|------------------|
| trtpn<br>PREOAD2 | 2 | 702<br>702 | 6.70<br>0.48 | 0.0013<br>0.4865 |
| BASE | 1 | 702 | 708.88 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLi<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 0.3088 | 0.1333<br>0.1877<br>0.1888 | 702<br>702<br>702 | 1.63<br>1.65<br>-2.88 | 0.1026<br>0.1004<br>0.0041 |
| | Least Squares Me | ans Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLi<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 - | 0.04381<br>0.05972<br>-0.9148 | 0.4796<br>0.6773<br>-0.1736 | | | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGINCL

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 708

Number of Observations

Number of Observations Read 718 Number of Observations Used 708 Number of Observations Not Used 10

Covariance Parameter Estimates

Cov Parm Estimate Residual 6.1783

Fit Statistics

-2 Res Log Likelihood 3305.5 AIC (Smaller is Better) AICC (Smaller is Better) 3307.5 3307.5 BIC (Smaller is Better) 3312.0

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 703 Intercept 1.7636 0.2019 8.74 < .0001 0.05 trtpn 1 0.3762 0.2295 703 1.64 0.1015 0.05 trtpn 0.9219 0.2651 703 3.48 0.0005 0.05 3 trtpn PREOAD2 0.09470 0.1995 703 0.47 0.6352 0.05 Metformin PREOAD2 Metformin + OAD BASE -0.8554 0.02759 703 -31.01 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 324 of 412 | |

Parameter Code=P9PGINCL

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.3672<br>-0.07428<br>0.4014 | 2.1600<br>0.8267<br>1.4424 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -0.2970 | 0.4864 |
| BASE | | | -0.9096 | -0.8013 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 703 | 6.15 | 0.0022 |
| PREOAD2 | 1 | 703 | 0.23 | 0.6352 |
| BASE | 1 | 703 | 961.45 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | | 0.1322<br>0.1874<br>0.1870 | 703<br>703<br>703 | 1.89<br>4.24<br>-0.68 | 0.0592<br><.0001<br>0.4996 |
| | Least Squares Mear | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | 0.00972<br>0.4276<br>-0.4935 | 0.5095<br>1.1636<br>0.2409 | | | |

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 325 of 412 Statistical document Page:

Prandial increment after 26 weeks of treatment - 9-point self-measured plasma glucose profile - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=P9PGIU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3 trtpn PREOAD2

Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 847.22

Fit Statistics

-2 Res Log Likelihood 6865.6 AIC (Smaller is Better) AICC (Smaller is Better) 6867.6 6867.6 BIC (Smaller is Better) 6872.1

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error Intercept 36.0789 2.7508 713 13.12 <.0001 0.05 2.99 trtpn 1 7.9719 2.6645 713 0.0029 0.05 15.3852 trtpn 3.0818 713 < .0001 0.05 3 trtpn PREOAD2 -4.2304 2.3209 713 -1.82 0.0688 0.05 Metformin PREOAD2 Metformin + OAD BASE -0.8250 0.02899 713 -28.46 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 326 of 412 | |

Parameter Code=P9PGIU

The Mixed Procedure

# Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 30.6782<br>2.7408<br>9.3347 | 41.4796<br>13.2031<br>21.4356 |
| PREOAD2<br>PREOAD2<br>BASE | Metformin<br>Metformin + OAD | | -8.7870<br>-0.8819 | 0.3263 |

## Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|------------|---------------|------------------|
| trtpn<br>PREOAD2 | 2 | 713<br>713 | 12.47<br>3.32 | <.0001<br>0.0688 |
| BASE | ī | 713 | 809.82 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 3.8331 | 1.5341<br>2.1769<br>2.1779 | 713<br>713<br>713 | -2.33<br>1.76<br>-5.30 | 0.0199<br>0.0787<br><.0001 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -6.5921<br>-0.4409<br>15.8279 | -0.5682<br>8.1070<br>-7.2763 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIALE | Status: | Final | |
| Statistical document | | Page: | 327 of 412 | |

# 22: Fasting insulin after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=INS\_TO\_S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 690

Number of Observations

Number of Observations Read 720 Number of Observations Used 690 Number of Observations Not Used 30

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.3923

Fit Statistics

-2 Res Log Likelihood 1329.8
AIC (Smaller is Better) 1331.8
AICC (Smaller is Better) 1331.8
BIC (Smaller is Better) 1336.3

Solution for Fixed Effects

Planned

Treatment Pre Trial for anti-Diabetic Standard Period Effect Estimate t Value Pr > |t|treatment2 01 (N) Error Alpha 0.7793 685 <.0001 0.05 Intercept 0.1511 5.16 0.05867 trtpn -0.6006 685 -10.24 <.0001 0.05 trtpn -0.8995 0.06772 685 -13.28 <.0001 0.05 0 trtpn PREOAD2 0.1397 0.05082 685 0.0061 0.05 Metformin 2.75 PREOAD2 Metformin + OAD 0.7857 base log 0.03686 685 21.32 <.0001 0.05


Fasting insulin after 26 weeks of treatment - supportive statistical analysis - full analysis set Parameter Code=INS\_TO\_S

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 0.4825<br>-0.7158<br>-1.0325 | 1.0760<br>-0.4854<br>-0.7666 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | 0.03996 | 0.2395 |
| base log | | | 0.7133 | 0.8581 |

# Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 685 | 92.97 | <.0001 |
| PREOAD2 | 1 | 685 | 7.56 | 0.0061 |
| base log | 1 | 685 | 454.43 | <.0001 |

## Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLi | work.ADATA2 | 3.3323 | 0.03368 | 685 | 98.94 | <.0001 | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | 3.0334 | 0.04766 | 685 | 63.65 | <.0001 | 0.05 |
| trtpn | LSMeans, Lira | WORK.ADATA2 | 3.9329 | 0.04800 | 685 | 81.94 | <.0001 | 0.05 |

# Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | IDegLira | 3.2662 | 3.3984 | 28.0031 | 26.2112 | 29.9174 |
| trtpn | LSMeans, | IDeg | 2.9398 | 3.1270 | 20.7677 | 18.9125 | 22.8049 |
| trtpn | LSMeans, | Lira | 3.8387 | 4.0272 | 51.0568 | 46.4650 | 56.1022 |

# Least Squares Means Estimates

| | | | | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | | Margins | Estimate | Error | DF | t Value | Pr > t |
| trtpn | Treatment ratio. | TDegLira - TDeg | WORK ADATA2 | 0.2989 | 0.05834 | 685 | 5.12 | < .0001 |

# Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | 0.1844 | 0.4135 | 1.3484 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 1.2025 | 1.5120 |

| | -4148<br>Trial Report<br>Il document | CONFIDENTIAL | Vers<br>Statu<br>Page | us: | 329 | 1.0<br>Final<br>of 412 |
|---|---|---|---|---|---|---|
| Fasting | Fasting insulin after 26 weeks of treatment - supportive statistical analysis - full analysis set | | | | | |
| Paramet | er Code=INS_TO_S | | | | | |
| The Mix | ed Procedure | | | | | |
| | | Least Squares Mean | s Estimates | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF t Va | lue Pr > t |
| trtpn | Treatment ratio, IDegI | Lira - Lira WORK.ADATA2 | -0.6006 | 0.05867 | 685 -10 | .24 <.0001 |
| | | Least Squares Means Est | imates | | | |
| Effect | Label | Alpha | Lower | Upper | Exponentia | ted |
| trtpn | Treatment ratio, IDegI | Lira - Lira 0.05 | -0.7158 | -0.4854 | 0.5 | 185 |
| | Least Squ | ares Means Estimates | | | | |
| Effect | Label | Exponentiat<br>Low | | entiated<br>Upper | | |
| trtpn | Treatment ratio, IDegI | Lira - Lira 0.48 | 88 | 0.6154 | | |

Date:

16 December 2019 | Novo Nordisk

NN9068

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIALE | Status: | Final | |
| Statistical document | | Page: | 330 of 412 | |

# 23: Fasting C-peptide after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C74736S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 717

Number of Observations

Number of Observations Read 720 Number of Observations Used 717 Number of Observations Not Used 3

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.2604

Fit Statistics

-2 Res Log Likelihood 1088.9
AIC (Smaller is Better) 1090.9
AICC (Smaller is Better) 1090.9
BIC (Smaller is Better) 1095.4

Solution for Fixed Effects

Planned

Treatment Pre Trial for anti-Diabetic Standard Period Effect Estimate DF t Value Pr > |t| treatment2 01 (N) Error Alpha 0.04809 712 0.0002 0.05 Intercept -0.1787 -3.72 trtpn -0.5435 0.04666 712 -11.65 <.0001 0.05 trtpn -0.8717 0.05399 712 -16.15 <.0001 0.05 0 trtpn PREOAD2 0.1591 712 0.0001 0.05 Metformin 0.04070 3.91 PREOAD2 Metformin + OAD 0.8438 base log 0.04307 712 19.59 <.0001 0.05

# NN9068 | Date: 16 December 2019 | Novo Nordisk NN9068-4148 | Confidential | Version: 1.0 | Status: Final |  |

Fasting C-peptide after 26 weeks of treatment - supportive statistical analysis - full analysis set Parameter Code=C74736S

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | -0.2731<br>-0.6351<br>-0.9777 | -0.08427<br>-0.4519<br>-0.7657 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | 3 | 0.07922 | 0.2391 |
| base log | riccioimill OAD | | 0.7592 | 0.9283 |

# Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 712 | 134.44 | <.0001 |
| PREOAD2 | 1 | 712 | 15.28 | 0.0001 |
| base log | 1 | 712 | 383.88 | <.0001 |

## Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | WORK.ADATA2 | -1.1571 | 0.02694 | 712 | -42.95 | <.0001 | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | -1.4853 | 0.03825 | 712 | -38.83 | <.0001 | 0.05 |
| trtpn | LSMeans, Lira | WORK.ADATA2 | -0.6136 | 0.03808 | 712 | -16.12 | <.0001 | 0.05 |

# Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | IDeg | -1.2100 | -1.1042 | 0.3144 | 0.2982 | 0.3315 |
| trtpn | LSMeans, | | -1.5604 | -1.4102 | 0.2264 | 0.2100 | 0.2441 |
| trtpn | LSMeans, | | -0.6884 | -0.5389 | 0.5414 | 0.5024 | 0.5834 |

# Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | 0.3282 | 0.04678 | 712 | 7.02 | <.0001 |

# Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | 0.2364 | 0.4200 | 1.3885 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 1.2666 | 1.5220 |

| | 4148<br>Frial Report<br>I document | CONFIDENTIAL | Version:<br>Status:<br>Page: | | 1.0<br>inal<br>412 |
|---|---|---|---|---|---|
| Fasting C-peptide after 26 weeks of treatment - supportive statistical analysis - full analysis set | | | | | |
| Paramet | er Code=C74736S | | | | |
| The Mix | ed Procedure | | | | |
| | | Least Squares Mea | ns Estimates | | |
| Effect | Label | Margins | Standa<br>Estimate Err | | Pr > t |
| trtpn | Treatment ratio, IDegLi | ra - Lira WORK.ADATA | 2 -0.5435 0.046 | 66 712 -11.65 | <.0001 |
| | I | east Squares Means Es | timates | | |
| Effect | Label | Alpha | Lower Uppe | r Exponentiated | |
| trtpn | Treatment ratio, IDegLi | ra - Lira 0.05 | -0.6351 -0.451 | 9 0.5807 | |
| | Least Squa | res Means Estimates | | | |
| Effect | Label | Exponentia<br>Lo | ted Exponentiate<br>wer Uppe | | |
| trtpn | Treatment ratio, IDegLi | ra - Lira 0.5 | 299 0.636 | 4 | |

Date:

16 December 2019 | Novo Nordisk

NN9068


Fasting C-peptide after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=CPEPTI\_U

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 717

Number of Observations

Number of Observations Read 720 Number of Observations Used 717 Number of Observations Not Used 3

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.2604

Fit Statistics

-2 Res Log Likelihood 1088.9
AIC (Smaller is Better) 1090.9
AICC (Smaller is Better) 1090.9
BIC (Smaller is Better) 1095.4

Solution for Fixed Effects

Planned Treatment for Period Pre Trial anti-Diabetic Standard 01 (N) Pr > |t| Effect Estimate DF t Value treatment2 Error Alpha Intercept -0.00601 0.04562 712 -0.13 0.8952 0.05 trtpn 1 -0.5435 0.04666 712 -11.65 <.0001 0.05 trtpn 2 -0.8717 0.05399 712 -16.15 <.0001 0.05 trtpn PREOAD2 3 0 0.1591 0.04070 712 3.91 0.0001 0.05 Met.formin PREOAD2 Metformin + OAD 0.8438 0.04307 712 19.59 <.0001 0.05 base log

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Fasting C-peptide after 26 weeks of treatment - supportive statistical analysis - full analysis set Parameter Code=CPEPTI\_U

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | -0.09558<br>-0.6351<br>-0.9777 | 0.08356<br>-0.4519<br>-0.7657 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | Ü | 0.07922 | 0.2391 |
| base log | Meclormin ( OAD | | 0.7592 | 0.9283 |

# Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 712 | 134.44 | <.0001 |
| PREOAD2 | 1 | 712 | 15.28 | 0.0001 |
| base log | 1 | 712 | 383.88 | <.0001 |

## Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | WORK.ADATA2 | -0.05188 | 0.02694 | 712 | -1.93 | 0.0545 | 0.05 |
| trtpn | LSMeans, | | WORK.ADATA2 | -0.3801 | 0.03825 | 712 | -9.94 | <.0001 | 0.05 |
| trtpn | LSMeans, | | WORK.ADATA2 | 0.4917 | 0.03808 | 712 | 12.91 | <.0001 | 0.05 |

## Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | -0.1048 | 0.001007 | 0.9494 | 0.9005 | 1.0010 |
| trtpn | LSMeans, | | -0.4552 | -0.3050 | 0.6838 | 0.6343 | 0.7371 |
| trtpn | LSMeans, | | 0.4169 | 0.5664 | 1.6350 | 1.5172 | 1.7619 |

# Least Squares Means Estimates

| | | | | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | | Margins | Estimate | Error | DF | t Value | Pr > t |
| trtpn | Treatment ratio. | TDegLira - TDeg | WORK ADATA2 | 0.3282 | 0.04678 | 712 | 7.02 | < .0001 |

# Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | 0.2364 | 0.4200 | 1.3885 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 1.2666 | 1.5220 |

| | 4148<br>Frial Report<br>I document | CONFIDENTIAL | Version<br>Status:<br>Page: | | 1.0<br>Final<br>335 of 412 | |
|---|---|---|---|---|---|---|
| Fasting | Fasting C-peptide after 26 weeks of treatment - supportive statistical analysis - full analysis set | | | | | |
| Paramet | Parameter Code=CPEPTI_U | | | | | |
| The Mix | The Mixed Procedure | | | | | |
| | Least Squares Means Estimates | | | | | |
| Effect | Label | Margins | St<br>Estimate | andard<br>Error DF | t Value Pr > t | I |
| trtpn | Treatment ratio, IDegLi | ra - Lira WORK.ADATA | 2 -0.5435 0 | 0.04666 712 | -11.65 <.000 | 1 |
| | I | east Squares Means Es | timates | | | |
| Effect | Label | Alpha | Lower | Upper Expone | entiated | |
| trtpn | Treatment ratio, IDegLi | ra - Lira 0.05 | -0.6351 -0 | 0.4519 | 0.5807 | |
| | Least Squa | res Means Estimates | | | | |
| Effect | Label | Exponentia<br>Lo | | iated<br>Upper | | |
| trtpn | Treatment ratio, IDegLi | ra - Lira 0.5 | 5299 0 | 0.6364 | | |

Date:

16 December 2019 | Novo Nordisk

NN9068
| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIALE | Status: | Final | |
| Statistical document | | Page: | 336 of 412 | |

## 24: Fasting glucagon after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C74859P

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 716

Number of Observations

Number of Observations Read 720
Number of Observations Used 716
Number of Observations Not Used 4

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.2508

Fit Statistics

-2 Res Log Likelihood 1061.4
AIC (Smaller is Better) 1063.4
AICC (Smaller is Better) 1063.4
BIC (Smaller is Better) 1068.0

Solution for Fixed Effects

Planned

Treatment Pre Trial for anti-Diabetic Standard Period Effect Estimate DF t Value Pr > |t| treatment2 01 (N) Error Alpha 0.09730 <.0001 711 18.56 0.05 Intercept 1.8063 -0.03470 trtpn 0.04578 711 -0.76 0.4487 0.05 trtpn 0.02292 0.05309 711 0.43 0.6661 0.05 trtpn PREOAD2 0.06368 711 0.1122 0.05 Metformin 0.04004 1.59 PREOAD2 Metformin + OAD 0.4190 base log 0.02777 711 15.09 <.0001 0.05

## NN9068 NN9068-4148 Clinical Trial Report Statistical document Date: 16 December 2019 Version: 1.0 Status: Final 

Fasting glucagon after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C74859P

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.6153<br>-0.1246<br>-0.08132 | 1.9973<br>0.05519<br>0.1272 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -0.01494 | 0.1423 |
| base_log | | | 0.3645 | 0.4736 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 711 | 0.85 | 0.4276 |
| PREOAD2 | 1 | 711 | 2.53 | 0.1122 |
| base log | 1 | 711 | 227.65 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | WORK.ADATA2 | 3.1465 | 0.02643 | 711 | 119.04 | <.0001 | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | 3.2042 | 0.03766 | 711 | 85.08 | <.0001 | 0.05 |
| trtpn | LSMeans, Lira | WORK.ADATA2 | 3.1812 | 0.03737 | 711 | 85.13 | <.0001 | 0.05 |

### Least Squares Means Estimates

| Effect | Label | Lower | Upper | Exponentiated | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|---|---|
| trtpn | LSMeans, | 3.0946 | 3.1984 | 23.2554 | 22.0793 | 24.4942 |
| trtpn | LSMeans, | 3.1302 | 3.2781 | 24.6348 | 22.8790 | 26.5253 |
| trtpn | LSMeans, | 3.1079 | 3.2546 | 24.0766 | 22.3734 | 25.9094 |

### Least Squares Means Estimates

| | | | | | | Standard | L . | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Label | | | Margins | Estimate | Error | DF | t Value | Pr > t |
| trtnn | Treatment ratio | TDegLira - | TDea | WORK ADATA? | -0 05762 | 0 04601 | 711 | -1 25 | 0 2108 |

#### Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | -0.1479 | 0.03270 | 0.9440 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.8625 | 1.0332 |

| | 4148<br>Frial Report<br>I document | CONFIDENTIA | Versi<br>Statu<br>Page | ıs: | | 1.0<br>nal<br>112 |
|---|---|---|---|---|---|---|
| Fasting | glucagon after 26 weeks | of treatment - supp | ortive statist | ical analys | sis - full ana | ysis set |
| Parameter Code=C74859P | | | | | | |
| The Mix | The Mixed Procedure | | | | | |
| | Least Squares Means Estimates | | | | | |
| Effect | Label | Margins | Estimate | Standard<br>Error | DF t Value | Pr > t |
| trtpn | Treatment ratio, IDegLi | ra - Lira WORK.ADAT | A2 -0.03470 | 0.04578 | 711 -0.76 | 0.4487 |
| | I | east Squares Means E | stimates | | | |
| Effect | Label | Alpha | Lower | Upper | Exponentiated | |
| trtpn | Treatment ratio, IDegLi | ra - Lira 0.05 | -0.1246 | 0.05519 | 0.9659 | |
| | Least Squa | res Means Estimates | | | | |
| Effect | Label | Exponenti<br>L | ated Expone<br>ower | ntiated<br>Upper | | |
| trtpn | Treatment ratio, IDegLi | ra - Lira 0. | 8829 | 1.0567 | | |

Date:

16 December 2019 | Novo Nordisk

NN9068

NN9068
NN9068-4148
Clinical Trial Report
Statistical document

Date: 16 December 2019
Version: 1.0
Status: Final


### 25: HOMA-B after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=HOMA BCS

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 690

Number of Observations

Number of Observations Read 720 Number of Observations Used 690 Number of Observations Not Used 30

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.3530

Fit Statistics

-2 Res Log Likelihood 1257.7
AIC (Smaller is Better) 1259.7
AICC (Smaller is Better) 1259.7
BIC (Smaller is Better) 1264.2

Solution for Fixed Effects

Planned

Treatment Pre Trial for anti-Diabetic Standard Period Effect Estimate t Value Pr > |t| treatment2 01 (N) Error DF Alpha <.0001 0.05 Intercept 1.9156 0.1653 685 11.59 -0.02107 trtpn 0.05561 685 -0.38 0.7049 0.05 trtpn -0.3761 0.06411 685 -5.87 < .0001 0.05 3 0 trtpn PREOAD2 0.2495 Metformin 0.04821 685 5.18 <.0001 0.05 PREOAD2 Metformin + OAD 0.6704 base log 0.03092 685 21.68 <.0001 0.05

## NN9068 | Date: 16 December 2019 | Novo Nordisk NN9068-4148 | CONFIDENTIAL | Version: 1.0 | Clinical Trial Report | Status: Final |  |

HOMA-B after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=HOMA\_BCS

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.5911<br>-0.1303<br>-0.5020 | 2.2402<br>0.08811<br>-0.2503 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | 0.1549 | 0.3442 |
| base_log | 1100101111 / 0/10 | | 0.6097 | 0.7311 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 685 | 24.13 | <.0001 |
| PREOAD2 | 1 | 685 | 26.79 | <.0001 |
| base log | 1 | 685 | 470.21 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, I | IDeģ | WORK.ADATA2 | 5.4547 | 0.03195 | 685 | 170.72 | <.0001 | 0.05 |
| trtpn | LSMeans, I | | WORK.ADATA2 | 5.0996 | 0.04518 | 685 | 112.88 | <.0001 | 0.05 |
| trtpn | LSMeans, I | | WORK.ADATA2 | 5.4757 | 0.04548 | 685 | 120.41 | <.0001 | 0.05 |

#### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | 5.3919 | 5.5174 | 233.85 | 219.63 | 248.99 |
| trtpn | LSMeans, | | 5.0109 | 5.1883 | 163.96 | 150.04 | 179.16 |
| trtpn | LSMeans, | | 5.3865 | 5.5650 | 238.83 | 218.43 | 261.13 |

### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | 0.3551 | 0.05533 | 685 | 6.42 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | Alpha | Lower | Upper | Exponentiated | |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | 0.2464 | 0.4637 | 1.4263 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio | , IDegLira - IDeg | 1.2795 | 1.5900 |

| NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Version:<br>Status:<br>Page: | 1.0<br>Final<br>341 of 412 | |
|---|---|---|---|---|
| HOMA-B after 26 weeks of treatment - supportive statistical analysis - full analysis set | | | | |
| Parameter Code=HOMA_BCS | | | | |
| The Mixed Procedure | | | | |
| Least Squares Means Estimates | | | | |
| Effect Label | Margins Estin | Standard<br>nate Error | DF t Value Pi | c > t |
| trtpn Treatment ratio, IDegLi | ra - Lira WORK.ADATA2 -0.02 | 2107 0.05561 | 685 -0.38 | 0.7049 |
| L | east Squares Means Estimates | | | |
| Effect Label | Alpha Lower | Upper | Exponentiated | |
| trtpn Treatment ratio, IDegLi | ra - Lira 0.05 -0.1303 | 0.08811 | 0.9791 | |
| Least Squa | res Means Estimates | | | |
| Effect Label | Exponentiated E<br>Lower | Exponentiated<br>Upper | | |
| trtpn Treatment ratio, IDegLi | ra - Lira 0.8779 | 1.0921 | | |

Date:

16 December 2019 | Novo Nordisk

NN9068

NN9068 Date: 16 December 2019 Novo Nordisk

NN9068-4148 Version: 1.0
Clinical Trial Report Status: Final
Statistical document 

## 26: HDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C105587S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used 2

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.02087

Fit Statistics

-2 Res Log Likelihood -710.3
AIC (Smaller is Better) -708.3
AICC (Smaller is Better) -708.3
BIC (Smaller is Better) -703.8

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect Estimate t Value Pr > |t| treatment2 01 (N) Error DF Alpha 3.54 0.0004 0.05 Intercept 0.04221 0.01193 713 trtpn -0.00377 0.01320 713 -0.29 0.7751 0.6777 0.05 trtpn 0.006356 0.01529 713 0.42 0.05 3 trtpn PREOAD2 -0.03054 Metformin 0.01155 713 -2.64 0.0084 0.05 PREOAD2 Metformin + OAD 0.8509 base log 0.02184 713 38.97 <.0001 0.05

## NN9068 NN9068-4148 Clinical Trial Report Statistical document Date: 16 December 2019 Version: 1.0 Status: Final 

HDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C105587S

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 0.01879<br>-0.02970<br>-0.02365 | 0.06564<br>0.02215<br>0.03637 |
| PREOAD2<br>PREOAD2<br>base log | Metformin<br>Metformin + OAD | | -0.05321<br>0.8080 | -0.00787<br>0.8937 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 713 | 0.29 | 0.7458 |
| PREOAD2 | 1 | 713 | 7.00 | 0.0084 |
| base log | 1 | 713 | 1518.36 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, I | IDeğ | WORK.ADATA2 | 0.1331 | 0.007616 | 713 | 17.47 | <.0001 | 0.05 |
| trtpn | LSMeans, I | | WORK.ADATA2 | 0.1432 | 0.01083 | 713 | 13.22 | <.0001 | 0.05 |
| trtpn | LSMeans, I | | WORK.ADATA2 | 0.1368 | 0.01078 | 713 | 12.69 | <.0001 | 0.05 |

## Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | 0.1181 | 0.1480 | 1.1423 | 1.1254 | 1.1595 |
| trtpn | LSMeans, | | 0.1219 | 0.1644 | 1.1539 | 1.1297 | 1.1787 |
| trtpn | LSMeans, | | 0.1157 | 0.1580 | 1.1466 | 1.1226 | 1.1712 |

### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | -0.01013 | 0.01324 | 713 | -0.77 | 0.4444 |

#### Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | -0.03612 | 0.01586 | 0.9899 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio | , IDegLira - IDeg | 0.9645 | 1.0160 |

| NN9068-4148<br>Clinical Trial Report<br>Statistical document | | CONFIDEN | TIAL | Version:<br>Status:<br>Page: | | 1.0<br>nal<br>112 |
|---|---|---|---|---|---|---|
| HDL cho | HDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set | | | | | |
| Parameter Code=C105587S | | | | | | |
| The Mixed Procedure | | | | | | |
| Least Squares Means Estimates | | | | | | |
| Effect | Label | Margin | s Estimat | Standard<br>te Error | DF t Value | Pr > t |
| trtpn | Treatment ratio, IDe | egLira - Lira WORK.A | DATA2 -0.0037 | 77 0.01320 | 713 -0.29 | 0.7751 |
| | | Least Squares Mean | s Estimates | | | |
| Effect | Label | Alpha | Lower | Upper | Exponentiated | |
| trtpn | Treatment ratio, IDe | egLira - Lira 0.05 | -0.02970 | 0.02215 | 0.9962 | |
| | Least S | Squares Means Estimat | es | | | |
| Effect | Label | Expone | ntiated Exp<br>Lower | oonentiated<br>Upper | | |
| trtpn | Treatment ratio, IDe | egLira - Lira | 0.9707 | 1.0224 | | |

Date:

16 December 2019 | Novo Nordisk

NN9068

## NN9068 | Date: 16 December 2019 | Novo Nordisk NN9068-4148 | CONFIDENTIAL | Version: 1.0 | Clinical Trial Report | Status: Final | Statistical document |  |

HDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=HDL SU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used 2

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.02087

Fit Statistics

-2 Res Log Likelihood -710.3
AIC (Smaller is Better) -708.3
AICC (Smaller is Better) -708.3
BIC (Smaller is Better) -703.8

Solution for Fixed Effects

Planned Treatment for Period Pre Trial anti-Diabetic Standard 01 (N) Effect Estimate DF t Value Pr > |t| treatment2 Error Alpha Intercept 0.5871 0.08405 713 6.99 <.0001 0.05 trtpn 1 -0.00377 0.01320 713 -0.29 0.7751 0.05 trtpn 2 0.006356 0.01529 713 0.42 0.6777 0.05 trtpn PREOAD2 0 -0.03054 0.01155 713 -2.64 0.0084 0.05 Met.formin PREOAD2 Metformin + OAD 0.8509 0.02184 713 38.97 <.0001 0.05 base log

## NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

 $\label{eq:hdl_substitute} \mbox{HDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set} \\ \mbox{Parameter Code=HDL\_SU}$ 

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 0.4221<br>-0.02970<br>-0.02365 | 0.7521<br>0.02215<br>0.03637 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -0.05321 | -0.00787 |
| base log | | | 0.8080 | 0.8937 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 713 | 0.29 | 0.7458 |
| PREOAD2 | 1 | 713 | 7.00 | 0.0084 |
| base log | 1 | 713 | 1518.36 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | IDeğ | WORK.ADATA2 | 3.7866 | 0.007616 | 713 | 497.19 | <.0001 | 0.05 |
| trtpn | LSMeans, | | WORK.ADATA2 | 3.7967 | 0.01083 | 713 | 350.56 | <.0001 | 0.05 |
| trtpn | LSMeans, | | WORK.ADATA2 | 3.7903 | 0.01078 | 713 | 351.64 | <.0001 | 0.05 |

#### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | 3.7716 | 3.8015 | 44.1045 | 43.4500 | 44.7690 |
| trtpn | LSMeans, | | 3.7754 | 3.8180 | 44.5536 | 43.6163 | 45.5111 |
| trtpn | LSMeans, | | 3.7692 | 3.8115 | 44.2713 | 43.3443 | 45.2182 |

### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | -0.01013 | 0.01324 | 713 | -0.77 | 0.4444 |

#### Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | -0.03612 | 0.01586 | 0.9899 |

| Effect | Label | | | | | Exponentiated<br>Lower | Exp | onentiated<br>Upper |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment | ratio, | IDegLira | _ | IDea | 0.9645 | | 1.0160 |

| | -4148<br>Гrial Report<br>I document | CONFIDENTIAL | Version:<br>Status:<br>Page: | 1.0<br>Final<br>347 of 412 |
|---|---|---|---|---|
| HDL cho | lesterol after 26 weeks | of treatment - support | tive statistical analy | ysis – full analysis set |
| Parameter Code=HDL_SU | | | | |
| The Mixed Procedure | | | | |
| Least Squares Means Estimates | | | | |
| Effect | Label | Margins | Standard<br>Estimate Error | DF t Value Pr > t |
| trtpn | Treatment ratio, IDegL: | ira - Lira WORK.ADATA2 | 2 -0.00377 0.01320 | 713 -0.29 0.7751 |
| | : | Least Squares Means Est | timates | |
| Effect | Label | Alpha | Lower Upper | Exponentiated |
| trtpn | Treatment ratio, IDegL | ira - Lira 0.05 - | -0.02970 0.02215 | 0.9962 |
| | Least Squa | ares Means Estimates | | |
| Effect | Label | Exponentiat<br>Lov | ted Exponentiated<br>wer Upper | |
| trtpn | Treatment ratio, IDegL | ira - Lira 0.9 | 707 1.0224 | |

NN9068

Date:

16 December 2019 | Novo Nordisk

NN9068
NN9068-4148
Clinical Trial Report
Statistical document

Date: 16 December 2019
Version: 1.0
Status: Final


## 27: LDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C105588S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 717

Number of Observations

Number of Observations Read 720 Number of Observations Used 717 Number of Observations Not Used 3

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.09670

Fit Statistics

-2 Res Log Likelihood 383.1
AIC (Smaller is Better) 385.1
AICC (Smaller is Better) 385.1
BIC (Smaller is Better) 389.7

Solution for Fixed Effects

Planned

Treatment Pre Trial for anti-Diabetic Standard Period Effect Estimate t Value Pr > |t| treatment2 01 (N) Error Alpha 7.56 0.05 Intercept 0.2751 0.03638 712 <.0001 -0.04478 trtpn 0.02840 712 -1.58 0.1153 0.05 trtpn 0.01832 0.03293 712 0.56 0.5783 0.05 3 0 trtpn PREOAD2 0.001663 Metformin 0.02477 712 0.07 0.9465 0.05 PREOAD2 Metformin + OAD base log 0.6341 0.03134 712 20.24 <.0001 0.05

## NN9068 | Date: 16 December 2019 | Novo Nordisk NN9068-4148 | CONFIDENTIAL | Version: 1.0 | Clinical Trial Report | Status: Final |  |

LDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C105588S

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 0.2037<br>-0.1005<br>-0.04634 | 0.3465<br>0.01098<br>0.08297 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -0.04697 | 0.05030 |
| base log | | | 0.5726 | 0.6956 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 712 | 2.84 | 0.0593 |
| PREOAD2 | 1 | 712 | 0.00 | 0.9465 |
| base log | 1 | 712 | 409.47 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, II | Değ | WORK.ADATA2 | 0.7677 | 0.01642 | 712 | 46.75 | <.0001 | 0.05 |
| trtpn | LSMeans, II | | WORK.ADATA2 | 0.8308 | 0.02336 | 712 | 35.57 | <.0001 | 0.05 |
| trtpn | LSMeans, L | | WORK.ADATA2 | 0.8125 | 0.02318 | 712 | 35.05 | <.0001 | 0.05 |

#### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | 0.7354 | 0.7999 | 2.1548 | 2.0864 | 2.2254 |
| trtpn | LSMeans, | | 0.7849 | 0.8766 | 2.2951 | 2.1922 | 2.4028 |
| trtpn | LSMeans, | | 0.7669 | 0.8580 | 2.2534 | 2.1532 | 2.3584 |

### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | -0.06309 | 0.02858 | 712 | -2.21 | 0.0276 |

#### Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | -0.1192 | -0.00698 | 0.9389 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.8876 | 0.9930 |

| | 4148<br>Frial Report<br>I document | CONFID | ENTIAL | Version:<br>Status:<br>Page: | | 1.0<br>nal<br>412 |
|---|---|---|---|---|---|---|
| LDL cho | LDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set | | | | | |
| Paramet | Parameter Code=C105588S | | | | | |
| The Mix | ed Procedure | | | | | |
| Least Squares Means Estimates | | | | | | |
| Effect | Label | Marg | ins Estima | Standard<br>te Error | DF t Value | Pr > t |
| trtpn | Treatment ratio, IDe | gLira - Lira WORK | .ADATA2 -0.044 | 78 0.02840 | 712 -1.58 | 0.1153 |
| | | Least Squares Me | ans Estimates | | | |
| Effect | Label | Alp | ha Lower | Upper | Exponentiated | |
| trtpn | Treatment ratio, IDe | gLira - Lira 0. | 05 -0.1005 | 0.01098 | 0.9562 | |
| | Least So | quares Means Estim | ates | | | |
| Effect | Label | Expo | nentiated Exp | ponentiated<br>Upper | | |
| trtpn | Treatment ratio, IDe | gLira - Lira | 0.9044 | 1.0110 | | |

Date:

16 December 2019 | Novo Nordisk

NN9068


LDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=LDL SU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 717

Number of Observations

Number of Observations Read 720 Number of Observations Used 717 Number of Observations Not Used 3

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.09670

Fit Statistics

-2 Res Log Likelihood 383.1
AIC (Smaller is Better) 385.1
AICC (Smaller is Better) 385.1
BIC (Smaller is Better) 389.7

Solution for Fixed Effects

Planned Treatment for Period Pre Trial anti-Diabetic Standard 01 (N) Effect Estimate t Value Pr > |t| treatment2 Error DF Alpha Intercept 1.6119 0.1434 712 11.24 <.0001 0.05 trtpn 1 -0.04478 0.02840 712 -1.58 0.1153 0.05 trtpn 2 0.01832 0.03293 712 0.56 0.5783 0.05 trtpn PREOAD2 0 0.001663 0.02477 712 0.07 0.9465 0.05 Met.formin PREOAD2 Metformin + OAD 0.6341 0.03134 712 20.24 <.0001 0.05 base log

## NN9068 NN9068-4148 Clinical Trial Report Statistical document Date: 16 December 2019 Version: 1.0 Status: Final 

 $\label{local_local_local_local_local} \mbox{LDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set} \\ \mbox{Parameter Code=LDL\_SU}$ 

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.3303<br>-0.1005<br>-0.04634 | 1.8935<br>0.01098<br>0.08297 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -0.04697 | 0.05030 |
| base log | | | 0.5726 | 0.6956 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 712 | 2.84 | 0.0593 |
| PREOAD2 | 1 | 712 | 0.00 | 0.9465 |
| base log | 1 | 712 | 409.47 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, ID | )eg | WORK.ADATA2 | 4.4212 | 0.01642 | 712 | 269.25 | <.0001 | 0.05 |
| trtpn | LSMeans, ID | | WORK.ADATA2 | 4.4843 | 0.02336 | 712 | 191.97 | <.0001 | 0.05 |
| trtpn | LSMeans, Li | | WORK.ADATA2 | 4.4660 | 0.02318 | 712 | 192.65 | <.0001 | 0.05 |

#### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | 4.3889 | 4.4534 | 83.1951 | 80.5558 | 85.9209 |
| trtpn | LSMeans, | | 4.4384 | 4.5301 | 88.6134 | 84.6413 | 92.7718 |
| trtpn | LSMeans, | | 4.4205 | 4.5115 | 87.0051 | 83.1340 | 91.0566 |

### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | -0.06309 | 0.02858 | 712 | -2.21 | 0.0276 |

#### Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | -0.1192 | -0.00698 | 0.9389 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.8876 | 0.9930 |

| NN9068-4148<br>Clinical Trial Report<br>Statistical document | | CC | ONFIDENTIAL | Sta | ersion:<br>atus:<br>ge: | F<br>353 of | 1.0<br>inal<br>412 |
|---|---|---|---|---|---|---|---|
| LDL cho | LDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set | | | | | | |
| Paramet | er Code=LDL_SU | | | | | | |
| The Mix | The Mixed Procedure | | | | | | |
| Least Squares Means Estimates | | | | | | | |
| Effect | Label | | Margins | Estimate | Standard<br>Error | DF t Value | Pr > t |
| trtpn | Treatment ratio, | IDegLira - Lira | WORK.ADATA2 | -0.04478 | 0.02840 | 712 -1.58 | 0.1153 |
| | | Least Squar | es Means Esti | mates | | | |
| Effect | Label | | Alpha | Lower | Upper | Exponentiated | |
| trtpn | Treatment ratio, | IDegLira - Lira | 0.05 - | 0.1005 | 0.01098 | 0.9562 | |
| | Lea | st Squares Means | Estimates | | | | |
| Effect | Label | | Exponentiate<br>Lowe | | nentiated<br>Upper | | |
| trtpn | Treatment ratio, | IDegLira - Lira | 0.904 | 4 | 1.0110 | | |

NN9068

Date:

16 December 2019 | Novo Nordisk

NN9068 Date: 16 December 2019 Vovo Nordisk
NN9068-4148 Version: 1.0
Clinical Trial Report Status: Final
Statistical document 

### 28: VLDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C105589S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used 2

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.1590

Fit Statistics

-2 Res Log Likelihood 739.1
AIC (Smaller is Better) 741.1
AICC (Smaller is Better) 741.1
BIC (Smaller is Better) 745.6

Solution for Fixed Effects

Planned

Treatment Pre Trial for anti-Diabetic Period Standard Effect Estimate t Value Pr > |t| treatment2 01 (N) Error DF Alpha 0.05 Intercept -0.1589 0.03205 713 -4.96 <.0001 trtpn -0.05191 0.03644 713 -1.42 0.1547 0.05 trtpn -0.1175 0.04219 713 -2.790.0055 0.05 3 0 trtpn PREOAD2 0.07176 Metformin 0.03185 713 2.25 0.0246 0.05 PREOAD2 Metformin + OAD base log 0.6564 0.02753 713 23.84 <.0001 0.05

## NN9068 | Date: 16 December 2019 | Novo Nordisk NN9068-4148 | CONFIDENTIAL | Version: 1.0 | Clinical Trial Report | Status: Final |  |

VLDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C105589S

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | -0.2218<br>-0.1235<br>-0.2003 | -0.09595<br>0.01963<br>-0.03468 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | Ü | 0.009229 | 0.1343 |
| base log | MECTOTHILL + OAD | | 0.6024 | 0.7105 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 713 | 3.90 | 0.0206 |
| PREOAD2 | 1 | 713 | 5.08 | 0.0246 |
| base log | 1 | 713 | 568.38 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | WORK.ADATA2 | -0.3405 | 0.02102 | 713 | -16.20 | <.0001 | 0.05 |
| trtpn | LSMeans, | | WORK.ADATA2 | -0.4061 | 0.02989 | 713 | -13.58 | <.0001 | 0.05 |
| trtpn | LSMeans, | | WORK.ADATA2 | -0.2885 | 0.02975 | 713 | -9.70 | <.0001 | 0.05 |

#### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | IDeg | -0.3817 | -0.2992 | 0.7114 | 0.6827 | 0.7414 |
| trtpn | LSMeans, | | -0.4647 | -0.3474 | 0.6663 | 0.6283 | 0.7065 |
| trtpn | LSMeans, | | -0.3470 | -0.2301 | 0.7493 | 0.7068 | 0.7944 |

### Least Squares Means Estimates

| | | | | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | | Margins | Estimate | Error | DF | t Value | Pr > t |
| trtpn | Treatment ratio. | TDeqLira - TDeq | WORK ADATA2 | 0.06560 | 0.03654 | 713 | 1.80 | 0.0730 |

#### Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | -0.00614 | 0.1373 | 1.0678 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.9939 | 1.1472 |

| | -4148<br>Гrial Report<br>I document | CONFIDENTIAL | Version:<br>Status:<br>Page: | 1<br>Fin<br>356 of 41 | ** |
|---|---|---|---|---|---|
| VLDL ch | VLDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set | | | | |
| Parameter Code=C105589S | | | | | |
| The Mixed Procedure | | | | | |
| Least Squares Means Estimates | | | | | |
| Effect | Label | Margins | Standard<br>Estimate Error | - | Pr > t |
| trtpn | Treatment ratio, IDegLi | ra - Lira WORK.ADATA2 | 2 -0.05191 0.0364 | 713 -1.42 | 0.1547 |
| | I | east Squares Means Est | timates | | |
| Effect | Label | Alpha | Lower Upper | Exponentiated | |
| trtpn | Treatment ratio, IDegLi | ra - Lira 0.05 | -0.1235 0.01963 | 0.9494 | |
| | Least Squa | res Means Estimates | | | |
| Effect | Label | Exponentiat<br>Lov | ted Exponentiated<br>wer Upper | | |
| trtpn | Treatment ratio, IDegLi | ra - Lira 0.88 | 1.0198 | | |

NN9068

Date:

16 December 2019 | Novo Nordisk


VLDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=VLDL\_SU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used 2

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.1590

Fit Statistics

-2 Res Log Likelihood 739.1
AIC (Smaller is Better) 741.1
AICC (Smaller is Better) 741.1
BIC (Smaller is Better) 745.6

Solution for Fixed Effects

Planned Treatment for Period Pre Trial anti-Diabetic Standard 01 (N) Effect Estimate t Value Pr > |t|treatment2 Error DF Alpha Intercept 1.0964 0.09974 713 10.99 <.0001 0.05 trtpn 1 -0.05191 0.03644 713 -1.42 0.1547 0.05 trtpn 2 -0.1175 0.04219 713 -2.79 0.0055 0.05 trtpn PREOAD2 3 0 0.07176 0.03185 713 2.25 0.0246 0.05 Met.formin PREOAD2 Metformin + OAD 0.6564 0.02753 713 23.84 <.0001 0.05 base log

## NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

VLDL cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=VLDL\_SU

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 0.9006<br>-0.1235<br>-0.2003 | 1.2922<br>0.01963<br>-0.03468 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | 0.009229 | 0.1343 |
| base log | IICCIOIMIII / OID | | 0.6024 | 0.7105 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 713 | 3.90 | 0.0206 |
| PREOAD2 | 1 | 713 | 5.08 | 0.0246 |
| base log | 1 | 713 | 568.38 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | WORK.ADATA2 | 3.3131 | 0.02102 | 713 | 157.61 | <.0001 | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | 3.2475 | 0.02989 | 713 | 108.63 | <.0001 | 0.05 |
| trtpn | LSMeans, Lira | WORK.ADATA2 | 3.3650 | 0.02975 | 713 | 113.11 | <.0001 | 0.05 |

#### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | 3.2718 | 3.3543 | 27.4688 | 26.3583 | 28.6262 |
| trtpn | LSMeans, | | 3.1888 | 3.3061 | 25.7247 | 24.2584 | 27.2797 |
| trtpn | LSMeans, | | 3.3066 | 3.4234 | 28.9324 | 27.2909 | 30.6726 |

### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | 0.06560 | 0.03654 | 713 | 1.80 | 0.0730 |

#### Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | -0.00614 | 0.1373 | 1.0678 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.9939 | 1.1472 |

| NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Version:<br>Status:<br>Page: | 1.0<br>Final<br>359 of 412 |
|---|---|---|---|
| VLDL cholesterol after 26 weeks | of treatment - supportive st | atistical analysis | - full analysis set |
| Parameter Code=VLDL_SU | | | |
| The Mixed Procedure | | | |
| Least Squares Means Estimates | | | |
| Effect Label | Margins Estim | Standard<br>ate Error | DF t Value Pr > t |
| trtpn Treatment ratio, IDegL: | ra - Lira WORK.ADATA2 -0.05 | 191 0.03644 7 | 13 -1.42 0.1547 |
| 1 | east Squares Means Estimates | | |
| Effect Label | Alpha Lower | Upper Ex | ponentiated |
| trtpn Treatment ratio, IDegL: | ra - Lira 0.05 -0.1235 | 0.01963 | 0.9494 |
| Least Squa | res Means Estimates | | |
| Effect Label | Exponentiated E<br>Lower | xponentiated<br>Upper | |
| trtpn Treatment ratio, IDegLi | ra - Lira 0.8839 | 1.0198 | |

NN9068

Date:

16 December 2019 | Novo Nordisk

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIALE | Status: | Final | |
| Statistical document | | Page: | 360 of 412 | |

### 29: Triglycerides after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C64812S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used 2

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.1843

Fit Statistics

-2 Res Log Likelihood 844.6
AIC (Smaller is Better) 846.6
AICC (Smaller is Better) 846.6
BIC (Smaller is Better) 851.2

Solution for Fixed Effects

Planned

Treatment Pre Trial for anti-Diabetic Standard Period Effect Estimate DF t Value Pr > |t| treatment2 01 (N) Error Alpha 0.03729 713 3.12 0.0019 0.05 Intercept 0.1162 -0.05449 trtpn 0.03922 713 -1.39 0.1652 0.05 trtpn -0.1254 0.04541 713 -2.76 0.0059 0.05 0 trtpn PREOAD2 0.07324 713 0.0333 0.05 Metformin 0.03435 2.13 PREOAD2 Metformin + OAD 0.6416 base log 0.02615 713 24.54 <.0001 0.05

## NN9068 NN9068-4148 Clinical Trial Report Statistical document Date: 16 December 2019 Version: 1.0 Status: Final 

Triglycerides after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C64812S

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 0.04296<br>-0.1315<br>-0.2145 | 0.1894<br>0.02252<br>-0.03622 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | 0.005797 | 0.1407 |
| base log | | | 0.5902 | 0.6929 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 713 | 3.84 | 0.0219 |
| PREOAD2 | 1 | 713 | 4.55 | 0.0333 |
| base log | 1 | 713 | 601.98 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, I | I Değ | WORK.ADATA2 | 0.4647 | 0.02263 | 713 | 20.53 | <.0001 | 0.05 |
| trtpn | LSMeans, I | | WORK.ADATA2 | 0.3938 | 0.03218 | 713 | 12.24 | <.0001 | 0.05 |
| trtpn | LSMeans, I | | WORK.ADATA2 | 0.5191 | 0.03202 | 713 | 16.21 | <.0001 | 0.05 |

### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | 0.4202 | 0.5091 | 1.5915 | 1.5223 | 1.6638 |
| trtpn | LSMeans, | | 0.3306 | 0.4570 | 1.4826 | 1.3918 | 1.5793 |
| trtpn | LSMeans, | | 0.4563 | 0.5820 | 1.6806 | 1.5782 | 1.7896 |

### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | 0.07089 | 0.03934 | 713 | 1.80 | 0.0720 |

#### Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | -0.00635 | 0.1481 | 1.0735 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.9937 | 1.1597 |

| | 4148<br>Frial Report<br>I document | CONFIDENTIAL | Version:<br>Status:<br>Page: | 1.0<br>Final<br>362 of 412 | |
|---|---|---|---|---|---|
| Triglyc | erides after 26 weeks of | treatment - supportiv | e statistical analysi | s - full analysis set | |
| Paramet | er Code=C64812S | | | | |
| The Mix | ed Procedure | | | | |
| | | Least Squares Mean | s Estimates | | |
| Effect | Label | Margins | Estimate Standard Error | DF t Value Pr > t | .1 |
| trtpn | Treatment ratio, IDegLi | ra - Lira WORK.ADATA2 | -0.05449 0.03922 | 713 -1.39 0.165 | 2 |
| | I | east Squares Means Est | imates | | |
| Effect | Label | Alpha | Lower Upper | Exponentiated | |
| trtpn | Treatment ratio, IDegLi | ra - Lira 0.05 | -0.1315 0.02252 | 0.9470 | |
| | Least Squa | res Means Estimates | | | |
| Effect | Label | Exponentiat<br>Low | | | |
| trtpn | Treatment ratio, IDegLi | ra - Lira 0.87 | 68 1.0228 | | |

NN9068

Date:

16 December 2019 | Novo Nordisk

## NN9068 NN9068-4148 Clinical Trial Report Statistical document Date: 16 December 2019 Version: 1.0 Status: Final 

Triglycerides after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=TRIG\_SU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used 2

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.1843

Fit Statistics

-2 Res Log Likelihood 844.6
AIC (Smaller is Better) 846.6
AICC (Smaller is Better) 846.6
BIC (Smaller is Better) 851.2

Solution for Fixed Effects

Planned Treatment for Period Pre Trial anti-Diabetic Standard 01 (N) Effect Estimate t Value Pr > |t| treatment2 Error DF Alpha Intercept 1.7251 0.1372 713 12.58 < .0001 0.05 trtpn 1 -0.05449 0.03922 713 -1.39 0.1652 0.05 trtpn 2 -0.1254 0.04541 713 -2.76 0.0059 0.05 trtpn PREOAD2 3 0 0.07324 0.03435 713 2.13 0.0333 0.05 Met.formin PREOAD2 Metformin + OAD 0.6416 0.02615 713 24.54 <.0001 0.05 base log

## NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Triglycerides after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=TRIG\_SU
The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.4558<br>-0.1315<br>-0.2145 | 1.9944<br>0.02252<br>-0.03622 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | - | 0.005797 | 0.1407 |
| base log | IICCICIMIII I OIID | | 0.5902 | 0.6929 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 713 | 3.84 | 0.0219 |
| PREOAD2 | 1 | 713 | 4.55 | 0.0333 |
| base log | 1 | 713 | 601.98 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | IDeg | WORK.ADATA2 | 4.9533 | 0.02263 | 713 | 218.87 | <.0001 | 0.05 |
| trtpn | LSMeans, | | WORK.ADATA2 | 4.8824 | 0.03218 | 713 | 151.71 | <.0001 | 0.05 |
| trtpn | LSMeans, | | WORK.ADATA2 | 5.0078 | 0.03202 | 713 | 156.38 | <.0001 | 0.05 |

#### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | 4.9089 | 4.9977 | 141.64 | 135.49 | 148.08 |
| trtpn | LSMeans, | | 4.8192 | 4.9456 | 131.95 | 123.87 | 140.55 |
| trtpn | LSMeans, | | 4.9449 | 5.0707 | 149.57 | 140.46 | 159.28 |

### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | 0.07089 | 0.03934 | 713 | 1.80 | 0.0720 |

#### Least Squares Means Estimates

| Effect | Label | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|
| trtpn | Treatment ratio, IDegLira - IDeg | 0.05 | -0.00635 | 0.1481 | 1.0735 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.9937 | 1.1597 |

| | -4148<br>Frial Report | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019 1.0 Final 365 of 412 | Novo Nordisk |
|---|---|---|---|---|---|
| Triglyc | erides after 26 weeks of tre | eatment - supportive | statistical analysi | s - full analysis se | t |
| Paramet | er Code=TRIG_SU | | | | |
| The Mix | ed Procedure | | | | |
| | | Least Squares Means | Estimates | | |
| Effect | Label | Margins | Estimate Standard Error | DF t Value Pr | > t |
| trtpn | Treatment ratio, IDegLira - | - Lira WORK.ADATA2 | -0.05449 0.03922 | 713 -1.39 0 | .1652 |
| | Least | : Squares Means Esti | mates | | |
| Effect | Label | Alpha | Lower Upper | Exponentiated | |
| trtpn | Treatment ratio, IDegLira - | - Lira 0.05 - | 0.1315 0.02252 | 0.9470 | |
| | Least Squares | Means Estimates | | | |
| Effect | Label | Exponentiate<br>Lowe | | | |
| trtpn | Treatment ratio, IDegLira - | - Lira 0.876 | 8 1.0228 | | |

NN9068
NN9068-4148
Clinical Trial Report
Statistical document

Date: 16 December 2019
Version: 1.0
Status: Final


## 30: Total cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C105586S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used 2

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.02679

Fit Statistics

-2 Res Log Likelihood -532.6
AIC (Smaller is Better) -530.6
AICC (Smaller is Better) -530.6
BIC (Smaller is Better) -526.0

Solution for Fixed Effects

Planned

Treatment Pre Trial for anti-Diabetic Period Standard Effect Estimate t Value Pr > |t| treatment2 01 (N) Error DF Alpha 0.05 Intercept 0.4849 0.04556 713 10.64 <.0001 trtpn -0.03161 0.01495 713 -2.11 0.0348 0.05 trtpn 0.003833 0.01736 713 0.22 0.8253 0.05 3 trtpn PREOAD2 0.01028 Metformin 0.01304 713 0.79 0.4307 0.05 PREOAD2 Metformin + OAD base log 0.6563 0.02899 713 22.64 <.0001 0.05

## NN9068 | Date: 16 December 2019 | Novo Nordisk NN9068-4148 | CONFIDENTIAL | Version: 1.0 | Clinical Trial Report | Status: Final |  |

Total cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set Parameter Code = C105586S

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 0.3955<br>-0.06095<br>-0.03025 | 0.5744<br>-0.00226<br>0.03791 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | Ü | -0.01533 | 0.03590 |
| base log | 1100101111111 1 0112 | | 0.5994 | 0.7133 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|------------|--------------|------------------|
| trtpn<br>PREOAD2 | 2 | 713<br>713 | 3.78<br>0.62 | 0.0232<br>0.4307 |
| base_log | 1 | 713 | 512.47 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | WORK.ADATA2 | 1.4372 | 0.008628 | 713 | 166.58 | <.0001 | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | 1.4727 | 0.01230 | 713 | 119.76 | <.0001 | 0.05 |
| trtpn | LSMeans, Lira | WORK.ADATA2 | 1.4688 | 0.01221 | 713 | 120.27 | <.0001 | 0.05 |

#### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | IDegLira | 1.4203 | 1.4542 | 4.2090 | 4.1383 | 4.2809 |
| trtpn | LSMeans, | IDeg | 1.4485 | 1.4968 | 4.3609 | 4.2569 | 4.4674 |
| trtpn | LSMeans, | Lira | 1.4449 | 1.4928 | 4.3442 | 4.2413 | 4.4496 |

### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | WORK.ADATA2 | -0.03544 | 0.01503 | 713 | -2.36 | 0.0186 |

#### Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | -0.06495 | -0.00593 | 0.9652 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.9371 | 0.9941 |

| NN9068<br>NN9068-4148<br>Clinical Trial<br>Statistical doc | Report | CC | ONFIDENTIAL | | rsion:<br>atus: | 16 Decem | 1.0 Final 68 of 412 |
|---|---|---|---|---|---|---|---|
| Total chole | Total cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set | | | | | | |
| Parameter C | Parameter Code=C105586S | | | | | | |
| The Mixed F | The Mixed Procedure | | | | | | |
| Least Squares Means Estimates | | | | | | | |
| Effect Lab | pel | | Margins | Estimate | Standard<br>Error | DF t V | alue Pr > t |
| trtpn Tre | eatment ratio, | IDegLira - Lira | WORK.ADATA2 | -0.03161 | 0.01495 | 713 - | 2.11 0.0348 |
| | | Least Squar | es Means Esti | mates | | | |
| Effect Lab | oel | | Alpha | Lower | Upper | Exponenti | ated |
| trtpn Tre | eatment ratio, | IDegLira - Lira | 0.05 -0 | .06095 | -0.00226 | 0. | 9689 |
| | Leas | st Squares Means | Estimates | | | | |
| Effect Lab | pel | | Exponentiate<br>Lowe | | nentiated<br>Upper | | |
| trtpn Tre | eatment ratio, | IDegLira - Lira | 0.940 | 9 | 0.9977 | | |


Total cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code= $T_CHOL_U$ 

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 718

Number of Observations

Number of Observations Read 720 Number of Observations Used 718 Number of Observations Not Used 2

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.02679

Fit Statistics

-2 Res Log Likelihood -532.6
AIC (Smaller is Better) -530.6
AICC (Smaller is Better) -530.6
BIC (Smaller is Better) -526.0

Solution for Fixed Effects

Planned Treatment for Period Pre Trial anti-Diabetic Standard 01 (N) Effect Estimate t Value Pr > |t| treatment2 Error DF Alpha Intercept 1.7405 0.1502 713 11.59 <.0001 0.05 trtpn 1 -0.03161 0.01495 713 -2.11 0.0348 0.05 trtpn 2 0.003833 0.01736 713 0.22 0.8253 0.05 trtpn PREOAD2 3 0 0.01028 0.01304 713 0.79 0.4307 0.05 Met.formin PREOAD2 Metformin + OAD 0.6563 0.02899 713 22.64 <.0001 0.05 base log

## NN9068 NN9068-4148 Clinical Trial Report Statistical document Date: 16 December 2019 Version: 1.0 Status: Final 

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.4457<br>-0.06095<br>-0.03025 | 2.0354<br>-0.00226<br>0.03791 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -0.01533 | 0.03590 |
| base log | | | 0.5994 | 0.7133 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 713 | 3.78 | 0.0232 |
| PREOAD2 | 1 | 713 | 0.62 | 0.4307 |
| base log | 1 | 713 | 512.47 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLira | WORK.ADATA2 | 5.0907 | 0.008628 | 713 | 590.03 | <.0001 | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | 5.1262 | 0.01230 | 713 | 416.87 | <.0001 | 0.05 |
| trtpn | LSMeans, Lira | WORK.ADATA2 | 5.1224 | 0.01221 | 713 | 419.42 | <.0001 | 0.05 |

#### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | 5.0738 | 5.1077 | 162.51 | 159.78 | 165.29 |
| trtpn | LSMeans, | | 5.1020 | 5.1503 | 168.37 | 164.36 | 172.49 |
| trtpn | LSMeans, | | 5.0984 | 5.1463 | 167.73 | 163.76 | 171.80 |

### Least Squares Means Estimates

| | | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Label | | Margins | Estimate Error DF t V | | t Value | Pr > t | | |
| trtnn | Treatment ratio | TDegLira - | TDea | WORK ADATA? | -0 03544 | 0 01503 | 713 | -2 36 | 0 0186 |

#### Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | -0.06495 | -0.00593 | 0.9652 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.9371 | 0.9941 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019 Novo Nordisk<br>1.0<br>Final<br>371 of 412 | | | | |
|---|---|---|---|--|--|--|--|
| Total cholesterol after 26 weeks of treatment - supportive statistical analysis - full analysis set | | | | | | | |
| Parameter Code=T_CHOL_U | | | | | | | |
| The Mixed Procedure | | | | | | | |
| Least Squares Means Estimates | | | | | | | |
| Effect Label | Margins | Estimate Standard Error | DF t Value Pr > t | | | | |
| trtpn Treatment ratio, I | IDegLira - Lira WORK.ADATA2 | -0.03161 0.01495 | 713 -2.11 0.0348 | | | | |
| Least Squares Means Estimates | | | | | | | |
| Effect Label | Alpha | Lower Upper | Exponentiated | | | | |
| trtpn Treatment ratio, I | IDegLira - Lira 0.05 -0 | .06095 -0.00226 | 0.9689 | | | | |
| Least Squares Means Estimates | | | | | | | |
| Effect Label | Exponentiate<br>Lowe | | | | | | |
| trtpn Treatment ratio, I | IDegLira - Lira 0.940 | 9 0.9977 | | | | | |
| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 372 of 412 | |

## 31: Free fatty acid after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=C80200S

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method Model-Based
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 717

Number of Observations

Number of Observations Read 720 Number of Observations Used 717 Number of Observations Not Used 3

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.3464

Fit Statistics

-2 Res Log Likelihood 1291.7 AIC (Smaller is Better) 1293.7 AICC (Smaller is Better) 1293.7 BIC (Smaller is Better) 1298.3

Solution for Fixed Effects

Planned

Treatment Pre Trial for anti-Diabetic Standard Period Effect Estimate DF t Value Pr > |t| treatment2 01 (N) Error Alpha -0.7292 0.06369 712 <.0001 0.05 Intercept -11.45 trtpn -0.3934 0.05383 712 -7.31 -7.68 <.0001 0.05 trtpn -0.4788 0.06237 712 <.0001 0.05 trtpn PREOAD2 -0.03614 712 -0.77 0.4410 0.05 Metformin 0.04688 PREOAD2 Metformin + OAD 0.2984 base log 0.05385 712 5.54 <.0001 0.05

# NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Free fatty acid after 26 weeks of treatment - supportive statistical analysis - full analysis set Parameter Code=C80200S

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | -0.8542<br>-0.4991<br>-0.6013 | -0.6041<br>-0.2877<br>-0.3564 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | 3 | -0.1282 | 0.05590 |
| base log | MECTOTIMIN + OND | | 0.1927 | 0.4042 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 712 | 35.68 | <.0001 |
| PREOAD2 | 1 | 712 | 0.59 | 0.4410 |
| base log | 1 | 712 | 30.71 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, IDegLir | WORK.ADATA2 | -1.3691 | 0.03102 | 712 | -44.14 | <.0001 | 0.05 |
| trtpn | LSMeans, IDeg | WORK.ADATA2 | -1.4546 | 0.04415 | 712 | -32.95 | <.0001 | 0.05 |
| trtpn | LSMeans, Lira | WORK.ADATA2 | -0.9757 | 0.04400 | 712 | -22.17 | <.0001 | 0.05 |

### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | -1.4300 | -1.3082 | 0.2543 | 0.2393 | 0.2703 |
| trtpn | LSMeans, | | -1.5413 | -1.3679 | 0.2335 | 0.2141 | 0.2546 |
| trtpn | LSMeans, | | -1.0621 | -0.8894 | 0.3769 | 0.3457 | 0.4109 |

### Least Squares Means Estimates

| | | | | | | Standard | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Label | | | Margins | Estimate | Error | DF | t Value | Pr > t |
| trtnn | Treatment ratio | TDeaLira - | TDea | WORK ADATA? | 0 08544 | 0 05397 | 712 | 1 58 | 0 1138 |

#### Least Squares Means Estimates

| Effect | Label | | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | -0.02052 | 0.1914 | 1.0892 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.9797 | 1.2109 |

| NN9068<br>NN9068-41<br>Clinical Tri<br>Statistical d | ial Report | CC | ONFIDENTIAL | | ersion:<br>atus: | 16 December 2019 Novo Nordisk<br>1.0<br>Final<br>374 of 412 | |
|---|---|---|---|---|---|---|---|
| Free fatt | Free fatty acid after 26 weeks of treatment - supportive statistical analysis - full analysis set | | | | | | |
| Parameter | Code=C80200S | | | | | | |
| The Mixed | d Procedure | | | | | | |
| Least Squares Means Estimates | | | | | | | |
| Effect L | Label | | Margins | Estimate | Standard<br>Error | DF t Value | Pr > t |
| trtpn T | Treatment ratio, | IDegLira - Lira | WORK.ADATA2 | -0.3934 | 0.05383 | 712 -7.31 | <.0001 |
| | | Least Squar | res Means Esti | mates | | | |
| Effect L | Label | | Alpha | Lower | Upper | Exponentiated | |
| trtpn T | Treatment ratio, | IDegLira - Lira | 0.05 - | 0.4991 | -0.2877 | 0.6748 | |
| | Leas | st Squares Means | Estimates | | | | |
| Effect L | Label | | Exponentiate<br>Lowe | | nentiated<br>Upper | | |
| trtpn T | Treatment ratio, | IDegLira - Lira | 0.607 | 1 | 0.7500 | | |


Free fatty acid after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=FFAU

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable aval\_log
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 717

Number of Observations

Number of Observations Read 720 Number of Observations Used 717 Number of Observations Not Used 3

Covariance Parameter Estimates

Cov Parm Estimate
Residual 0.3464

Fit Statistics

-2 Res Log Likelihood 1291.7 AIC (Smaller is Better) 1293.7 AICC (Smaller is Better) 1293.7 BIC (Smaller is Better) 1298.3

Solution for Fixed Effects

Planned Treatment for Period Pre Trial anti-Diabetic Standard Effect 01 (N) Estimate t Value Pr > |t| treatment2 Error DF Alpha Intercept 0.1442 712 11.19 <.0001 0.05 trtpn 1 -0.3934 0.05383 712 -7.31 < .0001 0.05 trtpn 2 -0.4788 0.06237 712 -7.68 <.0001 0.05 trtpn PREOAD2 0 -0.03614 0.04688 712 -0.77 0.4410 0.05 Met.formin PREOAD2 Metformin + OAD 0.2984 0.05385 712 5.54 <.0001 0.05 base log

# NN9068 | Date: 16 December 2019 | Novo Nordisk NN9068-4148 | Confidential | Version: 1.0 | Status: Final |  |

Free fatty acid after 26 weeks of treatment - supportive statistical analysis - full analysis set

Parameter Code=FFAU

The Mixed Procedure

Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 1.3304<br>-0.4991<br>-0.6013 | 1.8966<br>-0.2877<br>-0.3564 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | Ü | -0.1282 | 0.05590 |
| base log | riccioimili / OAD | | 0.1927 | 0.4042 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| trtpn | 2 | 712 | 35.68 | <.0001 |
| PREOAD2 | 1 | 712 | 0.59 | 0.4410 |
| base log | 1 | 712 | 30.71 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, ID | Değ | WORK.ADATA2 | 1.9702 | 0.03102 | 712 | 63.51 | <.0001 | 0.05 |
| trtpn | LSMeans, ID | | WORK.ADATA2 | 1.8847 | 0.04415 | 712 | 42.69 | <.0001 | 0.05 |
| trtpn | LSMeans, Li | | WORK.ADATA2 | 2.3636 | 0.04400 | 712 | 53.71 | <.0001 | 0.05 |

### Least Squares Means Estimates

| Effect | Label | | Lower | Upper | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|---|
| trtpn | LSMeans, | _ | 1.9093 | 2.0311 | 7.1720 | 6.7482 | 7.6223 |
| trtpn | LSMeans, | | 1.7981 | 1.9714 | 6.5847 | 6.0380 | 7.1809 |
| trtpn | LSMeans, | | 2.2772 | 2.4500 | 10.6289 | 9.7492 | 11.5880 |

### Least Squares Means Estimates

| | | | | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Label | | Margins | Estimate | Error | DF | t Value | Pr > t |
| trtpn | Treatment ratio. | TDeglira - TDeg | WORK ADATA2 | 0.08544 | 0.05397 | 712 | 1.58 | 0.1138 |

#### Least Squares Means Estimates

| Effect | Label | Alpha | Lower | Upper | Exponentiated | |
|---|---|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.05 | -0.02052 | 0.1914 | 1.0892 |

| Effect | Label | | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| trtpn | Treatment ratio, | IDegLira - IDeg | 0.9797 | 1.2109 |

| | -4148<br>Гrial Report<br>I document | CONFIDENTIAL | Version:<br>Status:<br>Page: | | 1.0<br>nal<br>12 |
|---|---|---|---|---|---|
| Free fa | Free fatty acid after 26 weeks of treatment - supportive statistical analysis - full analysis set | | | | |
| Paramet | Parameter Code=FFAU | | | | |
| The Mix | The Mixed Procedure | | | | |
| Least Squares Means Estimates | | | | | |
| Effect | Label | Margins | Standa<br>Estimate Erm | ard<br>cor DF t Value | Pr > t |
| trtpn | Treatment ratio, IDegL: | ira - Lira WORK.ADATA | 2 -0.3934 0.053 | 712 -7.31 | <.0001 |
| | 1 | Least Squares Means Es | timates | | |
| Effect | Label | Alpha | Lower Uppe | er Exponentiated | |
| trtpn | Treatment ratio, IDegL | ira - Lira 0.05 | -0.4991 -0.287 | 0.6748 | |
| | Least Squa | ares Means Estimates | | | |
| Effect | Label | Exponentia<br>Lo | ted Exponentiate<br>wer Uppe | | |
| trtpn | Treatment ratio, IDegL: | ira - Lira 0.6 | 0.750 | 00 | |

NN9068

Date:

16 December 2019 | Novo Nordisk

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 378 of 412 | |

## 32: Hypoglycaemic episodes - treatment emergent - confirmatory statistical analysis - full analysis set

Parameter Code=HYCNFSE

The GENMOD Procedure

Model Information

Data Set WORK.ANA\_DATA
Distribution Negative Binomial
Link Function
Dependent V

Dependent Variable Offset Variable AVAĹ Analysis Value logoff

Number of Observations Read Number of Observations Used Missing Values 713

Class Level Information

Levels Values Class 1 2 3 TRTPN

PREOAD2 Metformin Metformin + OAD

Parameter Information

Effect TRTPN PREOAD2 Parameter

Prm1 Intercept TRTPN 1
TRTPN 2
TRTPN 3
PREOAD2
PREOAD2 Prm2 Prm3 Prm4

Prm5 Metformin Prm6 Metformin + OAD

Iteration History For Parameter Estimates

| | | Log | | | | | |
|---|---|---|---|---|---|---|---|
| Iter | Ridge | Likelihood | Prm1 | Prm2 | Prm3 | Prm5 | Dispersion |
| 0 | 0 | -380.13843 | 4.8306049 | -0.036595 | -0.104861 | -0.051602 | 0.8802336 |
| 1 | 16 | -302.60682 | 4.5389129 | -0.1549 | -0.175903 | -0.142035 | 0.9183973 |
| 2 | 16 | -255.22114 | 4.2626473 | -0.251412 | -0.242057 | -0.226961 | 0.9503451 |
| 3 | 1 | -206.65271 | 2.8432976 | 0.1567368 | -0.10993 | -0.427447 | 0.0358785 |
| 4 | 1 | -202.3443 | 2.5892984 | 0.6980844 | 0.2589648 | -0.555308 | 0.0395708 |
| 5 | 1 | -200.99292 | 2.3670321 | 0.9318901 | 0.5113944 | -0.588845 | 0.043325 |
| 6 | 1 | -200.22341 | 2.198899 | 1.1100727 | 0.7072959 | -0.596857 | 0.0478977 |
| 7 | 1 | -199.73835 | 2.0671899 | 1.247524 | 0.8581409 | -0.59647 | 0.0535168 |
| 8 | 1 | -199.39683 | 1.9622075 | 1.3560667 | 0.9762753 | -0.593838 | 0.0605805 |
| 9 | 1 | -199.12347 | 1.8774354 | 1.443274 | 1.070397 | -0.590982 | 0.0697204 |
| 10 | 1 | -198.86994 | 1.8082494 | 1.5142491 | 1.1464569 | -0.588478 | 0.0819888 |
| 11 | 1 | -198.59526 | 1.751282 | 1.5725976 | 1.2086072 | -0.586426 | 0.0992653 |
| 12 | 1 | -198.24946 | 1.7040306 | 1.6209577 | 1.2598201 | -0.584788 | 0.1252315 |
| 13 | 1 | -197.74733 | 1.6646022 | 1.6613144 | 1.302261 | -0.583503 | 0.1680471 |
| 14 | 1 | -196.90293 | 1.6315452 | 1.695204 | 1.3374889 | -0.582535 | 0.2491751 |
| 15 | 1 | -195.23725 | 1.603746 | 1.7238705 | 1.3664613 | -0.581914 | 0.4401437 |
| 16 | 1 | -191.68986 | 1.5804119 | 1.7484509 | 1.389049 | -0.581882 | 1.0431561 |
| 17 | 1 | -187.56845 | 1.5611562 | 1.7700432 | 1.4034058 | -0.582981 | 2.7017295 |
| 18 | 0 | -186.76627 | 1.4976435 | 1.8401498 | 1.4556977 | -0.585191 | 6.8888986 |
| 19 | 0 | -186.39066 | 1.4866145 | 1.8515736 | 1.4690204 | -0.584467 | 5.1881713 |
| 20 | 0 | -186.38768 | 1.4871635 | 1.8506212 | 1.4690617 | -0.584092 | 5.0432744 |
| 21 | 0 | -186.38768 | 1.4871611 | 1.8506254 | 1.4690662 | -0.584093 | 5.0416978 |
| 2.2 | 0 | -186.38768 | 1.4871611 | 1.8506254 | 1.4690662 | -0.584093 | 5.0416978 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 379 of 412 | |

 ${\tt Hypoglycaemic\ episodes\ -\ treatment\ emergent\ -\ confirmatory\ statistical\ analysis\ -\ full\ analysis\ set}$ 

Parameter Code=HYCNFSE

The GENMOD Procedure

Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|---|---|---|---|
| Deviance Scaled Deviance Pearson Chi-Square Scaled Pearson X2 Log Likelihood Full Log Likelihood AIC (smaller is better) AICC (smaller is better) BIC (smaller is better) | 709<br>709<br>709<br>709 | 178.6787<br>178.6787<br>910.8445<br>910.8445<br>-186.3877<br>-197.5958<br>405.1916<br>405.2765<br>428.0391 | 0.2520<br>0.2520<br>1.2847<br>1.2847 |

Last Evaluation Of The Negative Of The Gradient and Hessian

| | Prm1 | Prm2 | Prm3 | Prm5 | Dispersion |
|------------|-----------|-----------|-----------|-----------|------------|
| Gradient | 4.5021E-9 | 8.37E-9 | 7.528E-10 | -1.755E-9 | 5.4659E-8 |
| Prm1 | 39.194138 | 26.152514 | 10.311714 | 9.5802638 | 0.0027883 |
| Prm2 | 26.152514 | 26.152514 | 0 | 6.9340316 | -0.018622 |
| Prm3 | 10.311714 | 0 | 10.311714 | 2.00561 | 0.0446241 |
| Prm5 | 9.5802638 | 6.9340316 | 2.00561 | 9.5802638 | 0.0038538 |
| Dispersion | 0.0027883 | -0.018622 | 0.0446241 | 0.0038538 | 0.2835077 |

Algorithm converged.

#### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidence | | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| Intercept | | 1 | 1.4872 | 0.6117 | 0.2882 | 2.6861 | 5.91 | 0.0151 |
| TRTPN | 1 | 1 | 1.8506 | 0.6363 | 0.6035 | 3.0978 | 8.46 | 0.0036 |
| TRTPN | 2 | 1 | 1.4691 | 0.6812 | 0.1338 | 2.8043 | 4.65 | 0.0310 |
| TRTPN | 3 | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 | | |
| PREOAD2 | Metformin | 1 | -0.5841 | 0.3726 | -1.3145 | 0.1463 | 2.46 | 0.1170 |
| PREOAD2 | Metformin + OAD | 0 | 0.0000 | 0.0000 | 0.0000 | 0.0000 | | |
| Dispersion | | 1 | 5.0417 | 1.8794 | 2.4281 | 10.4686 | | |

NOTE: The negative binomial dispersion parameter was estimated by maximum likelihood.

### TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|---|
| 1 | 3.0457 | 0.2142 | 14.22 | <.0001 | 0.05 | 2.6258 | 3.4656 | 21.0256 |
| 2 | 2.6642 | 0.3317 | 8.03 | <.0001 | 0.05 | 2.0141 | 3.3143 | 14.3562 |
| 3 | 1.1951 | 0.6135 | 1.95 | 0.0514 | 0.05 | -0.00724 | 2.3975 | 3.3039 |

TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Exponentiated Lower | Exponentiated<br>Upper |
|-----------------------------|---------------------|------------------------|
| 1 2 | 13.8162<br>7.4940 | 31.9969<br>27.5020 |
| 3 | 0.9928 | 10.9953 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 380 of 412 | |

Hypoglycaemic episodes - treatment emergent - confirmatory statistical analysis - full analysis set

Parameter Code=HYCNFSE

The GENMOD Procedure

#### Differences of TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| 1 | 2 | 0.3816 | 0.3688 | 1.03 | 0.3008 | 0.05 | -0.3412 | 1.1044 |
| 1 | 3 | 1.8506 | 0.6363 | 2.91 | 0.0036 | 0.05 | 0.6035 | 3.0978 |
| 2 | 3 | 1.4691 | 0.6812 | 2.16 | 0.0310 | 0.05 | 0.1338 | 2.8043 |

#### Differences of TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Planned<br>Treatment<br>(N) | Exponentiated | Exponentiated<br>Lower | Exponentiated Upper |
|---|---|---|---|---|
| 1 | 2 3 3 | 1.4646 | 0.7109 | 3.0173 |
| 1 | | 6.3638 | 1.8285 | 22.1486 |
| 2 | | 4.3452 | 1.1432 | 16.5153 |

#### Least Squares Means Estimates

| Effect | Label | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| TRTPN<br>TRTPN | IDegLira / IDeg<br>IDegLira / Lira | 0.3816<br>1.8506 | | 1.03<br>2.91 | | | -0.3412<br>0.6035 | 1.1044 |

| Effect | Label | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| TRTPN | IDegLira / IDeg | 1.4646 | 0.7109 | 3.0173 |
| TRTPN | IDegLira / Lira | 6.3638 | 1.8285 | 22.1486 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 381 of 412 | |

## 33: Hypoglycaemic episodes - treatment emergent - statistical sensitivity analysis - multiple imputation - full analysis set

ANA SORT=2 Parameter Code=HYCNFSE Planned Treatment (N)=1 Statement Number=1

The MIANALYZE Procedure

Estimate

Model Information

Data Set WORK.LSM MI2 Data Set WORK. Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----

Parameter Between 0.000963 0.044886 0.045849 2.26E6 Estimate

Variance Information (1000 Imputations)

Relative Fraction
Increase Missing Relative
Parameter in Variance Information Efficiency

0.021473 Estimate 0.021022 0.999979

Parameter Estimates (1000 Imputations)

95% Confidence Std Error Limits DF Estimate Minimum Maximum Parameter 0.214125 2.618397 3.457751 2.26E6

2.986481

3.203014

Parameter Estimates (1000 Imputations)

t for HO:

3.038074

Parameter Theta0 Parameter=Theta0 Pr > |t|14.19 <.0001 Estimate

#### NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

 $\mbox{Hypoglycaemic episodes - treatment emergent - statistical sensitivity analysis - multiple imputation - full analysis set \\$ 

ANA SORT=2 Parameter Code=HYCNFSE Planned Treatment (N)=2 Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSM MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.107840 0.110161 2.25E6 Estimate 0.002318

Variance Information (1000 Imputations)

Relative Fraction Missing

2.665038

Estimate

Relative Increase Information Parameter in Variance Efficiency 0.021518 0.021065 0.999979 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum 0.331905 2.014517 3.315560 2.25E6

2.592518

2.921904

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|0 8.03 <.0001 Estimate

#### NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

 $\mbox{Hypoglycaemic episodes - treatment emergent - statistical sensitivity analysis - multiple imputation - full analysis set \\$ 

ANA SORT=2 Parameter Code=HYCNFSE Planned Treatment (N)=3 Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSM MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance----Between Within Total DF Parameter 0.334826 0.373891 91512 Estimate 0.039026

Variance Information (1000 Imputations)

Relative

Fraction Missing Relative Increase Information Parameter in Variance Efficiency 0.116673 0.104502 0.999896 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence DF Parameter Estimate Std Error Limits Minimum Maximum 0.611466 -0.02079 2.376142 91512 1.003454 2.309467

Parameter Estimates (1000 Imputations)

1.177674

Estimate

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter 0 1.93 0.0541 Estimate

#### NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

 $\mbox{Hypoglycaemic episodes - treatment emergent - statistical sensitivity analysis - multiple imputation - full analysis set \\$ 

ANA SORT=2 Parameter Code=HYCNFSE Label=IDegLira / IDeg Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME MI2

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter 0.133550 0.136031 Estimate 0.002478 3E6

Variance Information (1000 Imputations)

Fraction Missing Relative

Relative Increase Parameter in Variance Information Efficiency 0.018575 0.018237 0.999982 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Parameter Estimate Std Error Limits DF Minimum Maximum 0.373036 0.368824 -0.34985 1.095918 3E6 0.121602 0.511817 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|

0 1.01 0.3118 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

 $\mbox{Hypoglycaemic episodes - treatment emergent - statistical sensitivity analysis - multiple imputation - full analysis set \\$ 

ANA SORT=3 Parameter Code=HYCNFSE Planned Treatment (N)=1 Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSM MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.045685 0.045994 2.22E7 Estimate 0.000309

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Information Parameter in Variance Efficiency 0.006760 0.006715 0.999993 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Estimate Std Error Limits

DF Parameter Minimum Maximum 0.214463 2.600497 3.441176 2.22E7 2.985600 3.127575 3.020836 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter Pr > |t|

0 14.09 <.0001 Estimate

#### NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

 $\mbox{Hypoglycaemic episodes - treatment emergent - statistical sensitivity analysis - multiple imputation - full analysis set \\$ 

ANA SORT=3 Parameter Code=HYCNFSE Planned Treatment (N)=2 Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSM MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter

0.108684 0.110788 2.77E6 Estimate 0.002102

Variance Information (1000 Imputations)

Relative Fraction Missing Increase

Relative Information Parameter in Variance Efficiency 0.019355 0.018989 0.999981 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence

DF Parameter Estimate Std Error Limits Minimum Maximum 0.332848 2.010241 3.314982 2.77E6 2.602009 2.921904 2.662611 Estimate

Parameter Estimates (1000 Imputations)

t for HO:

Theta0 Parameter=Theta0 Parameter Pr > |t|0 8.00 <.0001 Estimate

#### NN9068 Date: 16 December 2019 Novo Nordisk NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

 $\mbox{Hypoglycaemic episodes - treatment emergent - statistical sensitivity analysis - multiple imputation - full analysis set \\$ 

ANA SORT=3 Parameter Code=HYCNFSE Planned Treatment (N)=3 Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSM MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter 0.335631 0.374599 92316

Estimate 0.038929

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Information Parameter in Variance Efficiency 0.116104 0.104046 0.999896 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence Estimate Std Error Limits

DF Parameter Minimum Maximum 1.175999 0.612045 -0.02360 2.375601 92316 1.005759 2.300105 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Pr > |t| Parameter

0 1.92 0.0547 Estimate

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 **CONFIDENTIAL** Clinical Trial Report Status: Final Statistical document 

 $\mbox{Hypoglycaemic episodes - treatment emergent - statistical sensitivity analysis - multiple imputation - full analysis set \\$ 

ANA SORT=3 Parameter Code=HYCNFSE Label=IDegLira / Lira Statement Number=1

The MIANALYZE Procedure

Model Information

Data Set WORK.LSME MI3

Number of Imputations 1000

Variance Information (1000 Imputations)

-----Variance-----Between Within Total DF Parameter 0.363910 0.402410 109140 Estimate 0.038461

Variance Information (1000 Imputations)

Relative Fraction Missing

Relative Increase Information Parameter in Variance Efficiency 0.105795 0.095690 0.999904 Estimate

Parameter Estimates (1000 Imputations)

95% Confidence

DF Parameter Estimate Std Error Limits Minimum Maximum 0.634358 0.601505 3.088170 109140 0.750524 2.067895 1.844837 Estimate

Parameter Estimates (1000 Imputations)

t for HO: Theta0 Parameter=Theta0 Parameter

Pr > |t|0 2.91 0.0036 Estimate

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 389 of 412 | |

## 34: Hypoglycaemic episodes - treatment emergent - supportive statistical analysis - full analysis set

Parameter Code=HYCNFSES

The GENMOD Procedure

Model Information

Data Set WORK.ANA\_DATA
Distribution Negative Binomial
Link Function Log

Dependent Variable AVAL Analysis Value Offset Variable logoff

Number of Observations Read 720 Number of Observations Used 713 Missing Values 7

Class Level Information

Class Levels Values TRTPN 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Parameter Information

Parameter Effect TRTPN PREOAD2

 Prm1
 Intercept

 Prm2
 TRTPN
 1

 Prm3
 TRTPN
 2

 Prm4
 TRTPN
 3

 Prm5
 PREOAD2
 Metformin

 Prm6
 PREOAD2
 Metformin + OAD

Iteration History For Parameter Estimates

| | | Log | | | | | |
|---|---|---|---|---|---|---|---|
| Iter | Ridge | Likelihood | Prm1 | Prm2 | Prm3 | Prm5 | Dispersion |
| 0 | 0 | -353.06722 | 4.8066601 | -0.074818 | -0.131729 | -0.020934 | 0.861409 |
| 1 | 16 | -266.30919 | 4.49535 | -0.204286 | -0.209027 | -0.112915 | 0.8962711 |
| 2 | 16 | -210.74259 | 4.1900096 | -0.317233 | -0.284518 | -0.199872 | 0.9218333 |
| 3 | 16 | -173.55805 | 3.8503107 | -0.415706 | -0.366987 | -0.291605 | 0.9418687 |
| 4 | 1 | -143.6538 | 3.0355129 | -0.140169 | -0.327641 | -0.370119 | 0.8064204 |
| 5 | 1 | -135.39985 | 2.4869883 | 0.2781764 | -0.163044 | -0.420301 | 1.5551127 |
| 6 | 1 | -131.14278 | 2.0944005 | 0.6753206 | 0.0960382 | -0.432245 | 3.435585 |
| 7 | 0 | -128.32846 | 1.2717192 | 1.5420922 | 1.0071474 | -0.38109 | 8.3037715 |
| 8 | 0 | -127.62792 | 0.5784988 | 2.2398711 | 1.7079566 | -0.362035 | 6.2854472 |
| 9 | 0 | -127.59326 | 0.3486607 | 2.469668 | 1.937593 | -0.365232 | 6.226675 |
| 10 | 0 | -127.59288 | 0.3209942 | 2.4973578 | 1.9652698 | -0.365305 | 6.2291019 |
| 11 | 0 | -127.59288 | 0.3206337 | 2.4977184 | 1.9656304 | -0.365306 | 6.2291245 |
| 12 | 0 | -127.59288 | 0.3206337 | 2.4977184 | 1.9656304 | -0.365306 | 6.2291245 |

Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|--------------------------|-----|-----------|----------|
| Deviance | 709 | 123.9740 | 0.1749 |
| Scaled Deviance | 709 | 123.9740 | 0.1749 |
| Pearson Chi-Square | 709 | 1089.6976 | 1.5370 |
| Scaled Pearson X2 | 709 | 1089.6976 | 1.5370 |
| Log Likelihood | | -127.5929 | |
| Full Log Likelihood | | -132.8504 | |
| AIC (smaller is better) | | 275.7008 | |
| AICC (smaller is better) | | 275.7856 | |
| BIC (smaller is better) | | 298.5482 | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIALE | Status: | Final | |
| Statistical document | | Page: | 390 of 412 | |

Hypoglycaemic episodes - treatment emergent - supportive statistical analysis - full analysis set

Parameter Code=HYCNFSES

The GENMOD Procedure

Last Evaluation Of The Negative Of The Gradient and Hessian

| | Prm1 | Prm2 | Prm3 | Prm5 | Dispersion |
|------------|-----------|-----------|-----------|-----------|------------|
| Gradient | 5.7947E-8 | -5.49E-13 | 7.89E-13 | 1.6345E-8 | -6.43E-10 |
| Prm1 | 25.276692 | 18.132024 | 6.1824107 | 6.7687429 | 0.0081878 |
| Prm2 | 18.132024 | 18.132024 | 0 | 5.2170454 | -0.004494 |
| Prm3 | 6.1824107 | 0 | 6.1824107 | 1.2857398 | 0.0171082 |
| Prm5 | 6.7687429 | 5.2170454 | 1.2857398 | 6.7687429 | -0.006032 |
| Dispersion | 0.0081878 | -0.004494 | 0.0171082 | -0.006032 | 0.1016866 |

Algorithm converged.

### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidence | | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| Intercept<br>TRTPN<br>TRTPN<br>TRTPN | 1<br>2<br>3 | 1<br>1<br>1<br>0 | 0.3206<br>2.4977<br>1.9656<br>0.0000 | 1.0271<br>1.0462<br>1.0966<br>0.0000 | -1.6924<br>0.4472<br>-0.1836<br>0.0000 | 2.3337<br>4.5483<br>4.1148<br>0.0000 | 0.10<br>5.70<br>3.21 | 0.7549<br>0.0170<br>0.0730 |
| PREOAD2<br>PREOAD2<br>Dispersion | Metformin<br>Metformin + OAD | 1<br>0<br>1 | -0.3653<br>0.0000<br>6.2291 | 0.4505<br>0.0000<br>3.1372 | -1.2484<br>0.0000<br>2.3213 | 0.5178<br>0.0000<br>16.7154 | 0.66 | 0.4175 |

NOTE: The negative binomial dispersion parameter was estimated by maximum likelihood.

### TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|---|
| 1 | 2.6357 | 0.2536 | 10.39 | <.0001 | 0.05 | 2.1387 | 3.1327 | 13.9531 |
| 2 | 2.1036 | 0.4232 | 4.97 | <.0001 | 0.05 | 1.2741 | 2.9331 | 8.1957 |
| 3 | 0.1380 | 1.0245 | 0.13 | 0.8929 | 0.05 | -1.8700 | 2.1460 | 1.1480 |

TRTPN Least Squares Means

| Treatment (N) | Exponentiated Lower | Exponentiated Upper |
|---------------|---------------------|---------------------|
| 1 | 8.4884 | 22.9357 |
| 2 | 3.5755 | 18.7858 |
| 3 | 0.1541 | 8.5504 |

#### Differences of TRTPN Least Squares Means

| Planned<br>Treatment | Planned<br>Treatment | | Standard | | | | | |
|---|---|---|---|---|---|---|---|---|
| (N) | (N) | Estimate | | z Value | Pr > z | Alpha | Lower | Upper |
| 1 | 2 | 0.5321 | 0.4672 | 1.14 | 0.2547 | 0.05 | -0.3836 | 1.4478 |

#### Differences of TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Planned<br>Treatment<br>(N) | Exponentiated | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|
| 1 | 2 | 1.7025 | 0.6814 | 4.2537 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 391 of 412 | |

Hypoglycaemic episodes - treatment emergent - supportive statistical analysis - full analysis set Parameter Code=HYCNFSES

The GENMOD Procedure

#### Differences of TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| 1 2 | 3 | 2.4977 | 1.0462 | 2.39 | 0.0170 | 0.05 | 0.4472 | 4.5483 |
| | 3 | 1.9656 | 1.0966 | 1.79 | 0.0730 | 0.05 | -0.1836 | 4.1148 |

### Differences of TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Planned<br>Treatment<br>(N) | Exponentiated | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|
| 1 2 | 3 | 12.1547<br>7.1394 | 1.5639<br>0.8323 | 94.4701<br>61.2429 |

#### Least Squares Means Estimates

| Effect | Label | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| TRTPN<br>TRTPN | IDegLira / IDeg<br>IDegLira / Lira | | 0.4672<br>1.0462 | | 0.2547<br>0.0170 | | | 1.4478<br>4.5483 |

| Effect | Label | Exponentiated | Exponentiated<br>Lower | Exponentiated<br>Upper |
|---|---|---|---|---|
| TRTPN | IDegLira / IDeg | 1.7025 | 0.6814 | 4.2537 |
| TRTPN | IDegLira / Lira | 12.1547 | 1.5639 | 94.4701 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 392 of 412 | |

## 35: Nocturnal hypoglycaemic episodes - treatment emergent - supportive statistical analysis - full analysis set

Parameter Code=HYNOCSE

The GENMOD Procedure

Model Information

WORK.ANA\_DATA Data Set WORK.ANA\_DATA
Distribution Negative Binomial
Link Function Log
Dependent Variable AVAL
Offset Variable logoff Data Set

Analysis Value

Number of Observations Read Number of Observations Used Missing Values

Class Level Information

Levels Class Values

TRTPN 1 2

PREOAD2 Metformin Metformin + OAD

Parameter Information

Effect TRTPN PREOAD2 Parameter

Intercept
TRTPN 1
TRTPN 2
PREOAD2
PREOAD2 Prm1 Prm2 Prm3

Metformin Metformin + OAD Prm5

Iteration History For Parameter Estimates

| Iter | Ridge | Log<br>Likelihood | Prm1 | Prm2 | Prm4 | Dispersion |
|---|---|---|---|---|---|---|
| ICEI | Riage | HIREITHOOG | ETIIIT | FIIIZ | FIIIT | Dispersion |
| 0 | 0 | -243.64107 | 4.637979 | 0.0194619 | 0.0260575 | 0.8386892 |
| 1 | 16 | -184.26619 | 4.3981381 | -0.1288 | -0.045806 | 0.8662332 |
| 2 | 1 | -68.411958 | 2.935821 | -0.434955 | -0.206637 | 0.0121826 |
| 3 | 0.06 | -58.692105 | 2.1873247 | -0.320872 | -0.130925 | 0.0128597 |
| 4 | 0.06 | -57.230315 | 1.7003907 | -0.150367 | -0.025395 | 0.0151914 |
| 5 | 0.06 | -57.13682 | 1.5241268 | -0.041456 | 0.0331984 | 0.0206355 |
| 6 | 0.06 | -57.110943 | 1.4998604 | -0.020569 | 0.0424738 | 0.0343106 |
| 7 | 0.06 | -56.971669 | 1.4982316 | -0.018939 | 0.0431973 | 0.1151813 |
| 8 | 1 | -56.947602 | 1.4981784 | -0.018898 | 0.0432318 | 0.1298369 |
| 9 | 1 | -56.917385 | 1.4981527 | -0.018879 | 0.0432527 | 0.1485335 |
| 10 | 1 | -56.878466 | 1.4981399 | -0.018875 | 0.0432673 | 0.1731113 |
| 11 | 1 | -56.826753 | 1.4981338 | -0.018879 | 0.0432803 | 0.2066582 |
| 12 | 1 | -56.755364 | 1.4981313 | -0.018892 | 0.043295 | 0.2547 |
| 13 | 1 | -56.652094 | 1.498131 | -0.018915 | 0.0433146 | 0.32794 |
| 14 | 1 | -56.494193 | 1.4981321 | -0.018952 | 0.0433443 | 0.4491921 |
| 15 | 1 | -56.238368 | 1.4981344 | -0.019017 | 0.043395 | 0.6726469 |
| 16 | 1 | -55.810424 | 1.4981378 | -0.019144 | 0.0434916 | 1.1394896 |
| 17 | 1 | -55.147082 | 1.4981417 | -0.019409 | 0.0436941 | 2.2055893 |
| 18 | 1 | -54.385791 | 1.498142 | -0.019956 | 0.0441147 | 4.4431574 |
| 19 | 0 | -54.054726 | 1.498489 | -0.023739 | 0.0471084 | 38.111462 |
| 20 | 0 | -53.520173 | 1.4987877 | -0.02712 | 0.0502384 | 19.488384 |
| 21 | 0 | -53.506363 | 1.4984434 | -0.02461 | 0.0479554 | 17.083396 |
| 22 | 0 | -53.506335 | 1.4984612 | -0.024704 | 0.0480491 | 16.976997 |
| 23 | 0 | -53.506335 | 1.4984612 | -0.024704 | 0.0480488 | 16.976758 |


Nocturnal hypoglycaemic episodes - treatment emergent - supportive statistical analysis - full analysis set

Parameter Code=HYNOCSE

The GENMOD Procedure

Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|---|---|---|---|
| Deviance Scaled Deviance Pearson Chi-Square Scaled Pearson X2 Log Likelihood Full Log Likelihood AIC (smaller is better) AICC (smaller is better) | 530<br>530<br>530<br>530 | 45.8965<br>45.8965<br>488.5132<br>488.5132<br>-53.5063<br>-54.8926<br>117.7853<br>117.8610 | 0.0866<br>0.0866<br>0.9217<br>0.9217 |
| BIC (smaller is better) | | 134.8993 | |

Last Evaluation Of The Negative Of The Gradient and Hessian

| | Prm1 | Prm2 | Prm4 | Dispersion |
|---|---|---|---|---|
| Gradient<br>Prm1<br>Prm2 | 1.703E-12<br>8.6322112<br>5.7634921 | 3.889E-12<br>5.7634921<br>5.7634921 | -2.15E-12<br>2.8522502<br>2.1928143 | 5.95E-12<br>0.0009603<br>0.0011125 |
| Prm4<br>Dispersion | 2.8522502 | 2.1928143<br>0.0011125 | 2.8522502 | -0.000068<br>0.0048804 |

Algorithm converged.

#### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidenc | | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| Intercept<br>TRTPN<br>TRTPN | 1 2 | 1<br>1<br>0 | 1.4985<br>-0.0247<br>0.0000 | 0.6139<br>0.7309<br>0.0000 | 0.2952<br>-1.4573<br>0.0000 | 2.7017<br>1.4079<br>0.0000 | 5.96<br>0.00 | 0.0147<br>0.9730 |
| PREOAD2<br>PREOAD2<br>Dispersion | Metformin + OAD | 1<br>0<br>1 | 0.0480<br>0.0000<br>16.9768 | 0.7320<br>0.0000<br>14.3149 | -1.3866<br>0.0000<br>3.2518 | 1.4827<br>0.0000<br>88.6320 | 0.00 | 0.9477 |

NOTE: The negative binomial dispersion parameter was estimated by maximum likelihood.

#### TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|---|
| 1 | 1.4978 | 0.4256 | 3.52 | 0.0004 | 0.05 | 0.6635 | 2.3320 | 4.4718 |
| 2 | 1.5225 | 0.6226 | 2.45 | 0.0145 | 0.05 | 0.3021 | 2.7428 | 4.5836 |

TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Exponentiated Lower | Exponentiated<br>Upper |
|-----------------------------|---------------------|------------------------|
| 1 2 | 1.9417<br>1.3527 | 10.2987<br>15.5312 |

| NN9068<br>NN9068-414<br>Clinical Trial<br>Statistical doc | Report | | CONFID | ENTIAL | Date:<br>Version<br>Status<br>Page: | | | 2019 <b>Novo Nordisk</b> 1.0 Final f 412 |
|---|---|---|---|---|---|---|---|---|
| Nocturnal analysis s | hypoglycaemic<br>et | episodes - | treatment e | emergent - | supportive | statistica | al analysis | - full |
| Parameter | Code=HYNOCSE | | | | | | | |
| The GENMOD | Procedure | | | | | | | |
| | | Differen | ces of TRTE | PN Least S | quares Mean | S | | |
| Planned<br>Treatment<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper |
| 1 | 2 | -0.02470 | 0.7309 | -0.03 | 0.9730 | 0.05 | -1.4573 | 1.4079 |
| | Differen | ces of TRTPN | Least Squa | ares Means | | | | |
| Planned<br>Treatment<br>(N) | Planned<br>Treatment<br>(N) | Exponentiate | | nentiated<br>Lower | Exponent | iated<br>Upper | | |
| 1 | 2 | 0.97 | 56 | 0.2329 | 4 | .0873 | | |
| | | | Court Court | oo Moone | Estimata | | | |
| | | | Least Squar | | ESTIMATE | | | |
| Effect L | abel | Estimate | Standard<br>Error | - | e Pr > z | Alpha | Lower | Upper |
| TRTPN I | DegLira / IDe | g -0.02470 | 0.7309 | -0.0 | 3 0.973 | 0.05 | -1.4573 | 1.4079 |
| | | Least Square | s Means Est | imate | | | | |
| Effect L | abel | Exponent | | ponentiat<br>Low | | entiated<br>Upper | | |
| TRTPN I | DegLira / IDe | g 0 | .9756 | 0.23 | 29 | 4.0873 | | |

# NN9068 | Date: 16 December 2019 | Novo Nordisk NN9068-4148 | CONFIDENTIAL | Version: 1.0 | Clinical Trial Report | Status: Final |  |

 ${\tt Nocturnal\ hypoglycaemic\ episodes\ -\ treatment\ emergent\ -\ supportive\ statistical\ analysis\ -\ full\ analysis\ set}$ 

Parameter Code=HYNOCSES

The GENMOD Procedure

Model Information

Data Set WORK.ANA\_DATA
Distribution Negative Binomial
Link Function Log
Dependent Variable AVAL

Dependent Variable AVAL Analysis Value Offset Variable logoff

Number of Observations Read 540 Number of Observations Used 533 Missing Values 7

Class Level Information

Class Levels Values

TRTPN 2 1 2 PREOAD2 2 Metformin Metformin + OAD

Parameter Information

Parameter Effect TRTPN PREOAD2

 Prm1
 Intercept

 Prm2
 TRTPN
 1

 Prm3
 TRTPN
 2

 Prm4
 PREOAD2
 Metformin

 Prm5
 PREOAD2
 Metformin + OAD

Iteration History For Parameter Estimates

| Iter | Ridge | Log<br>Likelihood | Prm1 | Prm2 | Prm4 | Dispersion |
|---|---|---|---|---|---|---|
| 0 | 0 | -239.38395 | 4.6320803 | 0.0130252 | 0.0267412 | 0.8307234 |
| 1 | 16 | -178.5201 | 4.3885276 | -0.137679 | -0.045836 | 0.8568435 |
| 2 | 1 | -52.915 | 2.7724072 | -0.477285 | -0.213908 | 0.0055764 |
| 3 | 0.06 | -43.169463 | 1.9833211 | -0.422206 | -0.099201 | 0.0055064 |
| 4 | 0 | -41.402752 | 1.4086308 | -0.303289 | 0.0916114 | 0.0000105 |
| 5 | 0 | -41.279967 | 1.1755251 | -0.21786 | 0.2104166 | 3.6292E-6 |
| 6 | 0 | -41.278755 | 1.1467312 | -0.202954 | 0.2269668 | 1.4011E-6 |
| 7 | 0 | -41.278755 | 1.1463672 | -0.202723 | 0.227155 | 4.7003E-7 |
| 8 | 0 | -41.278755 | 1.1463672 | -0.202723 | 0.227155 | 4.7001E-7 |

#### Criteria For Assessing Goodness Of Fit

| Criterion | DF | Value | Value/DF |
|---|---|---|---|
| Deviance<br>Scaled Deviance | 530<br>530 | 66.5575<br>66.5575 | 0.1256<br>0.1256 |
| Pearson Chi-Square | 530 | 506.8188 | 0.1230 |
| Scaled Pearson X2 | 530 | 506.8188 | 0.9563 |
| Log Likelihood | | -41.2788 | |
| Full Log Likelihood | | -41.2788 | |
| AIC (smaller is better) | | 90.5575 | |
| AICC (smaller is better) | | 90.6333 | |
| BIC (smaller is better) | | 107.6716 | |


Nocturnal hypoglycaemic episodes - treatment emergent - supportive statistical analysis - full analysis set

Parameter Code=HYNOCSES

The GENMOD Procedure

Last Evaluation Of The Negative Of The Gradient and Hessian

| | Prm1 | Prm2 | Prm4 | Dispersion |
|------------|-----------|-----------|-----------|------------|
| Gradient | 1.7262E-7 | 3.2856E-8 | 1.7575E-8 | 0.0300508 |
| Prm1 | 8.000001 | 5 | 3 | -0.000228 |
| Prm2 | 5 | 5 | 1.8918351 | 0.0041442 |
| Prm4 | 3 | 1.8918351 | 3 | -0.004008 |
| Dispersion | -0.000228 | 0.0041442 | -0.004008 | 141409.99 |

Algorithm converged.

### Analysis Of Maximum Likelihood Parameter Estimates

| Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Confidenc | | Wald<br>Chi-Square | Pr > ChiSq |
|---|---|---|---|---|---|---|---|---|
| Intercept<br>TRTPN<br>TRTPN | 1 2 | 1<br>1<br>0 | 1.1464<br>-0.2027<br>0.0000 | 0.6373<br>0.7303<br>0.0000 | -0.1027<br>-1.6341<br>0.0000 | 2.3954<br>1.2287<br>0.0000 | 3.24<br>0.08 | 0.0720<br>0.7813 |
| PREOAD2<br>PREOAD2<br>Dispersion | Metformin + OAD | 1<br>0<br>1 | 0.2272<br>0.0000<br>0.0000 | 0.7303<br>0.0000<br>0.0027 | -1.2043<br>0.0000 | 1.6586<br>0.0000 | 0.10 | 0.7558 |

NOTE: The negative binomial dispersion parameter was estimated by maximum likelihood.

#### TRTPN Least Squares Means

| Treatment (N) | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|---|
| 1 2 | 1.0572 | 0.4560 | 2.32 | 0.0204 | 0.05 | 0.1636 | 1.9509 | 2.8784 |
| | 1.2599 | 0.5852 | 2.15 | 0.0313 | 0.05 | 0.1130 | 2.4069 | 3.5252 |

TRTPN Least Squares Means

| Treatment (N) | Exponentiated Lower | Exponentiated<br>Upper |
|---------------|---------------------|------------------------|
| 1 2 | 1.1777<br>1.1197 | 7.0348<br>11.0992 |

#### Differences of TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | z Value | Pr > z | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| 1 | 2 | -0.2027 | 0.7303 | -0.28 | 0.7813 | 0.05 | -1.6341 | 1.2287 |

#### Differences of TRTPN Least Squares Means

| Planned<br>Treatment<br>(N) | Planned<br>Treatment<br>(N) | Exponentiated | Exponentiated<br>Lower | Exponentiated Upper |
|---|---|---|---|---|
| 1 | 2 | 0.8165 | 0.1951 | 3.4168 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 397 of 412 | |

 ${\tt Nocturnal\ hypoglycaemic\ episodes\ -\ treatment\ emergent\ -\ supportive\ statistical\ analysis\ -\ full\ analysis\ set}$ 

Parameter Code=HYNOCSES

The GENMOD Procedure

Least Squares Means Estimate

Upper TRTPN IDegLira / IDeg -0.2027 0.7303 -0.28 0.7813 0.05 -1.6341 1.2287

Least Squares Means Estimate

Exponentiated Exponentiated Exponentiated Upper Effect Label TRTPN IDegLira / IDeg 0.8165 0.1951 3.4168

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 398 of 412 | |

# 36: Pulse after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=C49676X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 61.0988

Fit Statistics

-2 Res Log Likelihood 5001.9
AIC (Smaller is Better) 5003.9
AICC (Smaller is Better) 5003.9
BIC (Smaller is Better) 5008.5

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t|Alpha 39.7507 2.4558 0.7136 715 715 16.19 <.0001 0.05 Intercept trtpn -1.1609 -1.63 0.1042 0.05 -5.4522 0.8252 715 -6.61 <.0001 0.05 trtpn trtpn PREOAD2 Metformin -0.1803 0.6226 715 -0.29 0.7722 0.05 PREOAD2 Metformin + OAD 0.5538 0.03075 715 18.01 <.0001 0.05 BASE

# NN9068 Date: 16 December 2019 Vovo Nordisk NN9068-4148 Version: 1.0 Clinical Trial Report Status: Final Statistical document 

Pulse after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=C49676X

The Mixed Procedure

Effect Label

trtpn Treatment contrast, IDegLira - IDeg

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 34.9293<br>-2.5619<br>-7.0723 | 44.5720<br>0.2401<br>-3.8322 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -1.4025 | 1.0420 |
| BASE | riccioimili / OAD | | 0.4934 | 0.6142 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 715 | 25.41 | <.0001 |
| PREOAD2 | 1 | 715 | 0.08 | 0.7722 |
| BASE | 1 | 715 | 324.30 | <.0001 |

#### Least Squares Means Estimates

| | | | | | | ndard | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Label | | Margins | Estimat | te I | Error | DF | t Value | Pr > t | : Alpha |
| trtpn | | IDegLira | WORK.ADATA2 | | | 4115 | 715 | 197.44 | <.000 | |
| trtpn | LSMeans, | | WORK.ADATA2 | | | 5843 | 715 | 131.71 | | |
| trtpn | LSMeans, | Lira | WORK.ADATA2 | 82.408 | 34 0. | 5828 | 715 | 141.41 | <.000 | 0.05 |
| | | | Least S | quares Mea | ans Estir | nates | | | | |
| | | | | | | | Expon | entiated | Exponer | |
| Effect | Label | | Lower | Upper | Exponer | ntiated | | Lower | | Upper |
| trtpn | LSMeans, | IDegLira | 80.4396 | 82.0554 | 1. | 929E35 | | 8.6E34 | 4. | 327E35 |
| trtpn | LSMeans, | | | 78.1032 | | 2.64E33 | | 8.384E32 | | 314E33 |
| trtpn | LSMeans, | Lira | 81.2642 | 83.5525 | 6. | 159E35 | | 1.962E35 | 1. | 934E36 |
| | | | Least S | quares Mea | ans Estir | nates | | | | |
| | | | | | | | St | andard | | |
| Effect | Label | | | Marg: | ins | Estima | ite | Error | DF t | : Value |
| trtpn | Treatment | contrast. | IDegLira - I | Dea WORK | .ADATA2 | 4.29 | 914 | 0.7147 | 715 | 6.00 |
| | | , | | | | | | | . = - | |
| | | | Least S | quares Mea | ans Estir | nates | | | | |
| Effect | Label | | | D > | 1+1 7.3 | -1 | T | | | |
| EIIect | Label | | | Pr > | ITI A. | .pha | Lower | Upper | Exponer | itiated |
| trtpn | Treatment | contrast, | IDegLira - I | Deg <.0 | 0001 ( | 0.05 | 2.8882 | 5.6945 | 7 | 73.0660 |
| Least Squares Means Estimates | | | | | | | | | | |

Exponentiated Exponentiated

Upper

297.23

Lower

17.9611

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | NFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 De | 1.0<br>Final<br>400 of 412 | Novo Nordisk |
|---|---|---|---|---|---|
| Pulse after 26 weeks of treatment - change analysis set | e from baseline - | supportive st | atistical | analysis - | full |
| Parameter Code=C49676X | | | | | |
| The Mixed Procedure | | | | | |
| Least Squ | ares Means Estima | tes | | | |
| | | St | andard | | |
| Effect Label | Margins | Estimate | Error | DF t Va | lue |
| trtpn Treatment contrast, IDegLira - Lir | a WORK.ADATA2 | -1.1609 | 0.7136 | 715 -1 | .63 |
| Least Squ | ares Means Estima | tes | | | |
| Effect Label | Pr > t Alp | ha Lower | Upper | Exponentia | ted |
| trtpn Treatment contrast, IDegLira - Lir | a 0.1042 0. | 05 -2.5619 | 0.2401 | 0.3 | 132 |
| Least Squares Means | Estimates | | | | |
| Effect Label | Exponentiated<br>Lower | Exponentia<br>Ur | ated<br>oper | | |

trtpn Treatment contrast, IDegLira - Lira 0.07716 1.2714

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Pulse after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=C49676X

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 61.0988

Fit Statistics

-2 Res Log Likelihood 5001.9 AIC (Smaller is Better) AICC (Smaller is Better) 5003.9 5003.9 BIC (Smaller is Better) 5008.5

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 715 <.0001 Intercept 39.7507 2.4558 16.19 0.05 trtpn 1 -1.1609 0.7136 715 -1.63 0.1042 0.05 -6.61 trtpn -5.4522 0.8252 715 < .0001 0.05 3 trtpn PREOAD2 -0.1803 0.6226 715 -0.29 0.7722 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.4462 0.03075 715 -14.51 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 402 of 412 | |

Pulse after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=C49676X

The Mixed Procedure

### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn<br>PREOAD2 | Motformin | 1<br>2<br>3 | 34.9293<br>-2.5619<br>-7.0723 | 44.5720<br>0.2401<br>-3.8322 |
| PREOAD2<br>PREOAD2<br>BASE | Metformin<br>Metformin + OAD | | -1.4025<br>-0.5066 | 1.0420 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|------------|---------------|------------------|
| trtpn<br>PREOAD2 | 2 1 | 715<br>715 | 25.41<br>0.08 | <.0001<br>0.7722 |
| BASE | 1 | 715 | 210.49 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 4.1169<br>-0.1744<br>5.2778 | 0.4115<br>0.5843<br>0.5828 | 715<br>715<br>715 | 10.00<br>-0.30<br>9.06 | <.0001<br>0.7654<br><.0001 |
| | Least Squares Means | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | | 3.3090<br>-1.3215<br>4.1337 | 4.9248<br>0.9727<br>6.4220 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 403 of 412 | |

# 37: Systolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=SYSBPMEA

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 112.91

Fit Statistics

-2 Res Log Likelihood 5441.9
AIC (Smaller is Better) 5443.9
AICC (Smaller is Better) 5443.9
BIC (Smaller is Better) 5448.5

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t|Alpha 54.8951 3.5822 715 715 <.0001 0.05 15.32 Intercept trtpn 0.3202 0.9699 0.33 0.7414 0.05 2.3622 1.1218 715 2.11 0.0356 0.05 trtpn trtpn PREOAD2 Metformin -0.1735 0.8456 715 -0.21 0.8375 0.05 PREOAD2 Metformin + OAD 0.5459 0.02725 715 20.03 <.0001 0.05 BASE

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 404 of 412 | |

Systolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=SYSBPMEA

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 47.8622<br>-1.5840<br>0.1598 | 61.9280<br>2.2244<br>4.5646 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -1.8337 | 1.4867 |
| BASE | 110010111111 1 0111 | | 0.4924 | 0.5994 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 715 | 2.80 | 0.0613 |
| PREOAD2 | 1 | 715 | 0.04 | 0.8375 |
| BASE | 1 | 715 | 401.30 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha |
|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | 125.34<br>127.38<br>125.02 | 0.5593<br>0.7942<br>0.7922 | 715<br>715<br>715 | 224.09<br>160.38<br>157.81 | <.0001 | 0.05<br>0.05<br>0.05 |
| | | Least Sq | uares Means | Estimates | | | | |
| Effect | Label | Lower | Upper E | xponentiated | Expo | nentiated<br>Lower | Exponentia<br>Up | ted |
| trtpn<br>trtpn<br>trtpn | LSMeans, IDegLira<br>LSMeans, IDeg<br>LSMeans, Lira | | 126.44<br>128.94<br>126.57 | 2.717E54<br>2.094E55<br>1.972E54 | | 9.06E53<br>4.402E54<br>4.164E53 | 8.147<br>9.956<br>9.342 | E55 |
| | | Least Sq | uares Means | Estimates | | | | |
| Effect | Label | | Margins | Estima | | andard<br>Error | DF t Va | lue |
| trtpn | Treatment contrast | , IDegLira - IDe | eg WORK.AD | ATA2 -2.04 | 20 | 0.9715 | 715 -2 | .10 |
| Least Squares Means Estimates | | | | | | | | |
| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentia | ted |
| trtpn | Treatment contrast | , IDegLira - IDe | eg 0.035 | 9 0.05 - | 3.9492 | -0.1347 | 0.1 | .298 |
| | Lea | st Squares Mean | s Estimates | | | | | |

| Effect | Label | | | | | Exponentiated Lower | Exponentiated Upper |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment | contrast, | IDegLira | - I | Deg | 0.01927 | 0.8739 |

| NN9068<br>NN9068-4148<br>Clinical Trial Report<br>Statistical document | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 16 December 2019<br>1.0<br>Final<br>405 of 412 | Novo Nordisk |
|---|---|---|---|---|
| Systolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set | | | | |
| Parameter Code=SYSBPMEA | | | | |
| The Mixed Procedure | | | | |
| | Least Squares Means Estim | ates | | |
| Effect Label | Margins | Estimate Err | | alue |
| trtpn Treatment contrast, ID | egLira - Lira WORK.ADATA2 | 0.3202 0.96 | i99 715 C | .33 |

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - Lira 0.7414 0.05 -1.5840 2.2244 1.3774

Least Squares Means Estimates

Exponentiated Exponentiated Lower Upper

trtpn Treatment contrast, IDegLira - Lira 0.2052 9.2480

Effect Label

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final 406 of 412 Statistical document Page:

Systolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=SYSBPMEA

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 112.91

Fit Statistics

-2 Res Log Likelihood 5441.9 AIC (Smaller is Better) AICC (Smaller is Better) 5443.9 BIC (Smaller is Better) 5448.5

Solution for Fixed Effects

Planned

Treatment Pre Trial for Period anti-Diabetic Standard Effect 01 (N) Estimate DF t Value Pr > |t| Alpha treatment2 Error 15.32 Intercept 54.8951 3.5822 715 <.0001 0.05 trtpn 1 0.3202 0.9699 715 0.33 0.7414 0.05 0.0356 2.11 trtpn 2.3622 1.1218 715 0.05 3 trtpn PREOAD2 -0.1735 0.8456 715 -0.21 0.8375 0.05 Metformin Metformin + OAD PREOAD2 BASE -0.4541 0.02725 715 -16.66 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 407 of 412 | |

Systolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=SYSBPMEA

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 47.8622<br>-1.5840<br>0.1598 | 61.9280<br>2.2244<br>4.5646 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | | -1.8337 | 1.4867 |
| BASE | Metrormin + OAD | | -0.5076 | -0.4006 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 715 | 2.80 | 0.0613 |
| PREOAD2 | 1 | 715 | 0.04 | 0.8375 |
| BASE | 1 | 715 | 277.68 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -1.1778 | 0.5593<br>0.7942<br>0.7922 | 715<br>715<br>715 | -5.76<br>-1.48<br>-4.47 | <.0001<br>0.1386<br><.0001 |
| Least Squares Means Estimates | | | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -4.3179<br>-2.7371<br>-5.0953 | -2.1216<br>0.3816<br>-1.9846 | | | |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIALE | Status: | Final | |
| Statistical document | | Page: | 408 of 412 | |

# 38: Diastolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=DIABPMEA

The Mixed Procedure

Model Information

Data Set WORK.ADATA2
Dependent Variable AVAL
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method Profile
Fixed Effects SE Method
Degrees of Freedom Method Residual

Class Level Information

Class Levels Values trtpn 3 1 2 3

PREOAD2 2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1
Columns in X 7
Columns in Z 0
Subjects 1
Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used 0

Covariance Parameter Estimates

Cov Parm Estimate
Residual 50.4183

Fit Statistics

-2 Res Log Likelihood 4864.5 AIC (Smaller is Better) 4866.5 AICC (Smaller is Better) 4866.5 BIC (Smaller is Better) 4871.0

Solution for Fixed Effects

Planned Treatment Pre Trial for anti-Diabetic Period Standard Effect treatment2 01 (N) Estimate Error DF t Value Pr > |t| Alpha 33.7874 -0.2455 2.3740 715 715 <.0001 0.7049 0.05 14.23 Intercept trtpn 0.6479 -0.38 0.05 -0.8356 0.7496 715 -1.11 0.2653 0.05 trtpn trtpn PREOAD2 Metformin 0.6531 0.5681 715 1.15 0.2507 0.05 PREOAD2 Metformin + OAD 0.5735 0.02907 715 19.73 <.0001 0.05 BASE


Diastolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=DIABPMEA

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn | | 1<br>2<br>3 | 29.1266<br>-1.5175<br>-2.3072 | 38.4483<br>1.0265<br>0.6360 |
| PREOAD2<br>PREOAD2 | Metformin<br>Metformin + OAD | Ü | -0.4622 | 1.7685 |
| BASE | 110010111111111111111111111111111111111 | | 0.5165 | 0.6306 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------|-----------|-----------|---------|--------|
| trtpn | 2 | 715 | 0.67 | 0.5102 |
| PREOAD2 | 1 | 715 | 1.32 | 0.2507 |
| BASE | 1 | 715 | 389.16 | <.0001 |

#### Least Squares Means Estimates

| Effect | Label | | Margins | Est | imate | Stand<br>Er | lard<br>ror | DF | t Value | Pr > | · t | Alpha |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | LSMeans, IDe<br>LSMeans, IDe<br>LSMeans, Lir | eg | WORK.ADATA<br>WORK.ADATA<br>WORK.ADATA | 2 79 | 0.6002 | 0.5 | 737<br>308<br>293 | 715<br>715<br>715 | 212.99<br>148.86<br>150.86 | <. | 0001<br>0001<br>0001 | 0.05<br>0.05<br>0.05 |
| Least Squares Means Estimates | | | | | | | | | | | | |
| Effect | Label | | Lower | Upp | er E | Exponent | iated | Expon | entiated<br>Lower | Expo | nentia<br>Up | ted |
| trtpn<br>trtpn<br>trtpn | LSMeans, IDe<br>LSMeans, IDe<br>LSMeans, Lir | eg | 78.8664<br>77.9680<br>78.8066 | 80.33<br>80.05<br>80.88 | 21 | 2.0 | 15E34<br>59E34<br>48E34 | | 1.783E34<br>7.262E33<br>1.68E34 | | 7.737<br>5.837<br>1.342 | E34 |
| Least Squares Means Estimates | | | | | | | | | | | | |
| Effect | Label | | | M | Margins | 5 | Estimat | | andard<br>Error | DF | t Va | lue |
| trtpn | Treatment con | ntrast, | IDegLira - | IDeg W | ORK.AI | DATA2 | 0.590 | 1 | 0.6492 | 715 | 0 | .91 |

#### Least Squares Means Estimates

| Effect | Label | | Pr > t | Alpha | Lower | Upper | Exponentiated |
|---|---|---|---|---|---|---|---|
| trtpn | Treatment contrast, | IDegLira - IDeg | 0.3636 | 0.05 | -0.6844 | 1.8646 | 1.8042 |

| Effect | Label | | | | Exponentiated Lower | Exponentiated<br>Upper |
|---|---|---|---|---|---|---|
| trtpn | Treatment c | contrast, | IDegLira - | IDeg | 0.5044 | 6.4535 |

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 410 of 412 | |

Diastolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=DIABPMEA

The Mixed Procedure

Least Squares Means Estimates

Effect Label Margins Estimate Standard Error DF t Value trtpn Treatment contrast, IDegLira - Lira WORK.ADATA2 -0.2455 0.6479 715 -0.38

Least Squares Means Estimates

Effect Label Pr > |t| Alpha Lower Upper Exponentiated trtpn Treatment contrast, IDegLira - Lira 0.7049 0.05 -1.5175 1.0265 0.7823

Least Squares Means Estimates

Exponentiated Lower Upper trtpn Treatment contrast, IDegLira - Lira 0.2193 2.7913

#### NN9068 16 December 2019 Novo Nordisk Date: NN9068-4148 Version: 1.0 CONFIDENTIAL Clinical Trial Report Status: Final Statistical document 

Diastolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=DIABPMEA

The Mixed Procedure

Model Information

Data Set WORK.ADATA2 Dependent Variable CHG Covariance Structure Diagonal Estimation Method REML Residual Variance Method Fixed Effects SE Method Degrees of Freedom Method Profile Model-Based Residual

Class Level Information

Class Levels Values

1 2 3

trtpn PREOAD2 Metformin Metformin + OAD

Dimensions

Covariance Parameters 1 7 Columns in X Columns in Z 0 Subjects Max Obs per Subject 720

Number of Observations

Number of Observations Read 720 Number of Observations Used 720 Number of Observations Not Used

Covariance Parameter Estimates

Cov Parm Estimate Residual 50.4183

Fit Statistics

-2 Res Log Likelihood 4864.5 AIC (Smaller is Better) AICC (Smaller is Better) 4866.5 4866.5 BIC (Smaller is Better) 4871.0

Solution for Fixed Effects

Planned Treatment Pre Trial for Period anti-Diabetic Standard Effect treatment2 01 (N) Estimate DF t Value Pr > |t| Alpha Error <.0001 Intercept 33.7874 2.3740 715 14.23 0.05 trtpn 1 -0.2455 0.6479 715 -0.38 0.7049 0.05 0.2653 trtpn -0.8356 0.7496 715 -1.110.05 3 trtpn PREOAD2 0.6531 0.5681 715 1.15 0.2507 0.05 Metformin PREOAD2 Metformin + OAD BASE -0.4265 0.02907 715 -14.67 <.0001 0.05

| NN9068 | | Date: | 16 December 2019 | Novo Nordisk |
|---|---|---|---|---|
| Clinical Trial Report | CONTIDENTIAL | Status: | Final | |
| Statistical document | | Page: | 412 of 412 | |

Diastolic blood pressure after 26 weeks of treatment - change from baseline - supportive statistical analysis - full analysis set

Parameter Code=DIABPMEA

The Mixed Procedure

#### Solution for Fixed Effects

| Effect | Pre Trial<br>anti-Diabetic<br>treatment2 | Planned<br>Treatment<br>for<br>Period<br>01 (N) | Lower | Upper |
|---|---|---|---|---|
| Intercept<br>trtpn<br>trtpn<br>trtpn<br>trtpn<br>PREOAD2 | Metformin | 1<br>2<br>3 | 29.1266<br>-1.5175<br>-2.3072<br>-0.4622 | 38.4483<br>1.0265<br>0.6360<br>1.7685 |
| PREOAD2<br>BASE | Metformin + OAD | | -0.4835 | -0.3694 |

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|------------------|-----------|------------|--------------|------------------|
| trtpn<br>PREOAD2 | 2 1 | 715<br>715 | 0.67<br>1.32 | 0.5102<br>0.2507 |
| BASE | 1 | 715 | 215.17 | <.0001 |

| Effect | Label | Margins | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | WORK.ADATA2<br>WORK.ADATA2<br>WORK.ADATA2 | -0.9261 | 0.3737<br>0.5308<br>0.5293 | 715<br>715<br>715 | -0.90<br>-1.74<br>-0.17 | 0.3690<br>0.0815<br>0.8643 |
| | Least Squares Mean | s Estimates | | | | | |
| Effect | Label | Alpha | Lower | Upper | | | |
| trtpn<br>trtpn<br>trtpn | Change from baseline, IDegLira<br>Change from baseline, IDeg<br>Change from baseline, Lira | 0.05 | -1.0697<br>-1.9681<br>-1.1295 | 0.3978<br>0.1160<br>0.9486 | | | |